## Janssen Vaccines & Prevention B.V.\*

#### Clinical Protocol

#### **Protocol Title**

A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Assess the Efficacy and Safety of Ad26.COV2.S for the Prevention of SARS-CoV-2-mediated COVID-19 in Adults **Aged 18 Years and Older** 

#### **ENSEMBLE**

## Protocol VAC31518COV3001; Phase 3

#### **AMENDMENT 7**

## VAC31518 (JNJ-78436735)

\* Janssen Vaccines & Prevention B.V. is a Janssen pharmaceutical company of Johnson & Johnson and is hereafter referred to as the sponsor of the study. The sponsor is identified on the Contact Information page that accompanies the protocol.

United States (US) sites of this study will be conducted under US Food & Drug Administration Investigational New Drug (IND) regulations (21 CFR Part 312).

## **Regulatory Agency Identifier Number:**

IND: 22657

Approved **Status:** 15 April 2022 Date:

EDMS-RIM-50860, 10.0 EDMS number:

GCP Compliance: This study will be conducted in compliance with Good Clinical Practice, and applicable regulatory

requirements.

#### **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

## PROTOCOL AMENDMENT SUMMARY OF CHANGES TABLE

| DOCUMENT HISTORY | | |
|-------------------|-------------------|---|
| Document | Date | |
| Amendment 7 | This document | |
| Amendment 6 | 04 September 2021 | |
| Amendment 5 | 07 May 2021 | |
| Amendment 4 | 22 February 2021 | |
| Amendment 3 | 14 December 2020 | |
| Amendment 2 | 29 October 2020 | |
| Amendment 1 | 15 September 2020 | |
| Original Protocol | 22 July 2020 | • |

## **Amendment 7 (This document)**

#### **Overall Rationale for the Amendment:**

Following emergency use authorization (EUA) by the United States (US) Food and Drug Administration (FDA), the conditional marketing authorization by the European Commission, all participants were gradually unblinded and a single dose of Ad26.COV2.S was offered to enrolled participants who initially received placebo. Also, the epidemic continued, and new variants of concern emerged, national recommendations introduced booster vaccinations. The final analyses of the study that described the double-blind phase has been completed and the primary and secondary objectives have been met. Further efficacy evaluations of the open-label data have limitations, due to the loss of the placebo group, due to the loss of randomization, as many participants in the placebo groups in the studies did not cross over to Ad26.COV2.S (eg. they received another vaccine), and unblinding (eg, the participants' knowledge of the number and type of doses received or the timing since vaccination), which could have led to behavioral changes impacting the results. Operational challenges have impacted the feasibility of a strict follow-up of any COVID-19 episode and active follow-up cannot be sustained. Because of these reasons, the protocol has been amended to reduce the number of on-site visits and to change the requirements for COVID-19 episode reporting by applying a passive follow-up approach. Participants in the Immunogenicity Subset will continue with the on-site study visits. There are no changes to follow-up of safety endpoints, including the reporting of adverse events of special interest (AESIs). Two analyses are still planned for the study, a first analysis will be conducted for the open-label phase of the study (using the initially designed "active" follow-up of COVD-19 events) and a second end of study analysis is planned (using passive follow-up of COVID-19 events). The changes made to the clinical protocol VAC31518COV3001 as part of Protocol Amendment 7 are listed below, including the rationale of each change and a list of all applicable sections.

| Section Number and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| Synopsis 1.2 Schema 1.3 Schedules of Activities 2.1 Study Rationale 3 OBJECTIVES AND ENDPOINTS 4.1 Overall Design 4.4 End-of-study Definition 5.5 Criteria for Temporarily Delaying Administration of Study Vaccination 6.5 Booster Vaccination 6.10 Prestudy and Concomitant Therapy 8 STUDY ASSESSMENTS AND PROCEDURES 8.1.2 Procedures in the Event of (Suspected) COVID-19 8.1.3.4 Case Definition for Asymptomatic or Undetected COVID-19 8.1.3.6 Clinical Severity Adjudication Committee 8.2 Safety Assessments 8.2.1 Physical Examinations 8.2.2 Vital Signs 8.3.1 Time Period and Frequency for Collecting Adverse Event, Medically- attended Adverse Event, Adverse Events of Special Interest, and Serious Adverse Event Information 8.10 Assessment and Procedures Related to Booster Vaccination 9.2.4.2 All Participants 10.2 Appendix 2: Clinical Laboratory Tests 10.3.6 Committees Structure 10.4.1 Adverse Event Definitions and Classifications 10.7 Appendix 7: MRU Questionnaire 10.8 Appendix 8: Medically-attended COVID-19 (MA-COV) Form | The number of on-site study visits has been reduced and management of new suspected COVID-19 episodes has been changed from active to passive follow-up, defined as safety follow-up by the site at Month 18 and Month 24 to document COVID-19 participant-reported events as (S)AEs and MAAEs and to record concomitant therapies associated with COVID-19. eCOA has been decommissioned. No further booster doses will be provided. | With the cross-over vaccinations, the initial double-blind, randomized, placebo-controlled design of this study has been replaced with an open-label design, where the placebo group has been lost and received primary and booster vaccination (within or outside of the study). Finally, constant evolution of the COVID-19 pandemic has impacted the practical implementation of a strict follow-up of new suspected COVID-19 episodes. |
| Synopsis 3 OBJECTIVES AND ENDPOINTS 9.1 Statistical Hypotheses 9.7 Safety Analysis 9.8 Analysis of the Open-label Crossover Phase, Open-label Booster Vaccination Phase | The endpoints of the open-label cross-over phase and passive follow-up phase have been added and more clarification on the open-label booster phase has been provided. The scope and endpoints of the end of study analysis have been added. | To more clearly differentiate between the endpoints of the open-label cross-over phase and the booster phase. In addition, the changes in the follow-up of new suspected COVID-19 episodes come with endpoints specific to the follow-up phase. |
| 10.4.3 Severity Criteria | Instructions were added on grading severity of thrombocytopenia AEs with platelet counts between >140,000/μL and <150,000/μL. | Due to a discrepancy in what the FDA toxicity grading scale and the Brighton collaboration case definitions define as abnormal in terms of platelet counts. |

# Clinical Protocol VAC31518COV3001 Amendment 7

# VAC31518 (JNJ-78436735)

| Section Number and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| Throughout the protocol | Minor errors and inconsistencies | Correction of minor errors and |
| | were corrected, and minor | inconsistencies. Addition of |
| | clarifications were added throughout | minor clarifications. Alignment |
| | the protocol. | across sections in the protocol. |

# **TABLE OF CONTENTS**

| PROT | OCOL AMENDMENT SUMMARY OF CHANGES TABLE | <u>2</u> |
|---|---|---|
| TABL | E OF CONTENTS | 5 |
| LIST | OF IN-TEXT TABLES AND FIGURES | 8 |
| | PROTOCOL SUMMARY | |
| 1.1. | Synopsis | |
| 1.2. | Schema | |
| 1.3. | Schedules of Activities | |
| 1.3.1.<br>1.3.2. | Non-immunogenicity or Non-Booster Subset Participants (As of Amendment 7) Immunogenicity and Booster Subset Participants | 41 |
| 1.3.3. | | |
| 1.3.4. | ( ) ( ) | |
| 1.3.4. | , | |
| 1.3.4.2 | · | |
| 1.3.5. | Participants with a Suspected AESI | 60 |
| | INTRODUCTION | |
| 2.1. | Study Rationale | |
| 2.2. | Background | |
| 2.3. | Benefit-Risk Assessment | |
| 2.3.1 | Risks Related to Study Participation | |
| 2.3.2 | Benefits of Study Participation | |
| 2.3.3 | Benefit-Risk Assessment of Study Participation | |
| <b>3.</b> (3.1. | OBJECTIVES AND ENDPOINTS Double-blind Phase of the Study | |
| 3.1. | Open-label Active Phase | |
| 3.2.1. | Open-label Cross-over Phase | |
| 3.2.2. | Open-label Booster Phase | |
| 3.3. | Open-label Passive Follow-up Phase | |
| 4. | STUDY DESIGN | 93 |
| 4.1. | Overall Design | 93 |
| 4.2. | Scientific Rationale for Study Design | |
| 4.2.1. | Study-Specific Ethical Design Considerations | |
| 4.3. | Justification for Dose | 102 |
| 4.4. | End-of-study Definition | 102 |
| | STUDY POPULATION | |
| 5.1. | Inclusion Criteria | |
| 5.2. | Exclusion Criteria | |
| 5.3. | Lifestyle Considerations | |
| 5.4. | Screen Failures | |
| 5.5. | Criteria for Temporarily Delaying Administration of Study Vaccination | 110 |
| | STUDY VACCINATION AND CONCOMITANT THERAPY | |
| 6.1. | Study Vaccines Administered | |
| 6.2. | Preparation/Handling/Storage/Accountability | |
| 6.3. | Measures to Minimize Bias: Randomization and Blinding | |
| 6.4. | Unblinding and Open-label Phase | |
| 6.5. | Booster Vaccination Study Vaccine Compliance | |
| 6.6.<br>6.7. | Dose Modification | |
| 6.8. | Continued Access to Study Vaccine After the End of the Study | |
| 6.9. | Treatment of Overdose | |
| 0.0. | Troubilities of Overladde | 120 |

| 6.10.<br>6.11. | Prestudy and Concomitant Therapy | |
|---|---|---|
| | ISCONTINUATION OF STUDY VACCINATION AND PARTICIPANT ISCONTINUATION/WITHDRAWAL | 122 |
| | Discontinuation of Study Vaccination | |
| 7.1. | | |
| 7.2. | Participant Discontinuation/Withdrawal From the Study | |
| 7.2.1. | Withdrawal From the Use of Research Samples | |
| 7.3. | Lost to Follow-up | 124 |
| 8. S | TUDY ASSESSMENTS AND PROCEDURES | 125 |
| 8.1. | Efficacy and Immunogenicity Assessments | |
| 8.1.1. | Prespecified Criteria for Suspected COVID-19 Prior to Protocol Amendment 7 | 128 |
| 8.1.2. | Procedures in the Event of (Suspected) COVID-19 | 129 |
| 8.1.2.1. | · | |
| 8.1.2.2. | | |
| 8.1.3. | Efficacy Assessments | |
| 8.1.3.1. | | |
| 8.1.3.2. | | |
| 8.1.3.3. | | |
| 8.1.3.4. | | |
| 8.1.3.5. | | |
| 8.1.3.6. | | |
| 8.1.4. | Immunogenicity Assessments | |
| 8.2. | Safety Assessments | |
| 8.2.1. | Physical Examinations (Until Amendment 7) | |
| 8.2.2. | Vital Signs | |
| 8.2.3. | Pregnancy Testing | |
| 8.2.4. | Clinical Laboratory Assessments | |
| 8.3. | Adverse Events, Serious Adverse Events, Medically-attended Adverse Events, Adverse | 140 |
| 0.5. | Events of Special Interest, and Other Safety Reporting | 147 |
| 8.3.1. | Time Period and Frequency for Collecting Adverse Event, Medically-attended Adverse | 177 |
| 0.0.1. | Event, Adverse Events of Special Interest, and Serious Adverse Event Information | 147 |
| 8.3.2. | Method of Detecting Adverse Events, Medically-attended Adverse Events, Adverse | 177 |
| 0.0.2. | Events of Special Interest, and Serious Adverse Events | 150 |
| 8.3.3. | Follow-up of Adverse Events, Medically-attended Adverse Events, Adverse Events of | 100 |
| 0.0.0. | Special Interest, and Serious Adverse Events | 151 |
| 8.3.4. | Regulatory Reporting Requirements for Serious Adverse Events | |
| 8.3.5. | Pregnancy | |
| 8.3.6. | Disease-related Events and Disease-related Outcomes Not Qualifying as Adverse | 102 |
| | Events or Serious Adverse Events | 152 |
| 8.3.7. | Adverse Events of Special Interest | |
| 8.3.7.1. | | |
| 8.4. | Virology Assessments | |
| 8.5. | Biomarkers | |
| 8.6. | Medical Resource Utilization. | |
| 8.7. | Risk Factor Assessment | |
| 8.8. | Participant Medical Information Prior to, During and After the Study (Real-world Data) | |
| 8.9. | Assessment and Procedures After EUA or Approval/Licensure and Implementation of | |
| | Protocol Amendment 4 | |
| 8.10. | Assessment and Procedures Related to Booster Vaccination | 156 |
| 9. S | TATISTICAL CONSIDERATIONS | 157 |
| 9.1. | Statistical Hypotheses | |
| 9.2. | Sample Size Determination | |
| 9.2.1. | Efficacy (Total Sample Size) | |
| 9.2.2. | Immunogenicity Subset (Double-blind Phase) | |
| 9.2.3. | Immunogenicity Correlates (Correlates Subset) | |
| 0.2.0. | minutings marky controlates (controlates capacity) | .00 |

| 004 | O-feb. | 400 |
|---|---|---|
| 9.2.4.<br>9.2.4.1. | Safety | |
| | , and the state of | |
| 9.2.4.2. | · | |
| 9.3. | Populations for Analysis Sets | |
| 9.4. | Participant Information | |
| 9.5. | Efficacy Analyses | |
| 9.5.1. | Primary Endpoints Evaluation | |
| 9.5.1.1. | , | |
| 9.5.2. | Secondary Endpoints | 167 |
| 9.5.3. | Exploratory Endpoints | 168 |
| 9.5.4. | Other Analyses | 168 |
| 9.6. | Immunogenicity Analyses | 169 |
| 9.6.1. | Immunogenicity Subset | 169 |
| 9.6.2. | Correlates of Risk | 169 |
| 9.7. | Safety Analysis | |
| 9.8. | Analysis of the Open-label Cross-over Phase, Open-label Booster Vaccination Phase | |
| 0.0. | and Open-label Passive Follow-up Phase | 171 |
| 9.8.1. | Sample Size Determination of Immunogenicity Subset (Open-label Booster Vaccination Phase) | |
| 9.8.2. | Immunogenicity Correlates (Correlates Subset) | |
| 9.8.3. | Efficacy Analyses | |
| 9.9. | Interim Analysis and Committees | 1/3 |
| 9.10. | Analyses for Cohort Unblinded Due to Administration of an Authorized/Licensed COVID- | |
| | 19 Vaccine | 1/4 |
| 40 0 | UDDODTING DOCUMENTATION AND OPERATIONAL CONCIDERATIONS | 475 |
| | UPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | |
| 10.1. | Appendix 1: Abbreviations | |
| 10.2. | Appendix 2: Clinical Laboratory Tests | |
| 10.3. | Appendix 3: Regulatory, Ethical, and Study Oversight Considerations | |
| 10.3.1. | Regulatory and Ethical Considerations | |
| 10.3.2. | Financial Disclosure | |
| 10.3.3. | Informed Consent Process | |
| 10.3.4. | Data Protection | 185 |
| 10.3.5. | Long-term Retention of Samples for Additional Future Research | 186 |
| 10.3.6. | Committees Structure | 186 |
| 10.3.7. | Publication Policy/Dissemination of Clinical Study Data | 188 |
| 10.3.8. | Data Quality Assurance | 189 |
| 10.3.9. | Case Report Form Completion | |
| 10.3.10 | · | |
| 10.3.11 | | |
| 10.3.12 | | |
| 10.3.13 | | |
| 10.3.14 | | |
| 10.4. | Appendix 4: Adverse Events, Serious Adverse Events, Adverse Events of Special | 102 |
| 10.4. | Interest, Medically-attended Adverse Events, Product Quality Complaints, and Other | |
| | Safety Reporting: Definitions and Procedures for Recording, Evaluating, Follow-up, and | |
| | | 104 |
| 40.4.4 | Reporting | |
| 10.4.1. | Adverse Event Definitions and Classifications | |
| 10.4.2. | Attribution Definitions | |
| 10.4.3. | Severity Criteria | |
| 10.4.4. | Special Reporting Situations | |
| 10.4.5. | Procedures | |
| 10.4.6. | Product Quality Complaint Handling | |
| 10.4.7. | Contacting Sponsor Regarding Safety, Including Product Quality | |
| 10.5. | Appendix 5: Contraceptive Guidance and Collection of Pregnancy Information | |
| 10.6. | Appendix 6: Symptoms of Infection with Coronavirus-19 (SIC) | |
| 10.7. | Appendix 7: MRU Questionnaire | |
| 10.8. | Appendix 8: Medically-attended COVID-19 (MA-COV) Form | 210 |

| Figure 1: | Schematic Overview of Study VAC31518COV3001 | 36 |
|-----------|---------------------------------------------|-----|
| Figure 2: | Decision Tree for COVID-19 Procedures | 131 |

## 1. PROTOCOL SUMMARY

## 1.1. Synopsis

A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Assess the Efficacy and Safety of Ad26.COV2.S for the Prevention of SARS-CoV-2-mediated COVID-19 in Adults Aged 18 Years and Older

With protocol Amendment 4, an unblinding visit was introduced at which participants who initially received placebo in the double-blind phase, and consent, receive a single dose of Ad26.COV2.S vaccine. Following the unblinding, the study is conducted in an open-label fashion.

With protocol Amendment 6, the open-label phase of the study is extended to include an open-label booster vaccination with a single dose of Ad26.COV2.S.

As of Amendment 7, the number of on-site visits for participants who are not part of the Immunogenicity Subset or Booster Subset is reduced. For these participants, any outstanding Visits 8 and 9 are cancelled. In addition, any outstanding Visits 10 and 11 are replaced by a phone call. No further booster vaccination will be provided in the protocol. In addition, active follow-up of new suspected COVID-19 will be replaced by passive surveillance (ie, follow-up by the site at Month 18 and Month 24 to document COVID-19 participant-reported events as [S]AEs and MAAEs) and to record concomitant therapies associated with COVID-19. During these calls, the protocol required safety information (eg SAEs, AESIs, MAAEs 6 month post booster) are also collected.

This study is being conducted under the sponsorship of Janssen (Janssen Vaccines & Prevention B.V) in collaboration with the COVID-19 Response Team (formerly known as Operation Warp Speed [OWS]), which also encompasses the Biomedical Advanced Research and Development Authority (BARDA), the National Institutes of Health (NIH), and the COVID-19 Prevention Trials Network (COVPN).

Ad26.COV2.S (previously known as Ad26COVS1) is a monovalent vaccine composed of a recombinant, replication-incompetent adenovirus type 26 (Ad26) vector, constructed to encode the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) spike (S) protein.

Information about the disease, correlates of immunity, and safety issues concerning this new pandemic-causing virus are rapidly evolving. Therefore, it is critical to recognize that the approach outlined in this document might or will change as insights and discussions evolve.

#### **OBJECTIVES AND ENDPOINTS**

## 1. Double-blind phase

The primary and secondary objectives and endpoints of the main study (ie, the double blind phase) are:

| Objectives | Endpoints |
|---|---|
| Co-Primary | |
| To demonstrate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed <sup>a</sup> , moderate to severe/critical coronavirus disease-2019 (COVID-19) <sup>b</sup> , as compared to placebo, in SARS-CoV-2 seronegative adults | <ul> <li>First occurrence of molecularly confirmed<sup>a</sup>, moderate to severe/critical COVID-19<sup>b</sup>, with onset at least 14 days after double-blind vaccination (Day 15)</li> <li>First occurrence of molecularly confirmed<sup>a</sup>, moderate to severe/critical COVID-19<sup>b</sup>, with onset at least 28 days after double-blind vaccination (Day 29)</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Secondary <sup>e</sup> (The method used to perform hypothesis testing preserving the Statistical Analysis Plan [SAP]) Efficacy | ng the family wise error rate [FWER] will be specified in |
| To demonstrate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed <sup>a</sup> , severe/critical COVID-19 <sup>b</sup> , as compared to placebo | • First occurrence of molecularly confirmed <sup>a</sup> , severe/critical COVID-19 <sup>b</sup> , with onset at least 14 days after double-blind vaccination (Day 15) |
| | • First occurrence of molecularly confirmed <sup>a</sup> , severe/critical COVID-19 <sup>b</sup> , with onset at least 28 days after double-blind vaccination (Day 29) |
| To demonstrate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , as compared to placebo, in | First occurrence of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , with onset 1 day after double-blind vaccination |
| adults regardless of their serostatus | First occurrence of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , with onset at least 14 days after double-blind vaccination (Day 15) |
| | • First occurrence of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , with onset at least 28 days after double-blind vaccination (Day 29) |
| To evaluate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed moderate to severe/critical COVID-19 <sup>b</sup> as compared to placebo, with onset 1 day after study vaccination | First occurrence of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> with onset 1 day after double-blind vaccination |
| To assess the effect of Ad26.COV2.S on COVID-19 requiring medical intervention (based on objective criteria) compared to placebo | • First occurrence of COVID-19 requiring medical intervention (such as a composite endpoint of hospitalization, ICU admission, mechanical ventilation, and ECMO, linked to objective measures such as decreased oxygenation, X-ray or CT findings) and linked to any molecularly confirmed <sup>a</sup> , COVID-19 <sup>b,c</sup> at least 14 days after double-blind vaccination (Day 15) |
| | • First occurrence of COVID-19 requiring medical intervention and linked to any molecularly confirmed <sup>a</sup> , COVID-19 <sup>b,c</sup> at least 28 days after double-blind vaccination (Day 29) |
| To assess the effect of Ad26.COV2.S on SARS-CoV-2 viral ribonucleic acid (RNA) load compared to placebo for moderate to severe/critical COVID-19 <sup>b</sup> | Assessment of the SARS-CoV-2 viral load by quantitative reverse-transcriptase polymerase chain reaction (RT-PCR), in participants with molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> by serial viral load measurements during the course of a COVID-19 episode |
| To assess the effect of Ad26.COV2.S on molecularly confirmed <sup>a</sup> mild COVID-19 <sup>c</sup> | • First occurrence of molecularly confirmed <sup>a</sup> , mild COVID-19 <sup>c</sup> , at least 14 days after double-blind vaccination (Day 15) |
| | • First occurrence of molecularly confirmed <sup>a</sup> , mild COVID-19 <sup>c</sup> , at least 28 days after double-blind vaccination (Day 29) |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Objectives | Endpoints |
|---|---|
| To assess the effect of Ad26.COV2.S on COVID-19 as defined by the United States (US) Food and Drug Administration (FDA) harmonized case definition <sup>d</sup> | First occurrence of molecularly confirmed COVID-<br>19d at least 14 days after double-blind vaccination<br>(Day 15) |
| | First occurrence of molecularly confirmed COVID-<br>19 <sup>d</sup> at least 28 days after double-blind vaccination<br>(Day 29) |
| To assess the effect of Ad26.COV2.S on all molecularly confirmed <sup>a</sup> symptomatic COVID-19 <sup>b,c</sup> , as compared to placebo | Burden of disease (BOD) endpoint derived from the first occurrence of molecularly confirmed symptomatic COVID-19 <sup>b,c</sup> (meeting the mild, moderate or severe/critical COVID-19 case definition) with onset at least 14 days after double-blind vaccination (Day 15). |
| | BOD endpoint <sup>f</sup> derived from the first occurrence of molecularly confirmed <sup>a</sup> symptomatic COVID-19 <sup>b,c</sup> (meeting the mild, moderate or severe/critical COVID-19 case definition) with onset at least 28 days after double-blind vaccination (Day 29). |
| To assess the effect of Ad26.COV2.S on occurrence of confirmed asymptomatic or undetected infections with SARS-CoV-2, as compared to placebo | <ul> <li>Serologic conversions: between baseline (Day 1; pre-vaccination) and Day 29, between Day 29 and Day 71, between Day 71 and Month 6 /Unblinding Visit, and Month 18 after double-blind vaccination (approximately 12 months after initiation of the open-label phase of the study) using an enzymelinked immunosorbent assay (ELISA) and/or SARS-CoV-2 immunoglobulin assay that is dependent on the SARS-CoV-2 nucleocapsid (N) protein</li> <li>Asymptomatic infection detected by RT-PCR at the time of the Month 6 /Unblinding Visit</li> </ul> |
| To assess the efficacy of Ad26.COV2.S in the prevention of SARS-CoV-2 infection (both symptomatic and asymptomatic infections combined, that are serologically and/or molecularly confirmed <sup>a</sup> ), as compared to placebo | First occurrence of SARS-CoV-2 infection (serologically and/or molecularly confirmed <sup>a</sup> ) with onset at least 28 days after double-blind vaccination (Day 29) |
| Safety | |
| To evaluate safety in terms of serious adverse events (SAEs) adverse events of special interest (AESIs) (during the entire study), medically-attended adverse events (MAAEs; until 6 months after double-blind or open-label vaccination), and MAAEs leading to study discontinuation (during the entire study) for all participants | Occurrence and relationship of SAEs and AESIs (during the entire study), MAAEs (until 6 months after [double-blind or open-label] Ad26.COV2.S), and MAAEs leading to study discontinuation (during the entire study) for all participants following vaccination |
| In a subset of participants, to evaluate the safety and reactogenicity in terms of solicited local and systemic adverse events (AEs) during 7 days after double-blind vaccination, and in terms of unsolicited AEs during 28 days after double-blind vaccination | Occurrence, intensity, duration, and relationship of solicited local and systemic AEs during the 7 days following vaccination and of unsolicited AEs during the 28 days after double-blind vaccination |

| Objectives | Endpoints |
|---|---|
| Immunogenicity | |
| In a subset of participants, to evaluate the immunogenicity of Ad26.COV2.S, as compared to placebo | Analysis of antibodies binding to the SARS-CoV-2 S protein by ELISA |

<sup>&</sup>lt;sup>a</sup> Molecularly confirmed COVID-19 is defined as a positive SARS-CoV-2 viral RNA result by a central laboratory using a RT-PCR based or other molecular diagnostic test.

Exploratory objectives and endpoints, including correlates of protection, durability of protection, immunogenicity, and evaluation of efficacy in seropositive participants and/or participants with a SARS-CoV-2 positive RT-PCR or molecular test result, are included in the body of this protocol.

## **Hypotheses**

The study is designed to test the co-primary hypotheses of vaccine efficacy (VE) in the PP population. For both co-primary endpoints, the following hypothesis will be tested:

H0:  $VE \le 30\%$  versus H1: VE > 30% and each hypothesis will be evaluated at a 2.5% one-sided significance level.

The co-primary endpoints will evaluate

- the first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to the case definition, with onset at least 14 days after double-blind vaccination with Ad26.COV2.S versus placebo, in the PP population, including all events from both age groups, with and without comorbidities.
- the first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to
  the case definition, with onset at least 28 days after double-blind vaccination with Ad26.COV2.S
  versus placebo, in the PP population, including all events from both age groups, with and without
  comorbidities.

If testing for both primary endpoint hypotheses is successful, secondary objectives will be evaluated against a null hypothesis employing a lower limit VE>0%. The method to perform hypothesis testing of primary and secondary objectives preserving the FWER will be specified in the SAP. The FWER will be controlled at 2.5% one-sided significance level.

<sup>&</sup>lt;sup>b</sup> Per case definition for moderate to severe/critical COVID-19 as determined by the Clinical Severity Adjudication Committee (see below).

<sup>&</sup>lt;sup>c</sup> Per case definition for mild COVID-19 as determined by the Clinical Severity Adjudication Committee (see below).

<sup>&</sup>lt;sup>d</sup> Per US FDA harmonized case definition for COVID-19 (see below).

<sup>&</sup>lt;sup>e</sup> All secondary efficacy endpoint analyses will occur in the per-protocol (PP) analysis set, in seronegative participants unless otherwise indicated in the Statistical Analysis Plan (SAP).

<sup>&</sup>lt;sup>f</sup>For more information and the definition of the BOD endpoint, refer to the body of the protocol.

#### 2. Open-label active phase

A diagram showing the study phases is provided below:



## 2.1 Open-label Cross-over Phase

Participant will enter the open-label crossover phase on the day that the participant received the cross-over vaccination or is unblinded until the day that the participant completed the booster visit. There are 2 main cohorts in the open-label phase:

- Early vaccinated cohort: participants who were initially randomized to the Ad26.COV2.S group and received 1 dose of Ad26.COV2.S at Day 1 in the trial
- Late vaccinated cohort: participants who were initially randomized to the placebo group and who received 1 dose of Ad26.COV2.S after unblinding

The main objective of the open-label phase of the study is to evaluate the COVID-19 outcomes after an early vaccination and after a late vaccination. Efficacy evaluations may be performed if feasible, ie, if pre-specified criteria are met, as specified in the SAP.

The secondary and exploratory objectives and endpoints for the open-label phase of the study are:

| Objectives | Endpoints |
|---|---|
| The secondary safety objective of the double-blind | The secondary safety endpoint of the double-blind phase |
| phase (see secondary double-blind objective) | (see secondary double-blind endpoint) |
| To evaluate molecularly confirmed <sup>a</sup> , symptomatic | Incidence of symptomatic COVID-19 cases starting at |
| COVID-19 <sup>b</sup> | 28 days after last vaccination |
| To evaluate molecularly confirmed <sup>a</sup> , severe/critical | Incidence of severe/critical COVID-19 cases starting at |
| COVID-19 <sup>b</sup> | 28 days after last vaccination |
| To evaluate molecularly confirmed <sup>a</sup> COVID-19 <sup>b</sup> requiring medical intervention (based on objective criteria) | Incidence of COVID-19 cases requiring medical intervention, starting at 28 days after last vaccination |
| To evaluate COVID-19 related death | Insidence of COVID 10 related deaths starting at |
| 10 evaluate CO v ID-19 fetated death | Incidence of COVID-19 related deaths starting at 28 days after last vaccination |

| Objectives | Endpoints |
|---|---|
| To describe the severity of breakthrough infections | The severity of COVID-19 cases may be evaluated by the severity and number of symptoms (severity) of COVID-19 cases, ratio of severe/critical COVID-19 cases and ratio of long COVID-19 cases (duration of more than 28 days) |
| To estimate potential correlate of risk/efficacy in relation to the primary endpoint of the main study and serious disease, hospitalization, and death based on immune responses in breakthrough cases compared to non-infected participants. | Levels of immune responses (antibody titers) and RNA sequencing analysis as available for participants having COVID-19 compared to non-infected participants. |

<sup>&</sup>lt;sup>a</sup> Molecularly confirmed COVID-19 is defined as a positive SARS-CoV-2 viral RNA result by a central laboratory using a RT-PCR based or other molecular diagnostic test.

## 2.2 Open-label booster phase

Participants will enter the booster phase on the day that the participants completed the booster visit until consenting to Amendment 7 (or with the stop of the eCOA at each study site, which ever date comes first). There are 3 main cohorts, based on vaccination schedules received during the booster phase:

- Homologous boost cohort consists of following 2 groups:
  - o participants who were initially randomized to the Ad26.COV2.S group and received 1 dose of Ad26.COV2.S at Day 1 within the trial and a booster dose preferably within 6 to 12 months after the initial vaccination, with a minimum of 3 months after the initial vaccination with Ad26.COV.2.S
  - o participants who were initially randomized to the placebo group and who received 1 dose of Ad26.COV2.S after unblinding and a booster dose preferably within 6 to 12 months after the initial vaccination, with a minimum of 3 months after the last vaccination with Ad26.COV.2.S
- Heterologous boost cohort: participants who were initially randomized to the placebo group and who received an mRNA vaccination outside of the trial and an Ad26.COV2 booster dose preferably within 6 to 12 months after the initial vaccination, with a minimum of 3 months after the last outside vaccination
- Non-boost cohort: participants who received 1 Ad26.COV2.S vaccination, either at Day 1 or as a cross-over vaccination. These participants remain in this cohort until they receive the booster vaccination. Participants who opt not to receive a booster dose will continue in this cohort.

Data from participants who received a different sequence of vaccinations (eg, Ad26.COV2 prime vaccination and an outside booster) will be presented separately.

The main objective of the booster phase of the study is to evaluate the COVID-19 outcomes, safety, and immunogenicity of the different schedules that were assessed: homologous Ad26.COV2 booster schedule, 1-dose schedule, and heterologous booster schedule. All analyses are descriptive, efficacy evaluations may be done if feasible, ie, if pre-specified criteria are met, as described in the SAP.

<sup>&</sup>lt;sup>b</sup> Per case definition for moderate to severe/critical COVID-19 as determined by the Clinical Severity Adjudication Committee (see below).

The primary and secondary objectives and endpoints for the booster phase of the study are:

| Objectives | Endpoints |
|---|---|
| Primary Objective of the Booster Phase To assess the safety and reactogenicity of Ad26.COV2.S at the 5×10 <sup>10</sup> vp dose level administered | Solicited local and systemic AEs for 7 days after booster vaccination. |
| as homologous or heterologous booster vaccination in adults. | Unsolicited AEs for 28 days after booster vaccination. |
| | SAEs and AESIs from booster vaccination until end of the study. |
| To measure the primary endpoints previously utilized for the double-blind portion of the study in this unblinded booster portion of the trial during the time participants have and have not been boosted. | • Incidence of the primary endpoints utilized in the double-blind portion of the study, including moderate to severe/critical COVID-19 cases starting at 28 days by serostatus*, in the unblinded booster portion of the study (see definitions of terms in Section 10.1) during the times when they have and have not been boosted. |
| To measure the primary endpoints previously utilized for the double-blind portion of the study in participants infected with selected variants and the reference strain in this unblinded booster portion of the trial during the time participants have and have not been boosted. | Incidence of the primary endpoints (Day 28 after vaccination) in the main study as applicable as described in the first objective but for variants of concern and the reference strain. |
| Secondary Objectives of the Booster Phase | |
| To evaluate the secondary endpoints previously utilized for the double-blind portion of the study in this unblinded booster portion of the trial during the time participants have and have not been boosted. | Incidence of secondary endpoints (Day 28 after vaccination) from the double-blind portion of the study by serostatus* such as symptomatic severe/critical disease, hospitalization, and death. |
| To evaluate the primary and secondary endpoints utilized in the double-blind portion of the study in this unblinded booster portion of the trial in participants primed or boosted with Ad26.COV2.S, mRNA, inactivated, protein, and other adenovector-based vaccines during the time participants have and have not been boosted. | Description of the primary and secondary endpoints (Day 28 after vaccination), such as symptomatic, severe/critical disease, hospitalization, and death, in the double-blind portion of the study as applicable as described in the first primary objective and first secondary objective including variants of concern and reference variants. |
| To estimate a correlate of immunity (correlate of risk) in relation to the primary endpoint of the main study and serious disease, hospitalization, and death based on immune responses at Day 28 after booster vaccination in boosted compared to non-boosted participants. | • Serological response to vaccination and antibody titers (VNA) against the original strain, 28 days after Ad26.COV2.S (5×10 <sup>10</sup> vp dose level) single-dose booster vaccination. |
| To estimate potential correlate of risk/efficacy in relation to the primary endpoint of the main study and serious disease, hospitalization, and death based on immune responses in breakthrough cases compared to non-infected participants. | Levels of immune responses (antibody titers) and<br>RNA sequencing analysis as available. |

| Objectives | Endpoints |
|---|---|
| To compare the immune responses in the Heterologous and Homologous Booster Subsets 28 Days following booster dose administration. | Qualitative comparison of responses in terms of<br>binding, neutralizing antibody against Wuhan<br>reference strain and variants of interest utilizing<br>wtVNA and/or psVNA, depending on feasibility. |
| | Analysis of antibodies binding to the SARS- CoV-<br>2S protein by ELISA. |
| To evaluate SARS-CoV-2 infection (severe/critical, moderate to severe/critical, symptomatic, and asymptomatic infections, that are serologically and/or molecularly confirmed**) for the different cohorts | Incidence of SARS-CoV-2 infections (serologically and/or molecularly confirmed**). |
| To describe the severity of breakthrough infections. | The severity of COVID-19 cases may be evaluated<br>by the severity and number of symptoms (severity)<br>of COVID-19 cases and ratio of long COVID-19<br>cases (duration of more than 28 days) |
| To obtain samples to evaluate potential thromboembolic events following booster immunization by obtaining platelet counts and sufficient extra sera for specialized studies at the day of booster immunization and 28 days later. | Platelet count on the day of booster vaccination and 28 days after booster vaccination. Additional analysis on kept sera samples in case of potential thromboembolic events. |

<sup>\*</sup> Seronegative is defined as N-serology seronegative at the time of boosting or at the Year 1 visit if not boosted.

## 4. Open-label Passive follow-up phase

With Amendment 7, the active follow-up of new suspected COVID-19 is replaced by a passive follow-up. Participants will enter this phase on the day of consenting to Amendment 7 (or with the stop of the eCOA at each study site, which ever date comes first) until end of study.

In the passive follow-up phase, the same cohorts as from the booster phase are included, and all data will be descriptively presented by cohort depending on the vaccination schedule received during the follow-up. Since COVID-19 reporting changed from an active approach to a passive approach, the effectiveness evaluations may be limited and will be described in the SAP as applicable.

The secondary and exploratory objectives and endpoints for the passive follow-up phase of the study are:

| Objectives | Endpoints |
|---|---|
| The secondary safety objective of the double-blind phase (see double-blind objectives). | The secondary safety endpoint of the double-blind phase (see double-blind endpoints). |
| To evaluate COVID-19 in terms of (S)AEs MAAEs, hospitalizations and fatal AEs linked to COVID-19* | SAEs and AEs linked to COVID-19. |
| | MAAEs linked to COVID-19 |
| | SAEs linked to COVID-19 that require hospitalization |
| | Fatal AEs linked to COVID-19 |
| In the immunogenicity subset of participants: to evaluate the immunogenicity of Ad26.COV2.S at available timepoints | Analysis of antibodies binding to the SARS-CoV-<br>2 S protein by ELISA |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

<sup>\*\*</sup> Molecularly confirmed COVID-19 is defined as a positive SARS-CoV-2 viral RNA result by a central laboratory using a RT-PCR based or other molecular diagnostic test.

| Objectives | Endpoints |
|---|---|
| In the Heterologous and Homologous Booster Subsets: to compare the immune responses 28 days following booster dose administration | |

<sup>\*</sup> Refer to Section 8.3 for the safety follow up and COVID 19 reporting requirements as of Protocol Amendment 7.

#### **Case Definitions**

The Clinical Severity Adjudication Committee will review all cases in the study, except for cases already adjudicated as severe, as a supplement to the algorithm described in the SAP, as well as those requiring medical intervention (such as a composite endpoint of hospitalization, ICU admission, mechanical ventilation, and ECMO, linked to objective measures such as decreased oxygenation, X-ray or CT findings), including date of onset of cases, taking into account all available relevant information at the time of adjudication. As of Amendment 7, Clinical Severity Adjudication Committee may review all cases based on available data from the passive follow-up (eg, limited to COVID-19 AE/SAE data, CIOMS forms, local laboratory results). Details will be provided in the revised charter of the Clinical Severity Adjudication Committee. Readjudication will occur if new information becomes available. The last adjudication for a given case will determine the status of the case for analysis. The Clinical Severity Adjudication Committee's assessment will be considered the definitive classification of the case. The case review including severity assessments after implementation of Protocol Amendment 7 may change and will be reflected in the charter of the committee.

The criteria for suspected COVID-19 are described in the body of the protocol. As several of the prespecified criteria for suspected COVID-19 overlap with vaccine-related reactogenicity, investigators' clinical judgement is required to exclude vaccine-related events when assessing suspected COVID-19.

## Case Definition for Moderate to Severe/Critical COVID-19

For the co-primary endpoints (see above), all moderate and severe/critical COVID-19 cases will be considered.

#### Case Definition for Moderate COVID-19

• A SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample

#### AND at any time during the course of observationa:

# Any 1 of the following new or worsening signs or symptoms:

- Respiratory rate ≥20 breaths/minute
- Abnormal saturation of oxygen (SpO<sub>2</sub>) but still >93% on room air at sea level\*
- Clinical or radiologic evidence of pneumonia
- Radiologic evidence of deep vein thrombosis (DVT)
- Shortness of breath or difficulty breathing

# Any 2 of the following new or worsening signs or symptoms:

- Fever ( $\ge 38.0^{\circ}$ C or  $\ge 100.4^{\circ}$ F)
- Heart rate ≥90 beats/minute
- Shaking chills or rigors
- Sore throat
- Cough
- Malaise as evidenced by 1 or more of the following\*\*:
  - Loss of appetite
  - Generally unwell
  - Fatigue
  - Physical weakness
- Headache
- Muscle pain (myalgia)
- Gastrointestinal symptoms (diarrhea, vomiting, nausea, abdominal pain)\*\*
- New or changing olfactory or taste disorders
- Red or bruised looking feet or toes

OR

## Case Definition for Severe/Critical COVID-19

• A SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample

## AND any 1 of the following at any time during the course of observation<sup>a</sup>:

- Clinical signs at rest indicative of severe systemic illness (respiratory rate ≥30 breaths/minute, heart rate ≥125 beats/minute, oxygen saturation (SpO<sub>2</sub>) ≤93% on room air at sea level\*, or partial pressure of oxygen/fraction of inspired oxygen (PaO<sub>2</sub>/FiO<sub>2</sub>) <300 mmHg)
  - \* SpO<sub>2</sub> criteria will be adjusted according to altitude per the investigator judgement.
- Respiratory failure (defined as needing high-flow oxygen, non-invasive ventilation, mechanical ventilation, or extracorporeal membrane oxygenation [ECMO])
- Evidence of shock (defined as systolic blood pressure <90 mmHg, diastolic blood pressure <60 mmHg, or requiring vasopressors)
- Significant acute renal, hepatic, or neurologic dysfunction

<sup>\*</sup> SpO<sub>2</sub> criteria will be adjusted according to altitude per the investigator judgement.

<sup>\*\*</sup> Having 2 or more elements of a symptom (eg, vomiting and diarrhea or fatigue and loss of appetite) is counted only as 1 symptom for the case definition. To meet the case definition, a participant would need to have at least 2 different symptoms.

<sup>&</sup>lt;sup>a</sup> Until Amendment 7, participants will be asked to undertake the COVID-19 procedures until 14 days after symptom onset (COVID-19 Day 15) or until **resolution of the COVID-19 episode**, whichever comes last (see Section 8.1.2).

- Admission to the ICU
- Death

All cases meeting the severe/critical criteria will be adjudicated by the Clinical Severity Adjudication Committee to determine if the case is severe/critical in their judgement.

All cases meeting the moderate case definition and that include  $\geq 3$  signs and/or symptoms from the list of signs and symptoms will be evaluated by the Clinical Severity Adjudication Committee to determine if the case is severe/critical in their judgement.

Classification of a case as severe/critical by the Clinical Severity Adjudication Committee is considered definitive.

#### **Case Definition for Mild COVID-19**

• A SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample

## AND at any time during the course of observationa:

• One of the following symptoms: fever (≥38.0°C or ≥100.4°F), sore throat, malaise (loss of appetite, generally unwell, fatigue, physical weakness), headache, muscle pain (myalgia), gastrointestinal symptoms, cough, chest congestion, runny nose, wheezing, skin rash, eye irritation or discharge, chills, new or changing olfactory or taste disorders, red or bruised looking feet or toes, or shaking chills or rigors.

A case is considered mild when it meets the above case definition but not the moderate to severe/critical definition.

## **US FDA Harmonized Case Definition for COVID-19**

If a participant presents with symptoms as those listed by the US FDA harmonized case definition (see appendix to the protocol), the investigator (or designated medically trained clinician) should assess if these are suggestive of COVID-19:

- A SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample; **AND**
- COVID-19 symptoms consistent with those defined by the US FDA harmonized case definition at the time of finalization of this protocol: fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea.

## Case Definition for Asymptomatic or Undetected COVID-19

If a participant does not fulfil the criteria for suspected COVID-19 based on signs and symptoms which would classify them as mild, moderate, or severe by the protocol definitions

#### AND

• has a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample

<sup>&</sup>lt;sup>a</sup> Until Amendment 7, participants will be asked to undertake the COVID-19 procedures until 14 days after symptom onset (COVID-19 Day 15) or until **resolution of the COVID-19 episode**, whichever comes last (see Section 8.1.2).

OR

• develops a positive serology (non-S protein) test

Then, the participant will be considered to have experienced asymptomatic or undetected COVID-19.

Cases will be classified as being an "Asymptomatic SARS-CoV-2 infection" by the Clinical Severity Adjudication Committee utilizing the following guidelines as applicable, which are described in more detail in the charter for the committee.

- The definition of any case that is either RT-PCR positive that was previously RT-PCR negative or seropositive for N protein specific antibodies that was previously seronegative for N protein specific antibodies and is clinically asymptomatic will be considered as an asymptomatic COVID-19 case.
- The definition of clinically asymptomatic COVID-19 is defined as no clinical symptoms that would be classified as mild, moderate, or severe COVID-19 by the protocol case definition for symptoms independent of the SARS-CoV-2 N protein specific antibody seroconversion or RT-PCR results.

Potential asymptomatic cases that are identified by N protein specific SARS-CoV-2 seroconversion will all be examined by the Clinical Severity Adjudication Committee for the presence of any signs or symptoms and if found, to determine if they would still be classified as asymptomatic COVID-19. Cases which are moderate, severe, hospitalized, or fatal that are found by SARS-CoV-2 N protein specific antibody seroconversion will be utilized in a sensitivity analysis to determine, if any conclusions would be changed by adding to the primary case definition of a positive RT-PCR with appropriate signs and symptoms to those cases which were identified by SARS-CoV-2 N protein specific antibody seroconversion with appropriate signs and symptoms.

As of Amendment 7, severity assessment by the CSAC may still be performed and will be based on the data collected through the passive follow-up (eg, hospitalization reported in the context of SAEs). The scope of the severity review may change and will be described in the charter.

#### OVERALL DESIGN

This is a multicenter, randomized, double-blind, placebo-controlled, Phase 3, pivotal efficacy and safety study in adults  $\ge 18$  to < 60 years of age and  $\ge 60$  years of age. The efficacy, safety, and immunogenicity of Ad26.COV2.S will be evaluated in participants living in, or going to, locations with high risk for acquisition of SARS-CoV-2 infection after administration of study vaccine.

Following EUA, conditional licensure, or approval in any country for the single dose regimen, based on the VAC31518COV3001 primary analysis results described in an interim report, all participants from countries where Amendment 4 is approved by the Health Authority and IEC/IRB will be unblinded at the on-site Month 6/Unblinding Visit. The study will then be conducted in an open-label fashion. A final analysis of the double-blind phase will be performed, using the data collected prior to unblinding, when all participants have completed the Month 6/Unblinding Visit or discontinued earlier. Depending on the operational implementation of the Month 6/Unblinding Visit, as well as the stage of the pandemic, this analysis may be conducted when a minimum of 90% of the study population has been unblinded.

All participants will be invited for an on-site Month 6/Unblinding Visit and participants who initially received placebo in the double-blind phase will be offered a single dose of Ad26.COV2.S vaccine.

Initial immunogenicity and safety data (28 days post-Dose 1 data from Cohort 1a and available data from Cohort 3) from study VAC31518COV1001 have demonstrated that a single dose of Ad26.COV2.S at  $5 \times 10^{10}$  vp and  $1 \times 10^{11}$  vp induces an immune response that meets prespecified minimum criteria and had an acceptable safety profile. The sponsor has therefore decided to proceed with the single dose regimen at a  $5 \times 10^{10}$  virus particles (vp) dose level in this Phase 3 study.

With protocol Amendment 6, the open-label phase of the study is extended to include an open-label booster vaccination with a single dose of Ad26.COV2.S at the Year 1/Booster Visit (see also below). The combination of homologous or heterologous prime/boost vaccination will not be randomized, but depends on what participants received during the double-blind phase of the study as described in this protocol. The start date of the first cross-over unblinding visit (implemented with Amendment 4) and the date of first booster vaccine administration until 1-year follow-up of the last booster vaccination define the open-label booster vaccination phase of the study. This phase will be utilized to describe safety, immunogenicity, and efficacy during the time participants have and have not been boosted.

With Amendment 7, active follow-up of suspected COVID-19 will be replaced by passive surveillance (ie, follow-up by the site at Month 18 and Month 24 to document new COVID-19 participant-reported events as [S]AEs and MAAEs) and to record concomitant therapies associated with COVID-19, if available. During these calls, the protocol required safety information (eg SAEs, AESIs, MAAEs 6 month post booster) are also collected.

Participants will be randomized in parallel in a 1:1 ratio to receive Ad26.COV2.S or placebo intramuscularly (IM) as shown in the table below. Ad26.COV2.S will be administered at a dose level of 5×10<sup>10</sup> vp. At the Month 6/Unblinding Visit, participants who initially received placebo and signed an amended ICF will be offered a single dose of Ad26.COV2.S. vaccine at a dose level of 5×10<sup>10</sup> vp. At the Year 1/Booster Visit, all ongoing participants in the study who have previously received any COVID-19 vaccination(s) (as primary regimen or additional dose) with the Ad26.COV2.S vaccine, and/or an mRNA vaccine or another COVID-19 vaccine authorized for primary vaccination including protein, inactivated, and adenovector-based vaccines, will be offered a single booster dose of Ad26.COV2.S vaccine (5×10<sup>10</sup> vp) if the last vaccination was preferably 6 months but at least 3 months ago.

Table: Vaccination Schedule VAC31518COV3001

| Group | N | Day 1 | Month 6/Unblinding Visit* | Year 1/Booster Visit |
|---|---|---|---|---|
| 1 | 20,000 | Ad26.COV2.S (5×10 <sup>10</sup> vp) | - | Ad26.COV2.S (5×10 <sup>10</sup> vp) |
| 2 | 20,000 | Placebo | Ad26.COV2.S $(5\times10^{10} \text{ vp})$ | Ad26.COV2.S $(5\times10^{10} \text{ vp})$ |

EUA Emergency Use Authorization; N number of participants; vp virus particles.

Note: It is intended that a minimum of approximately 30% of recruited participants will be  $\ge$ 60 years of age and approximately 20% of recruited participants will be  $\ge$ 18 to <40 years of age.

The following enrollment strategy will be used:

- Stage 1a: Initially, approximately 2,000 participants ≥18 to <60 years of age without comorbidities that are associated with increased risk of progression to severe COVID-19 (including approximately 1,000 Ad26.COV2.S recipients and approximately 1,000 placebo recipients) will be enrolled, based on acceptable Day 29 safety and acceptable immunogenicity data, including Thelper 1/Thelper 2 (Th1/Th2), from the corresponding age group (Cohort 1a) of the first-in-human (FIH) study VAC31518COV1001.
- Stage 1b: After a vaccination pause (in the age group ≥18 to <60 years of age) to allow the Data Safety Monitoring Board (DSMB, also known as an Independent Data Monitoring Committee [IDMC]) to examine Day 3 safety data (ie, from Day 1 to Day 3; including safety data from the ongoing clinical studies), if no safety concerns are identified enrollment will proceed, expanding enrollment to include ≥18- to <60-year-old participants with and without comorbidities that are associated with increased risk of progression to severe COVID-19.

In Stage 1a and 1b combined, the enrollment of participants aged  $\ge$ 18 to <40 years will be limited to approximately 20% of the total study population.

<sup>\*</sup> All participants will be unblinded (informed whether they received placebo or Ad26.COV2.S) at the on site Month 6/ Unblinding Visit following EUA, conditional licensure or approval in any country and approval by regulatory and IEC/IRB and the study will continue as an open label study. Participants who received placebo on Day 1 will be offered to receive a single dose of Ad26.COV2.S 5×10<sup>10</sup> vp.

- Stage 2a: Initially, approximately 2,000 participants ≥60 years of age without comorbidities that are associated with increased risk of progression to severe COVID-19 will be enrolled (including approximately 1,000 Ad26.COV2.S recipients and approximately 1,000 placebo recipients). Considering the data from study VAC31518COV1001 (including data on elderly), Stage 2a will run in parallel with Stage 1a, unless this is not allowed per local Health Authority guidance.
- Stage 2b: After a vaccination pause (in the age group ≥60 years of age) to allow the DSMB to examine Day 3 safety data (ie, from Day 1 to Day 3;including safety data from Stage 1 and the ongoing clinical studies) from Stage 2a, if no safety concerns are identified in this population enrollment will proceed, expanding enrollment to include ≥60-year-old participants with and without comorbidities that are associated with increased risk of progression to severe COVID-19.

Stage 2 will enroll a minimum of approximately 30% of the total study population.

Comorbidities (or risk factors) that are or might be associated with an increased risk of progression to severe COVID-19<sup>a</sup> include: moderate to severe asthma; chronic lung diseases such as chronic obstructive pulmonary disease (COPD) (including emphysema and chronic bronchitis), idiopathic pulmonary fibrosis and cystic fibrosis; diabetes (including type 1 or type 2); serious heart conditions, including heart failure, coronary artery disease, congenital heart disease, cardiomyopathies, and pulmonary hypertension; moderate to severe high blood pressure; obesity (body mass index [BMI] ≥30 kg/m²); chronic liver disease, including cirrhosis; sickle cell disease; thalassemia; cerebrovascular disease; neurologic conditions (dementia); end stage renal disease; organ transplantation; cancer; human immunodeficiency virus (HIV) infection and other immunodeficiencies; hepatitis B infection; sleep apnea.

No additional participants will be recruited for the open-label phase.

The duration of individual participation, including screening, will be approximately 2 years and 1 month. If a participant is unable to complete the study, but has not withdrawn consent, an early exit visit will be conducted. The end-of-study is considered as the completion of the last visit for the last participant in the study.

Key efficacy assessments include the surveillance for COVID-19-like signs and symptoms, recording of COVID-19-related hospitalizations and complications, and the laboratory confirmation of SARS-CoV-2 infection by a molecular assay (based on RT-PCR) and by anti-SARS-CoV-2 serology. Immunogenicity assessments, and especially assessments of the humoral immune responses with emphasis on neutralizing and binding antibodies will also be performed. Key safety assessments during the double-blind phase will include the monitoring of solicited and unsolicited AEs in the Safety Subset only. Up to Amendment 7, all participants who received booster vaccination at the Year 1/Booster Visit will record solicited signs and symptoms in an e-Diary, if feasible. As of protocol Amendment 7, the collection of solicited AEs will stop. Up to Amendment 7, for a subset of participants, the e-Diary will be reviewed by the study personnel at the next visit, if feasible, and solicited AEs recorded. Unsolicited AEs will be recorded for all participants who received booster vaccination at the Year 1/Booster Visit. As of protocol Amendment 7, the collection of unsolicited AEs will stop.

In addition, key safety assessments throughout the study include the collection of SAEs and MAAEs in all participants.

Up to Amendment 7, the viral load of SARS-CoV-2 will be assessed in confirmed COVID-19 cases. Biomarkers correlating with SARS-CoV-2 infection and COVID-19 severity will also be studied. Medical

<sup>&</sup>lt;sup>a</sup>Centers for Disease Control and Prevention (CDC). Coronavirus Disease 2019 (COVID-19) Groups at Higher Risk for Severe Illness. https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/groups-at-higher-risk.html. (Accessed: 19 July 2020) In this study, former or current smoking/vaping and mild hypertension (according to the Toxicity Grading Scale in the body of this document) will not be considered as a comorbidity. Gestational diabetes was deleted from the list since it is not applicable as pregnant women were not allowed to enroll in the study.

resource utilization (MRU) following vaccination will be recorded for all participants with molecularly confirmed, symptomatic COVID-19.

Additional characteristics related to current work situation, living situation, and community interactions will be collected for risk factor analysis, if allowed per local regulations. Participants who consent to this will be interviewed on these aspects prior to vaccination on Day 1 and, at other timepoints, on changes compared to Day 1. For consenting participants in the US, medical data (electronic health records, claims and laboratory data from other care settings) from 5 years prior to study enrollment until 5 years after study completion may be accessed utilizing tokenization and matching procedures (ie, the generation of anonymous identifiers or "tokens" [hashed and encrypted combinations of identifying elements] to allow linking of participant data from different sources without compromising the participant's confidentiality). These data together with data collected as part of the study as specified in the Schedules of Activities, may be used for exploratory analyses to enhance our understanding of the impact of prior medical history on the response to immunization and the impact of immunization on efficacy and duration of efficacy as well as adverse events that may occur during and after completion of the study. Concomitant therapies associated with COVID-19 are also to be reported as of Amendment 7. The statistical analyses will be described in detail in a Statistical Analysis Plan.

As of Amendment 7, participants will continue to be required to report safety events, such as SAEs, AESIs, MAAEs. As mentioned above, participants who received booster vaccination will stop the reporting of solicited or unsolicited AEs as of Amendment 7. Finally, the active follow-up of new suspected COVID-19 episodes will be replaced by passive follow-up, defined as follow-up by the site at Month 18 and Month 24 to document COVID-19 participant-reported events as SAEs, AEs, or MAAEs.

Up to Amendment 7, until 1 year after the Month 6/Unblinding Visit, each participant will be asked at least twice a week, through the electronic clinical outcome assessment (eCOA), if they have experienced any new symptoms or health concerns that could be related to infection with SARS-CoV-2. As of 1-year after the Month 6/Unblinding Visit, until the end of the 2-year follow-up period, the frequency of this (suspected) COVID-19 surveillance (symptom check) through the eCOA may decrease to once every 2 weeks depending on epidemiology. All participants will be monitored for safety (including enhanced disease) for approximately 1 year after the Year 1/Booster Visit, ie, until the last study visit. Every effort will be made to document the status of all participants that are lost to follow-up due to not completing the eCOA and for whom hospitalization has not been recorded. As from Amendment 7, the eCOA will be decommissioned (passive follow-up approach). The eCOA will be stopped based on approval of protocol Amendment 7 at each study site.

Enrolled participants will be counselled on SARS-CoV-2 infection prevention each time that they have a contact with site staff, in line with local guidelines. At the time of study entry, each participant will need to indicate to the study site, in case they would get infected with SARS-CoV-2, the identity and location of their routine medical care physician and/or facility and the identity and location of where they would obtain emergency care and hospitalization if necessary. If this information is not available, a plan for where such care could be obtained should be developed. If a participant should have COVID-19 and their symptoms deteriorate, they will be instructed to go to the health care professional (HCP) or hospital that has been identified in advance.

Up to Amendment 7, any positive RT-PCR test result regardless if it is obtained outside the study or at a study visit will be considered a trigger to start COVID-19 procedures. All participants with COVID-19-like signs or symptoms meeting the prespecified criteria for suspected COVID-19 and all participants with at least 1 positive RT-PCR test for SARS-CoV-2 on COVID-19 Day 1-2 or Day 3-5 visits, should undertake the COVID-19 procedures until 14 days after symptom onset (COVID-19 Day 15) or until resolution of the COVID-19 episode, whichever comes last. However, participants with COVID-19-like signs or symptoms meeting the prespecified criteria for suspected COVID-19 should stop the COVID-19 procedures as soon as it is confirmed that both nasal swabs collected on COVID-19 Day 1-2 and Day 3-5 are negative for SARS-CoV-2. Resolution of the COVID-19 episode is defined as having 2 consecutive SARS-CoV-2

negative nasal swabs and 2 consecutive days with no COVID-19-related signs or symptoms. At the time of resolution of the COVID-19 episode, the collected information will be applied against the clinical case definition. As from Amendment 7, this active follow-up approach will no longer be pursued and will be replaced by passive follow-up. Passive follow-up of COVID-19 consists of recording of new COVID-19 episodes as SAEs, AEs, or MAAEs. The information of these AEs is collected during the scheduled phone calls with the participants. Positive COVID-19 laboratory findings should be reported in the eCRF, if available (eg, positive PCR results, positive nasal swab).

All necessary precautions (as per local regulation) should be taken to protect medical staff and other contacts of participants who are suspected to have COVID-19 until proven negative by molecular techniques or who are positive AND meet the prespecified criteria for suspected COVID-19 on COVID-19 Day 1-2 and Day 3-5 until they are no longer positive. In the event of a confirmed SARS-CoV-2 infection, the participant and participant's medical care provider will be notified, and the participant will be asked to adhere to the appropriate measures and restrictions as defined by local regulations.

A DSMB will be commissioned for this study.

#### NUMBER OF PARTICIPANTS

Overall, a target of approximately 40,000 adult participants ( $\geq$ 18- to <60-year-old and  $\geq$ 60-year-old, with and without relevant comorbidities) will be randomly assigned in this study. Efforts will be made to ensure good representation in terms of race, ethnicity, and gender.

It is intended that a minimum of approximately 30% of recruited participants will be  $\ge$ 60 years of age and approximately 20% of recruited participants will be  $\ge$ 18 to <40 years of age.

## INTERVENTION GROUPS AND DURATION

Participants will be vaccinated at the study site according to the schedules detailed above:

- Ad26.COV2.S supplied at a concentration of  $1\times10^{11}$  vp/mL in single-use vials, with an extractable volume of 0.5 mL, and dosed at  $5\times10^{10}$  vp
- Placebo: 0.9% sodium chloride (NaCl) solution

For blinding purposes, all participants will receive Ad26.COV2.S or placebo at Day 1 of the double-blind phase, using the same volume (ie, 0.5 mL). At the Month 6/Unblinding Visit, all placebo participants who have signed a new ICF will receive a single dose of Ad26.COV2.S, using the same dose level and the same volume (ie,  $5 \times 10^{10}$  vp per 0.5 mL). At the Year 1/Booster Visit, all participants who are eligible for booster vaccination, desire to receive a booster vaccination, and have signed a new ICF will receive a single dose of Ad26.COV2.S, using the same dose level and the same volume (ie,  $5 \times 10^{10}$  vp per 0.5 mL) as used for the primary regimen.

## **EFFICACY EVALUATIONS**

Up to Amendment 7, identification and molecular confirmation of SARS-CoV-2 infection and symptomatic COVID-19 will be performed throughout the study.

The occurrence of COVID-19-related hospitalization and COVID-19-related complications (such as but not limited to hyperinflammatory syndrome, pneumonia, neurological or vascular complications, severe

neurological or vascular events, acute respiratory distress syndrome, renal complications, sepsis, septic shock, death)<sup>a</sup> will be monitored throughout the study.

For the primary objective, all moderate to severe/critical COVID-19 cases will be considered.

As a secondary objective, VE in the prevention of asymptomatic SARS-CoV-2 infection and mild COVID-19 will be analyzed. For samples collected prior to implementation of Amendment 7: An immunologic test for SARS-CoV-2 seroconversion (ELISA and/or SARS-CoV-2 immunoglobulin assay) based on SARS-CoV-2 N protein, may be performed to identify cases of asymptomatic infection. This assay will be performed on samples obtained at Day 1 (pre-vaccination), Day 29, Day 71, Month 6 /Unblinding Visit, Year 1, and Month 18.

### IMMUNOGENICITY EVALUATIONS

Up to Amendment 7, blood will be collected from all non-Immunogenicity Subset (double-blind phase) participants for humoral immunogenicity assessments at Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, and Year 1.

For a total of approximately 400 participants in the Immunogenicity Subset (ie, 400 participants at sites with access to appropriate processing facilities), blood will be collected for analysis of humoral immune responses at Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, Year 1, Month 18, and Year 2 visit after double-blind vaccination, and additionally 28 days and 72 days after booster vaccination, if applicable.

Note: Those participants in the Immunogenicity Subset that transfer to the Homologous Booster Subset at the Year 1/Booster Visit (see below) will from that visit onwards follow the humoral immunogenicity sample schedule of the Homologous Booster Subset and discontinue the schedule of the Immunogenicity Subset.

Up to Amendment 7, for participants with suspected or confirmed COVID-19 (ie, meeting prespecified criteria on COVID-19 Day 1-2 and Day 3-5 and/or a SARS-CoV-2 positive sample on COVID-19 Day 1-2 or Day 3-5), blood will be collected on COVID-19 Day 3-5 and on COVID-19 Day 29 for immunogenicity assessments, including the assays summarized in the table below. As from Amendment 7, active follow-up will no longer be pursued and blood sampling for this purpose will no longer be performed.

#### **Booster Vaccination**

Up to Amendment 7, blood will be collected from all non-Subset participants who received booster vaccination for humoral immunogenicity assessments at the Year 1/Booster Visit and 28 days, 72 days, and 6 months after booster vaccination. A blood sample for transcriptomics will be collected from all participants 28 days after booster vaccination.

<u>Homologous Booster Subset:</u> The Homologous Booster Subset will include approximately 200 participants. This subset will include participants from the Immunogenicity Subset, who received Ad26.COV2.S in the double-blind phase or after cross-over, and subsequently received an Ad26.COV2.S booster vaccination in the study. This group may be augmented by other participants to replace participants who are not available. Participants in the Homologous Booster Subset will have a blood sample collected pre-booster vaccination, and 28 days, 72 days, 6 months, and 1 year post booster vaccination for humoral immunogenicity assessment.

\_

World Health Organization (WHO). Clinical management of severe acute respiratory infection (SARI) when COVID-19 is suspected. Interim guidance, 13 March 2020. https://www.who.int/docs/default-source/coronaviruse/clinical-management-of-novel-cov.pdf. Accessed 12 May 2020.

Heterologous Booster Subset: The Heterologous Booster Subset will include approximately 400 participants. This subset will include participants in the study who received placebo in the double-blind phase and have received primary vaccination with an mRNA vaccine or another authorized COVID-19 vaccine including protein, inactivated, and adenovector based vaccines outside the study, who subsequently remained in the study and subsequently received an Ad26.COV2.S booster vaccination in the study. Participants who already received an additional COVID-19 vaccination after the primary regimen outside the study will not be included in the Heterologous Booster Subset. Participants will be selected out of countries where these vaccines were authorized for emergency use or are licensed. Participants in the Heterologous Booster Subset will have blood collected pre-booster vaccination, and 28 days, 72 days, 6 months, and 1 year post booster vaccination for humoral immunogenicity assessment.

Additionally, approximately the first 60 eligible participants once operationally feasible of the Homologous Booster Subset and approximately the first 60 eligible participants once operationally feasible of the Heterologous Booster Subset will have blood collected pre-booster and 1 day and 28 days post booster vaccination for transcriptomics and cytokine/chemokine assessment.

#### Immunogenicity and Transcriptomic Assays

| Humoral Assays | Purpose |
|---|---|
| Supportive of Secondary Objectives | |
| SARS-CoV-2 binding antibodies to S protein (ELISA) | Analysis of antibodies binding to SARS-CoV-2 S protein |
| SARS-CoV-2 seroconversion based<br>on antibodies to N protein (ELISA<br>and/or SARS-CoV-2 Immunoglobulin<br>assay) | Analysis of antibodies binding to SARS-CoV-2 N protein |
| Supportive of Secondary and Explora | tory Objectives |
| SARS-CoV-2 neutralization (VNA) | Analysis of neutralizing antibodies against SARS-CoV-2 original strain and/or variants, using a live VNA and/or pseudovirion expressing S protein neutralization assay |
| SARS-CoV-2 binding antibodies to S protein (MSD) | Analysis of antibodies binding to the original and/or variants SARS-CoV-2 S protein (different than the assays supportive of the secondary objectives) and the receptor-binding domain (RBD) of SARS-CoV-2 S protein |
| Functional and molecular antibody characterization | Analysis of antibody characteristics including, but not limited to, avidity, crystallizable fragment (Fc)-mediated viral clearance, Fc characteristics, immunoglobulin (Ig) subclass, IgG isotype, antibody glycosylation, and assessment of antibody repertoire |
| Adenovirus neutralization (VNA) | Adenovirus neutralization assay to evaluate neutralizing antibody responses against the Ad26 vector |
| Binding antibodies to other coronaviruses (MSD) | Analysis of antibodies binding to coronaviruses other than SARS-CoV-2 |
| Cytokine profiling | Analysis of cytokines, chemokines, and other proteins of the innate or adaptive immune response in the serum or plasma |
| Transcriptomic Assay | Purpose |
| Supportive of Exploratory Objectives | |
| Gene expression analysis | Analysis of gene expression by RNA transcript profiling in unstimulated cells or whole blood |

Ad26 adenovirus type 26; ELISA enzyme linked immunosorbent assay; Fc crystallizable fragment; Ig(G) immunoglobulin (G); MSD Meso Scale Discovery; N nucleocapsid; RBD receptor binding domain; RNA ribonucleic acid; S spike; SARS CoV 2 severe acute respiratory syndrome coronavirus 2; VNA virus neutralization assay.

In areas where seroprevalence is predicted to be high, a screening serologic test for past or current infection with SARS-CoV-2 may be performed (in a local laboratory), at the discretion of the sponsor, to restrict the proportion of seropositive participants in the study. This does not apply to the open-label phase of the study.

A serologic test for past or current infection with SARS-CoV-2 may be performed for all participants at Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, Year 1/Booster Visit (prior to vaccination, if applicable), Year 1 + 28 days for participants who received booster vaccination, Year 1 + 72 days for participants who received booster vaccination, and Month 18 (24 weeks after Year 1 Visit). Samples for the serologic tests will be sent to a central laboratory for testing. Participants who test positive will be informed of the result by the study staff.

#### SAFETY EVALUATIONS

The first 2,000 participants in each of the 2 age groups will remain under observation at the study site for at least 30 minutes post-vaccination to monitor for the development of acute reactions. If at the time of the Day 3 safety review of the initial 2,000 participants no acute reactions have been observed in the age groups, the observation period at the study site may be reduced to at least 15 minutes post-vaccination for the remaining participants in the study.

For all participants (throughout the study regardless of any protocol amendment):

- (S)AEs that are related to study procedures or that are related to non-investigational sponsor products will be reported from the time a signed and dated informed consent form (ICF) is obtained until the end of the study/early withdrawal.
- Clinically relevant medical events not meeting the above criteria and occurring between signing of the ICF and moment of vaccination in the double-blind phase of the study will be collected on the Medical History electronic case report form (eCRF) page as pre-existing conditions. This does not apply to the open-label phase.
- All SAEs and all AEs leading to study discontinuation (regardless of the causal relationship) are to be reported from the moment of vaccination until completion of the participant's last study-related procedure, which may include contact for safety follow-up. The sponsor will evaluate any safety information that is spontaneously reported by an investigator beyond the time frame specified in the protocol.
- MAAEs are defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits will not be considered medically-attended visits. New onset of chronic diseases will be collected as part of the MAAEs. MAAEs are to be reported for all participants from the moment of each vaccination until 6 months after the vaccination (applicable for both the double-blind and open-label phases of the study), except for MAAEs leading to study discontinuation which are to be reported during the entire study.
- Special reporting situations, whether serious or non-serious, will be recorded from the time of each vaccination until 28 days post-vaccination (applicable for both the double-blind and open-label phases of the study).
- Suspected AESIs (thrombotic events and thrombocytopenia [defined as platelet count below  $150,000/\mu L^b$ ]) will be reported from the moment of vaccination until the end of the study/early

<sup>&</sup>lt;sup>a</sup> Vaccination with Ad26.COV2.S may interfere with some serologic assays utilized at local community health clinics/commercial laboratories, by seeking and identifying the spike protein in the vaccine and rendering a false positive result. For this reason, participants will be encouraged to not seek testing outside the study. If a participant requires testing outside of the protocol-mandated testing schedule, the site will guide them on the appropriate assay that identifies the viral nucleocapsid protein (and not the spike protein).

<sup>&</sup>lt;sup>b</sup> Updated Proposed Brighton Collaboration process for developing a standard case definition for study of new clinical syndrome X, as applied to Thrombosis with Thrombocytopenia Syndrome (TTS). 18 May 2021. https://brightoncollaboration.us/wp-content/uploads/2021/05/TTS-Interim-Case-Definition-v10.16.3-May-23-2021.pdf. Accessed: 02 September 2021.

withdrawal. An AESI Adjudication Committee with appropriate expertise will be established to evaluate each suspected AESI and determine whether it is a case of thrombosis with thrombocytopenia syndrome (TTS). From the time of local approval of protocol Amendment 5 onwards, TTS is considered an adverse event of special interest (AESI).

• All AEs will be followed until resolution or until clinically stable.

As of Amendment 7, for all participants:

- Active follow-up of suspected COVID-19 episodes will be replaced by passive surveillance: during follow-up calls by the site at Month 18 and Month 24, new COVID-19 participant-reported events are to be reported as SAEs, AE or MAAEs.
- Concomitant medications for these events should be reported.
- If a COVID-19 confirmatory laboratory or assay read-out is available, this should be reported in the eCRF (self-reported or as part of CIOMS form).

For participants in the Safety Subset (double-blind phase):

- Solicited AEs, collected through an e-Diary, will be recorded from the time of vaccination until 7 days post-vaccination.
- All other unsolicited AEs, whether serious or non-serious, will be recorded from the time of vaccination until 28 days post-vaccination.

Up to Amendment 7: For participants who received booster vaccination at the Year 1/Booster Visit:

• Solicited AEs, collected through an e-Diary, will be recorded from the time of vaccination until 7 days post-vaccination. All participants will collect signs and symptoms in the e-Diary, if feasible. For a subset of participants, ie, participants included in the Safety Subset of the double-blind phase and all participants who previously received a heterologous COVID-19 vaccination outside the study, the e-Diary will be reviewed by the study personnel and solicited AEs recorded in the eCRF, if feasible. All other unsolicited AEs, whether serious or non-serious, will be recorded from the time of vaccination until 28 days post-vaccination for all participants.

As of Amendment 7, solicited and unsolicited AE reporting will stop for all participants.

#### STATISTICAL METHODS

Note: The below is only applicable to the double-blind phase of the study unless mentioned otherwise.

### **Sample Size Calculation**

#### Efficacy (Total Sample Size)

The study target number of events (TNE) is determined using the following assumptions:

- a VE for molecularly confirmed, moderate to severe/critical SARS-CoV-2 infection of 60%.
- approximately 90% power to reject a null hypothesis of H0: VE<30%.
- type 1 error rate  $\alpha = 2.5\%$  to evaluate VE of the vaccine regimen (employing the sequential probability ratio test [SPRT] to perform a fully sequential design analysis; detailed in the methods section).
- a randomization ratio of 1:1 for active versus placebo.

Events for the co-primary endpoints are defined as first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to the case definition (see above) in the Per-protocol Efficacy

population at least 14 days after double-blind vaccination (Day 15) and at least 28 days after double-blind vaccination (Day 29) with study vaccine.

Under the assumptions above, the TNE to compare the active vaccine versus placebo equals 154, based on events in each active vaccination and placebo group, according to the primary endpoints case definition of moderate to severe/critical COVID-19.

If the primary hypotheses testing is successful, secondary objectives will be evaluated against a null hypothesis employing a lower limit VE>0%. The method to perform hypothesis testing of primary and secondary objectives preserving the FWER will be specified in the SAP. The FWER will be controlled at 2.5%.

Further details on the sample size calculation are provided in the body of the protocol.

The operating characteristics of the study design, statistical methods, study monitoring rules and efficacy evaluation specified in this protocol with the chosen event and sample sizes will be described in a separate modeling and simulation report and will be added to the SAP before the first participant is vaccinated.

No additional participants will be recruited for the open-label phase.

## Immunogenicity Correlates (Correlates Subset)

Correlates will be assessed in a subset where immune responses and transcriptome modifications are measured in all vaccine recipients who experience a SARS-CoV-2 event, and in random samples of vaccine recipients who have not been infected, in a 1:5 ratio. The goal of this case—control study is to assess correlates of risk of SARS-CoV-2 infection (and potential other secondary endpoints) in the vaccine group by comparing vaccine-induced immune responses and transcriptome modifications associated with COVID-19. Also, placebo participants will be included in this subset (placebo infected, seropositive [based on N protein] non-infected and seronegative non-infected), if feasible.

## Safety (Safety Subset)

Solicited and unsolicited AEs will be captured only in the Safety Subset, ie, approximately 6,000 participants ( $\sim$ 3,000 from the active group,  $\sim$ 3,000 from the placebo group; and including at least 2,000 from the older age group [ $\geq$ 60 years of age] if feasible).

#### **Populations for Analysis Sets**

For purposes of analysis, the following populations are defined:

- Full Analysis Set (FAS): All randomized participants with a documented study vaccine
  administration, regardless of the occurrence of protocol deviations and serostatus at enrollment.
  Analyses of safety will be performed on the FAS. Vaccine efficacy analyses can be repeated using the
  FAS.
- Safety Subset: subset of the FAS for the analysis of solicited and unsolicited AEs.
- **Per-protocol Efficacy (PP) population:** Participants in the FAS who receive study vaccine and who are seronegative at the time of vaccination and who have no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Participants who became aware of their study vaccine allocation will cease to be part of the PP population. The PA of VE will be based on the PP population. The PP will be the main analysis population for efficacy analyses.
- **Per-protocol Immunogenicity (PPI) population:** All randomized and vaccinated participants, including those who are part of the Immunogenicity Subset and for whom immunogenicity data are available, excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. In addition, for participants who experience a SARS-CoV-2 event

(molecularly confirmed), samples taken after the event and samples taken outside protocol windows will not be taken into account in the assessment of the immunogenicity. The PPI population is the primary immunogenicity population. For key tables, sensitivity immunogenicity analyses will also be performed on the FAS, including participants who are part of the Immunogenicity Subset for whom immunogenicity measures are available. Excluded samples might be taken into account as well in the sensitivity analysis. Analyses of vaccine immunogenicity and immune correlates of risk will be based on PPI.

The populations for the open label cross-over, booster and passive follow-up phase are described in the SAP. The list of major protocol deviations to be excluded from the efficacy for the double-blind analysis and/or immunogenicity analyses will be specified in the SAP and/or this list will be reported into the protocol deviation dataset of the clinical database before unblinding.

## **Efficacy Analyses**

The study will have the following timepoints for efficacy analyses:

- 1. The evaluation of the primary objective will be performed as soon as the TNE has been reached in the double-blind phase for both co-primary endpoints, or earlier based on sequential monitoring of both co-primary endpoints. Sponsor unblinding will occur but investigator and participants remain blinded until implementation of Amendment 4.
- 2. If an efficacy signal is triggered before the required 8-week follow-up after double-blind vaccination of 50% of participants is reached, an additional analysis will be performed when that follow-up timepoint is reached (8-week median follow-up timepoint). If the time between the efficacy signal and the required 8-week median follow-up is too short to make a difference in terms of preparing two analyses, then a single analysis will take place at the time of the 8-week median follow-up. The analysis at the time of the 8-week median follow-up is considered the primary analysis.
- 3. After the primary analysis, additional analyses to support health authority interactions will be planned, as deemed appropriate.
- 4. A final analysis of the double-blind phase of the study, including all double-blind data, will be performed when all participants have completed the Month 6/Unblinding Visit or discontinued earlier. Depending on the operational implementation of the Month 6/Unblinding Visit, as well as the stage of the pandemic, this analysis may be conducted when a minimum of 90% of the study population has been unblinded.

During the open-label phase, 2 analysis can be performed:

- 5. The open-label cross-over and booster analysis (active follow-up).
- 6. An end-of-study analysis is planned 1 year after a minimum of 90% of the enrolled study population have reached the Year 1/Booster Visit or discontinued earlier and will be conducted upon completion of the last active participant visit. Depending on the timing of approval of Amendment 7 across study sites, the open-label cross-over and booster analysis may be combined with the end-of-study analysis. At the end-of-study analysis, 90% of participants will have completed one year safety follow-up post booster; the remaining active boosted participants will have at least 6 months of safety follow-up.

Additional analyses may be conducted to support health authority interactions and/or based on public health demand in case of emerging variants.

#### **Primary Endpoints**

The study is designed to test the co-primary hypotheses of VE in the PP population. For both co-primary endpoints, the following hypothesis will be tested: H0:  $VE \le 30\%$  versus H1: VE > 30%. The co-primary endpoints will evaluate the first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to the case definition with onset at least 14 days after double-blind vaccination

(Day 15) and with onset at least 28 days after double-blind vaccination (Day 29) with Ad26.COV2.S versus placebo, separately, in the PP population, including all events from both age groups, with and without comorbidities.

Participants included in the seronegative analysis set are those participants with a negative SARS-CoV-2 serology test result at baseline.

## Evaluation of the Primary Endpoints

A fully sequential design with early stopping boundaries for efficacy based on the SPRT<sup>30</sup> will be used on the PP. The SPRT will control the type I error adjusting for the fully sequential approach. The decision rules for harm and non-efficacy are detailed in the protocol.

To that end, the boundaries are derived to achieve approximately 90% power to detect VE=60% using an alpha level of 2.5% against H0:VE≤30%.

To allow for durability assessment, sites and participants will continue the study and remain blinded until the final analysis.

A successful primary efficacy conclusion will require:

1. Establishing the hypothesis H1: VE>30% for each co-primary endpoint

#### **AND**

2. A favorable split vaccine: placebo for the subset of primary endpoints meeting the severe/critical COVID-19 case definition (expressed as a VE point estimate against severe/critical COVID-19 molecularly confirmed endpoints ≥50%) and a minimum of 5 events in the placebo group. This requirement needs to be met for severe/critical events with onset at least 14 days after double-blind vaccination and for severe/critical events with onset at least 28 days after double-blind vaccination

## AND

3. A VE of at least 50% for each co-primary endpoint.

To evaluate the primary null hypotheses: H0:  $VE \le 30\%$  versus H1: VE > 30% for the co-primary endpoints, the truncated sequential probability ratio test will be used based on accumulating event data for each co-primary endpoint. This boundary is set up using the fully sequential design and is derived in such a way to have approximately 90% power to detect a VE = 60% using a one-sided alpha=0.025 against H0:  $VE \le 30\%$ . For the evaluation of the favorable ratio against the severe/critical COVID-19 endpoints a sequential boundary corresponding to a VE point estimate  $\ge 50\%$  and a minimum of 5 events in the placebo group will be prespecified. The specific boundaries will be detailed in the SAP.

The monitoring can start as soon as the following conditions are met:

- 1. A minimum of 6 COVID-19 cases for the ≥60 years age group with onset at least 28 days after double-blind vaccination
- 2. At least 42 cases meeting the primary endpoint definition of moderate to severe/critical COVID-19 with onset at least 28 days after double-blind vaccination.
- 3. A subset of at least 5 cases meeting the primary endpoint definition of severe/critical COVID-19 with onset at least 28 days after double-blind vaccination.

No interim evaluation will be done, until those conditions are fulfilled. Monitoring for efficacy will not start before the above conditions 1-3 are met and will occur at least once a week by the SSG of the DSMB until the prespecified boundaries have been crossed.

The efficacy analysis will be triggered by either:

1. a) An interim evaluation if all prespecified efficacy boundaries have been met OR if 154 cases meeting the primary endpoint definition of moderate to severe/critical COVID-19 are observed for events with onset at least 28 days after double-blind vaccination.

AND

b) The above 3 conditions are met.

OR, alternatively,

- 2. If the prespecified non-efficacy boundary has been met (evaluating events with start 28 days after double-blind vaccination) or when the harm boundary has been crossed. The decision rules for harm and non-efficacy are detailed in Section 9.5.1.1.
- 3. If an efficacy signal is triggered before the required 8-week follow-up after double-blind vaccination of 50% of participants is reached (8-week median follow-up timepoint), an additional analysis will be performed when that follow-up timepoint is reached. If the time between the efficacy signal and the required 8-week median follow-up is too short to make a difference in terms of preparing two analyses, then a single analysis will take place at the time of the 8-week median follow-up. The analysis at the time of the 8-week median follow-up is considered the primary analysis.

If more than 154 primary endpoints are observed for events with onset at least 28 days after double-blind vaccination before the 3 conditions above are met, a single analysis will take place as soon as the conditions are met, using the full 2.5% one-sided significance level.

If the prespecified boundaries and above criteria are met, the SSG will inform the DSMB and if deemed appropriate by the DSMB, a meeting with the DSMB and Oversight Group will be set up to discuss the efficacy signal. Upon this meeting the sponsor representative on the Oversight Group can trigger internal decision procedures to initiate health authority interactions based on the outcome of the study.

The primary efficacy analysis will pool data across populations (both age groups with and without comorbidities) to evaluate the primary and secondary objectives. In addition, these will be supplemented with a subgroup analysis for age group (18 to <60 years,  $\geq$ 60 years) and comorbidities employing a descriptive summary, including 95% confidence intervals to describe the VE in each subpopulation. Depending on the recruited study population, the  $\geq$ 60 years subgroup may be further subcategorized ( $\geq$ 70 years,  $\geq$ 80 years).

In addition, to assess potential time-effects of VE, the Kaplan-Meier method will be used to plot the estimated cumulative incidence rates over time for the vaccine and placebo groups. This method will be used to estimate cumulative VE over time, defined as  $[(1 \text{ minus ratio (vaccine/placebo}) \text{ of cumulative incidence by time t)} \times 100\%]$ .

### Secondary Endpoints

All secondary endpoint analyses will occur in the PP analysis set, in seronegative participants unless otherwise indicated.

The multiple testing strategy and the timing of the hypothesis testing to evaluate the secondary objectives will be detailed in the SAP separately.

## **Immunogenicity Analyses**

No formal statistical testing of the immunogenicity data is planned. All immunogenicity analyses will be performed on the PPI set. Key tables might be repeated for the FAS (including samples that are excluded from the PPI analysis).

#### **Safety Analyses**

No formal statistical testing of safety data is planned. Safety data by vaccination group and based on the FAS will be analyzed descriptively. The analysis of solicited and unsolicited AEs will be restricted to a subset of the FAS (ie, the Safety Subset). For SAEs, AESIs, and MAAEs, the full FAS is considered. New onset of chronic disease will be collected as part of the MAAEs.

Safety endpoints following the open-label cross-over vaccination and following the booster vaccination will be descriptively summarized. Pooled safety analyses with other studies may also be performed.

# Analysis of the Open-label cross-over Phase, Open-label Booster Phase, and Passive Surveillance Phase

Safety, immunogenicity, and efficacy endpoints following cross-over and/or booster vaccination will be descriptively summarized by the different cohorts for the different phases (ie, for the open-label phase: early vaccinated cohort and late vaccinated cohort; ie, for the booster phase: 1-dose cohort, homologous booster cohort and the heterologous booster cohort).

Additional analyses may be conducted to support health authority interactions and/or based on public health demand in case of emerging variants.

If deemed feasible, efficacy of the booster vaccination may be explored by comparing efficacy data after boosting to data in the absence of booster, on the same primary regimen.

Feasibility will be assessed based on data availability as well as adjustments for potential confounding in the statistical analysis.

The following data sources will be explored:

- 1. If available, data of participants in the study who did not receive a booster and/or available data prior to boosting.
- 2. Data of individuals outside the study who received a similar primary regimen but did not receive a booster. It will be explored if external data (eg, real world evidence data, and/or published literature data) is available to that end for the countries enrolled in this trial.

For the statistical analysis, it will be explored if adjustment for potential confounding factors is feasible (based on risk factors identified in the analysis of the double-blind phase/and or literature) in each comparison. This may include, but not limit to age, presence of co-morbidities as well as the spatiotemporal evolution of variants and the epidemic. It is anticipated that comparative evaluation of efficacy against asymptomatic infections using real world evidence of data of individuals outside the study will not be feasible due to the difficulty of detecting asymptomatic infections in real world evidence.

Efficacy data may be compared following homologous versus heterologous booster vaccination. Efficacy data after primary vaccination until booster vaccination may be summarized (as immediate, early versus delayed, late vaccination).

Details will be provided in the SAP.

## **Interim Analyses and Committees**

The study will be formally monitored by a DSMB (also known as an IDMC). In general, the DSMB will monitor safety data on a regular basis to ensure the continuing safety of the participants. The DSMB will review unblinded data.

The DSMB will review Day 3 safety data (ie, from Day 1 to Day 3; including safety data from the ongoing clinical studies) from participants enrolled in Stage 1a and Stage 2a, before enrollment of participants in Stage 1b and Stage 2b, respectively. Vaccination of participants in the respective age groups will be paused during these safety reviews. Enrollment will not be paused during other safety reviews. The DSMB responsibilities, authorities, and procedures will be documented in the DSMB Charter.

Continuous monitoring for vaccine-associated enhanced disease will be performed through the SSG who will look at each of the diagnosed FAS COVID-19 events. Vaccine harm monitoring will be performed for severe/critical COVID-19/death endpoint based on the FAS. As these events will be monitored in real-time, and, after each confirmed respective case, the SSG will assess if a stopping boundary is reached. Specifically, monitoring for a higher rate of severe/critical disease or death in the vaccine group compared to the placebo group starts at the 5<sup>th</sup> event and at each additional event until the harm boundary is reached or until the efficacy analysis is triggered. If the stopping boundary is met, then the SSG immediately informs the Chair of the DSMB through secure communication procedures. At this point the DSMB will convene and provide a recommendation to the Oversight Group, which includes a sponsor representative as a core member. As such, the potential harm monitoring is in real-time, resulting in the earliest indication of harm possible as soon as data come in. In addition, the DSMB will formally monitor the SARS-CoV-2 events to conclude both non-efficacy and efficacy. The DSMB will evaluate in an unblinded fashion whether superiority is established for the co-primary endpoints or whether non-efficacy is shown based on a report provided by the SSG, when the prespecified boundaries have been crossed.

The study will also be monitored for operational non-efficacy to evaluate whether enough events to perform the PA can be collected within reasonable time. For that purpose, a monitoring rule will be set up to assess the probability that the minimal needed target number of primary endpoints events to be able to perform the PA in the PP set will be reached. For the double-blind phase of the study, two versions of the non-efficacy monitoring report will be generated. A report provided to the DSMB will contain unblinded events and a report provided to the sponsor will contain blinded events. While it is the primary responsibility of the sponsor to make decisions regarding study operations and modifications based on monitoring of study vaccine-blinded primary events from the study, the DSMB can evaluate the progress towards primary endpoints targets in the context of the study vaccine-unblinded data, and based on this review may recommend to the Oversight Group, which includes a sponsor representative as a core member, to complete the study early due to reaching a boundary for efficacy or non-efficacy to assess VE. During the open-label phase, the DSMB will continue to monitor safety.

The monitoring rules will be detailed in the DSMB Charter, with the statistical details in the SAP.

A final analysis of the double-blind phase will be performed when all participants have completed the Month 6/Unblinding Visit or discontinued earlier. Depending on the operational implementation of the Month 6/Unblinding Visit, as well as the stage of the pandemic, this analysis may be conducted when a minimum of 90% of the study population has been unblinded. This will provide an analysis of all endpoints for the blinded portion of the study. This analysis will also incorporate data collected after the EUA submission to the FDA. All data generated after the unblinding will be considered as part of an analytic plan devoted to the open-label phase. More details will be provided in the SAP. This analysis may be supplemented by independent measures of incidence and efficacy with real world data obtained in separate studies, to be described in a separate protocol.

The SAP will describe the planned analyses in greater detail.

## Unblinding due to availability of an authorized/licensed COVID-19 vaccine

In the double-blind-phase of the study, investigators may receive requests to unblind study participants who become eligible to receive an authorized/licensed COVID-19 vaccine if/when these become available. In these cases, the investigator will discuss with the participant available options and ramifications. If the participant is eligible for an authorized/licensed vaccine according to local immunization guidelines or

recommendation and if the participant wishes to proceed with the unblinding, the investigator will follow the unblinding procedures. The reason for the unblinding request should be documented. The name and date(s) of administration of the other COVID-19 vaccine should be recorded (see body of the protocol for more details).

When unblinding, if it is determined that the participant received the Ad26.COV2.S vaccine (and not placebo), the participant will be informed that there are no data on the safety of receiving two different COVID-19 vaccines. Unblinded participants, both in the double-blind and open-label phase, will be asked to continue to be followed in this study in line with the Schedule of Activities to the extent that they permit. Safety, efficacy, and immunogenicity evaluations will be identical for all participants, including participants that are unblinded to obtain an authorized/licensed COVID-19 vaccine and who remain in the study, including participants in the Safety Subset, if applicable and feasible. All data will be analyzed separately from the point of unblinding, for safety, efficacy, and immunogenicity analysis, as described in the Statistical Analysis Plan.

Prior to EUA, conditional licensure or approval in any country, participants who opt for enrollment in an Expanded Access Program or a Phase 3b study (eg, Sisonke/TOGETHER in South Africa) may be unblinded upon their request and will be encouraged to continue in study VAC31518COV3001. Study investigators should query participants to elicit and document such participation in other studies in the VAC31518COV3001 study record.

### 1.2. Schema

Figure 1: Schematic Overview of Study VAC31518COV3001



 $Active = Ad26.COV2.S; incl. = including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; rand. = randomization; Th = T-helper\ cell\ type\ 1/2 and the randomization including; LTFU = long-term\ follow-up; randomization including; LTFU = long-term\ follow-up; randomization including; LTFU = long-term\ follow-up; randomization including; LTFU = long-term\ follow-up; randomization including; long-term\ follow-up; randomization in$ 

<sup>&</sup>lt;sup>a</sup> At the time of protocol Amendment 1 writing, immunogenicity and safety data from Cohort 1a (≥18-≤55 years of age) and Cohort 3 (≥65 years of age) of study VAC31518COV1001 have become available. The data demonstrated that a single dose of Ad26.COV2.S at a dose level of 5×10<sup>10</sup> vp is sufficient to induce an acceptable immune response that meets prespecified minimum criteria and that the dose is considered safe. Stage 2a can therefore be enrolled in parallel to Stage 1a, unless this is not allowed per local Health Authority guidance.

<sup>\*</sup> Upon implementation of protocol Amendment 4, all participants will be unblinded and the study will continue as an open-label study. Participants who received placebo as vaccination 1 (Day 1) will be offered to receive Ad26.COV2.S at this Month 6/Unblinding Visit
\*\* Upon implementation of protocol Amendment 6, all ongoing participants who have previously received any COVID-19 vaccination(s) (as primary regimen or additional dose) with the Ad26.COV2.S vaccine and/or an mRNA vaccine or another for primary vaccination authorized COVID-19 vaccine including protein, inactivated, and adenovector based vaccines will be offered a single booster dose of Ad26.COV2.S vaccine (5×10<sup>10</sup> vp) at the Year 1/Booster Visit. Participants who choose to receive a booster vaccination with the Ad26.COV2.S vaccine (if recommended and available) or another authorized COVID-19 vaccine outside the study or choose not to receive a booster vaccination will not be withdrawn from the study and will be encouraged to remain in the study.

A screening phase of up to 28 days is included, however, screening may also be performed prior to randomization on the day of vaccination.

In Stage 1a and 1b combined, the enrollment of participants aged ≥18 to <40 years will be limited to approximately 20% of the total study population. Stage 2, including participants aged ≥60 years, will enroll a minimum of approximately 30% of the total study population. The analysis of the data will not be staggered: the primary analysis will be based on pooled data from both stages of the study.

Refer to Section 2.1 for details on initiation of study VAC31518COV3001 based on data from study VAC31518COV1001.

Refer to Section 2.2 for details about the VAC31518COV1001 study.

Refer to Section 5.2 for details on the relevant comorbidities.

#### 1.3. Schedules of Activities

As of Amendment 7, the number of on-site visits for participants who are not part of the Immunogenicity or Booster Subsets is reduced. For these participants, any outstanding Visits 8 and 9 are cancelled. In addition, any outstanding Visits 10 and 11 are replaced by a phone call. Also, active follow-up of suspected COVID-19 episodes for all participants is replaced by a passive surveillance approach.

All participants will be reconsented either at the upcoming study Visit 6 or at an unscheduled visit (whichever comes first) and may be performed on-site or by phone as per local informed consent process guidelines. Reconsenting at the study site should be performed as soon as operationally feasible and preferably within 4 weeks after protocol Amendment 7 approval. The eCOA stop will be done at the study site level based on approval of protocol Amendment 7.

No further booster doses will be administered under protocol Amendment 7, except if there is a medical reason that prevented a participant to receive the Ad26.COV2.S vaccine prior to acceptance of Amendment 7 or if there is a non-availability of other vaccines to the participant. The investigator should inform participants on the availability of other COVID-19 vaccines. It is expected that at least 90% of the active boosted participants will have a one-year safety follow-up. For the remaining active boosted participants may have a shorter follow-up, and the end of study visit may occur prior to the year 2 visit.

# 1.3.1. Non-immunogenicity or Non-Booster Subset Participants (As of Amendment 7)

| Phase | Study Period | | r Follow-up<br>e Calls | Early Exit<br>Phone Call |
|---|---|---|---|---|
| Visit number | 6ª | 7 (previously numbered as Visit 10) | 8 (previously numbered as Visit 11) | Exitb |
| Visit Timing | Primary Vac<br>+52 w | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Year 1<br>(Week 52) | Month 18<br>(24 weeks after Year 1 Visit) | Year 2<br>(52 weeks after Year 1 Visit) | |
| Visit Window | Preferably 6 months,<br>but at least 3 months<br>after last COVID-19<br>vaccination* | ±28 d | ±28 d <sup>n</sup> | |
| Informed consent for Amendment 7c | •# | | | |
| MAAE recording <sup>g</sup> | 6 | Continuous | | • |
| (S)AE recording <sup>h</sup> | | Continuous | | • |
| Passive follow up of COVID 19i | | Continuous | | • |
| Concomitant therapies <sup>j</sup> | Continuous | | | |

| Phase | Study Period | | ı Follow-up<br>e Calls | Early Exit<br>Phone Call |
|---|---|---|---|---|
| Visit number | 6ª | 7 (previously numbered as Visit 10) | 8 (previously numbered as Visit 11) | Exit <sup>b</sup> |
| Visit Timing | Primary Vac<br>+52 w | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Year 1<br>(Week 52) | Month 18<br>(24 weeks after Year 1 Visit) | Year 2<br>(52 weeks after Year 1 Visit) | |
| Visit Window | Preferably 6 months,<br>but at least 3 months<br>after last COVID-19<br>vaccination* | ±28 d | ±28 d <sup>n</sup> | |
| Activities below are only applicable to those that will receive a booster vaccination under special circumstances <sup>m</sup> | | No further booster vaccination is to be given | ven as of Protocol Amendment 7** | |
| Body temperature <sup>d</sup> | ●#,+ | | | |
| Urine pregnancy test <sup>e</sup> | ●#,+ | | | |
| Pre vaccination symptoms <sup>f</sup> | ●#,+ | | | |
| Vaccination | ●+ | | | |
| Clinical laboratory blood sample (whole blood), mL <sup>k,1</sup> | •# <del>,</del> +7 | | | |
| Approx. blood draw range per visit, mL | 7 ml | | | |

<sup>#</sup> pre vaccination

- a. If allowed by local regulations, study visit 6 may take place at the participant's home or other location in the event of ongoing SARS-CoV-2 transmission in the area of the participant. If possible and allowed per local regulation, visits can be performed by a phone call or a telemedicine contact. Except for the vaccination visit, assessments scheduled for the other visits may also be performed by a trained health care professional (HCP), if allowed per local regulations.
- b. For those participants who are unable to continue participation in the study up to Visit 8, but for whom consent is not withdrawn, an early exit visit will be conducted as soon as possible. Participants who wish to withdraw consent from participation in the study will be offered an optional visit for safety follow-up.
- c. Reconsenting may take place at the Year 1/Booster Visit or, if Visit 6 already occurred, at an unscheduled visit and may be performed on-site or by phone as per local regulations.
- d. Body temperature will be measured preferably via the oral route, or in accordance with the local standard of care.

<sup>\*</sup> ie, preferably within window of 100 to +170 days around Year 1, but no later than the expiry date of the Ad26.COV2.S vials available at your site.

<sup>\*\*</sup> Except if there is a medical reason that prevents a participant to receive the Ad26COV2.S vaccine prior to acceptance of Amendment 7 or if there is a non availability of other vaccines to the participant, but no later than the expiry date of the Ad26.COV2.S vials available at your site

<sup>&</sup>lt;sup>+</sup> applicable for participants who receive(d) a single dose of Ad26.COV2.S booster vaccination at the Year 1/Booster Visit under the conditions delineated in Section 6.5 (more details in Section 8.10) and for participants who receive(d) a booster vaccination outside of the study. Participants who choose to receive a booster vaccination outside of the study are encouraged to schedule their Year 1/Booster Visit prior to their booster vaccination, if feasible, and come in for the Year 1 + 28 Days visit within the specified visit window, if feasible, or as close as possible to the visit window. As of protocol amendment 7, some participants may still receive a booster, for those subjects, the follow up should be a least 6 months post vaccination, but the last visit can be shorter than 1 year post vaccination.

- e. For participants of childbearing potential only. Participants who are pregnant may receive booster vaccination with Ad26.COV2.S, if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (see Section 6.5).
- f. Investigator must check for acute illness or body temperature  $\ge 38.0^{\circ}\text{C}/100.4^{\circ}\text{F}$  at the time of each vaccination. If any of these events occur at the scheduled time for the booster vaccination, the Year 1/Booster Visit with active vaccine can be delayed within the preferred visit window.
- g. MAAEs are to be reported for all participants from the moment of each vaccination until 6 months after the booster vaccination, except for MAAEs leading to study discontinuation which are to be reported during the entire study. New onset of chronic diseases will be collected as part of the MAAEs.
- h. All (S)AEs related to study procedures or non-investigational sponsor products will be reported from the time a signed and dated ICF is obtained until the end of the study/early withdrawal. All other SAEs are to be reported from the moment of vaccination until completion of the participant's last study-related procedure. AEs leading to study discontinuation (regardless of the causal relationship) and AESIs are to be reported from the moment of vaccination until completion of the participant's last study-related procedure. Suspected AESIs are to be reported from the moment of vaccination until completion of the participant's last study-related procedure (see Section 8.3.1). Special reporting situations, whether serious or non-serious, are to be recorded from the time of booster vaccination until 28 days post-vaccination.
- i. From the moment the ICF for Amendment 7 is signed, the participant moves to the passive follow-up phase schedule. COVID-19 is to be reported as SAE, AE, or MAAE until study end (see Section 8.3.1 for the reporting of COVID-19 events as of protocol amendment 7). Ongoing COVID 19 episodes from the date of Amendment 7 approval will not be reported as SAEs, AEs, or MAAEs Participants may contact the site at any time in between scheduled visits to report COVID-19 episodes.
- j. Refer to Section 6.10 for collection and recording of concomitant therapies associated with SAEs, solicited and unsolicited AEs, suspected AESIs, and MAAEs and COVID-19 (S)AEs or COVID-19 MAAEs.
- k. To be collected pre-vaccination only from participants receiving Ad26.COV2.S as booster vaccination at Year 1/Booster Visit. Whole blood samples will be used for a complete blood count, including platelets, in a local laboratory or a substitute for local laboratory, depending on local feasibility towards turnaround time of sample processing. Serum samples will be derived from the whole blood sample and stored for potential future coagulation-related testing in a central laboratory if the participant experiences a suspected AESI (see Section 10.2, Appendix 2).
- 1. To be collected once operationally feasible.
- m. No further booster doses will be administered under protocol amendment 7, except if there was a medical reason that prevented a participant to receive the Ad26COV2.S vaccine prior to acceptance of amendment 7 or if there is a non-availability of other vaccines to the participant. The investigator should inform participants on the availability of other COVID-19 vaccines.
- n. The end-of-study analysis is planned 1 year after a minimum of 90% of the enrolled study population have reached the Year 1/Booster Visit or discontinued earlier and will be conducted upon completion of the last participant visit. Hence, the end of study visit may occur at an earlier timepoint for those 10% of remaining active participants. A minimum of 6 month safety follow-up should be done.

AE = adverse event; AESI = adverse event of special interest; approx.. = approximate; cont. = continuous; COVID-19 = coronavirus disease-2019; d = day(s); ICF = informed consent form; MAAE = medically-attended adverse event; SAE = serious adverse event; SARS-CoV-2 = severe acute respiratory syndrome coronavirus-2.

# 1.3.2. Immunogenicity and Booster Subset Participants

As of Amendment 7, no further subjects will be recruited in the booster subset, and no further booster vaccination will be provided unless there is a medical reason or if there is a non-availability of other vaccines to the participant.

| Visit Number | 6 | 7** | 8+ | 9+ | 10 | 11 | Exit <sup>a</sup> |
|---|---|---|---|---|---|---|---|
| Visit Timing | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+ 1 Day | Year 1 +28<br>Days (Week<br>56) | Year 1+72<br>Days (Week<br>62) | Month 18<br>(24 weeks<br>after Year 1<br>Visit) | Year 2<br>(52 weeks<br>after Year 1<br>Visit) | |
| Visit Window | Preferably 6 months, but at least 3 months after last COVID-19 vaccination* | +1 d | ±3 d | ±3 d | ±28 d | ±28 d <sup>t</sup> | |
| Visit Type | Safety and Immuno | Immuno | Safety and<br>Immuno | Safety and<br>Immuno | Safety and<br>Immuno | Safety and<br>Immuno | Early<br>Exit |
| Phase | Study Period | Long-term<br>Follow-up | Phase | Study<br>Period | Long-term<br>Follow-up | Phase | Study<br>Period |
| Informed consent for Amendment 7 <sup>b</sup> | •# | | | | | | |
| Vital signs <sup>c</sup> | | | | 7 | | | |
| Body temperature <sup>d</sup> | •# | | •+ | •+ | • | • | <b>●</b> e |
| Urine pregnancy test <sup>f</sup> | <b>_#</b> .+ | | | | | | |
| Biomarker RNAseq blood sample /<br>transcriptomics (PAXgene tubes,<br>whole blood), mL <sup>g</sup> | | | •+,r2.5 | | | | |
| Pre vaccination symptoms <sup>h</sup> | •# | | | | | , | |
| Vaccination <sup>s</sup> | •+ | | | | | | |
| Post vaccination observationi | •+ | | | | | | |
| MAAE recording | | Contin | nuous | | | | |
| (S)AE recording <sup>k</sup> | | Contin | uous | | | | |
| Passive surveillance of COVID 19 <sup>1</sup> | | Contin | nuous | | | | |
| Concomitant therapies <sup>m</sup> | | Conti | nuous | | | | |
| Clinical laboratory blood sample (whole blood), mL <sup>n</sup> | <b>●#</b> ,+,x7 | | | | | | |

| Visit Number | 6 | 7 <sup>++</sup> | 8+ | 9+ | 10 | 11 | Exita |
|---|---|---|---|---|---|---|---|
| Visit Timing | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+ 1 Day | Year 1 +28<br>Days (Week<br>56) | Year 1 +72<br>Days (Week<br>62) | Month 18<br>(24 weeks<br>after Year 1<br>Visit) | Year 2<br>(52 weeks<br>after Year 1<br>Visit) | |
| Visit Window | Preferably 6 months, but at least 3 months after last COVID-19 vaccination* | +1 d | ±3 d | ±3 d | ±28 d | ±28 d <sup>t</sup> | |
| Visit Type | Safety and Immuno | Immuno | Safety and<br>Immuno | Safety and<br>Immuno | Safety and<br>Immuno | Safety and<br>Immuno | Early<br>Exit |
| Phase | Study Period | Long-term<br>Follow-up | Phase | Study<br>Period | Long-term<br>Follow-up | Phase | Study<br>Period |
| IMMUNOGENICITY SUBSET | | | | | | | |
| Humoral immunogenicity (serum), mL <sup>p,o</sup> | ●15 | | ● <sup>+,</sup> r15 | ● <sup>+,</sup> r15 | ●15 | ●15 | ●15 |
| HOMOLOGOUS AND HETEROLO | OGOUS BOOSTER SUBSET | | | | | | |
| Humoral immunogenicity (serum), mL <sup>q</sup> | ●#15 | | ●15 | ●15 | ●15 | ●15 | ●15° |
| SUBSET OF HOMOLOGOUS ANI | HETEROLOGOUS BOOSTER SUBSETS | | | | | | |
| Blood cytokine/chemokine assessment | ●#5 | ●5 | | | | | |
| Biomarker RNAseq blood sample/<br>transcriptomics (PAXgene tubes,<br>whole blood), mL <sup>g</sup> | •#2.5 | ●2.5 | | | | | |
| Approx. blood draw range per visit, mL <sup>r</sup> | 10.0 29.5 | 0.0 7.5 | 0.0 29.5 | 0.0 15.0 | 10.0 15.0 | 0.0 15.0 | 10 15 |
| Approx. cumulative blood draw range, mL <sup>r</sup> | 62.0 101.5 | 62.0 109.0 | 62.0 138.5 | 62.0 153.5 | 72.0 168.5 | 72.0-183.5 | |
| Activities below are only applicable to those that will receive a booster vaccination under special circumstances <sup>m</sup> | No further boo | ester vaccination | is to be given as | of Protocol Ame | ndment 7** | | |
| Urine pregnancy test <sup>f</sup> | <b>⊕</b> #,+ | | | | | | |
| Pre vaccination symptoms <sup>h</sup> | •# | | | | | | |
| Vaccinations | • | | | | | | |
| Post vaccination observation <sup>i</sup> | • | | | | | | |
| Clinical laboratory blood sample (whole blood), mL <sup>n</sup> | ● <sup>#,+,r</sup> 7 | | | | | | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

- a. For those participants who are unable to continue participation in the study up to Visit 11, but for whom consent is not withdrawn, an early exit visit will be conducted as soon as possible. Participants who wish to withdraw consent from participation in the study will be offered an optional visit for safety follow-up. This includes the safety assessments of the early exit visit (no blood sampling for immunogenicity).
- b. Reconsenting may take place at the Year 1/Booster Visit or, if Visit 6 already occurred, at an unscheduled visit and may be performed on-site or by phone as per local regulations.
- c. Vital signs may be measured at the discretion of the investigator. Under special circumstances such as high altitude, the investigator should assess baseline respiratory rate and other vital signs, as appropriate. Blood pressure is to be graded by the investigator using the toxicity grading scale in Appendix 9.
- d. Body temperature will be measured preferably via the oral route, or in accordance with the local standard of care.
- e. If within 7 days of the vaccination.
- f. For participants of childbearing potential only. Participants who are pregnant may receive booster vaccination with Ad26.COV2.S, if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (see Section 6.5).
- g. Blood sample for exploration of biomarkers correlating with SARS-CoV-2 infection and COVID-19 severity.
- h. Investigator must check for acute illness or body temperature ≥38.0°C/100.4°F at the time of each vaccination. If any of these events occur at the scheduled time for the booster vaccination, the Year 1/Booster Visit with active vaccine can be delayed within the preferred visit window.
- i. Participants in the study will be closely observed for at least 15 minutes post-vaccination. Participants will be allowed to leave the study site after it is documented that the post-vaccination observation period is complete.
- j. MAAEs are to be reported for all participants from the moment of each vaccination until 6 months after the booster vaccination, except for MAAEs leading to study discontinuation which are to be reported during the entire study. New onset of chronic diseases will be collected as part of the MAAEs.
- k. All (S)AEs related to study procedures or non-investigational sponsor products will be reported from the time a signed and dated ICF is obtained until the end of the study/early withdrawal. All other SAEs are to be reported from the moment of vaccination until completion of the participant's last study-related procedure. AEs leading to study discontinuation (regardless of the causal relationship) are to be reported from the moment of vaccination until completion of the participant's last study-related procedure. Suspected AESIs are to be reported from the moment of vaccination until completion of the participant's last study-related procedure (see Section 8.3.1). Special reporting situations, whether serious or non-serious, are to be recorded from the time of booster vaccination until 28 days post-vaccination.
- 1. From the moment the ICF for Amendment 7 is signed, the participant moves to the passive surveillance phase schedule. COVID-19 is to be reported as SAE, AE, or MAAE until study end (see Section 8.3.1 for the reporting of COVID-19 events as of protocol amendment 7). Participants may contact the site at any time in between scheduled visits to report COVID-19 episodes.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

<sup>#</sup> pre vaccination

<sup>\*</sup> ie, preferably within window of 100 to +170 days around Year 1, but no later than the expiry date of the Ad26.COV2.S vials available at your site.

<sup>\*\*</sup> Except if there is a medical reason that prevents a participant to receive the Ad26COV2.S vaccine prior to acceptance of Amendment 7 or if there is a non availability of other vaccines to the participant, but no later than the expiry date of the Ad26.COV2.S vials available at your site

<sup>&</sup>lt;sup>+</sup> applicable for participants who receive(d) a single dose of Ad26.COV2.S booster vaccination at the Year 1/Booster Visit under the conditions delineated in Section 6.5 (more details in Section 8.10) and for participants who receive(d) a booster vaccination outside of the study. Participants who choose to receive a booster vaccination outside of the study are encouraged to schedule their Year 1/Booster Visit prior to their booster vaccination, if feasible, and come in for the Year 1 + 28 Days and Year 1 + 72 Days visits within the specified visit window, if feasible, or as close as possible to the visit window.

<sup>&</sup>lt;sup>++</sup> only applicable for approximately the first 60 eligible participants once operationally feasible of the Homologous Booster Subset (approximately 15 per subgroup [1a, 1b, 2a, and 2b]) and approximately the first 60 eligible participants once operationally feasible of the Heterologous Booster Subset (approximately 15 per subgroup [primary vaccination with mRNA vaccine, protein vaccine, adenovector vaccine, and inactivated vaccine]) (see Section 8.1.4).

- m. Refer to Section 6.10 for collection and recording of concomitant therapies associated with SAEs, solicited and unsolicited AEs, suspected AESIs, and MAAEs and new COVID-19 (S)AEs or COVID-19 MAAEs.
- n. Whole blood samples will be used for a complete blood count, including platelets, in a local laboratory or a substitute for local laboratory, depending on local feasibility towards turnaround time of sample processing. Serum samples will be derived from the whole blood sample and stored for potential future coagulation-related testing in a central laboratory if the participant experiences a suspected AESI (see Section 10.2, Appendix 2).
- o. Blood samples for immunogenicity will only be taken if the early exit visit is at least 10 days after the previous immunogenicity blood draw.
- p. Blood sample for humoral immunity at Year 1/Booster Visit (prior to booster vaccination), Month 18, and Year 2, and additionally 28 days and 72 days after booster vaccination, if applicable, may also include sample for sero-confirmation of SARS-CoV-2 infection. Samples will be collected for 400 participants at selected sites.
- q. Blood sample for humoral immunity at the Year 1/Booster Visit (pre-vaccination) and 28 days, 72 days, 6 months, and 1 year after booster vaccination, may also include sample for sero-confirmation of SARS-CoV-2 infection. Samples will be collected for 600 participants at selected sites.
- r. The approximate blood volume collected depends on which one of the immunogenicity or booster subgroups the participant is in.
- s. No further booster doses will be administered under protocol amendment 7, except if there was a medical reason that prevented a participant to receive the Ad26COV2.S vaccine prior to acceptance of amendment 7 or if there is a non-availability of other vaccines to the participant. The investigator should inform participants on the availability of other COVID-19 vaccines.
- t. The end-of-study analysis is planned 1 year after a minimum of 90% of the enrolled study population have reached the Year 1/Booster Visit or discontinued earlier and will be conducted upon completion of the last participant visit. Hence, the end of study visit may occur at an earlier timepoint for those 10% of remaining active participants. A minimum of 6 month safety follow-up should be done.

AE = adverse event; AESI = adverse event of special interest; approx.. = approximate; cont. = continuous; COVID-19 = coronavirus disease-2019; d = day(s); ICF = informed consent form; MAAE = medically-attended adverse event; SAE = serious adverse event; SARS-CoV-2 = severe acute respiratory syndrome coronavirus-2; vac = vaccination; w = week(s).

# 1.3.3. All Participants (Prior to Amendment 7)

| Phase | Screening <sup>a</sup> | | Study Period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number <sup>b</sup> | 1 | 2 | 3 | 4 | 5 | 6 | 7** | 8+ | 9+ | 10 | 11 | Exite |
| Visit Timing | | Vac | Vac<br>+ 28 d | Vac<br>+ 70 d | Vac + 24 w/ Post EUA, conditional licensure or approval in any country | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Day -28 to 1 | Day 1 | Day 29 | Day 71 | Month 6<br>(Week 24)/<br>Unblinding Visit | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+ 1 Day | Year 1<br>+28<br>Days<br>(Week<br>56) | Year 1<br>+72<br>Days<br>(Week<br>62) | Month 18<br>(24 weeks<br>after Year<br>1 Visit) | Year 2<br>(52<br>weeks<br>after<br>Year 1<br>Visit) | |
| Visit Window | | | ±3 d | ±3 d | As soon as possible<br>post Day 71 visit** | Preferably 6 months, but at least 3 months after last COVID-19 vaccination*** | +1 d | ±3 d | ±3 d | ±28 d | ±28 d | |
| Visit Type | Screening | Vaccination | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and Immuno | Safety and<br>Immuno | Immuno | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and<br>Immuno | Safety<br>and<br>Immuno | Early<br>Exit |
| Informed consent <sup>d</sup> | • | | | | • | • | | | | | | |
| Inclusion/exclusion | • | <b>●</b> e | | | | | | | | | | |
| criteria | | - | | | | | | | | | | |
| Demographics Risk factor | • | | | | | | | | | | | |
| assessment <sup>f</sup> | | • | | • | • | • | | | | | | |
| Optional consent to | | | | | | | g | | | | | I |
| access medical data | | | | 1 | Т | T | 1 | 1 | 1 | Т | 1 | 1 |
| Relevant medical | | | | | | | | | | | | |
| history <sup>h</sup> /prestudy<br>therapies <sup>i</sup> | • | | | | | | | | | | | |
| Body weight and | | | 1 | | | | 1 | 1 | | | | |
| height | • | | | | | | | | | | | |
| Vital signs <sup>j</sup> | • | | | | | | | | | | | |
| Body temperature <sup>k</sup> | • | • | • | • | • | • | 1 | •+ | •+ | • | • | <b>●</b> 1 |
| Urine pregnancy | - | | | | - | | | | - | | - | |
| test <sup>m</sup> | • | • | | | <b>●*</b> ,kk | ●+,kk | | | | | | |

| Phase | Screeninga | Study Period | | | | | | | | Long-term<br>up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number <sup>b</sup> | 1 | 2 | 3 | 4 | 5 | 6 | 7** | 8+ | 9+ | 10 | 11 | Exite |
| Visit Timing | | Vac | Vac<br>+ 28 d | Vac<br>+ 70 d | Vac + 24 w/ Post EUA, conditional licensure or approval in any country | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Day -28 to 1 | Day 1 | Day 29 | Day 71 | Month 6<br>(Week 24)/<br>Unblinding Visit | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+ 1 Day | Year 1<br>+28<br>Days<br>(Week<br>56) | Year 1<br>+72<br>Days<br>(Week<br>62) | Month 18<br>(24 weeks<br>after Year<br>1 Visit) | Year 2<br>(52<br>weeks<br>after<br>Year 1<br>Visit) | |
| Visit Window | | | ±3 d | ±3 d | As soon as possible<br>post Day 71 visit** | Preferably 6 months, but at least 3 months after last COVID-19 vaccination*** | +1 d | ±3 d | ±3 d | ±28 d | ±28 d | |
| Visit Type | Screening | Vaccination | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and Immuno | Safety and<br>Immuno | Immuno | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and<br>Immuno | Safety<br>and<br>Immuno | Early<br>Exit |
| Pulse oximetry | | • | | | | | | | | | | |
| Randomization | | • | | | | | | | | | | |
| Nasal sample<br>collection for<br>SARS CoV 2<br>testing <sup>n</sup> | | • | | | •11 | | | | | | | |
| Biomarker RNAseq<br>blood sample /<br>transcriptomics<br>(PAXgene tubes,<br>whole blood), mL° | | ●2.5 | ●2.5 | | | | | •+,ss2.5 | | | | |
| Blood sample collection for screening serological test for anti SARS CoV 2 antibody MRU questionnaire (baseline version) <sup>q</sup> | <b>●</b> P | • | | | | | | | | | | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Phase | Screeninga | | Study Period | | | | | | | | Follow- | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number <sup>b</sup> | 1 | 2 | 3 | 4 | 5 | 6 | 7** | 8+ | 9+ | 10 | 11 | Exite |
| Visit Timing | | Vac | Vac<br>+ 28 d | Vac<br>+ 70 d | Vac + 24 w/ Post EUA, conditional licensure or approval in any country | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Day -28 to 1 | Day 1 | Day 29 | Day 71 | Month 6<br>(Week 24)/<br>Unblinding Visit | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+ 1 Day | Year 1<br>+28<br>Days<br>(Week<br>56) | Year 1<br>+72<br>Days<br>(Week<br>62) | Month 18<br>(24 weeks<br>after Year<br>1 Visit) | Year 2<br>(52<br>weeks<br>after<br>Year 1<br>Visit) | |
| Visit Window | | | ±3 d | ±3 d | As soon as possible<br>post Day 71 visit** | Preferably 6 months, but at least 3 months after last COVID-19 vaccination*** | +1 d | ±3 d | ±3 d | ±28 d | ±28 d | |
| Visit Type | Screening | Vaccination | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and Immuno | Safety and<br>Immuno | Immuno | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and<br>Immuno | Safety<br>and<br>Immuno | Early<br>Exit |
| Pre vaccination | | • | | | •* | • | | | | | | |
| symptoms <sup>r</sup> | | _ | | | - | - | | | | | | |
| eCOA training and set up <sup>s</sup> | | • | | | | | | | | | | |
| Distribution of thermometer | | • | | | | | | | | | | |
| Distribution of | | • | | | | | | | | | | |
| pulse oximeter <sup>t</sup> Distribution of MA | | | | | | | | | | | | |
| COV form <sup>u</sup> | | • | | | | | | | | | | |
| Training and distribution: nasal swab kit and saliva recipients | | • | | | | | | | | | | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S. Status: Approved, Date: 15 April 2022

| Phase | Screening <sup>a</sup> | | | 2 | Long-term<br>up | | 5 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit numberb | 1 | 2 | 3 | 4 | 5 | 6 | 7** | 8+ | 9+ | 10 | 11 | Exite |
| Visit Timing | | Vac | Vac<br>+ 28 d | Vac<br>+ 70 d | Vac + 24 w/ Post EUA, conditional licensure or approval in any country | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Day -28 to | Day 1 | Day 29 | Day 71 | Month 6<br>(Week 24)/<br>Unblinding Visit | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+1 Day | Year 1<br>+28<br>Days<br>(Week<br>56) | Year 1<br>+72<br>Days<br>(Week<br>62) | Month 18<br>(24 weeks<br>after Year<br>1 Visit) | Year 2<br>(52<br>weeks<br>after<br>Year 1<br>Visit) | |
| Visit Window | | | ±3 d | ±3 d | As soon as possible<br>post Day 71 visit** | Preferably 6 months, but at least 3 months after last COVID-19 vaccination*** | +1 d | ±3 d | ±3 d | ±28 d | ±28 d | |
| Visit Type | Screening | Vaccination | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and Immuno | Safety and<br>Immuno | Immuno | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and<br>Immuno | Safety<br>and<br>Immuno | Early<br>Exit |
| Symptoms of Infection with Coronavirus 19 (SIC), including body temperature measured by the participant (ePROs to be completed by the participant in the eCOA) <sup>v</sup> | | • | | | | | | | | | | |
| Vaccination | | • | | | •* | •+ | | | | | | |
| Post vaccination observation <sup>w</sup> | | • | | | •* | •+ | | | | | | , |
| (Suspected) COVID 19 surveillance (symptom check) <sup>x</sup> | | | | | | Continuous | | | | | | |
| MAAE recordingy | | | | | | Continuous | | | | | | |
| (S)AE recording <sup>z</sup> | 1 | | | | | Continuous | | | | | | • |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Phase | Screeninga | Study Period | | | | | | | | Long-term Follow-<br>up | | č |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number <sup>b</sup> | 1 | 2 | 3 | 4 | 5 | 6 | 7** | 8+ | 9+ | 10 | 11 | Exite |
| Visit Timing | | Vac | Vac<br>+ 28 d | Vac<br>+ 70 d | Vac + 24 w/ Post EUA, conditional licensure or approval in any country | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Day -28 to<br>1 | Day 1 | Day 29 | Day 71 | Month 6<br>(Week 24)/<br>Unblinding Visit | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+1 Day | Year 1<br>+28<br>Days<br>(Week<br>56) | Year 1<br>+72<br>Days<br>(Week<br>62) | Month 18<br>(24 weeks<br>after Year<br>1 Visit) | Year 2<br>(52<br>weeks<br>after<br>Year 1<br>Visit) | |
| Visit Window | | | ±3 d | ±3 d | As soon as possible post Day 71 visit** | Preferably 6 months, but at least 3 months after last COVID-19 vaccination*** | +1 d | ±3 d | ±3 d | ±28 d | ±28 d | |
| Visit Type | Screening | Vaccination | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and Immuno | Safety and<br>Immuno | Immuno | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and<br>Immuno | Safety<br>and<br>Immuno | Early<br>Exit |
| Concomitant therapies <sup>aa</sup> | | | | | | Continuous | | | | | | • |
| Clinical laboratory<br>blood sample<br>(whole blood),<br>mL <sup>bb</sup> | | | | | ●#7 | •+,ss7 | | ●+,ss7 | | | | |
| Humoral<br>immunogenicity<br>(serum), mL (non<br>Subset<br>Participants) <sup>cc</sup> | | ●10 | ●10 | ●10 | ● <sup>mm</sup> 10 | ●≈10 | | •+,ss10 | •+,ss10 | ●10 | | ● <sup>dd</sup> 10 |
| IMMUNOGENICITY | SUBSET ON | ILY | | | | | 3. | | | | | |
| Humoral<br>immunogenicity<br>(serum), mL <sup>ee,oo</sup> | | ●15 | ●15 | ●15 | ●#15 | ●15 | i e | ●+,ss15 | ●+,ss15 | ●15 | ●15 | ● <sup>dd</sup> 15 |
| HOMOLOGOUS AN | D HETEROL | OGOUS BOO | STER SUB | SET ONLY | 7 | 2 | 3b. | | | | | t e |
| Humoral<br>immunogenicity<br>(serum), mL <sup>ff</sup> | | | | | | <b>•</b> #15 | | ●15 | ●15 | ●15 | ●15 | ● <sup>dd</sup> 15 |

 $CONFIDENTIAL-FOIA\ Exemptions\ Apply\ in\ U.S.$ 

| Phase | Screeninga | | Study Period | | | | | | | | Follow- | 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit numberb | 1 | 2 | 3 | 4 | 5 | 6 | 7** | 8+ | 9+ | 10 | 11 | Exite |
| Visit Timing | | Vac | Vac<br>+ 28 d | Vac<br>+ 70 d | Vac + 24 w/ Post EUA, conditional licensure or approval in any country | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Day -28 to 1 | Day 1 | Day 29 | Day 71 | Month 6<br>(Week 24)/<br>Unblinding Visit | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+1 Day | Year 1<br>+28<br>Days<br>(Week<br>56) | Year 1<br>+72<br>Days<br>(Week<br>62) | Month 18<br>(24 weeks<br>after Year<br>1 Visit) | Year 2<br>(52<br>weeks<br>after<br>Year 1<br>Visit) | |
| Visit Window | | | ±3 d | ±3 d | As soon as possible post Day 71 visit** | Preferably 6 months, but at least 3 months after last COVID-19 vaccination*** | +1 d | ±3 d | ±3 d | ±28 d | ±28 d | |
| Visit Type | Screening | Vaccination | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and Immuno | Safety and<br>Immuno | Immuno | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and<br>Immuno | Safety<br>and<br>Immuno | Early<br>Exit |
| SUBSET OF HOMO | LOGOUS AN | D HETEROLO | OGOUS BO | OSTER SU | JBSET ONLY** | | ** | | | | | |
| Blood<br>cytokine/chemokine<br>assessment | | | | | | ●5 | ●5 | ●5 | | | | |
| Biomarker RNAseq<br>blood sample/<br>transcriptomics<br>(PAXgene tubes,<br>whole blood), mL° | | | | | | ●2.5 | ●2.5 | ●2.5 | | | | |
| SAFETY SUBSET O | NLY | | | | | | | | | | | |
| Solicited AE<br>recording <sup>gg</sup> | | Cont +7d | | | | | | | | | | •1 |
| Unsolicited AE<br>recordinghh | | Cont + | 28 d | | | | | | | | | ● ii |
| Ruler training and<br>distribution of<br>ruler <sup>ij</sup> | | • | | | | | | | | | | |
| Participant e Diary review | | | • | | | | | | | | | |

| Phase | Screeninga | Study Period | | | | | | 3 | Long-term<br>up | | .5 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit numberb | 1 | 2 | 3 | 4 | 5 | 6 | 7** | 8+ | 9+ | 10 | 11 | Exite |
| Visit Timing | | Vac | Vac<br>+ 28 d | Vac<br>+ 70 d | Vac + 24 w/ Post EUA, conditional licensure or approval in any country | Primary Vac<br>+52 w | Booster<br>+1 d | Booster<br>+28 d | Booster<br>+72 d | Booster<br>+24 w | Booster<br>+52 w | |
| Visit Day/Week | Day -28 to 1 | Day 1 | Day 29 | Day 71 | Month 6<br>(Week 24)/<br>Unblinding Visit | Year 1<br>(Week 52)/<br>Booster Visit | Year 1<br>+1 Day | Year 1<br>+28<br>Days<br>(Week<br>56) | Year 1<br>+72<br>Days<br>(Week<br>62) | Month 18<br>(24 weeks<br>after Year<br>1 Visit) | Year 2<br>(52<br>weeks<br>after<br>Year 1<br>Visit) | |
| Visit Window | | | ±3 d | ±3 d | As soon as possible<br>post Day 71 visit** | Preferably 6 months, but at least 3 months after last COVID-19 vaccination*** | +1 d | ±3 d | ±3 d | ±28 d | ±28 d | |
| Visit Type | Screening | Vaccination | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and Immuno | Safety and<br>Immuno | Immuno | Safety<br>and<br>Immuno | Safety<br>and<br>Immuno | Safety and<br>Immuno | Safety<br>and<br>Immuno | Early<br>Exit |
| PARTICIPANTS WE | O RECEIVE | THE BOOS | TER VACO | CINATION | | | • | | | | | |
| Solicited AE<br>recording <sup>pp</sup> | | | | | | Cont +7 6 | d | | | | | •1 |
| Unsolicited AE<br>recording <sup>qq</sup> | | | | | | Con | t +28 d | | | | | ⊕ ii |
| Ruler training and<br>distribution of<br>ruler <sup>rr</sup> | | | | | | • | | | | | | |
| Participant e Diary review <sup>pp</sup> | | | | | | | | • | | | | |
| Approx. blood draw<br>range per visit,<br>mL <sup>nn</sup> | | 12.5 17.5 | 12.5<br>17.5 | 10.0<br>15.0 | 17.0 22.0 | 10.0 29.5 | 0.0 7.5 | 0.0<br>29.5 | 0.0<br>15.0 | 10.0 15.0 | 0.0<br>15.0 | 10 15 |
| Approx. cumulative<br>blood draw range,<br>mL <sup>nn</sup> | | 12.5 17.5 | 25.0<br>35.0 | 35.0<br>50.0 | 52.0 72.0 | 62.0 101.5 | 62.0<br>109.0 | 62.0<br>138.5 | 62.0<br>153.5 | 72.0 168.5 | 72.0-<br>183.5 | |

<sup>\*</sup> applicable for participants who initially received placebo, who will be offered a single dose of Ad26.COV2.S at the Month 6/Unblinding Visit under the conditions delineated in Section 6.4 (more details in Section 8.9).

<sup>\*\*</sup> ie, preferably within a window of 106 to +28 days around Month 6.

- \*\*\* ie, preferably within window of 100 to +170 days around Year 1, but no later than the expiry date of the Ad26.COV2.S vials available at your site.
- <sup>+</sup> applicable for participants who receive(d) a single dose of Ad26.COV2.S booster vaccination at the Year 1/Booster Visit under the conditions delineated in Section 6.5 (more details in Section 8.10) and for participants who receive(d) a booster vaccination outside of the study. Participants who choose to receive a booster vaccination outside of the study are encouraged to schedule their Year 1/Booster Visit prior to their booster vaccination, if feasible, and come in for the Year 1 + 28 Days and Year 1 + 72 Days visits within the specified visit window, if feasible, or as close as possible to the visit window.
- <sup>++</sup> only applicable for approximately the first 60 eligible participants once operationally feasible of the Homologous Booster Subset (approximately 15 per subgroup [1a, 1b, 2a, and 2b]) and approximately the first 60 eligible participants once operationally feasible of the Heterologous Booster Subset (approximately 15 per subgroup [primary vaccination with mRNA vaccine, protein vaccine, adenovector vaccine, and inactivated vaccine]) (see Section 8.1.4).
- a. Screening will be performed within 28 days prior to the study vaccination or on the day of vaccination. If screening is performed on the day of vaccination (recommended), Visit 1 and Visit 2 will coincide on Day 1. In that case, assessments should only be done once. Screening must be completed and all eligibility criteria must be fulfilled prior to randomization and vaccination.
- b. If allowed by local regulations, study visits may take place at the participant's home or other location in the event of ongoing SARS-CoV-2 transmission in the area of the participant. If possible and allowed per local regulation, visits can be performed by a phone call or a telemedicine contact. Except for the screening and vaccination visits, assessments scheduled for the other visits may also be performed by a trained health care professional (HCP), if allowed per local regulations.
- c. For those participants who are unable to continue participation in the study up to Visit 11, but for whom consent is not withdrawn, an early exit visit will be conducted as soon as possible. Participants who wish to withdraw consent from participation in the study will be offered an optional visit for safety follow-up. This includes the safety assessments of the early exit visit (no blood sampling for immunogenicity).
- d. Signing of the ICF should be done before any study-related procedure. The ICF can be signed remotely prior to the Screening Visit. Downloading of an application to the participant's eDevice, to access materials for enrollment and study information, is not considered a study-related procedure. Participants entering the open-label phase are required to sign a new ICF at the Month 6/Unblinding Visit. All participants are required to sign a new ICF at the Year 1/Booster Visit. At the Month 6/Unblinding Visit and at the time of booster vaccination (Year 1/Booster Visit), if applicable, all participants will be counselled about the importance of continuing other public health measures to limit the spread of disease including social distancing, wearing a mask, and hand-washing (see Sections 8.9 and 8.10).
- e. Check clinical status again before study vaccination.
- f. If allowed by local regulations and if the participant consents, he/she will be interviewed on characteristics related to his/her current work situation, living situation, and community interactions on Day 1 (see Appendix 12) and, at other timepoints, on changes compared to Day 1. These data will be used for risk factor analysis.
- g. For US participants only, at Day 29 or any time thereafter, the participant will be asked for optional consent to allow access to their medical data (electronic health records, claims, laboratory data from other care settings) from 5 years prior to study enrollment until 5 years after study completion utilizing tokenization and matching procedures (see Section 4.2, and Section 8.8). Participants will be informed that consent can be withdrawn at any given time. The sponsor will then remove the token generated and any associated linked real-world data (see Section 4.2.1).
- h. Only relevant medical history is to be collected, in particular: congenital abnormalities, history of cancer, history of immunodeficiency or conditions treated with immunomodulators, major psychiatric illness, major cardiovascular or lung diseases, history of an allergy to vaccination, ongoing comorbidities, history of any medical conditions known to be associated with an increased risk of progression to severe COVID-19, and history of hepatitis B or hepatitis C infection. Participants with stable/well-controlled HIV infection are allowed to enroll in the study (see Section 5.1). These participants will be encouraged to have HIV RNA viral load and CD4 cell count assessed at least twice a year and to provide these data for inclusion in the eCRF.
- i. Prestudy therapies are only to be recorded for participants with relevant comorbidities and participants aged ≥60 years. For these participants, all prestudy therapies (excluding vitamins, herbal supplements; non-pharmacologic therapies such as electrical stimulation, acupuncture, special diets, and exercise regimens) administered up to 30 days before vaccination must be recorded at screening.

- j. Vital signs may be measured at the discretion of the investigator. Under special circumstances such as high altitude, the investigator should assess baseline respiratory rate and other vital signs, as appropriate. Blood pressure is to be graded by the investigator using the toxicity grading scale in Appendix 9.
- k. Body temperature will be measured preferably via the oral route, or in accordance with the local standard of care.
- 1. If within 7 days of the vaccination.

- m. For participants of childbearing potential only. At the Month 6/Unblinding Visit, participants who are pregnant and received placebo during the double-blind phase, may be vaccinated with Ad26.COV2.S, if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (see Section 6.4). Participants who are pregnant may receive booster vaccination with Ad26.COV2.S, if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (see Section 6.5).
- n. Diagnostic molecular RT-PCR or other molecular diagnostic test for SARS-CoV-2 infection (from nasal swab collected prior to vaccination on Day 1) will be performed at a central laboratory on a retrospective basis. These baseline results will not be available in real time, and thus cannot be used to inform participants at time of enrollment.
- o. Blood sample for exploration of biomarkers correlating with SARS-CoV-2 infection and COVID-19 severity.
- p. In areas where seroprevalence is predicted to be high, a screening serologic test for past or current infection with SARS-CoV-2 may be performed (in a local laboratory), at the discretion of the sponsor, to restrict the proportion of seropositive participants in the study. This does not apply to the open-label phase of the study.
- q. MRU over the last 3 months before vaccination will be collected by interview with the participant and recorded in the eCRF.
- r. Investigator must check for acute illness or body temperature ≥38.0°C/100.4°F at the time of each vaccination. If any of these events occur within 24 hours prior to the planned vaccination in the double-blind phase, the vaccination can be rescheduled as long as this is within the allowed window. If the vaccination visit cannot be rescheduled within the allowed window or the contraindications to vaccination persist, the sponsor should be contacted for further guidance. If, at the start of the open-label phase, any of the above listed events occur at the scheduled time for the vaccination, the Month 6/Unblinding Visit with active vaccine can be delayed up to 28 days following unblinding. If any of the above listed events occur at the scheduled time for the booster vaccination, the Year 1/Booster Visit with active vaccine can be delayed within the preferred visit window.
- s. Participants will complete the eCOA using an application on their own eDevice (smartphone or tablet) if their device is compatible with the application or using the web portal.
  - All eCOA assessments should be conducted/completed before any tests, procedures, or other consultations to prevent influencing participant responses. If a participant is unable to complete the eCOA, a study staff member or the participant's caregiver can collect information on the participant's behalf as detailed in Section 8.1.2.
- t. All participants will be provided a pulse oximeter at baseline to measure blood oxygen saturation and pulse rate during a COVID-19 episode (see Section 1.3.4).
- u. The Medically-attended COVID-19 form (Appendix 8) will be provided to the participant at the vaccination visit and should be completed by the medical care provider or the study site personnel during medical visits for COVID-19 or COVID-19 complications.
- v. The SIC questionnaire asks the participant if he/she had any of the prespecified signs or symptoms (see Appendix 6) during the past 24 hours (including highest temperature in the last 24 hours), and (when applicable) to rate the severity.
- w. The first 2,000 participants in each of the 2 age groups will be closely observed for at least 30 minutes post-vaccination to monitor for the development of acute reactions. If at the time of the Day 3 safety review of the initial 2,000 participants no acute reactions have been observed in the age groups, the remaining participants in the study will be closely observed for at least 15 minutes post-vaccination. For participants in the Safety Subset (double-blind phase), any solicited local (at injection site) and systemic AEs, unsolicited AEs, SAEs, and concomitant therapies will be documented by study-site personnel following this observation period. Participants will be allowed to leave the study site after it is documented that the post-vaccination observation period is complete.
- x. Until 1 year after the Month 6/Unblinding Visit, each participant will be asked at least twice a week, through the eCOA, if they have experienced any new symptoms or health concerns that could be related to infection with SARS-CoV-2. As of 1-year after the Month 6/Unblinding Visit, through the end of the 2-year follow-up period, the frequency of this (suspected) COVID-19 surveillance (symptom check) through the eCOA may decrease to once every 2 weeks depending on

epidemiology. Sites should reach out to a participant if the participant fails to complete the surveillance question upon any of these reminders. The questionnaire will be accessible on the eCOA platform in between scheduled reminders and participants will be encouraged to answer the surveillance question in the eCOA as soon as possible after the onset of COVID-19-like symptoms. Every effort will be made to document the status of all participants that are lost to follow-up due to not completing the eCOA and for whom hospitalization has not been recorded.

If a participant develops COVID-19-like signs and symptoms, refer to Section 1.3.4 and Section 8.1.2.

Enrolled participants will be counselled on SARS-COV-2 infection prevention each time that they have a contact with site staff, in line with local guidelines. At the time of study entry, each participant will need to indicate to the study site, in case they would get infected with SARS-CoV-2, the identity and location of their routine medical care physician and/or facility and the identity and location of where they would obtain emergency care and hospitalization if necessary. If this information is not available, a plan for where such care could be obtained should be developed. If a participant should have COVID-19 and their symptoms deteriorate, they will be instructed to go to the HCP or hospital that has been identified in advance.

- y. MAAEs are to be reported for all participants from the moment of each vaccination until 6 months after the vaccination (applicable for both the double-blind and open-label phases of the study), except for MAAEs leading to study discontinuation which are to be reported during the entire study. New onset of chronic diseases will be collected as part of the MAAEs.
- z. All (S)AEs related to study procedures or non-investigational sponsor products will be reported from the time a signed and dated ICF is obtained until the end of the study/early withdrawal. All other SAEs are to be reported from the moment of vaccination until completion of the participant's last study-related procedure. AEs leading to study discontinuation (regardless of the causal relationship) are to be reported from the moment of vaccination until completion of the participant's last study-related procedure. Applicable from the time of local approval of protocol Amendment 5 onwards: Suspected AESIs are to be reported from the moment of vaccination until completion of the participant's last study-related procedure (see Section 8.3.1). Special reporting situations, whether serious or non-serious, are to be recorded from the time of each vaccination until 28 days post-vaccination (applicable for both the double-blind and open-label phases of the study). Participants will be reminded once a month to contact the study site in case of an SAE.
- aa. Refer to Section 6.10 for collection and recording of concomitant therapies associated with SAEs, solicited and unsolicited AEs, suspected AESIs, and MAAEs.
- bb. To be collected pre-vaccination only from participants receiving Ad26.COV2.S (after unblinding and/or as booster vaccination at Year 1/Booster Visit) and 28 days post booster vaccination (if applicable). Whole blood samples will be used for a complete blood count, including platelets, in a local laboratory or a substitute for local laboratory, depending on local feasibility towards turnaround time of sample processing. Serum samples will be derived from the whole blood sample and stored for potential future coagulation-related testing in a central laboratory if the participant experiences a suspected AESI (see Section 10.2, Appendix 2).
- cc. Blood sample for humoral immunity at Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, Year 1/Booster Visit (pre-vaccination, if applicable), Year 1 + 28 days for participants who received booster vaccination, Year 1 + 72 days for participants who received booster vaccination, and Month 18 (24 weeks after Year 1 Visit), also includes sample for sero-confirmation of SARS-CoV-2 infection.
- dd. Blood samples for immunogenicity will only be taken if the early exit visit is at least 10 days after the previous immunogenicity blood draw.
- ee. Blood sample for humoral immunity at Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, Year 1/Booster Visit (prior to booster vaccination, if applicable), Month 18, and Year 2, and additionally 28 days and 72 days after booster vaccination, if applicable, also includes sample for sero-confirmation of SARS-CoV-2 infection. Samples will be collected for 400 participants at selected sites.
- ff. Enrollment into the Homologous Booster Subset and Heterologous Booster subset will start once operationally feasible. Blood sample for humoral immunity at the Year 1/Booster Visit (pre-vaccination) and 28 days, 72 days, 6 months, and 1 year after booster vaccination, also includes sample for sero-confirmation of SARS-CoV-2 infection. Samples will be collected for 600 participants at selected sites.
- gg. A subset of participants (N=6,000; Safety Subset) will record solicited signs and symptoms (including body temperature) in an e-Diary via the eCOA from the time of vaccination until 7 days after double-blind vaccination.

- hh. All other unsolicited AEs will be reported for the vaccination from the time of vaccination until 28 days after double-blind vaccination. In order to perform the safety assessment after 2,000 participants have been vaccinated in Stages 1a and 2a, participants will be asked to reach out to the study site as soon as possible in case they experience a serious or severe adverse event.
- ii. If within 28 days of the vaccination.
- ij. A ruler to measure local injection site reactions will be distributed to each participant in the Safety Subset.
- kk. To be repeated pre-vaccination if previous test was >1 day ago. Participants who originally received placebo and will not be receiving the Ad26.COV2.S vaccine under EUA, do not need to complete a pregnancy test.
- 11. To be repeated pre-vaccination if previous sample was >3 days ago.
- mm. To be repeated pre-vaccination if previous sample was >5 days ago.
- nn. The approximate blood volume collected depends on whether the participant is in one of the immunogenicity subgroups and/or received Ad26.COV2.S booster vaccination at the Year 1/Booster Visit.
- oo. Those participants in the Immunogenicity Subset that transfer to the Homologous Booster Subset at the Year 1/Booster Visit will from that visit onwards follow the humoral immunogenicity sample schedule of the Homologous Booster Subset and discontinue the schedule of the Immunogenicity Subset.
- pp. All participants will collect solicited signs and symptoms (including body temperature) in an e-Diary via the eCOA from the time of booster vaccination until 7 days after booster vaccination, if feasible. The diary will be reviewed by the study personnel and solicited AEs recorded for a subset of participants included in the Safety Subset of the double-blind phase and all participants who received a heterologous prime or booster vaccination outside the study, if feasible. After the signing of informed consent of Amendment 7, no further solicited symptoms will be collected.
- qq. Unsolicited AEs will be recorded for all participants from time of booster vaccination until 28 days after booster vaccination. After signing informed consent of Amendment 7, no futher unsolicited symptoms will be collected.
- rr. A ruler to measure local injection site reactions will be distributed to all participants, if feasible.
- ss. To be collected once operationally feasible.

AE = adverse event; AESI = adverse event of special interest; approx... = approximate; cont. = continuous; COVID-19 = coronavirus disease-2019; d = day(s); eCOA = electronic clinical outcome assessment; eCRF = electronic case report form; ePRO = electronic patient-reported outcome; EUA = Emergency Use Authorization; ICF = informed consent form; MAAE = medically-attended adverse event; MRU = medical resource utilization; SAE = serious adverse event; SARS-CoV-2 = severe acute respiratory syndrome coronavirus-2; SIC = Symptoms of Infection with Coronavirus-19; vac = vaccination; w = week(s).

# 1.3.4. Participants With (Suspected) COVID-19

## 1.3.4.1. Passive Follow-up (As of Amendment 7)

As of Amendment 7, active follow-up of suspected COVID-19 episodes will be replaced by a passive follow-up approach.

New suspected COVID-19 episodes will be participant-reported and will not include any laboratory sampling. Site staff will collect information on the new COVID-19 episodes at scheduled time points and report these as SAEs, AEs, or MAAEs, as applicable. Participants may contact the site at any time in between scheduled visits to report COVID-19 episodes. Concomitant therapies related to these events are to be reported, as well as any confirmatory COVID-19 laboratory information, if available.

Guidance on (S)AE coding may be provided.

Some participants will have an ongoing COVID-19 event at time of signing the informed consent of protocol amendment 7. Also, under protocol amendment 7, the eCOA will be decommissioned. Hence participant will stop using the eCOA as of the consent visit. The outstanding activities planned for the follow-up of COVID-19 events will also end on that date for the participants (eg no further samples, no MRU completion, no MA-COV completion, no further visit in the context of the COVID-19 follow-up). The eCOA will be stopped based on approval of protocol Amendment 7 at each study site.

## 1.3.4.2. Active Follow-up (Prior to Amendment 7)

| Timing relative to onset of signs and symptoms | COVID<br>-19 | | /ID-19<br>/ 3-5 <sup>a</sup> | 2-day cy<br>repeate | | COVID<br>-19<br>Day 29<br>(±7 d) <sup>f,g</sup> |
|---|---|---|---|---|---|---|
| | Day 1-2 | Part 1 | Part 2 <sup>b</sup> | 1 <sup>st</sup> day of cycle | 2 <sup>nd</sup> day<br>of cycle | |
| Location | Homeh | Site or<br>Home <sup>i,j</sup> | Site or<br>Home <sup>i,j</sup> | Home <sup>j</sup> | Home <sup>j</sup> | Site or<br>Home <sup>i,j</sup> |
| Participant to contact study site with any health concerns/participant notifies the site of becoming aware of a positive RT-PCR test | • | | | | | |
| Site to contact participant if COVID-19 signs or symptoms are recorded in eCOA | • | | | | | |
| Confirmation of suspected COVID-19 using prespecified criteria | <b>●</b> <sup>k</sup> | •¹ | | | | |
| Nasal swab sample (collected by the participant at home) <sup>m</sup> | ● <sup>n</sup> | | | • | | |
| Nasal swab sample (collected by qualified study staff) | | •0 | | | | |
| Saliva sample (collected by the participant) <sup>p</sup> | | | • | | • | |
| Humoral immunity (serum), mL | | | ●15 | | | ●15 <sup>q</sup> |
| Biomarker RNAseq blood sample (PAXgene tubes, whole blood), mL <sup>r</sup> | | | ●2.5 | | | ●2.5 |

| In case of signs and symptoms: Symptoms of Infection with Coronavirus-19 (SIC), including highest body temperature over the last 24 hours measured by the participant <sup>s</sup> (ePROs to be completed by the participant in the eCOA) | | | Daily | | <b>●</b> <sup>t</sup> |
|---|---|---|---|---|---|
| In case of no signs or symptoms: (Suspected) COVID-19 surveillance (symptom check) | At least twice a week | | • | | |
| Risk factor assessment <sup>u</sup> | 6 | | • | | |
| Vital signs <sup>v</sup> | | • | 2 80 08 | | • |
| Targeted physical examination | | • | 2 80 08 | | • |
| Pulse oximetry by site staff | | • | 2 80 08 | | • |
| Pulse oximetry by the participant (ePRO to be completed by the participant in the eCOA) <sup>w</sup> | n | | 3 times a a | lav | |
| T disc oximed y by the participant (of its to be completed by the participant in the ecori) | 10 | | o mineo di d | | |
| Medical history (including recent flu or pneumococcal vaccination) and description of COVID-19 episode (collected by interview with the participant) | | | • | | • |
| Medical history (including recent flu or pneumococcal vaccination) and description of | | | • | | • |
| Medical history (including recent flu or pneumococcal vaccination) and description of COVID-19 episode (collected by interview with the participant) | | | • | | • |
| Medical history (including recent flu or pneumococcal vaccination) and description of COVID-19 episode (collected by interview with the participant) MRU questionnaire (collected by interview with the participant) <sup>x</sup> Capture medical information from medical visits for COVID-19 or COVID-19 complications | | | • | uous | • |

- a. The visit at COVID-19 Day 3-5 should be scheduled 2 to 4 days after symptoms onset/positive RT-PCR test from outside the study.
- b. Only applicable for participants that meet the prespecified criteria for suspected COVID-19 (Section 8.1.1) on COVID-19 Day 1-2 and COVID-19 Day 3-5 or who have a positive test result for SARS-CoV-2 on COVID-19 Days 1-2 or 3-5 visits.
- c. Participants should be encouraged by the site to collect nasal swabs and saliva samples as indicated in the Schedule of Activities. If the participant is unable or unwilling to collect all samples as requested, the participant should still complete the other COVID-19 assessments, including the visit at COVID-19 Day 29.
- d. As soon as it is confirmed that both nasal swabs (collected on COVID-19 Day 1-2 and COVID-19 Day 3-5) are negative for SARS-CoV-2, the participant will not undertake any further COVID-19 procedures and will fall back to the default Schedule of Activities, until the end of the study/early withdrawal.
- e. Participants should undertake the COVID-19 procedures until 14 days after symptom onset (COVID-19 Day 15) or until resolution of the COVID-19 episode, whichever comes last. Resolution of a COVID-19 episode is defined as having 2 consecutive SARS-CoV-2 negative nasal swabs and 2 consecutive days with no COVID-19-related signs or symptoms. Once past COVID-19 Day 15, participants should stop the collection of nasal swabs and saliva samples as soon as 2 consecutive nasal samples are SARS-CoV-2 negative, but (if still symptomatic at that time) should continue completing the ePROs (including SIC, body temperature, and pulse oximetry) in the eCOA until 2 consecutive days with no COVID-19-related signs or symptoms (Section 8.1.1).
- f. Only applicable for participants that have at least 1 SARS-CoV-2 positive nasal swab collected on COVID-19 Day 1-2 or Day 3-5. COVID-19 Day 29 should still be performed even if the nasal swabs results are still pending.
- g. The visit on COVID-19 Day 29 can be combined with a regular study visit if within the applicable visit windows.
- h. The COVID-19 Day 1-2 nasal swab can be collected at the study site (or hospital or other location, if needed), if preferred by the participant.
- i. All COVID-19 Day 3-5 and Day 29 assessments may be performed by a trained HCP at the participant's home, if allowed per local and/or institutional regulations.
- j. If a participant has a positive test result for SARS-CoV-2 infection and/or depending on the medical status of the participant, the participant may be requested to remain at home and not visit the study site. If necessary, study-site personnel or a trained HCP will visit the participant at home (or at the hospital or other location, if needed), if allowed by local regulations. Under these circumstances, the participant will be contacted by the site at least once per week and the participant's medical care provider will be notified.
- k. In case of COVID-19 like symptoms, based on the information collected through the SIC, the site will reach out to the participant at the latest on COVID-19 Day 2 (the day after the day of symptom onset) to assess whether the reported signs and symptoms qualify as a suspected COVID-19 episode using prespecified criteria

- (Section 8.1.1). As several of the prespecified criteria for suspected COVID-19 overlap with vaccine-related reactogenicity, investigators' clinical judgement is required to exclude vaccine-related events. In case the participant would actively reach out to the site already on COVID-19 Day 1, the site should already make a first assessment on COVID-19 Day 1 to check whether the reported signs and symptoms qualify as a suspected COVID-19 episode using prespecified criteria (Section 8.1.1).
- In case of COVID-19 like symptoms, the site will interview the participant to assess whether the reported signs and symptoms still qualify as a suspected COVID-19 episode using prespecified criteria (Section 8.1.1).
- m. A nasal swab should be collected from the participant at home (using available material for home swabs provided by the study staff) as soon as the prespecified criteria for suspected COVID-19 are met and, in case of COVID-19 like symptoms, preferably on the day of symptom onset or the day thereafter (COVID-19 Day 1-2). The sample collected on COVID-19 Day 1-2 should be transferred to the study site, as arranged by the study site, as soon as possible after collection, preferably within 24 hours. Nasal swabs should also be collected once every 2 days until 14 days after symptoms onset (COVID-19 Day 15) or until resolution of the COVID-19 episode, whichever comes last. These samples should be transferred to the study site, as arranged by the study site, within 3 days after collection. Details are provided in the laboratory manual. If the participant requires assistance, a trained HCP can help the participant to collect the nasal swabs. If 2 consecutive nasal swabs negative for SARS-CoV-2 are not available due to operational reasons (eg, delays in results availability), participants may cease collection of nasal swabs and saliva samples after COVID-19 Day 29, provided they have 2 consecutive days with no COVID-19-related signs and symptoms. In these cases, participants may be asked to resume sample collection if nasal sample results—once available—do not present with 2 consecutive negative swabs for SARS-CoV-2.
- n. The nasal swab should be collected and pulse oximetry should be started as soon as possible after it has been confirmed that the prespecified criteria for suspected COVID-19 (Section 8.1.1) are met.
- o. For participants with suspected COVID-19, confirmation of SARS-CoV-2 infection by RT-PCR or other molecular diagnostic test performed at a central laboratory will be used for the analysis of the case definition. All nasal swabs will also be tested by a local laboratory for case management.
- p. Saliva samples should be collected from the participant (using recipients provided by the study staff). The samples should be transferred to the study site, as arranged by the study site, within 3 days after collection. Details are provided in the laboratory manual. If the participant requires assistance, a trained HCP can help the participant to collect the saliva samples.
- q. Blood sample for humoral immunity also includes sample for sero-confirmation of SARS-CoV-2 infection (antibody).
- r. Blood sample for exploration of biomarkers correlating with SARS-CoV-2 infection and COVID-19 severity.
- s. Participants should complete the (suspected) COVID-19 surveillance (symptom check). In case of COVID-19 like signs and symptoms, participants should be encouraged by the site to complete the SIC (Appendix 6) daily, preferably in the evening around the same time each day, starting on the first day they experience symptoms. Sites should remind the participant to complete the SIC, unless special circumstances occur such as hospitalization or ventilation, in which case the reason for not completing the SIC should be recorded by site staff in the clinical database If signs and symptoms are still ongoing on COVID-19 Day 3-5, collection of SIC will be continued until AT LEAST 14 days after onset UNLESS both COVID-19 Day 1-2 and COVID-19 Day 3-5 are both negative. If either of the swabs is positive or the result is unknown AND the participant is beyond 14 days after onset of symptoms, the SIC can be stopped after 2 days without signs and symptoms.
  - If a participant is unable to complete the eCOA, a study staff member or the participant's caregiver can collect information on the participant's behalf as detailed in Section 8.1.2.
  - Participant should measure body temperature daily (oral route preferred, or in accordance with the local standard of care) and record the highest temperature in the last 24 hours.
- t. If the participant does not have symptoms at that time, he/she will only need to complete the (suspected) COVID-19 surveillance (symptom check).
- u. If allowed by local regulations and if the participant consents, he/she will be interviewed on characteristics related to their current work situation, living situation, and community interactions (See Appendix 12). These data will be used for risk factor analysis.
- v. Includes measurement of vital signs (preferably supine systolic and diastolic blood pressure, heart rate, and respiratory rate [after at least 5 minutes rest] and body temperature). It is recommended that vital signs are measured before collection of nasal swabs and blood draws.

- w. In case of COVID-19 like symptoms, the participant will be asked to measure blood oxygen saturation and pulse rate at home 3 times a day (preferably in the morning, at lunch time, and in the evening). The results will be recorded by the participant in the eCOA.
- x. Data collected as part of the MRU will be recorded in the eCRF.
- y. The MA-COV form (Appendix 8) will be provided to the participant at the vaccination visit and should be completed by the medical care provider or the study site personnel during medical visits for COVID-19 or COVID-19 complications.

Upon closure of the COVID-19 episode and procedures, all participants will fall back to the default Schedule of Activities, until the end of the study/early withdrawal. If the participant experiences new signs or symptoms suggesting possible COVID-19 at a later point in time, the participant would re-start the COVID-19 procedures from COVID-19 Day 1 onwards.

COVID-19 = coronavirus disease-2019; eCOA = electronic clinical outcome assessment; eCRF = electronic case report form; ePRO = electronic patient-reported outcome; MA-COV = medically-attended COVID-19; MRU = medical resource utilization; SARS-CoV-2 = severe acute respiratory syndrome coronavirus-2; SIC = Symptoms of Infection with Coronavirus-19.

## 1.3.5. Participants with a Suspected AESI

The medical management of thrombotic events with thrombocytopenia is different from the management of isolated thromboembolic diseases. Study site personnel and/or treating physicians should follow available guidelines for treatment of thrombotic thrombocytopenia (eg, from the American Society of Hematology<sup>2</sup>, British Society of Haematology Expert Haematology Panel<sup>10</sup>, and the CDC<sup>15</sup>). The use of heparin may be harmful and alternative treatments may be needed. Consultation with a hematologist is strongly recommended. Management of the participant should not be delayed by decision-making of the AESI Adjudication Committee. In the event of a suspected thrombotic event or TTS, laboratory assessments (to be performed locally) are required to facilitate diagnosis and determine treatment options, including but not limited to platelet count and anti- platelet factor 4 (PF4) tests.

Additional blood samples should be collected for central laboratory testing as detailed below. However, results of central laboratory testing may not be available to guide immediate treatment decisions.

In the event of a suspected thrombotic event or TTS, laboratory assessments are required to facilitate diagnosis and determine treatment options, including but not limited to platelet count and anti-PF4 tests. Additional blood samples should be collected for testing requested by the sponsor as detailed below. However, results of central laboratory testing may not be available to guide immediate treatment decisions.

| Timing relative to onset of suspected AESI | AESI<br>Day 1ª | AESI<br>Day 29 <sup>b</sup> |
|---|---|---|
| Visit Window | | ±7 d |
| Site to report suspected AESI <sup>c</sup> | • | |
| Clinical lab blood sample (whole blood), mL <sup>d</sup> | <b>●</b> 15 | • 15 |
| AESI form <sup>e</sup> Continuous | | tinuous |
| Concomitant therapies <sup>f</sup> | • | • |

- a. Day 1 refers to first awareness of the event, which might be later than the date of onset. Every effort should be made to report as much information as possible about the event to the sponsor in a reasonable timeframe. The investigator should contact the sponsor for input on the feasibility of collecting blood samples, including the need for additional samples based on the nature of the event.
- b. Day 29 is to be calculated relative to the actual day of onset of the event. If the event is not resolved on Day 29, subsequent follow-up assessments can be performed at unscheduled visits as needed until resolution of the event.
- c. Suspected AESIs must be reported to the sponsor within 24 hours of awareness irrespective of seriousness (ie, serious and non-serious AEs) or causality assessment (see Section 8.3.7).
- d. Whole blood samples will be used for a platelet count (as part of a complete blood count, if applicable) in a local laboratory or substitute for local laboratory, depending on local feasibility towards turnaround time of sample processing. Serum and plasma samples will be derived from the whole blood sample for coagulation-related testing in a central laboratory (see Section 10.2, Appendix 2). For the follow-up visit, the volume of blood to be collected may vary depending on the clinical evaluation of the case.
- e. Medical information on local case management will be collected. Upon becoming aware of the suspected AESI, study site personnel should provide information on an ongoing basis. See Section 8.3.7 and Section 10.13, Appendix 13 for further details.
- f. Refer to Section 6.10 for collection and recording of concomitant therapies associated with a suspected AESI.

AESI = adverse event of special interest; CDC = Centers for Disease Control and Prevention; PF4 = platelet factor 4; TTS = thrombosis with thrombocytopenia syndrome

## 2. INTRODUCTION

Ad26.COV2.S (previously known as Ad26COVS1) is a monovalent vaccine composed of a recombinant, replication-incompetent adenovirus type 26 (Ad26) vector, constructed to encode the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) spike (S) protein.

Unless clearly specified otherwise, this section presents information available at the time of the writing of the initial protocol, dated 22 July 2020. At that time, the Ad26.COV2.S Investigator's Brochure (IB) Edition 1.0 and its Addendum 1 were in place.<sup>41,42</sup>

Information about the disease, correlates of immunity, and safety issues concerning this new pandemic-causing virus are rapidly evolving. Therefore, it is critical to recognize that the approach outlined in this document might or will change as insights and discussions evolve.

For the most comprehensive nonclinical and clinical information regarding Ad26.COV2.S, refer to the latest version of the IB and its addenda (if applicable) for Ad26.COV2.S.

The term "study vaccine" throughout the protocol, refers to Ad26.COV2.S or placebo as defined in Section 6.1. The term "sponsor" used throughout this document refers to the entities listed in the Contact Information page(s), which will be provided as a separate document. The term "participant" throughout the protocol refers to the common term "subject." The "unblinding visit" refers to the Month 6 visit that starts the open-label phase of the study, as described in Section 2.1.

Study VAC31518COV3001 is being conducted under the sponsorship of Janssen (Janssen Vaccines & Prevention B.V) in collaboration with the coronavirus disease-2019 (COVID-19) Response Team (formerly known as OWS), which also encompasses the Biomedical Advanced Research and Development Authority (BARDA), the National Institutes of Health (NIH), and the COVID-19 Prevention Trials Network (COVPN).

#### **COVID-19 Vaccine and Considerations**

Currently, there are no available vaccines for the prevention of COVID-19. The development of a safe and effective COVID-19 vaccine is considered critical to contain the current outbreak and help prevent future outbreaks.

Although the quantitative correlate of protection against SARS-CoV-2 infection has not yet been identified, neutralizing antibody responses against the severe acute respiratory syndrome coronavirus (SARS-CoV) and Middle East respiratory syndrome coronavirus (MERS-CoV) S protein have been associated with protection against experimental SARS-CoV and MERS-CoV infection in nonclinical models. Recent studies suggest that SARS-CoV-2 has several similarities to SARS-CoV based on the full-length genome phylogenetic analysis and the putatively similar cell entry mechanism and human cell receptor usage. Therefore, a neutralizing antibody response against the SARS-CoV-2 S protein may also have a protective effect.

#### **Adenoviral-vectored Vaccines**

Recombinant, replication-incompetent adenoviral vectors are attractive candidates for expression of foreign genes for a number of reasons. The adenoviral genome is well characterized and comparatively easy to manipulate. Adenoviruses exhibit broad tropism, infecting a variety of dividing and non-dividing cells. The adenoviral vaccine (AdVac®) vector platform, developed by Crucell Holland B.V. (now Janssen Vaccines & Prevention B.V.) allows for high-yield production of replication-incompetent adenovirus vectors, eg, Ad26, with desired inserts. The adenovirus E1 region is deleted to render the vector replication-incompetent and create space for transgenes, with viral replication taking place in cells that complement for the E1 deletion in the virus genome. Ad26 has been selected as a potential vaccine vector because there is substantial nonclinical and clinical experience with Ad26-based vaccines that demonstrate their capacity to elicit strong humoral and cellular immune responses and their acceptable safety profile, irrespective of the antigen transgene (see also Section 2.3.1).

The immunogenicity profile of adenoviral vectors is illustrated by data obtained following the immunization of adults with Ad26-vectored human immunodeficiency virus (HIV) vaccines (Ad26.ENVA.01, Ad26.Mos.HIV, and Ad26.Mos4.HIV), an Ad26-vectored Ebola virus vaccine (Ad26.ZEBOV), Ad26-vectored respiratory syncytial virus (RSV) vaccines (Ad26.RSV.FA2 and Ad26.RSV.preF), an Ad26-vectored Zika virus vaccine (Ad26.ZIKV.001), and an Ad26-vectored malaria vaccine (Ad26.CS.01). Antigen-specific antibody responses are observed in almost all participants after 1 dose, in both naïve and pre-immune individuals (RSV). These antibodies may persist for a year or more (RSV) after a single-dose in pre-immune participants. They have functional properties of neutralization (RSV, Zika), crystallizable fragment (Fc)-mediated antibody-dependent cellular cytotoxicity (ADCC) and antibody-dependent cellular phagocytosis (HIV, malaria). Furthermore, these data support an immunogenicity profile with emphasis on T-helper cell type 1 (Th1) responses and demonstrate predominantly interferon gamma (IFN-γ) and tumor necrosis factor alpha (TNF-α) production in CD4<sup>+</sup> and CD8<sup>+</sup> T cells. 4,43,53

#### Ad26.COV2.S Candidate Vaccine

The aim of the COVID-19 vaccine clinical development program is to develop a safe and effective vaccine for the prevention of COVID-19. The initial effort will be to rapidly demonstrate safety and immunogenicity in adults aged ≤55 years in study VAC31518COV1001, in order to initiate the efficacy study VAC31518COV3001 in this age group as soon as possible, and to evaluate safety and immunogenicity in older adults aged ≥65 years. The candidate vaccine to be assessed in this study is Ad26.COV2.S, which is a recombinant, replication-incompetent Ad26 encoding a prefusion stabilized variant of the SARS-CoV-2 S protein. The parental S protein sequence was derived from a SARS-CoV-2 clinical isolate (Wuhan, 2019; whole genome sequence NC\_045512). The selection of antigen was based on previous work on the SARS-CoV and MERS-CoV candidate vaccines. <sup>22,33,54</sup> The S protein is the major surface protein on coronaviruses and is responsible for binding to the host cell receptor and mediating the fusion of host and viral membranes, thereby facilitating virus entry into the cell. <sup>81</sup>

## SARS-CoV-2 Virology and COVID-19 Disease Burden

SARS-CoV-2 is an enveloped, positive-sense, single-stranded ribonucleic acid (RNA) betacoronavirus. <sup>26,74</sup> It was first identified following reports of a cluster of acute respiratory illness cases in Wuhan, Hubei Province, China in December 2019. <sup>49</sup> Early epidemiological investigations suggested that the majority of early cases were linked to a seafood market, with patients infected through zoonotic or environmental exposure, followed by the subsequent spread of infection by human-to-human transmission among close contacts. <sup>49</sup> However, there is some controversy about the initial origin of the virus. <sup>27</sup> Genomic sequencing was performed on bronchoalveolar lavage fluid samples collected from patients with viral pneumonia admitted to hospitals in Wuhan, which identified a novel RNA virus from the family Coronaviridae. <sup>50,74</sup> Phylogenetic analysis of the complete viral genome revealed that the virus, SARS-CoV-2, is part of the subgenus Sarbecovirus of the genus Betacoronavirus, and is most closely related (approximately 88% identity) to a group of SARS-CoV-like coronaviruses previously sampled from bats in China. <sup>50</sup>

SARS-CoV-2 has spread rapidly and globally since its emergence. The World Health Organization (WHO) declared that the outbreak constituted a public health emergency of international concern on 30 January 2020, and declared the outbreak to be a pandemic on 11 March 2020.<sup>71,72</sup> As of 1 June 2020, approximately 6,680,000 cases of COVID-19 and approximately 375,000 COVID-19-related deaths have been reported.<sup>44</sup>

Symptoms of infection may appear from 2 to 14 days following exposure, with the clinical manifestations ranging from mild symptoms to severe illness or death.<sup>11</sup> Severe clinical presentations have been reported in as many as 20% to 25% of laboratory-confirmed cases. 32 In a study of 99 patients in a single center in Wuhan with SARS-CoV-2 infection confirmed by real-time reverse-transcriptase polymerase chain reaction (RT-PCR), the most commonly reported clinical manifestations were fever (83%), cough (82%), shortness of breath (31%), and muscle aches (11%).<sup>21</sup> In chest X-rays and computed tomographic (CT) scans, 75% of patients showed bilateral pneumonia and 14% of patients showed diffuse mottling and ground-glass opacities. In a further study of 138 patients with novel coronavirus-induced pneumonia in a single center in Wuhan, common symptoms included fever (98.6%), fatigue (69.6%), and dry cough (59.4%). 64 Lymphopenia occurred in 70.3% of patients, and chest CT scans showed bilateral patchy shadows or ground-glass opacities in the lungs of all patients. Thirty-six patients (26%) were transferred to the intensive care unit (ICU) because of complications, including acute respiratory distress syndrome, arrhythmia, and shock. Subsequent United States (US) Centers for Disease Control and Prevention (CDC) descriptions of COVID-19 clinical case definitions<sup>11</sup> and Janssen-sponsored interviews with COVID-19-experienced clinicians have included signs and symptoms of respiratory distress such as blue lips, extreme shortness of breath and dyspnea, persistent cough, deep vein thrombosis (DVT), Kawasaki-like disease, discoloration of feet and toes, chills, shaking chills, loss of sense of taste and smell, signs of stroke, disorientation, inability to respond or understand verbal communication, among others.

At present, it appears that individuals aged ≥65 years, especially those with comorbid diseases, are subject to the highest incidence of morbidity and mortality. <sup>36</sup> In contrast, a study of 2,143 children aged <18 years in China with laboratory-confirmed (34.1%) or suspected (65.9%) COVID-19

indicated that the clinical manifestations of the disease may be less severe in children than adults, with approximately 94% of cases being asymptomatic, mild, or moderate.<sup>29</sup> However, young children, particularly infants, were susceptible to severe disease, with the highest proportion of severe and critical cases by age group reported for children aged <1 year (10.6% of cases in this age group). A study of 149,082 COVID-19 cases reported in the US was consistent with these findings.<sup>18</sup> Only 1.7% of these cases occurred in persons aged <18 years although this age group accounts for 22% of the US population. Furthermore, relatively few pediatric COVID-19 cases were hospitalized, indicating that COVID-19 might have a mild course among younger patients. Hospitalization was most common among pediatric patients aged <1 year and those with underlying conditions. Recent (April-May 2020) reports describe several cases of multisystem inflammatory syndrome (MIS) in children with Kawasaki disease-like features (ie, fever, laboratory markers of inflammation, severe illness requiring hospitalization, multisystem organ involvement). Most of these children had tested positive for current or recent SARS-CoV-2 infection or were linked to a COVID-19 case. It is currently unknown if MIS is specific to children or if it may also occur in adults.<sup>13,69</sup>

The identification of SARS-CoV-2 follows the emergence of 2 other novel betacoronaviruses capable of causing severe human disease over the past 18 years: SARS-CoV and MERS-CoV, which have nucleotide sequence identity with SARS-CoV-2 of approximately 79% and 50%, respectively. The first known cases of severe acute respiratory syndrome (SARS) occurred in Southern China in November 2002. The etiological agent, SARS-CoV, is believed to be an animal virus that crossed the species barrier to humans followed by human-to-human transmission, leading to SARS cases in >25 countries. The MERS-CoV was isolated from a patient in Saudi Arabia who died of severe pneumonia and multi-organ failure in June 2012. MERS-CoV is considered to be a zoonotic virus capable of nonsustained human-to-human transmission. Since 2012, sporadic cases and community and health-care-associated clusters of infected individuals have been reported in the Middle East.

Patients with SARS or MERS present with various clinical features, ranging from asymptomatic or mild respiratory illness to fulminant severe acute respiratory disease with extrapulmonary manifestations. Both diseases have predominantly respiratory manifestations, but extrapulmonary features may occur in severe cases. By July 2003, the international spread of SARS-CoV resulted in 8,098 SARS cases and 774 deaths (case- fatality rate: 10%) with substantial social, economic and health service disruption in some affected countries. The case-fatality rate of MERS-CoV infections is estimated to be 35%.

It is not known if SARS-CoV-2 will remain as a worldwide pandemic. It is also not known if immunity is acquired after symptomatic or asymptomatic SARS-CoV-2 infection and how long it might last. Currently, the only preventive measures that have been employed with some success have been social distancing and quarantine after contact tracing and testing. Test and treat approaches await an effective proven safe therapy that can be implemented on a mass scale. It is generally believed that an effective vaccine will be 1 of the most important tools to help control this highly contagious respiratory virus.

## 2.1. Study Rationale

The sponsor is developing a COVID-19 vaccine based on a human replication-incompetent Ad26 vector encoding the SARS-CoV-2 S protein. The S protein is the major surface protein of coronaviruses. Different animal models have been used for the evaluation of candidate coronavirus vaccines against SARS-CoV (2003 outbreak), and the common conclusion that has emerged from the evaluation of several different vaccines is that the viral S protein is the only significant target for neutralizing antibodies 11,61,77,80 and the only viral protein that can elicit protective immunity in animal models. 67,12,60,75 Based on these findings, the S protein was selected as the sponsor's candidate vaccine antigen.

At the time of protocol Amendment 1 writing, initial immunogenicity and safety data (28 days post-Dose 1 data from Cohort 1a and available data from Cohort 3) from study VAC31518COV1001 have become available and demonstrate that a single dose of Ad26.COV2.S at  $5\times10^{10}$  virus particles (vp) and  $1\times10^{11}$  vp induces an immune response that meets prespecified minimum criteria and had an acceptable safety profile. These data support the sponsor's decision to proceed with the single dose regimen at a  $5\times10^{10}$  vp dose level in this Phase 3 study.

Vaccine-associated enhanced disease has been described in some animal models for SARS and MERS in which candidate vaccines induced a Th2 biased immune response, <sup>1,8,28,39,40</sup> but proof of human SARS- or MERS-vaccine-associated enhanced disease does not exist as these candidate vaccines were never tested for efficacy nor used in outbreak situations. The Ad26 vector was chosen due to its ability to induce humoral and strong cellular responses with a Th1 immune phenotype. <sup>3,5,25,53,56,57,59,68,70,76</sup> This type 1 polarity of the immune response is thought to minimize the risk of enhanced disease after SARS-CoV-2 infection.

Study VAC31518COV3001 will include  $\geq$ 18- to <60-year-old participants and participants  $\geq$ 60 years of age.

Study VAC31518COV3001 will start with enrollment in Stage 1 (≥18- to <60-year-old participants) based on all available safety and reactogenicity data, and all relevant and available immunogenicity data from Cohort 1a (adults ≥18 to ≤55 years) of the first-in-human (FIH) study with the vaccine candidate (Ad26.COV2.S; study VAC31518COV1001; see Section 2.2), immunogenicity data (including Th1 responses) from non-human primates (NHPs), and efficacy in hamsters and NHPs and all other relevant data. Immunogenicity data from Cohort 1a of study VAC31518COV1001 will include virus neutralization assay (VNA), enzyme-linked immunosorbent assay (ELISA) and Th1/Th2 response data.

Because the data from study VAC31518COV1001 (including data on elderly) demonstrated that Ad26.COV2.S at  $5\times10^{10}$  vp is both immunogenic and safe, Stage 2a (participants  $\geq$ 60 years of age) of study VAC31518COV3001 will start enrolling in parallel to Stage 1a, unless this is not allowed per local Health Authority guidance.

Within Stage 1a and Stage 2a, enrollment will be restricted to participants without comorbidities that are associated with increased risk of progression to severe COVID-19 as described below.

The study will start by enrolling approximately 2,000 participants ( $\geq$ 18- to <60-year-old) without comorbidities that are associated with increased risk of progression to severe COVID-19 (including approximately 1,000 Ad26.COV2.S recipients and approximately 1,000 placebo recipients) (Stage 1a of the study), then vaccination will be paused to allow the Data Safety Monitoring Board (DSMB) to examine Day 3 safety data (ie, from Day 1 to Day 3; including safety data from the ongoing clinical studies). If no safety concerns are identified, enrollment will proceed, expanding enrollment to  $\geq$ 18- to <60-year-old participants with and without comorbidities that are associated with increased risk of progression to severe COVID-19 (Stage 1b) (see Section 1.2 [Figure 1] for a schematic overview of the study and Section 5.2 for the list of relevant comorbidities).

In parallel to Stage 1a, in Stage 2 of the study, approximately 2,000 adults ≥60 years of age without comorbidities that are associated with increased risk of progression to severe COVID-19 will be enrolled (Stage 2a; including approximately 1,000 Ad26.COV2.S recipients and approximately 1,000 placebo recipients). Following enrollment of these initial 2,000 participants in Stage 2a, further vaccination in Stage 2 of the study will be paused to allow the DSMB to examine Day 3 safety data (ie, from Day 1 to Day 3; including safety data from Stage 1 and the ongoing clinical studies). Upon confirmation that there are no safety concerns in this population or in the Stage 1 population up to that point, enrollment will proceed, including participants aged ≥60 years with and without comorbidities that are associated with increased risk of progression to severe COVID-19 (Stage 2b) (see Section 1.2 [Figure 1] for a schematic overview of the study and Section 5.2 for the list of relevant comorbidities).

The total sample size for the study (including  $\geq 18$ - to <60-year-old and  $\geq 60$ -year-old participants, and participants with and without comorbidities that are associated with increased risk of progression to severe COVID-19) will be approximately 40,000 participants. It is intended that a minimum of approximately 30% of recruited participants will be  $\geq 60$  years of age and approximately 20% of recruited participants will be  $\geq 18$  to <40 years of age.

Refer to Section 9.2.1 for details about the sample size determination.

Following EUA, conditional licensure, or approval in any country, a single dose of Ad26.COV2.S will be offered to enrolled participants who initially received placebo, where Amendment 4 is approved by the local Health Authority and IEC/IRB, resulting in de facto unblinding of participants and investigators. Of note, after the primary analysis, sponsor personnel except individuals directly in contact with study investigators are already unblinded according to the study protocol. All participants will be encouraged to remain in the study and continue to be followed for efficacy/effectiveness, safety and immunogenicity as originally planned up to 2 years after double-blind vaccination. This will allow assessment of the duration of protection and immunogenicity of a single dose of Ad26.COV2.S by comparing 2 groups vaccinated approximately 4 to 6 months apart.

As of implementation of protocol Amendment 6, all ongoing participants in the study who have previously received any COVID-19 vaccination(s) (as primary regimen or additional dose) with the Ad26.COV2.S vaccine, and/or an mRNA vaccine or another COVID-19 vaccine authorized

for primary vaccination including protein, inactivated, and adenovector based vaccines will be offered a single booster dose of Ad26.COV2.S vaccine (5×10<sup>10</sup> vp) if the last vaccination was preferably 6 months but at least 3 months ago. Participants who choose to receive a booster vaccination with the Ad26.COV2.S vaccine (if recommended and available) or another authorized COVID-19 vaccine outside the study or choose not to receive a booster vaccination will not be withdrawn from the study and will be encouraged to remain in the study.

Following EUA approval, Ad26.COV2.S EUA, conditional licensure, or approval in any country of COVID-19 vaccines, all participants were gradually unblinded and a single dose of Ad26.COV2.S was offered to enrolled participants who initially received placebo. Also, the epidemic continued, and new variants of concern emerged, national recommendations introduced booster vaccination. The final analyses of the study that described the double-blind phase have been completed and the primary objective has been met. Further efficacy evaluations of the open-label data have limitations, due to the loss of the placebo group, due to the loss of randomization, as many participants in the placebo groups in the studies did not cross over to Ad26.COV2.S (eg., because they received another vaccine), and the participants' knowledge of the number of doses received or the timing since vaccination, which could have led to behavioral changes impacting the results. Operational challenges have impacted the feasibility of a strict follow-up of any COVID-19 episode and active surveillance cannot be sustained. Because of these reasons, the protocol has been amended to reduce the need of on-site visits and to change the requirements for COVID-19 episode reporting by applying a passive surveillance approach. Participants in the Immunogenicity Subset will continue with the on-site study visits. There are no changes to follow-up of safety endpoints, including the reporting of adverse events of special interest (AESIs). Two analyses are planned for the study: a first analysis will be conducted for the open-label phase of the study (using the initially designed "active" follow-up of COVID-19 events) and a second end-of-study analysis is planned (using passive follow-up of COVID-19 events).

## 2.2. Background

## **Nonclinical Pharmacology**

Nonclinical studies were performed to test the immunogenicity of different vaccine candidates, leading to the selection of the current vaccine for this development program. In addition, VE of Ad26.COV2-S has been shown in Syrian hamsters and NHP. Details are provided in the IB.<sup>41,42</sup>

## **Nonclinical Safety**

#### **Biodistribution**

To assess distribution, persistence, and clearance of the Ad26 viral vector platform, intramuscular (IM) biodistribution studies have been conducted in rabbits using an Ad26-based HIV vaccine, Ad26.ENVA.01, and an Ad26-based RSV vaccine, Ad26.RSV.preF. In the available biodistribution studies, the Ad26 vector did not widely distribute following IM administration in rabbits. Ad26 vector deoxyribonucleic acid (DNA) was primarily detected at the site of injection, draining lymph nodes and (to a lesser extent) the spleen. Clearance of the Ad26 vector from the tissues was observed. Both Ad26 vectors showed a comparable biodistribution despite carrying

different antigen transgenes. These data further indicate that the Ad26 vector does not replicate and/or persist in the tissues following IM injection. These platform data are considered sufficient to inform on the biodistribution profile of Ad26.COV2.S for which the same Ad26 vector backbone is used.

## **Toxicology**

The sponsor has significant nonclinical experience with Ad26-vectored vaccines using various transgenes encoding HIV, RSV, Ebola virus, filovirus, human papilloma virus, Zika, influenza (universal flu [Uniflu]), and malaria antigens. To date, more than 10 Good Laboratory Practice (GLP) combined repeated dose toxicology and local tolerance studies have been performed in rabbits (and 1 study in rats), testing the nonclinical safety of various homologous and heterologous regimens with Ad26-based vaccines at full human doses up to 1.2×10<sup>11</sup> vp. No adverse effects have been observed in these studies. The vaccine-related effects observed were similar across studies, considered to be reflective of a physiological response to the vaccines administered, and seem to be independent of the antigen transgene. Overall, there were no safety signals detected in any of the available GLP toxicology studies with Ad26-based vaccines up to the highest dose tested (1.2×10<sup>11</sup> vp). In a combined embryo-fetal and pre- and postnatal development GLP study in female rabbits with another Ad26-based vaccine (Ad26.ZEBOV, encoding an Ebola virus antigen), there was no maternal or developmental toxicity observed following maternal exposure during the premating and gestation period. A repeated dose and local tolerance GLP study, and a combined embryo-fetal and pre- and postnatal development GLP study with Ad26.COV2.S are planned to run in parallel with study VAC31518COV1001.

### **Clinical Studies**

At the time of initial protocol writing, no clinical data with the Ad26.COV2.S vaccine were available. As of 10 September 2020, a single injection of Ad26.COV2.S has been administered to 805 adult participants, aged 18 and older.

The FIH study VAC31518COV1001 will be ongoing at the time of initiation of study VAC31518COV3001. Study VAC31518COV1001 is a randomized, double-blind, placebo-controlled, Phase 1/2a multicenter study in adults aged  $\geq 18$  to  $\leq 55$  years and aged  $\geq 65$  years. The safety, reactogenicity, and immunogenicity of Ad26.COV2.S will be evaluated at 2 dose levels  $(5\times10^{10} \text{ vp})$  and  $1\times10^{11} \text{ vp}$ , administered IM as a single-dose or 2-dose schedule, with a single booster vaccination administered in 1 cohort.

The safety, reactogenicity, and immunogenicity will be evaluated in a cohort of adults aged  $\geq$ 18 to  $\leq$ 55 years (Cohort 1). Safety, reactogenicity, and immunogenicity will also be evaluated in an expanded cohort in this age group (Cohort 2). In addition, safety, reactogenicity, and immunogenicity will be evaluated in a cohort of adults aged  $\geq$ 65 years (Cohort 3). Overall, a target of 1,045 adult participants in these 2 age groups will be randomly assigned in this study.

The study includes the following cohorts (Table 1):

#### 1. Cohort 1:

- a. Cohort 1a: 375 participants (75 participants per group) aged ≥18 to ≤55 years who will be randomized in parallel in a 1:1:1:1:1 ratio to 1 of 5 vaccination groups.
- b. Cohort 1b: 25 participants (5 participants per group) aged ≥18 to ≤55 years who will be enrolled at the Beth Israel Deaconess Medical Center (BIDMC) and randomized in parallel in a 1:1:1:1:1 ratio to 1 of 5 vaccination groups. Additional exploratory immunogenicity evaluations (eg, epitope mapping, passive transfer, and certain analyses of functional and molecular antibody characteristics) will be performed for Cohort 1b.
- 2. Cohort 2: 270 participants aged ≥18 to ≤55 years will be randomized to receive Ad26.COV2.S (240 participants) or a placebo (30 participants) in the primary regimen. Cohort 2 will include an evaluation of a single booster vaccination.
- 3. Cohort 3: 375 participants (75 participants per group) aged ≥65 years who will be randomized in parallel in a 1:1:1:1:1 ratio to 1 of 5 vaccination groups.

| | | es of Study VAC31518COV1001 | |
|---|---|---|---|
| Cohort 1a (Adult | ts ≥18 to ≤55 yea | ars) | |
| Group | N | Day 1 (Vaccination 1) | Day 57 (Vaccination 2) |
| 1 | 75 | Ad26.COV2.S 5×10 <sup>10</sup> vp | Ad26.COV2.S 5×10 <sup>10</sup> vp |
| 2 | 75 | Ad26.COV2.S 5×10 <sup>10</sup> vp | Placebo |
| 3 | 75 | Ad26.COV2.S 1×10 <sup>11</sup> vp | Ad26.COV2.S 1×10 <sup>11</sup> vp |
| 4 | 75 | Ad26.COV2.S 1×10 <sup>11</sup> vp | Placebo |
| 5 | 75 | Placebo | Placebo |
| Cohort 1b (Adul | ts ≥18 to ≤55 yea | urs) <sup>a</sup> | |
| Group | N | Day 1 (Vaccination 1) | Day 57 (Vaccination 2) |
| 1 | 5 | Ad26.COV2.S 5×10 <sup>10</sup> vp | Ad26.COV2.S 5×10 <sup>10</sup> vp |
| 2 | 5 | Ad26.COV2.S 5×10 <sup>10</sup> vp | Placebo |
| 3 | 5 | Ad26.COV2.S 1×10 <sup>11</sup> vp | Ad26.COV2.S 1×10 <sup>11</sup> vp |
| 4 | 5 | Ad26.COV2.S 1×10 <sup>11</sup> vp | Placebo |
| 5 | 5 | Placebo | Placebo |
| Cohort 2a (Adult | ts ≥18 to ≤55 yea | rs) | |
| Group | N | Day 1 (Vaccination 1) b | Day 57 b |
| 1-4 | 120 | Ad26.COV2.S 5×10 <sup>10</sup> vp <sup>c</sup> | No vaccination |
| 5 | 15 | Placebo | No vaccination |
| Cohort 2b (Adul | ts ≥18 to ≤55 yea | urs) | |
| Group | N | Day 1 (Vaccination 1) b | Day 57 (Vaccination 2) b |
| 1-4 | 120 | Ad26.COV2.S 5×10 <sup>10</sup> vp | Ad26.COV2.S 5×10 <sup>10</sup> vp |
| 5 | 15 | Placebo | Placebo |
| Cohort 3 (Adults | s ≥65 years) | | |
| Group | $\mathbf{N}$ | Day 1 (Vaccination 1) | Day 57 (Vaccination 2) |
| 1 | 75 | Ad26.COV2.S 5×10 <sup>10</sup> vp | Ad26.COV2.S 5×10 <sup>10</sup> vp |
| 2 | 75 | Ad26.COV2.S 5×10 <sup>10</sup> vp | Placebo |
| 3 | 75 | Ad26.COV2.S 1×10 <sup>11</sup> vp | Ad26.COV2.S 1×10 <sup>11</sup> vp |
| 4 | 75 | Ad26.COV2.S 1×10 <sup>11</sup> vp | Placebo |
| 5 | 75 | Placebo | Placebo |
| Total | 1,045 | | |

a. Cohort 1b comprises 5 participants in each group who will be enrolled at Beth Israel Deaconess Medical Center (BIDMC) and for whom additional exploratory immunogenicity analyses will be performed.

At the time of protocol Amendment 1 writing, initial immunogenicity and safety data (28 days post-Dose 1 data from Cohort 1a and available data from Cohort 3) from study VAC31518COV1001 have demonstrated that a single dose of Ad26.COV2.S at  $5\times10^{10}$  vp and  $1\times10^{11}$  vp induces an immune response that meets prespecified minimum criteria and had an acceptable safety profile. The sponsor has therefore decided to proceed with the single dose regimen at a  $5\times10^{10}$  vp dose level in this Phase 3 study.

For more detailed information about the clinical experience with Ad26.COV2.S,refer to the IB. 42

b. Study vaccine will be administered as a single dose (Day 1) or 2 dose (Day 1 and Day 57) primary regimen. Cohort 2 will also include an evaluation of a single booster vaccination at 6, 12, or 24 months after completion of the primary single dose or 2 dose primary regimen.

c. Revised per VAC31518COV1001 protocol Amendment 6, dated 19 September 2020.

N number of participants; vp virus particles.

## Clinical Safety Experience With Ad26-based Vaccines

As described above, replication-incompetent Ad26 is being used as a vector in the development of vaccine candidates against diseases such as malaria, RSV, HIV, Ebola virus, Zika virus, and filovirus.

As of 01 July 2020, Ad26-based vaccines had been administered to approximately 90,000 participants in ongoing and completed studies, including more than 76,000 participants in an ongoing Ebola vaccine study in the Democratic Republic of the Congo (VAC52150EBL3008/DRC-EB-001) and an ongoing immunization campaign in Rwanda (UMURINZI Ebola Vaccine Program campaign).

The sponsor's clinical AdVac® safety database report (V5.0, dated 10 April 2020, cut-off date 20 December 2019) describes integrated safety data from 26 completed clinical studies using Ad26-based vaccines for which the database was locked for final analysis. In these 26 studies, 4,224 adult participants were vaccinated with an Ad26-based vaccine and 938 adult participants received a placebo. A total of 6,004 Ad26-based vaccine doses were administered to adults. Most adult participants (3,557 out of 4,224; 84.2%) received Ad26-based vaccine at a dose level of  $5\times10^{10}$  vp, while 284 adult participants (6.7%) received Ad26-based vaccine at the  $1\times10^{11}$  vp dose level (the highest dose level tested).

As of 01 July 2020, more than 85,000 participants were enrolled in ongoing studies and the ongoing immunization campaign in Rwanda (UMURINZI Ebola Vaccine Program campaign). However, their safety data were not included in the AdVac® safety database report V5.0 because the studies were still blinded, the studies were unblinded but their analysis took place after the AdVac® safety database report cut-off date, or the study data were not integrated in the Ad26-based vaccine database used for the report.

Overall, the Ad26-based vaccines were well tolerated irrespective of the antigen transgene, without significant safety issues identified to date. See Section 2.3.1 for a summary of data from the AdVac® safety database report.

Ad26-based Vaccines in Adults Aged 60 Years and Older

In the RSV vaccine clinical development program, Ad26.RSV.preF has been evaluated in studies in participants aged  $\geq$ 60 years, including the Phase 1 studies VAC18193RSV1003 and VAC18193RSV1005, Phase 1/2a study VAC18193RSV1004, Phase 2a study VAC18193RSV2003, and Phase 2b study VAC18193RSV2001. Up to a cut-off date of 24 April 2020, approximately 3,700 participants aged  $\geq$ 60 years have received an Ad26.RSV.preF-based regimen in completed and ongoing studies. An acceptable safety and reactogenicity profile in participants aged  $\geq$ 60 years has been reported for the Ad26.RSV.preF-based regimens assessed in these studies, and no safety concerns have been raised to date.

Th1/Th2 Profile of Ad26-based Vaccines in Clinical Studies

In the 1960s, a formalin-inactivated RSV vaccine was associated with enhanced respiratory disease (ERD) in young children, characterized by an increased rate of RSV-mediated, severe lower

respiratory tract infection in the vaccinated individuals compared with the control group. 23,35,45,46 Although the mechanisms for ERD are not fully understood, it is thought that FI-RSV may have: 1) failed to induce adequate neutralizing antibody titers; 2) led to an overproduction of binding antibodies promoting immune complex deposition and hypersensitivity reactions; 3) failed to induce adequate numbers of memory CD8+ T cells important for viral clearance; and 4) induced a Th2-skewed type T-cell response. 55 Vaccine-induced ERD has also been described for SARS-CoV and MERS-CoV in animal models, 42 but proof of human SARS-CoV or MERS-CoV vaccineassociated enhanced disease does not exist as these candidate vaccines were never tested for efficacy nor used in outbreak situations. For SARS and MERS, the mechanism of enhanced disease observed in mice has been associated with a Th2-mediated eosinophilic infiltration in the lung, which is reminiscent of ERD effects observed after RSV infection of mice immunized with FIRSV. Similar to RSV vaccines, enhanced disease has been shown for whole-inactivated SARS-CoV vaccines, as well as subunit vaccines inducing a Th2-type immune response, which can be rescued by formulating vaccines in Th1-skewing adjuvants. In addition to a Th1-biased immune response, also induction of a high proportion of neutralizing antibodies compared with virus binding antibodies is desirable to prevent predisposition to enhanced disease as observed for RSV vaccines. While vaccine-associated enhanced disease was observed in nonclinical studies with experimental SARS and MERS vaccines, it is not a given that the same risk applies to COVID-19 vaccines. To the sponsor's knowledge, antibody-related COVID-19 disease enhancement has not been observed in nonclinical models yet. Antibodies against the receptor-binding domain of SARS-CoV-2 were shown not to enhance in vitro infectivity. Repeated SARS-CoV-2 challenge of NHP or NHP studies with Th2 biasing COVID-19 vaccines that would be expected to predispose to enhanced disease did not show any signs of enhanced disease. In addition, disease enhancement was not observed in NHP immunized with ChAdOx1 encoding SARS-CoV-2 S protein prior to challenge with SARS-CoV-2.42

The immunogenicity profile of adenoviral vectors, with particular emphasis on Th1 responses, is illustrated by data obtained from immunization of adults with Ad26-vectored HIV vaccines (Ad26.ENVA.01 and Ad26.Mos.HIV) and Ad26-vectored Ebola vaccine (Ad26.ZEBOV). These data show predominantly IFN-γ and TNF-α production in CD4<sup>+</sup> and CD8<sup>+</sup> T cells.<sup>3,4,5</sup> In the RSV vaccine clinical development program, Ad26.RSV.preF is being evaluated in healthy RSV-seropositive toddlers aged 12 to 24 months (Phase 1/2a study VAC18194RSV2001). Safety data from the PA at 28 days after the second study vaccination revealed no safety concerns following Ad26.RSV.preF dosing at 5×10<sup>10</sup> vp or a placebo. The immunogenicity of a single immunization with Ad26.RSV.preF in RSV-seropositive toddlers aged 12 to 24 months, including favorable Th1 bias, was confirmed. In a further study of Ad26.RSV.preF in RSV-seronegative toddlers aged 12 to 24 months (Phase 1/2a study VAC18194RSV2002), initial safety data have not revealed concerns after Ad26.RSV.preF dosing.

### 2.3. Benefit-Risk Assessment

More detailed information about the known and expected benefits and risks of Ad26.COV2.S may be found in the IB.<sup>42</sup>
## 2.3.1 Risks Related to Study Participation

The following potential risks of Ad26.COV2.S will be monitored during the study and are specified in the protocol.

#### Risks Related to Ad26.COV2.S

No clinical data with Ad26.COV2.S are available at the time of finalization of the initial VAC31518COV3001 protocol.

For emerging clinical data and the most comprehensive nonclinical information regarding Ad26.COV2.S, refer to the latest version of the IB and its addenda (if applicable).

Sites should advise participants that side effects include fever as well as injection site pain, headache, fatigue, myalgia, and nausea per the current ICF; however, the occurrence of fever appears to be more common in younger adults and can be severe. This is based on information from study VAC31518COV1001 that became available at the time of protocol Amendment 1 writing.

Anaphylaxis is considered an important identified risk for Ad26.COV2.S. Individuals should be observed by a healthcare provider after vaccination per protocol requirements. Refer to the latest version of the IB and its addenda (if applicable) for further details.

Thrombosis in combination with thrombocytopenia (thrombosis with thrombocytopenia syndrome [TTS]), in some cases accompanied by bleeding, has been observed very rarely following vaccination with Ad26.COV2.S. Reports include severe cases of venous thrombosis at unusual sites such as cerebral venous sinus thrombosis (CVST), splanchnic vein thrombosis and arterial thrombosis, in combination with thrombocytopenia. These cases occurred approximately 1-2 weeks following vaccination, mostly in women under 60 years of age. Thrombosis in combination with thrombocytopenia can be fatal. The exact physiology of TTS is unclear. TTS is considered an important identified risk for Ad26.COV2.S. Participants should be instructed to seek immediate medical attention if they develop symptoms such as shortness of breath, chest pain, leg swelling, persistent abdominal pain, severe or persistent headaches, blurred vision, and skin bruising and/or petechiae beyond the site of vaccination. The medical management of thrombosis with thrombocytopenia is different from the management of isolated thromboembolic diseases. Study site personnel and/or treating physicians should follow available guidelines for treatment of thrombotic thrombocytopenia (eg, from the American Society of Hematology<sup>2</sup>, British Society of Haematology - Expert Haematology Panel<sup>10</sup>, and the CDC<sup>15</sup>). The use of heparin may be harmful and alternative treatments may be needed. Consultation with a hematologist is strongly recommended. Management of the participant should not be delayed by decision-making of the AESI Adjudication Committee. Refer to the latest version of the IB and its addenda (if applicable) for further details. Due to the possibility of the occurrence of TTS after vaccination with Ad26.COV2.S, additional reporting and data collection procedures have been included in the study

for thrombotic events, thrombocytopenia, and TTS (see Section 8.3.7 and Section 8.3.7.1), which may facilitate diagnosis and clinical management of the event.

## Risks Related to Ad26.COV2.S Administration after Previous Vaccination Ad26.COV2.S

Preliminary safety data of an Ad26.COV2.S booster administered at the 5×10<sup>10</sup> vp dose level ≥6 months post-primary single-dose Ad26.COV2.S (5×10<sup>10</sup> vp) vaccination indicate that the safety and reactogenicity of a second Ad26.COV2.S dose is acceptable and in line with the safety and reactogenicity observed after the first Ad26.COV2.S dose. There is no indication of increased reactogenicity upon administration of a second dose of Ad26.COV2.S and no safety concerns have been observed.

# Risks Related to Ad26.COV2.S Administration after Previous Vaccination with a Different COVID-19 Vaccine

To date, no clinical data are available for Ad26.COV2.S vaccination after previous vaccination with a different COVID-19 vaccine.

#### Risks Related to Adenoviral-vectored Vaccines

The clinical AdVac® safety database (report version 5.0, dated 10 April 2020, cut-off date 20 December 2019) contains pooled safety data from 26 Janssen-sponsored clinical studies with Ad26 vaccine candidates: Ad26.ZEBOV (Ebola; 10 studies), Ad26.ENVA.01, Ad26.Mos.HIV and Ad26.Mos4.HIV (HIV; 8 studies), Ad26.CS.01 (malaria; 1 study), Ad26.RSV.FA2 and Ad26.RSV.preF (RSV; 6 studies), and Ad26.Filo (filovirus; 1 study). In these studies, 4,224 adult participants and 650 children received at least 1 vaccination with an Ad26-based vaccine. The AdVac® safety database report includes data only from studies for which the database has been locked for the final analysis; therefore, of the studies including an Ad26.RSV.preF-based regimen mentioned in Section 2.2, only data for approximately 230 participants aged ≥60 years from studies VAC18193RSV1003, VAC18193RSV1005, and VAC18193RSV2003 were included.

Overall, the Ad26-based vaccines were well tolerated, without significant safety issues identified.

The majority of solicited local and systemic AEs were of mild or moderate severity and usually started within 1 to 2 days after vaccination. Most of the events resolved within 1 to 3 days.

In adults, the most frequently reported solicited local AE was injection site pain (56.9% of Ad26 participants, compared with 22.5% of placebo participants). All other solicited local AEs were experienced by less than 25% of adult participants. The most frequently experienced solicited local AE in children was injection site pain, reported in 13.9% of children aged 1-3 years, 29.8% of children aged 4 to 11 years, and 24.8% of children aged 12 to 17 years after vaccination with an Ad26-based vaccine. For placebo, these percentages were 29.2% in children aged 4 to 11 years and 14.3% in children aged 12 to 17 years. No children aged 1 to 3 years have received placebo.

Severe injection site pain was experienced by 1.0% of adult Ad26 participants and 0.8% of children aged 4 to 11 years. No children in the other 2 age groups and no placebo participants experienced severe injection site pain.

There was a trend toward an increase in the frequency of some local AEs with an increase in Ad26 dose, ie, injection site pain (18.7% of participants at the  $0.8\times10^{10}$  vp dose level, 38.7% of participants at the  $2\times10^{10}$  vp dose level, 52.0% of participants at the  $5\times10^{10}$  vp dose level, and 77.1% of participants at the  $1\times10^{11}$  vp dose level), and to a lesser extent injection site swelling (6.7%, 2.7%, 9.3%, and 17.6%, respectively). Injection site warmth was not collected at the  $0.8\times10^{10}$  vp and the  $2\times10^{10}$  vp dose level. The frequency of injection site warmth at the  $5\times10^{10}$  vp and the  $1\times10^{11}$  vp dose level was 19.5%, and 26.7%, respectively. This trend needs to be interpreted with caution since the participants in the lower dose groups ( $0.8\times10^{10}$  vp and  $2\times10^{10}$  vp dose level) were all from a single study (VAC52150EBL3002), and the majority of the participants in the highest dose group ( $1\times10^{11}$  vp dose level) were also from a single study (VAC18193RSV2003).

The most frequently reported solicited systemic AEs (ie, reported in more than 30% of participants) for adult Ad26 participants were malaise (53.8%), fatigue (48.3%), headache (45.7%), and myalgia (38.3%), all of which were more frequent for Ad26 participants compared with placebo (36.4%, 30.7%, 30.0%, and 17.7% of placebo participants, respectively). Most of these events were considered related to the study vaccine. Pyrexia (9.9%) and vaccine-related pyrexia (9.0%) were also reported more frequently after administration of an Ad26-based vaccine compared with placebo (3.5% and 2.9%, respectively).

Solicited systemic AEs reported in  $\geq 10\%$  of children aged 1 to 3 years were decreased appetite (13.9%), decreased activity (13.2%), pyrexia (11.1%), and irritability (10.4%). The most frequently reported solicited systemic AEs in children aged 4 to 11 years (reported in  $\geq 15\%$  of Ad26 participants) were headache (23.6%; no data are available for the placebo group in this age group), and decreased activity (18.5%) and irritability (17.6%), which were both reported in 4.2% (N 1) of placebo participants. The most frequently reported solicited systemic AEs in children aged 12 to 17 years (reported in  $\geq 15\%$  of Ad26 participants) were headache (34.6%) and fatigue (24.0%), compared to 33.3% and 19.0% of placebo participants, respectively. Most of the frequently experienced solicited systemic AEs in children were considered related to the study vaccine.

The majority of solicited systemic AEs were of mild or moderate severity. For adults, 6.5% of Ad26 participants and 2.0% of placebo participants reported severe solicited systemic AEs, mostly malaise and fatigue. Other severe solicited systemic AEs were reported in less than 3% of adult Ad26 participants.

There was a trend toward an increase in the frequency of solicited systemic AEs with an increase in Ad26 dose (35.3% at the  $0.8 \times 10^{10}$  vp dose level, 49.3% at the  $2 \times 10^{10}$  vp dose level, 64.5% at the  $5 \times 10^{10}$  vp dose level, and 70.4% at the  $1 \times 10^{11}$  vp dose level). The frequency of severe solicited systemic AEs also tended to increase with higher Ad26 dose, ie, 1.3% of participants at the  $0.8 \times 10^{10}$  vp and the  $2 \times 10^{10}$  vp dose level, 5.3% of participants at the  $5 \times 10^{10}$  vp dose level, and 14.4% of participants at the  $1 \times 10^{11}$  vp dose level. This trend needs to be interpreted with caution since the participants in the lower dose groups  $(0.8 \times 10^{10}$  vp and  $2 \times 10^{10}$  vp dose level) were all from a single study (VAC52150EBL3002), and the majority of the participants in the highest dose group  $(1 \times 10^{11}$  vp dose level) were also from a single study (VAC18193RSV2003).

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

The most frequently reported unsolicited AE in adult Ad26 participants was upper respiratory tract infection (5.3% vs. 7.0% in adult placebo participants). The most frequently reported unsolicited AEs considered related to the vaccine were neutropenia (1.0% of adult Ad26 participants vs. 0.5% of adult placebo participants) and dizziness (0.7% vs. 0.2%, respectively).

For Ad26, the most frequently reported unsolicited AE in children was malaria, a reported in 36.8% of children aged 1 to 3 years, in 19.0% of children aged 4 to 11 years, and in 10.6% of children aged 12 to 17 years. One child in the 12 to 17 years group (4.8%) experienced malaria after placebo vaccination. There were no other children in the placebo groups who experienced malaria. The most frequently reported related unsolicited AE was hypernatremia (1.6% of children aged 4 to 11 years [vs. 4.2% with placebo] and 2.4% of children aged 12 to 17 years [vs. 4.8% with placebo]). No AEs in children aged 1 to 3 years were considered related to the vaccine.

#### **General Risks Related to Vaccination**

In general, IM injection may cause local itching, warmth, pain, tenderness, erythema/redness, induration, swelling, arm discomfort, or bruising of the skin. Participants may exhibit general signs and symptoms associated with IM injection of a vaccine and/or placebo, including fever, chills, rash, myalgia, nausea/vomiting, headache, dizziness, arthralgia, general itching, and fatigue. These side effects will be monitored but are generally short-term. Instructions regarding use of antipyretic medication can be found in Section 6.10.

Syncope can occur in association with administration of injectable vaccines. Syncope can be accompanied by falls. Procedures should be in place to avoid falling injury. If syncope develops, participants should be observed until the symptoms resolve. Fear of injection might lead to fainting and fast breathing.

Participants may have an allergic reaction to the vaccination. An allergic reaction may cause a rash, urticaria, or even anaphylaxis (see above risks related to Ad26.COV2.S). Severe reactions are rare. Participants with a known or suspected allergy, or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine), will be excluded from the study.

After vaccination, participants will remain at the study site for close observation by study staff to monitor for the development of any acute reactions. The first 2,000 participants in each of the 2 age groups will remain under observation at the study site for at least 30 minutes after vaccination to monitor for the development of acute reactions. If at the time of the Day 3 safety review of the initial 2,000 participants no acute reactions have been observed in the age groups, the observation period at the study site may be reduced to at least 15 minutes for the remaining participants in the study. Necessary emergency equipment and medications must be available in the study site to treat severe allergic reactions.

а

<sup>&</sup>lt;sup>a</sup>This was expected as the pediatric studies were conducted in malaria-endemic regions. The imbalance in the frequency of malaria between Ad26 participants and placebo participants can largely be explained by the fact that the active control group of study VAC52150EBL3001 was not included in the pooling.

# **Pregnancy and Birth Control**

The effect of the study vaccine on a fetus or on nursing baby is unknown.

Given the limited number of incident pregnancies in the clinical studies with Ad26-based vaccines in the AdVac® safety database report (HIV vaccine: 20 pregnancies in participants and 10 in partners of participants; Ebola vaccine: 32 pregnancies in participants and 13 in partners of participants), it is not possible at present to draw firm conclusions on the safety of the vaccines when administered around the time of conception or prior to the initiation of the pregnancies. There is currently no concerning pattern of AEs in the pregnancies initiated around the time of vaccination or after exposure to the Ad26-based vaccines in the Janssen vaccines clinical development programs.

Participants of childbearing potential will be required to agree to practicing an acceptable effective method of contraception and agree to remain on such a method of contraception from providing consent until 3 months after receiving study vaccine (see Section 5.1). Use of condoms is not considered as an acceptable contraceptive barrier method due to the failure rate of female and male condoms. Participants who are pregnant at screening will be excluded from the double-blind phase of the study. Participants who are pregnant at their Month 6/Unblinding Visit and received placebo during the double-blind phase, may be vaccinated with Ad26.COV2.S if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (see Section 6.4). Participants who are pregnant may receive booster vaccination with Ad26.COV2.S, if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus. Participants who become pregnant during the study will remain in the study and will continue to undergo all procedures for surveillance and follow-up of COVID-19 and all safety follow-up as outlined in the protocol for all participants. Participants who are breastfeeding are allowed to participate in the study.

#### **Risks from Blood Draws**

Blood draws may cause pain, tenderness, bruising, bleeding, dizziness, vasovagal response, syncope, and rarely, infection at the site where the blood is taken.

#### Risks from Collection of Nasal Swab Samples

Collection of a nasal swab sample may cause a nosebleed.

Participants are asked to perform the nasal swab samples themselves at home or to seek assistance from a trained health care professional (HCP). Assistance with the collection of nasal swab samples bears the risk of potentially infecting the assistant.

#### Theoretical Risk of Enhanced Disease

Vaccine-associated enhanced disease has been described for SARS-CoV and MERS-CoV in some animal models<sup>1,8,28,39,40</sup>, and is associated with non-neutralizing antibodies and a Th2-skewed immune response. In contrast, the Ad26-based vaccines have been shown to induce a clear Th1-skewed immune response and generate potent neutralizing antibody responses in both humans

and animal models (see Section 2.2). Participants in the present study will be informed of the theoretical risk of disease enhancement in the informed consent form (ICF). As a risk mitigation strategy, all enrolled participants will be intensively monitored (up to Amendment 7) during the conduct of the study to rapidly diagnose COVID-19 and refer for treatment, if applicable. In case of any new symptoms or health concerns that could be related to infection with SARS-CoV-2, participants will be evaluated for acquisition of molecularly confirmed COVID-19 and severity will be assessed using the case definitions specified in Section 8.1.3 by the investigator. The subset of cases with potential for severe disease will be assessed by the Clinical Severity Adjudication Committee (see Section 8.1.3.6), as part of the primary and secondary endpoints (see Section 3). All participants will be monitored for safety (including enhanced disease) for approximately 1 year after the Year 1/Booster Visit, ie, until the last study visit. In addition, as detailed in Section 9.8, the statistical support group (SSG) will monitor the number and severity of molecularly confirmed COVID-19 cases in the Ad26.COV2.S and placebo groups to identify an imbalance between groups if it occurs. The SSG will inform the DSMB as soon as an imbalance between groups is detected. A prespecified threshold (imbalance above a certain percentage and/or number of cases) that will trigger notification of the DSMB will be described in the SAP.

#### **Unknown Risks**

There may be other risks that are not known. If any significant new risks are identified, the investigators and participants will be informed.

# 2.3.2 Benefits of Study Participation

Participants may benefit from clinical testing and physical examination.

The efficacy, immunogenicity and safety data to date support a favorable benefit-risk profile for Ad26.COV2.S in the proposed indication, ie, active immunization to prevent COVID-19 caused by SARS-CoV-2 in adults ≥18 years of age. The overall benefit and risk balance for individual participants is ongoing.

Preliminary immunogenicity and safety data for a Ad26.COV2.S booster dose ( $5 \times 10^{10}$  vp) at  $\ge 6$  months post-primary single-dose Ad26.COV2.S administration and efficacy data for a  $2^{nd}$  dose of Ad26.COV2.S 2-3 months post-primary single-dose Ad26.COV2.S administration support a favorable benefit-risk profile.

## 2.3.3 Benefit-Risk Assessment of Study Participation

Based on the available data and proposed safety measures, the overall benefit-risk assessment for this clinical study is considered acceptable for the following reasons:

• Only participants who meet all inclusion criteria and none of the exclusion criteria (specified in Section 5) will be allowed to participate in this study. The selection criteria include adequate provisions to minimize the risk and protect the well-being of participants in the study.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

• Safety will be closely monitored throughout the study:

In general, safety evaluations will be performed at scheduled visits during the study, as indicated in the Schedules of Activities.

The first 2,000 participants in each of the 2 age groups will remain under observation at the study site for at least 30 minutes after vaccination to monitor for the development of acute reactions. If at the time of the Day 3 safety review of the initial 2,000 participants no acute reactions have been observed in the age groups, the observation period at the study site may be reduced to at least 15 minutes for the remaining participants in the study. Necessary emergency equipment and medications must be available in the study site to treat severe allergic reactions. Participants in the Safety Subset will use an e-Diary to document solicited signs and symptoms. Details are provided in Section 8.3.

The investigator or the designee will document unsolicited AEs for participants in the Safety Subset, and SAEs and medically-attended adverse events (MAAEs) for all participants as indicated in Section 8.3 and Appendix 4.

Suspected AESIs (thrombotic events and thrombocytopenia [defined as platelet count below  $150,000/\mu L]^9$ ) must be reported to the sponsor within 24 hours of awareness. From the time of local approval of protocol Amendment 5 onwards, TTS is considered an AESI (Section 8.3.7). Suspected AESIs will be followed up as described in the Schedule of Activities in Section 1.3.5. Refer to Section 10.14 Appendix 14 for a list of thrombotic events to be reported to the sponsor as suspected AESIs.

Any clinically significant abnormalities (including those persisting at the end of the study/early withdrawal) will be followed by the investigator until resolution or until clinically stable.

A DSMB will be established to monitor safety data on an ongoing basis to ensure the continuing safety of the participants enrolled in this study. This committee will review interim unblinded data. The DSMB responsibilities, authorities, and procedures will be documented in the DSMB Charter. The DSMB will also review Day 3 safety data (ie, from Day 1 to Day 3; including safety data from the ongoing clinical studies) from participants enrolled in Stages 1a and Stage 2a, before enrollment of participants in Stages 1b and Stage 2b, respectively. Additional ad hoc review may be performed further to the occurrence of any SAE leading to a study pausing situation as outlined in Section 6.11, or at request of the sponsor's medical monitor or designee. During the open-label phase, the DSMB will continue to monitor safety.

• Several safety measures are included in this protocol to minimize the potential risk to participants, including the following:

The study will use the following enrollment strategy to mitigate the risks for participants at increased risk of progression to severe COVID-19:

In Stage 1 (double-blind phase), the study will enroll ≥18- to <60-year-old participants (Stage 1 of the study) based on immunogenicity and safety data from Cohort 1a of study VAC31518COV1001 (see details in Section 2.1). In Stage 1a, approximately 2,000 participants without comorbidities that are associated with increased risk of progression to severe COVID-19 will be enrolled (including

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

approximately 1,000 Ad26.COV2.S recipients and approximately 1,000 placebo recipients), then vaccination will be paused to allow the DSMB to examine Day 3 safety data (ie, from Day 1 to Day 3; including safety data from the ongoing clinical studies). If no safety concerns are identified, enrollment will proceed, including ≥18-to <60-year-old participants with and without comorbidities that are associated with increased risk of progression to severe COVID-19 (Stage 1b) (see Section 1.2 [Figure 1] for a schematic overview of the study and Section 5.2 for the list of relevant comorbidities).

In Stage 2 (double-blind phase) of the study, approximately 2,000 adults ≥60 years of age without comorbidities that are associated with increased risk of progression to severe COVID-19 will be enrolled (Stage 2a; including approximately 1,000 Ad26.COV2.S recipients and approximately 1,000 placebo recipients) (see details in Section 2.1). Considering the data from study VAC31518COV1001 (including data on elderly), Stage 2a will be enrolled in parallel with Stage 1a, unless this is not allowed per local Health Authority guidance. Following enrollment of the initial 2,000 participants aged ≥60 years (Stage 2a), further vaccination in Stage 2 of the study will be paused to allow the DSMB to examine Day 3 safety data (ie, from Day 1 to Day 3; including safety data from Stage 1 and the ongoing clinical studies). Upon confirmation that there are no safety concerns in this population or in the Stage 1 population up to that point, enrollment will proceed, including participants aged ≥60 years with and without comorbidities that are associated with increased risk of progression to severe COVID-19 (Stage 2b) (see Section 1.2 [Figure 1] for a schematic overview of the study and Section 5.2 for the list of relevant comorbidities).

Up to Protocol Amendment 7: Participants will be intensively monitored in this study to rapidly diagnose COVID-19 and refer for treatment, if applicable. This will mitigate the theoretical potential risk for vaccine-associated enhanced disease when immunized individuals are infected with the virus. The induction of neutralizing antibody and the Th1 response induced by this vaccine in animals also mitigates this risk.

There are prespecified rules for participants in Stages 1a and 2a, that if met would result in pausing of further vaccinations (see Section 6.11), preventing exposure of new participants to study vaccine until the DSMB reviews all safety data (see Committees Structure in Appendix 3 [Section 10.3.6]).

Study vaccinations will be discontinued in participants for the reasons included in Section 7.

Contraindications to vaccination are included in Section 5.5.

After the EUA, conditional licensure, or approval in any country, the study will be conducted in the open-label fashion. All enrolled participants who initially received placebo will be offered to receive a single dose of Ad26.COV2.S and will continue to be monitored for safety as mentioned in Section 8.3. At the Month 6/Unblinding Visit, all participants will be counselled about the importance of continuing other public health

measures to limit the spread of disease including social distancing, wearing a mask, and hand-washing (Section 8.9).

Ninety% of the participants who receive a booster vaccination will be monitored for safety until 1 year post booster vaccination as mentioned in Section 8.3. The remaining 10% of subjects will be monitored for safety at least 6 months. At the Year 1/Booster Visit, all participants will be counselled about the importance of continuing other public health measures to limit the spread of disease including social distancing, wearing a mask, and hand-washing (Section 8.10).

## 3. OBJECTIVES AND ENDPOINTS

# 3.1. Double-blind Phase of the Study

| Objectives | Endpoints |
|---|---|
| Co-Primary | |
| To demonstrate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , as compared to placebo, in SARS-CoV-2 seronegative adults | <ul> <li>First occurrence of molecularly confirmed<sup>a</sup>, moderate to severe/critical COVID-19<sup>b</sup>, with onset at least 14 days after double-blind vaccination (Day 15)</li> <li>First occurrence of molecularly confirmed<sup>a</sup>, moderate to severe/critical COVID-19<sup>b</sup>, with onset at least 28 days after double-blind vaccination (Day 29)</li> </ul> |
| Secondarye | |
| (The method used to perform hypothesis testing prespecified in the Statistical Analysis Plan [SAP]) | serving the family-wise error rate [FWER] will be |
| Efficacy | |
| To demonstrate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed <sup>a</sup> , severe/critical COVID-19 <sup>b</sup> , as compared to placebo | <ul> <li>First occurrence of molecularly confirmed<sup>a</sup>, severe/critical COVID-19<sup>b</sup>, with onset at least 14 days after double-blind vaccination (Day 15)</li> <li>First occurrence of molecularly confirmed<sup>a</sup>, severe/critical COVID-19<sup>b</sup>, with onset at least 28 days after double-blind vaccination (Day 29)</li> </ul> |
| To demonstrate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , as compared to placebo, in adults regardless of their serostatus | <ul> <li>First occurrence of molecularly confirmed<sup>a</sup>, moderate to severe/critical COVID-19<sup>b</sup>, with onset 1 day after double-blind vaccination</li> <li>First occurrence of molecularly confirmed<sup>a</sup>, moderate to severe/critical COVID-19<sup>b</sup>, with onset 14 days after double-blind vaccination (Day 15)</li> </ul> |
| | • First occurrence of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , with onset at least 28 days after double-blind vaccination (Day 29) |

| Objectives | Endpoints |
|---|---|
| To evaluate the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed moderate to severe/critical COVID-19 <sup>b</sup> as compared to placebo, with onset 1 day after study vaccination | First occurrence of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> with onset 1 day after double-blind vaccination |
| To assess the effect of Ad26.COV2.S on COVID-19 requiring medical intervention (based on objective criteria) compared to placebo | • First occurrence of COVID-19 requiring medical intervention (such as a composite endpoint of hospitalization, ICU admission, mechanical ventilation, and ECMO, linked to objective measures such as decreased oxygenation, X-ray or CT findings) and linked to any molecularly confirmed <sup>a</sup> , COVID-19 <sup>b,c</sup> at least 14 days after double-blind vaccination (Day 15) |
| | • First occurrence of COVID-19 requiring medical intervention and linked to any molecularly confirmed <sup>a</sup> , COVID-19 <sup>b,c</sup> at least 28 days after double-blind vaccination (Day 29) |
| To assess the effect of Ad26.COV2.S on SARS-CoV-2 viral RNA load compared to placebo for moderate to severe/critical COVID-19 <sup>b</sup> | Assessment of the SARS-CoV-2 viral load by quantitative RT-PCR, in participants with molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> by serial viral load measurements during the course of a COVID-19 episode |
| To assess the effect of Ad26.COV2.S on molecularly confirmed <sup>a</sup> , mild COVID-19 <sup>c</sup> | • First occurrence of molecularly confirmed <sup>a</sup> , mild COVID-19 <sup>c</sup> , at least 14 days after double-blind vaccination (Day 15) |
| | • First occurrence of molecularly confirmed <sup>a</sup> , mild COVID-19 <sup>c</sup> , at least 28 days after double-blind vaccination (Day 29) |
| To assess the effect of Ad26.COV2.S on COVID-<br>19 as defined by the US FDA harmonized case<br>definition <sup>d</sup> | • First occurrence of molecularly confirmed <sup>a</sup> COVID-19 <sup>d</sup> at least 14 days after double-blind vaccination (Day 15) |
| | • First occurrence of molecularly confirmed <sup>a</sup> COVID-19 <sup>d</sup> at least 28 days after double-blind vaccination (Day 29) |
| To assess the effect of Ad26.COV2.S on all molecularly confirmed <sup>a</sup> symptomatic COVID 19 <sup>b,c</sup> , as compared to placebo | • Burden of disease (BOD) endpoint (see Section 9.5.2) derived from the first occurrence of molecularly confirmed symptomatic COVID-19 <sup>c</sup> (meeting the mild, moderate or severe/critical COVID-19 case definition) with onset at least 14 days after double-blind vaccination (Day 15). |
| | BOD endpoint (see Section 9.5.2) derived from<br>the first occurrence of molecularly confirmed <sup>a</sup><br>symptomatic COVID-19 <sup>c</sup> (meeting the mild,<br>moderate or severe/critical COVID-19 case) |

| Objectives | Endpoints |
|---|---|
| | definition) with onset at least 28 days after double-blind vaccination (Day 29). |
| To assess the effect of Ad26.COV2.S on occurrence of confirmed asymptomatic or undetected infections with SARS-CoV-2, as compared to placebo | • Serologic conversions: between baseline (Day 1; pre-vaccination) and Day 29, between Day 29 and Day 71, between Day 71 and Month 6/Unblinding Visit, and Month 18 after double-blind vaccination (approximately 12 months after initiation of the open-label phase of the study) using an ELISA and/or SARS-CoV-2 immunoglobulin assay that is dependent on the SARS-CoV-2 nucleocapsid (N) protein |
| | • Asymptomatic infection detected by RT-PCR at the time of the Month 6/Unblinding Visit |
| To assess the efficacy of Ad26.COV2.S in the prevention of SARS-CoV-2 infection (both symptomatic and asymptomatic infections combined, that are serologically and/or molecularly confirmed <sup>a</sup> ), as compared to placebo | First occurrence of SARS-CoV-2 infection (serologically and/or molecularly confirmed <sup>a</sup> ) with onset at least 28 days after double-blind vaccination (Day 29) |
| Safety | |
| To evaluate safety in terms of SAEs and AESIs (during the entire study), MAAEs (until 6 months after double-blind or open-label vaccination), and MAAEs leading to study discontinuation (during the entire study) for all participants | Occurrence and relationship of SAEs and AESIs (during the entire study), MAAEs (until 6 months after [double-blind or open-label] Ad26.COV2.S), and MAAEs leading to study discontinuation (during the entire study) for all participants following vaccination |
| In a subset of participants, to evaluate the safety and reactogenicity in terms of solicited local and systemic AEs during the 7 days after double-blind vaccination, and in terms of unsolicited AEs during the 28 days after double-blind vaccination | Occurrence, intensity, duration and relationship of solicited local and systemic AEs during the 7 days following vaccination and of unsolicited AEs during the 28 days after double-blind vaccination |
| Immunogenicity | |
| In a subset of participants, to evaluate the immunogenicity of Ad26.COV2.S, as compared to placebo | Analysis of antibodies binding to the SARS-CoV-2 S protein by ELISA |
| Exploratory | |
| To evaluate the long term durability of the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , by comparing 2 groups vaccinated approximately 4 to 6 months apart | First occurrence of molecularly confirmed <sup>a</sup> , moderate to severe/critical COVID-19 <sup>b</sup> , defined as having an onset of at least: • 1 day after Ad26.COV2.S • 14 days after Ad26.COV2.S • 28 days after Ad26.COV2.S. |
| To assess the effect of Ad26.COV2.S on occurrence of confirmed asymptomatic or undetected infections with SARS-CoV-2, as compared to placebo from Day 1 to Day 29 | Serologic conversion between baseline (Day 1; pre-vaccination) and Day 29 after double-blind vaccination using an ELISA and/or SARS-CoV-2 |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Objectives | Endpoints |
|---|---|
| | immunoglobulin assay that is dependent on the SARS-CoV-2 nucleocapsid (N) protein |
| To assess the effect of Ad26.COV2.S on SARS-CoV-2 viral RNA load compared to placebo for mild COVID-19° | Assessment of the SARS-CoV-2 viral load by quantitative RT-PCR, in participants with molecularly confirmed <sup>a</sup> , mild COVID-19 <sup>c</sup> by serial viral load measurements during the course of a COVID-19 episode |
| To assess the effect of Ad26.COV2.S on health care utilization (such as hospitalization, ICU admission, ventilator use) linked to any molecularly confirmed COVID-19, as compared | • Health care utilization (such as hospitalization, ICU admission, ventilator use) linked to any molecularly confirmed COVID-19 at least 14 days after double-blind vaccination (Day 15) |
| to placebo | Health care utilization (such as hospitalization, ICU admission, ventilator use) linked to any molecularly confirmed COVID-19 at least 28 days after double-blind vaccination (Day 29) |
| To assess the efficacy of Ad26.COV2.S in the prevention of SARS-CoV-2 infection in participants with comorbidities associated with increased risk of progression to severe COVID-19, as compared to placebo | First occurrence of SARS-COV-2 infection (serologically and/or molecularly confirmed <sup>a</sup> ) in participants with comorbidities associated with increased risk of progression to severe COVID-19 with onset at least 28 days after double-blind vaccination (Day 29) |
| To explore the effect of Ad26.COV2.S on other potential complications of COVID-19 (linked to any respiratory disease and linked to any molecularly confirmed COVID-19) not previously described, as compared to placebo | • First occurrence of potential complications of COVID-19 linked to any respiratory disease and linked to any molecularly confirmed COVID-19, with onset at least 14 days after double-blind vaccination (Day 15) |
| | • First occurrence of potential complications of COVID-19 linked to any respiratory disease and linked to any molecularly confirmed COVID-19, with onset at least 28 days after double-blind vaccination (Day 29) |
| To explore the effect of Ad26.COV2.S on all-cause mortality, as compared to placebo | Deaths occurring at least 14 days after double-<br>blind vaccination (Day 15) |
| | • Deaths occurring at least 28 days after double-blind vaccination (Day 29) |
| To evaluate the immune response in participants with COVID-19 in relation to risk of development of COVID-19, protection induced by Ad26.COV2.S, and risk of accelerated disease | Assessment of the correlation of humoral immune responses with emphasis on neutralizing, binding and functional antibodies, as well as gene transcript profiling (RNA sequencing), with the risk of COVID-19 and protection induced by the study vaccine |
| In a subset of participants to further assess the humoral immune response to Ad26.COV2.S, as compared to placebo | Humoral immunogenicity endpoints: Functional and molecular antibody characterization including, but not limited to avidity, Fc-mediated viral clearance, Fc characteristics, Ig subclass, IgG isotype, antibody glycosylation, and assessment of antibody repertoire |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

84

| Objectives | Endpoints |
|---|---|
| | Adenovirus neutralization as measured by VNA |
| | Analysis of antibodies to S and the receptor-<br>binding domain (RBD) of the SARS-CoV-2 S<br>protein |
| | Original and/or emerging SARS-CoV-2 virus lineage neutralization as measured by virus neutralization assay (VNA; wild-type virus and/or pseudovirion expressing SARS-CoV-2 S protein) |
| | Passive transfer: analysis of immune mediators correlating with protection against experimental SARS-CoV-2 challenge in a suitable animal model. |
| To explore changes in the SARS-CoV-2 genome | Development of SARS-CoV-2 variants |
| To examine efficacy for moderate/severe and severe disease as well as medical utilization or death in the vaccine and placebo groups for variant strains that have been identified | Occurrence of moderate/severe or severe COVID-19, medical utilization, or death for each of the circulating viral variants, identified by S-gene sequencing |
| To evaluate patient-reported outcomes (PROs) in relation to the presence of SARS-CoV-2 infection and the presence, severity and duration of COVID-19 signs and symptoms in participants who received Ad26.COV2.S, as compared to placebo | Presence, severity and duration of COVID-19 signs and Symptoms; Confirmation of SARS-CoV-2 infection by molecular testing |
| To assess the difference in severity of cases in participants who received Ad26.COV2.S as compared to placebo | Reduction in severity of COVID-19 signs and Symptoms |
| To assess the impact of pre-existing humoral immunity against coronaviruses other than SARS-CoV-2 at baseline on Ad26.COV2.S vaccine immunogenicity | Analysis of antibodies binding to coronaviruses other than SARS-CoV-2 by ELISA |
| To assess the incidence of co-infection of COVID-19 and other respiratory pathogens and to assess the effect of the vaccine during such co-infections as well as to estimate the incidence of other respiratory pathogens during the study period. | Analysis of broad respiratory pathogens panel in the nasal swabs collected during a confirmed COVID-19 episode and in a subset of nasal swab samples from participants with a symptomatic infection. |
| To examine the degree of frailty in terms of balance in participants receiving Ad26.COV2.S vs placebo, the effect of degree of frailty on vaccine efficacy, and the degree of frailty in cases occurring in the Ad26.COV2.S vs placebo group. | Utilization of the frailty index as a measure of frailty prior to double-blind vaccination comparing the Ad26.COV2.S vs placebo group and as a measure to compare cases in the Ad26.COV2.S vaccine vs placebo group. |

| Endpoints |
|------------------------------------------------------|
| Utilization of tokenization and matching |
| procedures for exploratory analysis of participant's |
| medical data prior to, during, and following |
| participation in the study (real-world data). |
| Analysis will be performed to relate real-world |
| data to vaccine immune responses, efficacy and |
| duration of protection, and AEs (see Section 4.2 |
| and Section 8.8). |

<sup>&</sup>lt;sup>a</sup> Molecularly confirmed COVID-19 is defined as a positive SARS-CoV-2 viral RNA result by a central laboratory using a RT-PCR based or other molecular diagnostic test.

Refer to Section 8, Study Assessments and Procedures for evaluations related to endpoints.

#### **HYPOTHESES**

The study is designed to test the co-primary hypotheses of VE in the per-protocol (PP) population. For both co-primary endpoints the following hypothesis will be tested:

H0: VE  $\leq$ 30% versus H1: VE >30% and each hypothesis will be evaluated at a 2.5% one-sided significance level.

The co-primary endpoints will evaluate:

- the first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to the case definition (Section 8.1.3.1), with onset at least 14 days after double-blind vaccination with Ad26.COV2.S versus placebo, in the PP population, including all events from both age groups, with and without comorbidities.
- the first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to the case definition (Section 8.1.3.1), with onset at least 28 days after double-blind vaccination with Ad26.COV2.S versus placebo, in the PP population, including all events from both age groups, with and without comorbidities.

If testing for both primary endpoint hypotheses are successful, secondary objectives will be evaluated against a null hypothesis employing a lower limit VE>0%. The method to perform hypothesis testing of primary and secondary objectives preserving the FWER will be specified in the SAP. The FWER will be controlled at 2.5%.

Details are described in Section 9.

<sup>&</sup>lt;sup>b</sup> Per case definition for moderate to severe/ critical COVID-19 (see Section 8.1.3.1) as determined by the Clinical Severity Adjudication Committee (see Section 8.1.3.6).

<sup>&</sup>lt;sup>c</sup> Per case definition for mild COVID-19 (see Section 8.1.3.2) as determined by the Clinical Severity Adjudication Committee (see Section 8.1.3.6).

<sup>&</sup>lt;sup>d</sup> Per case definition for COVID-19 according to the US FDA harmonized case definition (see Section 8.1.3.3)

<sup>&</sup>lt;sup>e</sup> All secondary efficacy endpoint analyses will occur in the Per-Protocol (PP) analysis set, in seronegative participants unless otherwise indicated in the SAP.

## 3.2. Open-label Active Phase

# 3.2.1. Open-label Cross-over Phase

Participants will enter the open-label cross-over phase on the day that the participant received the cross-over vaccination or are unblinded until the day that the participant completed the booster visit. There are 2 main cohorts in the open label phase:

- Early vaccinated cohort: participants who were initially randomized to the Ad26.COV2.S group and received 1 dose of Ad26.COV2.S at day 1 in the trial
- Late vaccinated cohort: participants who were initially randomized to the placebo group and who received 1 dose of Ad26.COV2.S after unblinding

The main objective of the open-label phase of the study is to evaluate the COVID-19 outcomes after an early vaccination and after a late vaccination. Efficacy evaluations may be performed if feasible, ie, if pre-specified criteria are met, and will be specified in the SAP.

The exploratory objectives and endpoints for the open-label phase of the study are:

| Objectives | Endpoints |
|---|---|
| The secondary safety objective of the double-blind phase | See double-blind endpoint |
| To evaluate molecularly confirmed <sup>a</sup> , symptomatic COVID-19 <sup>b</sup> | Incidence of symptomatic COVID-19 cases starting at 28 days after last vaccination |
| To evaluate molecularly confirmed <sup>a</sup> , severe/critical COVID-19 <sup>b</sup> | Incidence of severe/critical COVID-19 cases starting at 28 days after last vaccination |
| To evaluate confirmed <sup>a</sup> COVID-19 <sup>b</sup> requiring medical intervention (based on objective criteria) | Incidence of COVID-19 cases requiring medical intervention, starting at 28 days after last vaccination |
| To evaluate COVID-19 related death | Incidence of COVID-19 related deaths starting at 28 days after last vaccination |
| To describe the severity of breakthrough infections | The severity of COVID-19 cases may be evaluated by the severity and number of symptoms (severity) of COVID-19 cases, ratio of severe/critical COVID-19 cases and ratio of long COVID-19 cases (duration of more than 28 days) |
| To estimate potential correlate of risk/efficacy in relation to the primary endpoint of the main study and serious disease, hospitalization, and death based on immune responses in breakthrough cases compared to non-infected participants. | Levels of immune responses (antibody titers) and RNA sequencing analysis as available for participants having COVID-19 compared to non-infected participants. |

<sup>&</sup>lt;sup>a</sup> Molecularly confirmed COVID-19 is defined as a positive SARS-CoV-2 viral RNA result by a central laboratory using a RT-PCR based or other molecular diagnostic test.

<sup>&</sup>lt;sup>b</sup> Per case definition for moderate to severe/critical COVID-19 as determined by the Clinical Severity Adjudication Committee (see below).

## 3.2.2. Open-label Booster Phase

Participants will enter the booster phase on the day that the participants completed the booster visit until consenting to Amendment 7 (or with the stop of the eCOA at each study site, which ever date comes first). There are 3 main cohorts based on vaccination schedules received in the booster phase:

- Homologous boost cohort consists of following 2 groups:
  - o participants who were initially randomized to the Ad26.COV2.S group and received 1 dose of Ad26.COV2.S at day 1 within the trial and a booster dose preferably within 6 to 12 months after the initial vaccination, with a minimum of 3 months after the initial vaccination with Ad26.COV2.S
  - o participants who were initially randomized to the placebo group and who received 1 dose of Ad26.COV2.S after unblinding and a booster dose preferably within 6 to 12 months after the initial vaccination, with a minimum of 3 months after the last vaccination with Ad26.COV.2.S
- Heterologous boost cohort: participants who were initially randomized to the placebo group and who received an mRNA vaccination outside of the trial and an Ad26.COV2 booster dose preferably within 6 to 12 months after the initial vaccination, with a minimum of 3 months after the last outside vaccination
- Non-boost cohort: participants who received 1 Ad26.COV2.S vaccination, either at Day 1 or as a cross-over vaccination. These participants remain in this cohort until they receive the booster vaccination. Participants who opt not to receive a booster dose will continue in this cohort.

Data from participants who received a different sequence of vaccinations (eg, Ad26.COV2 prime vaccination and an outside booster) will be presented separately.

The main objective of the booster phase of the study is to evaluate the COVID-19 outcomes, safety, and immunogenicity of the different schedules that were assessed: homologous Ad26.COV2 booster schedule, 1-dose schedule, heterologous booster schedule. All analyses are descriptive, efficacy evaluations may be done if feasible, ie, if pre-specified criteria are met, and will be described in the SAP.

The primary, secondary, and exploratory objectives and endpoints for the booster phase of the study are:

| Objectives | Endpoints |
|---|---|
| Primary (Booster Phase) | |
| To assess the safety and reactogenicity of Ad26.COV2.S at the 5×10 <sup>10</sup> vp dose level administered as homologous or heterologous booster vaccination in adults. | |
| | SAEs and AESIs from booster vaccination until end of the study. |

| Endpoints |
|---|
| • Incidence of primary endpoints utilized in the double-blind portion of the study, including moderate to severe/critical COVID-19 cases starting at 28 days by serostatus*, in the unblinded booster portion of the study (see definitions of terms in Section 10.1) during the times when they have and have not been boosted. |
| • Incidence of primary endpoints (Day 28 after vaccination) in the main study as applicable as described in the first objective but for variants of concern and the reference variants. |
| • Incidence of secondary endpoints (Day 28 after vaccination) from the double-blind portion of the study by serostatus* such as symptomatic severe/critical disease, hospitalization, and death. |
| Description of the primary and secondary endpoints (Day 28 after vaccination), such as symptomatic, severe/critical disease, hospitalization, and death, in the double-blind portion of the study as applicable as described in the first primary objective and first secondary objective including variants of concern and reference variants. |
| • Serological response to vaccination and antibody titers (VNA) against the original strain, 28 days after Ad26.COV2.S (5×10 <sup>10</sup> vp dose level) single-dose booster vaccination. |
| Levels of immune responses (antibody titers) and RNA sequencing analysis as available. |
| Qualitative comparison of responses in terms of binding, neutralizing antibody against Wuhan reference strain and variants of interest utilizing wtVNA and/or psVNA, depending on feasibility. |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Objectives | Endpoints |
|---|---|
| | Analysis of antibodies binding to the SARS-<br>CoV-2S protein by ELISA. |
| To evaluate SARS-CoV-2 infection (severe/critical, moderate to severe/critical, moderate, symptomatic, and asymptomatic infections, that are serologically and/or molecularly confirmed**) for the different cohorts | Incidence of SARS-CoV-2 infections (serologically and/or molecularly confirmed**). |
| To describe the severity of SARS.COV2.S infections | The severity of COVID-19 cases may be evaluated by the severity and number of symptoms (severity) of COVID-19 cases, ratio of severe/critical COVID-19 cases and ratio of long COVID-19 cases (duration of more than 28 days) |
| To obtain samples to evaluate potential thromboembolic events following booster immunization by obtaining platelet counts and sufficient extra sera for specialized studies at the day of booster immunization and 28 days later. | Platelet count on the day of booster vaccination and 28 days after booster vaccination. Additional analysis on kept sera samples in case of potential thromboembolic events. |
| Exploratory (Booster Phase) | |
| To measure the primary and secondary endpoints previously utilized in the double-blind portion of the study for all participants who have received any SARS-CoV-2 booster vaccine outside the study within the past month, are N-serology seronegative*, and remained in the unblinded booster portion of the study during the time when they have and have not been boosted. To utilize this data to explore estimates of efficacy comparing boosted to unboosted periods and by utilization of real-world data control groups constructed of vaccinees that are not boosted, if feasible. | Estimation of the primary and secondary endpoints in the main study, as applicable, and described above. |
| To measure moderate to severe/critical and severe/critical endpoints as defined for the double-blind portion of the study in participants who were N ELISA sero-negative and those who were N ELISA sero-positive at the time they received their booster. To utilize this data to compare rates of these endpoints in participants who are seropositive vs those that are seronegative* at the time they received their booster. | Describe rates of infection for moderate to severe/critical as defined and determined by the protocol in boosted participants who are N-serology seropositive versus those that are N-serology seronegative* at the time of booster vaccination. |
| An attempt to estimate the duration of protection following booster vaccination with Ad26.COV2.S for the primary and secondary endpoints will be made as outlined in the SAP. | Estimation of the primary and selected secondary endpoints in the main study as applicable. |

| Objectives | Endpoints |
|---|---|
| To estimate if there is a relationship between efficacy and the time period between priming COVID-19 vaccination regimen and Ad26.COV2.S booster vaccination. | • Estimation of the primary and selected secondary endpoints in the main study as applicable. |
| To compare the immune responses in the Heterologous and Homologous Booster Subsets compared to the immune responses observed in the VAC31518COV2008 boosting study and in this study after primary vaccination. | • Qualitative comparison of responses in terms of binding (S and/or RBD), neutralizing antibody against Wuhan reference and variants of interest utilizing wVNA and/or psVNA, depending on feasibility. |
| To analyze for signs of inflammation, coagulation pathway disorders, and markers of potential correlates of protection in a subset of participants from the Heterologous and Homologous Booster Subsets at baseline (prior to booster vaccination), 1 day, and 28 days after booster vaccination, depending on feasibility. | • mRNA sequencing immediately after immunization up to 28 days after vaccination analyzed in participants who received booster vaccination compared to responses after primary immunization following immunization of cross-over participants from the placebo group at unblinding in VAC31518COV3001 and VAC31518COV2008 for differences in gene expression. |
| | • Cytokine profiling: Analysis of cytokines, chemokines, and other proteins of the innate or adaptive immune response in the serum or plasma. |
| To further assess the humoral immune response to Ad26.COV2.S, in participants from the | Exploratory analyses may include, but are not limited to, the following assays: |
| Homologous and Heterologous Booster Subsets | • SARS-CoV-2 neutralization as assessed by alternative SARS-CoV-2 neutralization assays (VNA). |
| | Adenovirus neutralization. |
| | • Functional and molecular antibody characterization including Fc-mediated viral clearance, avidity, Fc characteristics, Ig subclass and IgG isotype. |
| | • Epitope-specificity characterization of antibodies. |
| | • Passive transfer: Analysis of immune mediators correlating with protection against experimental SARS-CoV-2 challenge in a suitable animal model. |

<sup>\*</sup> Seronegative is defined as N-serology seronegative at the time of boosting or at the Year 1 visit if not boosted

\*\* Molecularly confirmed COVID-19 is defined as a positive SARS-CoV-2 viral RNA result by a central laboratory
using a RT-PCR based or other molecular diagnostic test.

# 3.3. Open-label Passive Follow-up Phase

With Amendment 7, the active follow up of suspected COVID-19 episodes is replaced by a passive follow-up. Participants will enter this phase on the day of consenting to Amendment 7 (or with the stop of the eCOA at each study site, which ever comes first) until end of study.

In the passive follow-up phase, the same cohorts as from the booster phase are included, and all data will be descriptively presented by cohort depending on the vaccination schedule received during the follow-up phase. Since COVID-19 reporting changed from an active approach to a passive approach, the evaluations will be limited. Efficacy evaluations may be performed if feasible and will be described in the SAP as applicable.

The secondary and exploratory objectives and endpoints for the passive follow-up phase of the study are:

| Objectives | Endpoints |
|---|---|
| The secondary safety objective of the double-blind phase (see double-blind objectives). | The secondary safety endpoint of the double-<br>blind phase (see double-blind endpoints). |
| Exploratory | |
| To evaluate COVID-19 in terms of (S)AEs | SAEs and AEs linked to COVID-19 |
| MAAEs, hospitalizations and fatal AEs linked to COVID-19* | MAAEs linked to COVID-19 |
| | SAEs linked to COVID-19 that require hospitalization |
| | Fatal AEs linked to COVID-19 |
| In the immunogenicity subset of participants: to evaluate the immunogenicity of Ad26.COV2.S at available timepoints | Analysis of antibodies binding to the SARS-CoV-2 S protein by ELISA |
| In the Heterologous and Homologous Booster Subsets: to compare the immune responses 28 days | Analysis of antibodies binding to the SARS-<br>CoV-2 S protein by ELISA |
| following booster dose administration | <ul> <li>Qualitative comparison of responses in terms<br/>of binding, neutralizing antibody against<br/>Wuhan reference strain and variants of<br/>interest utilizing wtVNA and/or psVNA,<br/>depending on feasibility.</li> </ul> |
| In the Heterologous and Homologous Booster Subsets: to compare the immune responses compared to the immune responses observed in the VAC31518COV2008 boosting study and in this study after primary vaccination | Qualitative comparison of responses in terms of binding (S and/or RBD), neutralizing antibody against Wuhan reference and variants of interest utilizing wtVNA and/or psVNA, depending on feasibility. |
| In a subset of participants from the Heterologous and Homologous Booster Subsets: to analyze for signs of inflammation, coagulation pathway disorders, and markers of potential correlates of protection at baseline (prior to booster vaccination), 1 day, and 28 days after booster vaccination, depending on feasibility. | mRNA sequencing immediately after immunization up to 28 days after vaccination analyzed in participants who received booster vaccination compared to responses after primary immunization following immunization of cross-over participants from the placebo group at unblinding in VAC31518COV3001 |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Objectives | Endpoints |
|---|---|
| | VAC31518COV2008 for differences in gene expression. |
| | Cytokine profiling: Analysis of cytokines, chemokines, and other proteins of the innate or adaptive immune response in the serum or plasma. |
| In the Homologous and Heterologous Booster Subsets: to further assess the humoral immune | Exploratory analyses may include, but are not limited to, the following assays: |
| response to Ad26.COV2.S | • SARS-CoV-2 neutralization as assessed by alternative SARS-CoV-2 neutralization assays (VNA). |
| | Adenovirus neutralization. |
| | • Functional and molecular antibody characterization including Fc-mediated viral clearance, avidity, Fc characteristics, Ig subclass and IgG isotype. |
| | • Epitope-specificity characterization of antibodies. |
| | Passive transfer: Analysis of immune mediators correlating with protection against experimental SARS-CoV-2 challenge in a suitable animal model. |

<sup>\*</sup> Refer to Section 8.3 for the safety follow-up and COVID-19 reporting requirements as of Amendment 7.

#### 4. STUDY DESIGN

# 4.1. Overall Design

This is a multicenter, randomized, double-blind, placebo-controlled, Phase 3, pivotal efficacy and safety study in adults  $\ge$ 18 to <60 years of age and  $\ge$ 60 years of age. The efficacy, safety, and immunogenicity of Ad26.COV2.S will be evaluated in participants living in, or going to, locations with high risk for acquisition of SARS-CoV-2 infection after administration of study vaccine.

Following EUA, conditional licensure, or approval in any country for a single dose regimen, based on the VAC31518COV3001 study interim results, all participants from countries where protocol Amendment 4 is approved by the local Health Authority and IEC/IRB will be unblinded at the on-site Month 6/Unblinding Visit. The study will then be conducted in an open-label fashion. A final analysis of the double-blind phase will be performed, using the data collected prior to unblinding, when all participants have completed the Month 6/Unblinding Visit or discontinued earlier. Depending on the operational implementation of the Month 6/Unblinding Visit, as well as the stage of the pandemic, this analysis may be conducted when a minimum of 90% of the study population has been unblinded.

All participants will be invited for an on-site Month 6/Unblinding Visit and will undergo the procedures in the Schedule of Activities in Section 1.3. Participants who initially received placebo in the double-blind phase and consent will receive a single dose of Ad26.COV2.S vaccine under the conditions delineated in Section 6.4.

Initial immunogenicity and safety data (28 days post-Dose 1 data from Cohort 1a and available data from Cohort 3) from study VAC31518COV1001 have demonstrated that a single dose of Ad26.COV2.S at  $5\times10^{10}$  vp and  $1\times10^{11}$  vp induces an immune response that meets prespecified minimum criteria and had an acceptable safety profile. The sponsor has therefore decided to proceed with the single dose regimen at a  $5\times10^{10}$  vp dose level in this Phase 3 study.

With protocol Amendment 6, the open-label phase of the study is extended to include an open-label booster vaccination with a single dose of Ad26.COV2.S at the Year 1/Booster Visit (see also below). The combination of homologous or heterologous prime/boost vaccination will not be randomized, but depends on what participants received during the double-blind phase of the study as described in this protocol. The start date of the first cross-over unblinding visit (implemented with Amendment 4) and the date of first booster vaccine administration until 1-year follow-up of the last booster vaccination define the open-label booster vaccination phase of the study. This phase will be utilized to describe safety, immunogenicity, and efficacy during the time participants have and have not been boosted.

With Amendment 7, active follow-up of suspected COVID-19 episodes will be replaced by passive follow-up (ie, follow-up by the site at Month 18 and Month 24 to document new COVID-19 participant-reported events as safety endpoints [SAEs, AEs, MAAEs] and to record concomitant therapies associated with COVID-19).

The study will consist of a screening phase of up to 28 days, a 62-week study period (including the administration of 1 dose of study vaccine [on Day 1], after randomization, unblinding and, for consenting participants, cross-over vaccination at the Month 6/Unblinding Visit, and, for consenting participants, Ad26.COV2.S booster vaccination at the Year 1/Booster Visit), and a long-term follow-up period until the Year 2 Visit (52 weeks after the Year 1/Booster Visit). The duration of individual participation, including screening, will be approximately 2 years and 1 month. If a participant is unable to complete the study, but has not withdrawn consent, an early exit visit will be conducted. The end-of-study is considered as the completion of the last visit for the last participant in the study (see Section 4.4).

Participants will be randomized in parallel in a 1:1 ratio to receive Ad26.COV2.S or placebo intramuscularly (IM) as shown in Table 2. Ad26.COV2.S will be administered at a dose level of  $5\times10^{10}$  vp.

At the Month 6/Unblinding Visit, participants who initially received placebo and signed a new ICF will be offered a single dose of Ad26.COV2.S at a dose level of 5×10<sup>10</sup> vp.

As of implementation of protocol Amendment 6, all ongoing participants in the study who have previously received any COVID-19 vaccination(s) (as primary regimen or additional dose) with

the Ad26.COV2.S vaccine, and/or an mRNA vaccine or another COVID-19 vaccine authorized for primary vaccination including protein, inactivated, and adenovector-based vaccines will be offered a single booster dose of Ad26.COV2.S vaccine (5×10<sup>10</sup> vp) at the Year 1/Booster Visit under the conditions delineated in Section 6.5.

Table 2: Vaccination Schedule VAC31518COV3001

| Group | N | Day 1 | Month 6/Unblinding<br>Visit* | Year 1/Booster Visit |
|---|---|---|---|---|
| 1 | 20,000 | Ad26.COV2.S (5×10 <sup>10</sup> vp) | - | Ad26.COV2.S (5×10 <sup>10</sup> vp) |
| 2 | 20,000 | Placebo | Ad26.COV2.S $(5\times10^{10} \text{ vp})$ | Ad26.COV2.S $(5\times10^{10} \text{ vp})$ |

EUA Emergency Use Authorization; N number of participants; vp virus particles.

Note: It is intended that a minimum of approximately 30% of recruited participants will be  $\ge$ 60 years of age and approximately 20% of recruited participants will be  $\ge$ 18 to <40 years of age.

The following enrollment strategy will be used in the double-blind phase:

- Stage 1a: Initially, approximately 2,000 participants (≥18- to <60-year-old) without comorbidities that are associated with increased risk of progression to severe COVID-19 (including approximately 1,000 Ad26.COV2.S recipients and approximately 1,000 placebo recipients) will be enrolled based on acceptable Day 29 safety and acceptable immunogenicity data, including Th1/Th2, from the corresponding age group (Cohort 1a) of the FIH study VAC31518COV1001 (see Section 2.2 for more details).
- Stage 1b: After a vaccination pause (in the age group ≥18 to <60 years of age), to allow the DSMB (also known as an independent data monitoring committee [IDMC]) to examine Day 3 safety data (ie, from Day 1 to Day 3; including safety data from the ongoing clinical studies) from Stage 1a, if no safety concerns are identified enrollment will proceed, expanding enrollment to include ≥18- to <60-year-old participants with and without comorbidities that are associated with increased risk of progression to severe COVID-19 (see Section 1.2 [Figure 1] for a schematic overview of the study and Section 5.2 for the list of relevant comorbidities).

In Stage 1, the enrollment of participants aged  $\geq$ 18 to <40 years will be limited to approximately 20% of the total study population.

• Stage 2a: Initially, approximately 2,000 participants ≥60 years of age without comorbidities that are associated with increased risk of progression to severe COVID-19 will be enrolled (including approximately 1,000 Ad26.COV2.S recipients and approximately 1,000 placebo recipients). Considering the data from study VAC31518COV1001 (including data on elderly), Stage 2a will be enrolled in parallel with Stage 1a, unless this is not allowed per local Health Authority guidance.

<sup>\*</sup> All participants will be unblinded (informed whether they received placebo or Ad26.COV2.S) at the on site Month 6/
Unblinding Visit following EUA, conditional licensure, or approval in any country and approval of protocol Amendment 4
by the local Health Authority and IEC/IRB the study will continue as an open label study. Participants who received placebo
on Day 1 will be offered to receive a single dose of Ad26.COV2.S 5×10<sup>10</sup> vp under conditions delineated in Section 6.4.
Investigators are encouraged to consider current local public health guidance for determining the scheduling priority of
participants when feasible, eg, participants with co morbidities and/or of specific age groups can be scheduled prior to
participants without co morbidities if this is in line with local guidance. This should be done in a blinded way, ensuring that
participants who were not previously unblinded for other reasons are not unblinded until the Month 6/Unblinding Visit.

• Stage 2b: After a vaccination pause (in the age group ≥60 years of age) to allow the DSMB to examine Day 3 safety data (ie, from Day 1 to Day 3; including safety data from Stage 1 and the ongoing clinical studies) from Stage 2a, if no safety concerns are identified in this population, enrollment will proceed, expanding enrollment to include ≥60 year-old participants with and without comorbidities that are associated with increased risk of progression to severe COVID-19 (see Section 1.2 [Figure 1] for a schematic overview of the study and Section 5.2 for the list of relevant comorbidities).

Stage 2 will enroll a minimum of approximately 30% of the total study population.

Overall, a target of approximately 40,000 adult participants ( $\geq$ 18- to <60-year-old and  $\geq$ 60-year-old, with and without relevant comorbidities) will be randomly assigned in this study. Efforts will be made to ensure good representation in terms of race, ethnicity, and gender.

All participants will be actively and passively followed for acute molecularly confirmed, symptomatic COVID-19, regardless of severity. Molecularly confirmed COVID-19 is defined as a positive SARS-CoV-2 viral RNA result by a central laboratory using a RT-PCR based or other molecular diagnostic test. With Amendment 7, new COVID-19 episodes will be monitored through passive follow-up.

The primary objective will be evaluated in real-time manner through sequential testing of accumulating primary endpoints through the SSG and DSMB. Only if both co-primary endpoints have crossed the sequential boundary, the DSMB will discuss the signal with the Oversight Group. As soon as a decision is reached, the sponsor representative on the Oversight Group will initiate internal decision procedures to trigger health authority interactions based on the outcome of the study. Sponsor personnel will be unblinded at the time of the primary analysis. If an efficacy signal is triggered before the required 8-week follow-up after double-blind vaccination for 50% of participants is reached, selected sponsor personnel will be unblinded at the time of the snapshot analysis. Further details are described in Section 9.5.1.

In the open-label phase, participants who initially received placebo and consent will receive a single dose of Ad26.COV2.S. No additional participants will be recruited for the open-label phase. With Amendment 6, the open-label phase of the study was extended to include an open-label booster vaccination with a single dose of Ad26.COV2.S. As of Amendment 7, no further booster vaccinations will be provided with the following exceptions: 1) participants who could not receive a booster vaccination prior to implementation of Amendment 7 due to medical reasons or 2) participants who cannot receive a booster vaccination outside of this study may still receive a booster vaccination up to the expiry date of the vaccine. These participants will be followed for less than 1 year after booster vaccination but for a minimum of 6 months.

Key efficacy assessments include the surveillance for COVID-19-like signs and symptoms, recording of COVID-19-related hospitalizations and complications, and the laboratory confirmation of SARS-CoV-2 infection by a molecular assay (based on RT-PCR) and by anti-SARS-CoV-2 serology (see Section 8.1.2). Immunogenicity assessments, and especially assessments of the humoral immune responses with emphasis on neutralizing and binding antibodies will also be performed (see Section 8.1.4). Key safety assessments during the double-

blind phase will include the monitoring of solicited and unsolicited AEs in the Safety Subset only. Up to Amendment 7, all participants who received booster vaccination at the Year 1/Booster Visit will record solicited signs and symptoms, collected through an e-Diary. As of protocol Amendment 7, the collection of solicited AEs will stop. Up to Amendment 7, for a subset of participants, the e-Diary will be reviewed by the investigator at the next visit, if feasible. Unsolicited AEs will be recorded for all participants who received booster vaccination at the Year 1/Booster Visit. As of protocol Amendment 7, the collection of unsolicited AEs will stop.

In addition, key safety assessments throughout the study include the collection of SAEs and MAAEs in all participants (see Section 8.3).

Up to Amendment 7, the viral load of SARS-CoV-2 will be assessed in confirmed COVID-19 cases (see Section 8.4). Biomarkers correlating with SARS-CoV-2 infection and COVID-19 severity will also be studied (see Section 8.5). Medical resource utilization (MRU) following vaccination will be recorded for all participants with molecularly confirmed, symptomatic COVID-19 (see Section 8.6).

Additional characteristics related to current work situation, living situation, and community interactions, from participants who consent to this, will be collected for risk factor analysis, if allowed per local regulations. Participants who consent to this will be interviewed on these aspects prior to vaccination on Day 1 and, at other timepoints, on changes compared to Day 1 (See Appendix 12). For consenting participants in the US, medical data (electronic health records, claims, laboratory data from other settings) from 5 years prior to study enrollment until 5 years after study completion may be accessed utilizing tokenization and matching procedures (See Section 4.2 and Section 8.8). These data together with prior medical history data collected at study entry may be used for exploratory analyses to enhance our understanding of the potential impact of prior medical history on the response to immunization and the impact of immunization on efficacy and duration of efficacy as well as adverse events that may occur during and after completion of the study.

The first 2,000 participants in each of the 2 age groups will be closely observed at the study site for at least 30 minutes post-vaccination to monitor for the development of acute reactions. If at the time of the Day 3 safety review of the initial 2,000 participants no acute reactions have been observed in the age groups, the observation period at the study site may be reduced to at least 15 minutes post-vaccination for the remaining participants in the study. For participants in the Safety Subset, solicited local (at injection site) and systemic AEs, unsolicited AEs, SAEs, and concomitant therapies will be documented by study-site personnel following this observation period. Participants in the Safety Subset (double-blind phase) will also record solicited signs and symptoms in an e-Diary for 7 days post-vaccination. The reporting periods of unsolicited AEs, MAAEs, SAEs, and special reporting situations are detailed in Section 8.3. Reporting periods for concomitant therapy are outlined in Section 6.10. Concomitant therapies associated with COVID-19 are also to be reported as of Amendment 7. The statistical analyses will be described in detail in a Statistical Analysis Plan.

Under protocol amendment 7, the protocol described safety follow-up will continue for all participants (eg SAEs, MAAEs, AESIs - please refer to Section 8.3.1). As mentioned above, participants who received booster vaccination will stop the reporting of solicited or unsolicited AEs as of Amendment 7. Finally, the management of suspected COVID-19 episodes has been changed from active to passive follow-up, defined as follow-up by the site at Month 18 and Month 24 to document new COVID-19 participant-reported events as SAEs, AEs, or MAAEs (see Section 8.3.3).

All participants will be followed-up until implementation of protocol amendment 7 to monitor for signs and symptoms of COVID-19 (to determine duration of protection) and to monitor for safety (including enhanced disease). As of protocol amendment 7, COVID-19 events will be followed through a passive follow-up and sites are instructed to report these events as (S)AE or MAAEs. The approach for the analysis of this long-term follow-up cohort for safety and VE will be provided in detail in the analytic plan. Participants in the Immunogenicity Subset will additionally be followed-up for long-term immunogenicity. Up to amendment 7, participants will also be monitored for complications potentially associated with COVID-19 (such as but not limited to hyperinflammatory syndrome, pneumonia, neurological or vascular complications, severe pneumonia, severe neurological or vascular events, acute respiratory distress syndrome, renal complications, sepsis, septic shock, death)<sup>71</sup>, and for MRU (such as rates of ICU admission, ventilator use).

Until 1 year after the Month 6/Unblinding Visit, each participant will be asked at least twice a week, through the electronic clinical outcome assessment (eCOA), if they have experienced any new symptoms or health concerns that could be related to infection with SARS-CoV-2. As of 1-year after the Month 6/Unblinding Visit, until the end of the 2-year follow-up period, the frequency of this surveillance question through the eCOA may decrease to once every 2 weeks depending on epidemiology. All participants will be monitored for safety (including enhanced disease) for approximately 1 year after the Year 1/Booster Visit, ie, until the last study visit. Every effort will be made to document the status of all participants that are lost to follow-up due to not completing the eCOA and for whom hospitalization has not been recorded. As from Amendment 7, the eCOA will be decommissioned (passive follow-up approach). The eCOA will be stopped based on approval of protocol Amendment 7 at each study site.

Enrolled participanICFts will be counselled on SARS-COV-2 infection prevention each time that they have a contact with site staff, in line with local guidelines. At the time of study entry, each participant will need to indicate to the study site, in case they would get infected with SARS-CoV-2, the identity and location of their routine medical care physician and/or facility and the identity and location of where they would obtain emergency care and hospitalization if necessary. If this information is not available, a plan for where such care could be obtained should be developed. If a participant should have COVID-19 and their symptoms deteriorate, they will be instructed to go to the HCP or hospital that has been identified in advance.

Up to Amendment 7, any positive RT-PCR test regardless if it is obtained outside the study or at a study visit will be considered a trigger to start COVID-19 procedures. All participants with COVID-19-like signs or symptoms meeting the prespecified criteria for new suspected

 $CONFIDENTIAL-FOIA\ Exemptions\ Apply\ in\ U.S.$ 

COVID-19<sup>a</sup> (see Section 8.1.1) and all participants with at least one positive RT-PCR test for SARS-CoV-2 on COVID-19 Day 1-2 or Day 3-5 visits, should undertake the COVID-19 procedures (see Section 8.1.2 and Section 1.3) until 14 days after symptom onset (COVID-19 Day 15) or until resolution of the COVID-19 episode, whichever comes last. However, participants with COVID-19-like signs or symptoms meeting the prespecified criteria for suspected COVID-19<sup>a</sup> should stop the COVID-19 procedures as soon as it is confirmed that both nasal swabs collected on COVID-19 Day 1-2 and Day 3-5 are negative for SARS-CoV-2. Resolution of the COVID-19 episode is defined as having 2 consecutive SARS-CoV-2 negative nasal swabs and 2 consecutive days with no COVID-19-related signs or symptoms. At the time of resolution of the COVID-19 episode, the collected information will be applied against the clinical case definition (Sections 8.1.3.1, 8.1.3.2, and 8.1.3.3).

As of Amendment 7, active follow-up of suspected COVID-19 episodes will be replaced by passive follow-up.

Site staff and participants will not be blinded as to the outcome of the molecular test results from the local (hospital) laboratory and the baseline molecular test results from the central laboratory. Their routine HCP can obtain external diagnostics, including RT-PCR or other molecularly confirmed viral tests, as medically needed.

The occurrence of molecularly confirmed COVID-19, all complications associated with COVID-19, and concomitant therapies associated with COVID-19 will be captured in the electronic case report form (eCRF) for the duration of the study. Up to Amendment 7, every effort will be made to capture medical information from any medical visits (eg, visits to the primary care providers, emergency department/urgent care clinic visits, etc.) related to COVID-19 or its complications via the medically-attended COVID-19 form (MA-COV form) (see Appendix 8). As of Amendment 7, the MA-COV and the MRU forms are no longer to be completed.

All necessary precautions (as per local regulation) should be taken to protect medical staff and other contacts of participants who are suspected to have COVID-19 until proven negative by molecular techniques or who are positive until they are no longer positive. In the event of a confirmed SARS-CoV-2 infection, the participant and participant's medical care provider will be notified, and the participant will be asked to adhere to the appropriate measures and restrictions as defined by local regulations.

Additional study procedures and assessments for immunogenicity and safety (reactogenicity and unsolicited AE) will be performed in subsets of participants (see Section 8.1.4 and Section 8.3).

A DSMB will be commissioned for this study. Refer to Section 9.8 and Appendix 3 for more details.

A diagram of the study design is provided in Section 1.2.

\_

<sup>&</sup>lt;sup>a</sup> As several of the prespecified criteria for suspected COVID-19 overlap with vaccine-related reactogenicity, investigators' clinical judgement is required to exclude vaccine-related events when assessing suspected COVID-19.

# 4.2. Scientific Rationale for Study Design

#### **Vector Selection**

The rationale behind the selection of the Ad26 vector is described in Section 2.

#### **Dose Selection**

The rationale behind the selection of the dose is described in Section 4.3.

### Blinding, Control, Study Phase/Periods, Vaccine Groups

A placebo control will be used to establish the frequency and magnitude of changes in clinical and immunological endpoints that may occur in the absence of active vaccine. Randomization will be used to minimize bias in the assignment of participants to vaccine groups, to increase the likelihood that known and unknown participant attributes (eg, demographic and baseline characteristics) are evenly balanced across vaccine groups, and to enhance the validity of statistical comparisons across vaccine groups. Blinded study vaccine will be used to reduce potential bias during data collection and evaluation of study endpoints.

Blinding will be guaranteed by the preparation of the study vaccine by an unblinded pharmacist or other qualified study-site personnel with primary responsibility for study vaccine preparation and dispensing, and by the administration of vaccine in a masked syringe by a blinded study vaccine administrator. Participants will be randomly assigned to 1 of the groups based on a computer-generated randomization schedule prepared before the study by or under the supervision of the sponsor and using the interactive web response system (IWRS) (see also Section 6.3).

When EUA, conditional licensure, or approval is granted in any country and upon implementation of protocol Amendment 4, all participants will be invited for an on-site Month 6/Unblinding Visit and will be unblinded at that visit. Participants who initially received placebo, will be offered to receive a single dose of Ad26.COV.2 vaccine. All participants will be requested to provide a blood sample and nasal swab, which will require a new informed consent.

#### **Biomarker Collection (Up to Amendment 7)**

For participants with a positive test result for SARS-CoV-2 infection, biomarker analysis (PAXgene, RNAseq) may be performed to explore potentially informative biomarkers, eg, those associated with severe COVID-19.

#### Medical Resource Utilization Data Collection (Up to Amendment 7)

Prophylaxis of COVID-19 with Ad26.COV2.S may reduce the need for and duration of supportive care (eg, hospitalization, oxygen supplementation). The study will evaluate the impact of Ad26.COV2.S versus placebo on the development and clinical course of COVID-19.

## Participant Medical Information Prior to, During and After the Study (Real-world Data)

Real-world data plays a critical role in improving understanding of factors that may influence response to immunization and the effectiveness and safety of a vaccine product during and after completion of the study. This may be important to gain insight into duration of efficacy and

incidence of adverse events after study completion. This may be especially important in the event that efficacy of Ad26.COV2.S or another vaccine is shown and follow-up in a randomized manner is compromised.

To allow the linking of participant records from different sources, ie, data collected as part of the study as specified in the Schedules of Activities and longitudinal real-world data (from 5 years prior to enrollment in the study until 5 years after study completion) such as electronic health records, claims, and laboratory data from other care settings, without compromising the participant's confidentiality, tokenization and matching procedures will be utilized **for US participants only**. The tokenization process starts with each data provider generating a token behind the firewall via a proprietary software. Personal information such as names and dates of birth from study participants are removed from real-world data sources and replaced with encrypted, one-way, hashed identifiers then further encrypted using asymmetric keys in compliance with Health Insurance Portability and Accountability Act (HIPAA). This encrypted anonymized information is sent for matching to the anonymized participant master index. While it is not possible to reverse the hash, source-specific tokens can be decrypted and re-encrypted so that records can be linked across sources. The result of the process is a unique anonymized identifier for each participant, which can be used to link participant records across sources (real world data and study data).

## 4.2.1. Study-Specific Ethical Design Considerations

Potential participants will be fully informed of the risks and requirements of the study and, during the study, participants will be given any new information that may affect their decision to continue participation. They will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only participants who are fully able to understand the risks, benefits, and potential AEs of the study, and provide their consent voluntarily will be enrolled.

The primary ethical concern is that this study will be performed in adult participants who will receive no direct benefit from participation in the study, except for participant reimbursement for the time and inconveniences that may arise from participation in the study. See Section 2.3 for details on potential and known benefits and risks, and for the safety measures taken to minimize risk to participants.

Another ethical concern is the use of placebo vaccine and maintaining the study blind during the double-blind phase of the study while the active study vaccine may prevent a serious disease. The study design, with continuous evaluation of efficacy, addresses that concern as much as possible. The sponsor will offer the active study vaccine to placebo recipients, with the implementation of Amendment 4. See Section 6.8 for details. In addition, the sponsor will offer a single booster dose of Ad26.COV2.S vaccine (5×10<sup>10</sup> vp) at the Year 1/Booster Visit booster to all ongoing participants who have previously received any COVID-19 vaccination(s) (as primary regimen or additional dose) with the Ad26.COV2.S vaccine and/or an mRNA vaccine or another for primary vaccination authorized COVID-19 vaccine including protein, inactivated, and adenovector based vaccines with the implementation of Amendment 6.

The total blood volume to be collected is considered to be an acceptable amount of blood to be collected over this time period from the population in this study based upon the US Department of Health and Human Services Office for Human Research Protections, and US Food and Drug Administration (FDA) guidelines of 550 mL in any 8-week period.<sup>64</sup>

For participants in the US who consent to the optional collection of real-world medical data, the sponsor is committed to protect their data and privacy. Tokenization and matching procedures will be utilized to allow for those participant's medical data to be obtained without violation of participant confidentiality (See Section 4.2). Participants will be informed that consent to this part of the study is completely optional and that they can withdraw their consent at any given time. In case of withdrawal of consent, the sponsor will remove the token generated and any associated linked real-world data. Participation in or withdrawal from this optional part of the study will not affect the participation in the main study.

# 4.3. Justification for Dose

The dose level of Ad26.COV2.S to be assessed in the present study  $(5\times10^{10} \text{ vp})$  is based on experience with other Ad26-vectored vaccines administered to adults in clinical studies including Ad26.ZEBOV (Ebola virus program); Ad26.ENVA.01, Ad26.Mos.HIV, and Ad26.Mos4.HIV (HIV program); Ad26.CS.01 (malaria program); Ad26.RSV.FA2 and Ad26.RSV.preF (RSV program); and Ad26.ZIKV.001 (Zika virus program). Studies with Ad26.RSV.preF also included participants aged  $\geq$ 60 years. The dose level of  $5\times10^{10}$  vp is the most extensively tested dose to date and has shown to be well tolerated and immunogenic in these vaccine programs. Safety data from studies with other Ad26-based vaccines are summarized in Section 2.3.1.

The same dose level is also being assessed in study VAC31518COV1001, where initial immunogenicity and safety data (28 days post-Dose 1 data from Cohort 1a and available data from Cohort 3) have demonstrated that a single dose of Ad26.COV2.S at  $5\times10^{10}$  vp and  $1\times10^{11}$  vp induces an immune response that meets prespecified minimum criteria and had an acceptable safety profile. The sponsor has therefore decided to proceed with the single dose regimen at a  $5\times10^{10}$  vp dose level in this Phase 3 study.

Non-human primates immunized with a single-dose of Ad26.COV2.S (Study 20-14, dose level titration study) showed robust protection after intranasal and intratracheal challenge with SARS-CoV-2. Ad26.COV2.S at 5×10<sup>10</sup> vp provided complete protection in the lung in 5 of 5 animals, and in 5 of 6 animals in the upper respiratory tract. All control animals showed substantial viral load in both the lower and upper respiratory tract.

# 4.4. End-of-study Definition

#### **End-of-study Definition**

The end-of-study is considered as the completion of the last visit for the last participant in the study. The final data from each participating study site will be sent to the sponsor (or designee) after completion of the final participant visit at that study site, in the time frame specified in the Clinical Trial Agreement.

All participants should have their last study contact visit completed by 31 March 2023. The investigator (like for any lost to follow-up) should make three attempts to reach the participant for the last call, whereafter the participant is considered to have finished participation in the study. At that time point, 90% of the participants who receive a booster vaccination will have been monitored for safety for 1 year post the booster vaccination. The remaining 10% of the participants will have been monitored for safety at least for 6 months.

## **Study Completion Definition**

A participant will be considered to have completed the study if he or she has completed the assessments at the visit approximately 104 weeks after double-blind vaccination. Participants who prematurely discontinue study participation for any reason before completion of these assessments will not be considered to have completed the study.

#### 5. STUDY POPULATION

Screening for eligible participants will be performed within  $\leq$ 28 days before randomization and administration of the study vaccine, or on the day of the vaccination. Refer to Section 5.4 for conditions under which the repeat of any screening procedures are allowed.

The inclusion and exclusion criteria for enrolling participants in this study are described below. Some inclusion and exclusion criteria only apply to a particular stage (1a, 1b, 2a, and/or 2b), as indicated below. See Section 4.1 for more details about enrollment in the different stages. If there is a question about these criteria, the investigator must consult with the appropriate sponsor representative and resolve any issues before enrolling a participant in the study. Waivers are not allowed.

Once enrolled, all participants who received placebo during the double-blind phase will be eligible to receive vaccination with Ad26.COV2.S at the Month 6/Unblinding Visit if they agree and consent to receive the active vaccine and meet the criteria described in Section 6.4.

As of Amendment 6, all ongoing participants who have previously received any COVID-19 vaccination(s) (as primary regimen or additional dose) with the Ad26.COV2.S vaccine, and/or an mRNA vaccine or another COVID-19 vaccine authorized for primary vaccination including protein, inactivated, and adenovector based vaccines will be eligible to receive a 1-dose booster vaccination with Ad26.COV2.S at the  $5 \times 10^{10}$  vp dose level at the Year 1/Booster Visit if they agree and consent to receive the active vaccine and meet the criteria described in Section 6.5.

For a discussion of the statistical considerations of participant selection, refer to Section 9.2.

#### 5.1. Inclusion Criteria

Each potential participant must satisfy all of the following criteria to be enrolled in the study:

1. Criterion modified per Amendment 1:

- 1.1 Participants must provide consent indicating that he or she understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study.
- 2. Participant is willing and able to adhere to the prohibitions and restrictions specified in this protocol.
- 3. Stages 1a and 1b: Participant is  $\ge 18$  to < 60 years of age on the day of signing the ICF.

<u>Stages 2a and 2b:</u> Participant is  $\geq$ 60 years of age on the day of signing the ICF.

- 4. Criterion modified per Amendment 1:
  - 4.1. Criterion modified per Amendment 2:
  - 4.2 Criterion modified per Amendment 3:
  - 4.3 <u>Stages 1a and 2a:</u> In the investigator's clinical judgement, participant must be either in good or stable health, including a BMI <30 kg/m<sup>2</sup>.

Participants may have underlying illnesses (not associated with increased risk of progression to severe COVID-19<sup>a,17</sup> as specified in Exclusion Criterion 15), as long as their symptoms and signs are stable and well-controlled. If participants are on medication for a condition not part of the comorbidities listed in Exclusion Criterion 15, the medication dose cannot have been increased within 12 weeks preceding vaccination and expected to remain stable for the duration of the study. Participants will be included on the basis of relevant medical history and BMI measurement at screening.

Stages 1b and 2b: In the investigator's clinical judgement, participant may have a stable and well-controlled medical condition including comorbidities associated with an increased risk of progression to severe COVID-19 as specified in Exclusion Criterion 15 (eg, stable/well controlled -HIV infection)\*. If participants are on medication for a medical condition (including comorbidities associated with an increased risk of progression to severe COVID-19), the medication dose cannot have been increased within 12 weeks preceding vaccination and must be expected to remain stable for the duration of the study<sup>b</sup>. Participants will be included on the basis of relevant medical history and BMI measurement at screening.

- \* Stable/well-controlled HIV infection includes:
  - a. Documented CD4 cell count  $\geq$ 300 cells/ $\mu$ L within 6 months prior to screening.
  - b. Documented HIV viral load <50 copies/mL within 6 months prior to screening.
  - c. Participant must be on a stable anti-retroviral treatment (ART) for 6 months (unless the change is due to tolerability, in which case the regimen can be for only

\_

<sup>&</sup>lt;sup>a</sup>Per US CDC (Appendix 11). In this study, former or current smoking/vaping and mild hypertension (according to the Toxicity Grading Scale in Section 10.9) will not be considered as a comorbidity. In addition, for this study gestational diabetes was deleted from the list since it is not applicable as pregnant women were not allowed to enroll in the study.

<sup>&</sup>lt;sup>b</sup> No longer applicable as of Protocol Amendment 7.

the previous 3 months; changes in formulation are allowed; nationwide guidelines that require transition from one ART regimen to another are allowed) and the participant must be willing to continue his/her ART throughout the study as directed by his/her local physician.

Note: Participants with ongoing and progressive comorbidities associated with HIV infection will be excluded but comorbidities associated with HIV infection that have been clinically stable for the past 6 months are not an exclusion criterion.

Laboratory methods for confirming a diagnosis of HIV infection are: Any evidence (historic or current) from medical records, such as ELISA with confirmation with Western Blot or RT-PCR, or of a detectable viral load (country-specific regulatory approved tests). A laboratory result within 6 months of screening does not need to be repeated.

If a potential participant does not have HIV viral load and CD4 cell count data in his/her medical records from the last 6 months, they will be instructed to go to their local health care provider and obtain the necessary data for potential entry into the trial.

- 5. Criterion modified per Amendment 1:
  - 5.1 Contraceptive (birth control) use should be consistent with local regulations regarding the acceptable methods of contraception<sup>a</sup> for those participating in clinical studies.

Before randomization, participants must be either (as defined in Appendix 5):

- a. Not of childbearing potential
- b. Of childbearing potential and practicing an acceptable effective method of contraception and agrees to remain on such a method of contraception from providing consent until 3 months after administration of study vaccine. Use of hormonal contraception should start at least 28 days before the administration of study vaccine. The investigator should evaluate the potential for contraceptive method failure (eg, noncompliance, recently initiated) in relationship to the vaccination. Acceptable effective methods for this study include:
  - 1. hormonal contraception:
    - i. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
    - ii. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable)
  - 2. intrauterine device:
  - 3. intrauterine hormone-releasing system;

<sup>&</sup>lt;sup>a</sup> Use of condoms is not considered as an acceptable contraceptive barrier method due to the failure rate of female and male condoms. <sup>19</sup>

- 4. bilateral tubal occlusion/ligation procedure;
- 5. vasectomized partner (the vasectomized partner should be the sole partner for that participant);
- 6. sexual abstinence\*.

\*Sexual abstinence is considered an effective method **only** if defined as refraining from heterosexual intercourse from providing consent until 3 months after receiving study vaccine. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

- 6. All participants of childbearing potential must:
  - a. Have a negative highly sensitive urine pregnancy test at screening
  - b. Have a negative highly sensitive urine pregnancy test on the day of and prior to study vaccine administration.
- 7. Participant agrees to not donate bone marrow, blood, and blood products from the study vaccine administration until 3 months after receiving the study vaccine.
- 8. Must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study.
- 9. Must be able to read, understand, and complete questionnaires in the eCOA (ie, the COVID-19 signs and symptoms surveillance question, the e-Diary, and the electronic patient-reported outcomes (ePROs) [see Appendix 1 for definition of terms])<sup>a</sup>.

#### 5.2. Exclusion Criteria

Any potential participant who meets any of the following criteria will be excluded from participating in the study:

- 1. Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature ≥38.0°C (100.4°F) within 24 hours prior to the planned study vaccination; randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor.
- 2. Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine; refer to the IB).
- 3. Criterion modified per Amendment 1:
  - 3.1 Criterion modified per Amendment 2:
  - 3.2 Criterion modified per Amendment 3:
  - 3.3 Participant has abnormal function of the immune system resulting from:

<sup>&</sup>lt;sup>a</sup> Participants with visual impairment are eligible for study participation and may have caregiver assistance in completing the eCOA questionnaires.

- a. Clinical conditions (eg, autoimmune disease or potential immune mediated disease or known or suspected immunodeficiency, or participant on hemodialysis) expected to have an impact on the immune response of the study vaccine. Participants with clinical conditions stable under non-immunomodulator treatment (eg, autoimmune thyroiditis, autoimmune inflammatory rheumatic disease such as rheumatoid arthritis) may be enrolled at the discretion of the investigator. Non-immunomodulator treatment is allowed as well as steroids at a non-immunosuppressive dose or route of administration.
- b. Chronic or recurrent use of systemic corticosteroids within 6 months before administration of study vaccine and during the study. A substantially immunosuppressive steroid dose is considered to be ≥2 weeks of daily receipt of 20 mg of prednisone or equivalent.
  - Note: Ocular, topical or inhaled steroids are allowed.
- c. Administration of antineoplastic and immunomodulating agents or radiotherapy within 6 months before administration of study vaccine and during the study.
- 4. Criterion modified per Amendment 3:
  - 4.1 Participant received treatment with Ig in the 3 months or exogenous blood products (autologous blood transfusions are not exclusionary) in the 4 months before the planned administration of the study vaccine or has any plans to receive such treatment during the study.
- 5. Participant received or plans to receive:
  - a. Licensed live attenuated vaccines within 28 days before or after planned administration of study vaccine.
  - b. Other licensed (not live) vaccines within 14 days before or after planned administration of study vaccine.
- 6. Participant previously received a coronavirus vaccine.
- 7. Criterion modified per Amendment 1:
  - 7.1 Criterion modified per Amendment 2:
  - 7.2 Criterion modified per Amendment 3:
  - 7.3 Participant received an investigational drug (including investigational drugs for prophylaxis of COVID-19) within 30 days or used an invasive investigational medical device within 30 days or received investigational immunoglobulin (Ig) or monoclonal antibodies within 3 months, or received convalescent serum for COVID-19 treatment within 4 months or received an investigational vaccine (including investigational Adenoviral-vectored vaccines) within 6 months before the planned administration of the study vaccine or is currently enrolled or plans to participate in another investigational study during the course of this study. See also Section 6.10.

Note: Participation in an observational clinical study is allowed at the investigator's discretion; please notify the sponsor (or medical monitor) of this decision.

Efforts will be made to ensure inclusion of participants who have not been previously enrolled in coronavirus studies and to prevent participants from subsequently enrolling in other coronavirus studies during their participation in this study.

The use of any coronavirus vaccine (licensed or investigational) other than Ad26.COV2.S is disallowed at any time prior to vaccination (see also Exclusion Criterion 6) and during the study, except under the conditions described in Section 6.8.

- 8. Criterion modified per Amendment 1:
  - 8.1 Participant is pregnant or planning to become pregnant within 3 months after study vaccine administration.
- 9. Participant has a history of an underlying clinically significant acute or chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the wellbeing) or that could prevent, limit, or confound the protocol-specified assessments.
- 10. Participant has a contraindication to IM injections and blood draws, eg, bleeding disorders.
- 11. Criterion deleted per Amendment 1:
- 12. Criterion modified per Amendment 1:
  - 12.1 Participant has had major psychiatric illness which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures.
- 13. Participant cannot communicate reliably with the investigator.
- 14. Participant who, in the opinion of the investigator, is unlikely to adhere to the requirements of the study, or is unlikely to complete the full course of vaccination and observation.
- 15. Criterion modified per Amendment 1:
  - 15.1 Criterion modified per Amendment 2:

#### 15.2 **Stages 1a and 2a:**

• Participants with comorbidities that are or might be associated with an increased risk of progression to severe COVID-19<sup>a,17</sup>, ie, participants with moderate to severe asthma; chronic lung diseases such as chronic obstructive pulmonary disease (COPD) (including emphysema and chronic bronchitis), idiopathic pulmonary fibrosis and cystic fibrosis; diabetes (including type 1 or type 2); serious heart conditions, including heart failure, coronary artery disease, congenital heart disease, cardiomyopathies, and pulmonary hypertension; moderate to severe high blood pressure; obesity (body mass index [BMI] ≥30 kg/m²); chronic liver disease, including cirrhosis; sickle cell disease;

\_

<sup>&</sup>lt;sup>a</sup> Per US CDC (Appendix 11). In this study, former or current smoking/vaping and mild hypertension (according to the Toxicity Grading Scale in Section 10.9) will not be considered as a comorbidity. Gestational diabetes was deleted from the list since it is not applicable as pregnant women were not allowed to enroll in the study.
- thalassemia; cerebrovascular disease; neurologic conditions (dementia); end stage renal disease; organ transplantation; cancer; HIV infection and other immunodeficiencies; hepatitis B infection; and sleep apnea.
- Participants with a history of or current Parkinson's disease; seizures; ischemic strokes; intracranial hemorrhage; encephalopathy and meningoencephalitis.
- 16. <u>Stages 1a and 2a:</u> Participant has a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or other malignancies with minimal risk of recurrence).
- 17. Criterion Modified per Amendment 2:
  - 17.1 Participant has a history of acute polyneuropathy (eg, Guillain-Barré syndrome).
- 18. <u>Stages 1a and 2a:</u> Participant had surgery requiring hospitalization (defined as inpatient stay for longer than 24 hours or overnight stay), within 12 weeks before vaccination, or will not have fully recovered from surgery requiring hospitalization, or has surgery requiring hospitalization planned during the time the participant is expected to participate in the study or within 6 months after study vaccine administration.
- 19. <u>Stages 1a and 2a:</u> Participant has chronic active hepatitis B or hepatitis C infection per medical history.

*Note*: Investigators should ensure that all study enrollment criteria have been met prior to the study vaccination. If a participant's clinical status changes (including any available laboratory results or receipt of additional medical records) after screening but before the study vaccination is given such that he or she no longer meets all eligibility criteria, then the participant should be excluded from participation in the study. Section 5.4 describes options for retesting. The required documentation to support meeting the enrollment criteria is described under Source Documents in Appendix 3.

# 5.3. Lifestyle Considerations

Potential participants must be willing and able to adhere to the following lifestyle considerations during the course of the study to be eligible for participation:

- 1. Refer to Section 6.10 for details regarding prohibited and restricted therapy during the study.
- 2. Agree to follow all requirements that must be met during the study as noted in the inclusion and exclusion criteria (eg, contraceptive requirements).
- 3. Agree to follow requirements for the electronic completion of the COVID-19 signs and symptoms surveillance question in the eCOA.

### 5.4. Screen Failures

## Participant Identification, Enrollment, and Screening Logs

The investigator agrees to complete a participant identification and enrollment log to permit easy identification of each participant during and after the study, however, without referring to direct communication with participants. This document will be reviewed by the sponsor study-site contact for completeness.

The participant identification and enrollment log will be treated as confidential and will be filed by the investigator in the study file. To ensure participant confidentiality, no copy will be made. All reports and communications relating to the study will identify participants by participant identification and age at initial informed consent. In cases where the participant is not randomized into the study, the date seen and age at initial informed consent will be used.

In cases where a participant does not meet the criteria for participation in this study (screen failure), the main reason for non-eligibility is to be documented in the eCRF.

An individual who does not meet the criteria for participation in Stages 1a or 2a, but does meet the criteria for participation in Stages 1b or 2b, will not be considered a screening failure and can be enrolled in the appropriate stage, if enrollment occurs within the 28-day Screening window.

An individual who does not meet the criteria for participation in this study (screen failure) or individuals for whom the 28-day screening window is exceeded may be rescreened on 1 occasion only.

All participants who are rescreened will be assigned a new participant number, undergo the informed consent process, and then re-start a new screening phase.

# 5.5. Criteria for Temporarily Delaying Administration of Study Vaccination

The following events constitute a temporary contraindication to study vaccination:

- Clinically significant acute illness at the time of vaccination. This does not include minor illnesses, such as diarrhea or mild upper respiratory tract infection.
- Fever (body temperature ≥38.0°C/100.4°F) within 24 hours prior to the planned time of vaccination.
- An illness which in the judgement of the investigator may interfere with reactogenicity/Day 0-7 safety assessments.

If, at the start of the double-blind phase, any of these events occur at the scheduled time for the vaccination, randomization at a later date within the screening window is permitted at the discretion of the investigator and after consultation with the sponsor. If randomization cannot occur within the screening window, rescreening is required.

If, at the start of the open-label phase, any of the above listed events occur at the scheduled time for the vaccination, the Month 6/Unblinding Visit with active vaccine can be delayed up to 28 days

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

following unblinding. In addition, a urine pregnancy test (for participants of childbearing potential, according to the local guidelines) will be required for the Month 6/Unblinding Visit for participants who will be vaccinated at this visit. Participants who are pregnant at the Month 6/Unblinding Visit and received placebo during the double-blind phase may be vaccinated with Ad26.COV2.S, if allowed by local regulations, and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (See Section 6.4).

If any of the above listed events occur at the scheduled time for the booster vaccination, the Year 1/Booster Visit with active vaccine can be delayed within the preferred visit window, but not occur later than May 15, 2022. In addition, a urine pregnancy test (for participants of childbearing potential, according to the local guidelines) will be required for the Year 1/Booster Visit for participants who will be vaccinated at this visit. Participants who are pregnant at the Year 1/Booster Visit may receive booster vaccination with Ad26.COV2.S, if allowed by local regulations, and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (see Section 6.5).

As of Protocol Amendment 7, no further booster doses will be administered, except if there was a medical reason that prevented a participant to receive the Ad26COV2.S vaccine prior to acceptance of amendment 7 or if there is a non-availability of other vaccines to the participant. The investigator should inform participants on the availability of other COVID-19 vaccines.

### 6. STUDY VACCINATION AND CONCOMITANT THERAPY

# 6.1. Study Vaccines Administered

Ad26.COV2.S will be supplied at a concentration of  $1\times10^{11}$  vp/mL in single-use vials, with an extractable volume of 0.5 mL, and dosed at  $5\times10^{10}$  vp. Placebo is 0.9% NaCl.

For blinding purposes, all participants will receive Ad26.COV2.S or placebo at Day 1 of the double-blind phase (see Schedules of Activities), using the same volume (ie, 0.5 mL). At the Month 6/Unblinding Visit, all placebo participants who have signed a new ICF will receive a single dose of Ad26.COV2.S (Schedules of Activities, Section 1.3), using the same dose level and the same volume (ie,  $5 \times 10^{10}$  vp per 0.5 mL). At the Year 1/Booster Visit, all participants who are eligible for booster vaccination (see Section 6.5), desire to receive a booster vaccination, and have signed a new ICF will receive a single dose of Ad26.COV2.S (Schedules of Activities, Section 1.3), using the same dose level and the same volume (ie,  $5 \times 10^{10}$  vp per 0.5 mL) as used for the primary regimen.

Study vaccine will be administered by IM injection into the deltoid muscle, preferably of the non-dominant arm. If an injection cannot be given in the deltoids due to a medical or other contraindication (for example, tattooed upper arms rendering it difficult to assess site reactogenicity), use alternative locations such as the hip, thigh or buttocks (to be avoided in overweight participants). In all circumstances, IM injections in other locations than the upper arm are not considered protocol deviations.

Study vaccine administration must be captured in the source documents and the eCRF.

Ad26.COV2.S will be manufactured and provided under the responsibility of the sponsor. Refer to the IB for a list of excipients.<sup>42</sup>

Refer to the study site investigational product and procedures manual (SIPPM) and the Investigational Product Preparation Instructions (IPPI) for additional guidance on study vaccine administration.

# **Description of Interventions**

| Group Name | Group 1, Group 2 cross-over* participants, Booster Group 2 | |
|---|---|---|
| | Vaccination | |
| Intervention Name | Ad26.COV2.S (1×10 <sup>11</sup> vp/mL) | Placebo 0.9% Sodium Chloride |
| Type | Biologic/vaccine (1 dose) | Placebo (1 dose) |
| Dose Formulation | Single-use vials, with an extractable volume of 0.5 mL | Single-use vials, with an extractable volume of 0.5 mL |
| Unit Dose Strength(s) | Ad26.COV2.S at a concentration of 1×10 <sup>11</sup> vp/mL | 0.9% NaCl |
| Dosage Level(s) | <b>Day 1</b> : Ad26.COV2.S (5×10 <sup>10</sup> vp), Month 6/Unblinding | Day 1: Placebo |
| | Visit, Year 1/Booster Visit | |
| Route of Administration | IM injection | IM injection |
| Use | Experimental | Placebo-comparator |
| Investigational Medicinal Product (IMP) | Yes | Yes |
| Non-Investigational Medicinal | No | No |
| Product/Auxiliary Medicinal Product | | |
| (NIMP/AxMP) | | |
| Sourcing | Provided centrally by the sponsor | Provided centrally by the sponsor |
| Packaging and Labeling | The study vaccines will be packaged and labeled according to good manufacturing practices and local regulations. The | |
| | study vaccines will not be packed in individual participant kits, 1 kit will be used by multiple participants. Each kit | |
| | will contain single-use vials. | |
| | Not in child resistant packaging | |

IM = intramuscular; vp = virus particles

<sup>\*</sup>Cross-over refers to participants who initially received placebo and were administered a single dose of Ad26.COV2.S vaccine at the Month 6/Unblinding Visit.

# 6.2. Preparation/Handling/Storage/Accountability

## Preparation/Handling/Storage

All study vaccine must be stored in a secured location with no access for unauthorized personnel and at controlled temperatures as indicated on the clinical labels. If study vaccine is exposed to temperatures outside the specified temperature range, all relevant data will be sent to the sponsor to determine if the affected supplies can be used or will be replaced. The affected study vaccine must be quarantined and not used until further instruction from the sponsor is received.

Refer to the study SIPPM and the IPPI for additional guidance on study vaccine preparation, handling, and storage.

In the double-blind phase, an unblinded study-site pharmacist, or other qualified individual, who will have no other study function following vaccination, will prepare the appropriate vials and syringes, labeled with the participant's identification number, and provide the syringes for the study vaccine in a blinded manner to the blinded vaccine administrator (a trained and qualified study nurse, medical doctor, or otherwise qualified HCP) who will perform the injection.

At the Month 6/Unblinding Visit, all participants will be unblinded to their study vaccine allocation. Participants, who initially received placebo, will be offered to receive a single dose of Ad26.COV2.S vaccine. Vaccination at the Month 6/Unblinding Visit will be performed by a trained and qualified study nurse, medical doctor, or otherwise qualified HCP.

Within the window of the Year 1/Booster Visit, eligible participants can choose to receive a single booster dose of Ad26.COV2.S vaccine. Vaccination at the Year 1/Booster Visit will be performed by a trained and qualified study nurse, medical doctor, or otherwise qualified HCP.

### **Accountability**

The investigator is responsible for ensuring that all study vaccine received at the site is inventoried and accounted for throughout the study. The study vaccine administered to the participant must be documented on the vaccine accountability form. All study vaccine will be stored and disposed of according to the sponsor's instructions. Study-site personnel must not combine contents of the study vaccine containers.

Study vaccine must be handled in strict accordance with the protocol and the container label and must be stored at the study site in a limited-access area or in a locked cabinet under appropriate environmental conditions. Unused study vaccine must be available for verification by the sponsor's unblinded site monitor during on-site monitoring visits. The return to the sponsor of unused study vaccine will be documented on the vaccine accountability form. When the study site is an authorized destruction unit and study vaccine supplies are destroyed on-site, this must also be documented on the vaccine accountability form.

Potentially hazardous materials containing hazardous liquids, such as needles and syringes should be disposed of immediately in a safe manner and therefore will not be retained for vaccine accountability purposes.

Study vaccine should be dispensed under the supervision of the investigator or a qualified member of the study-site personnel, or by a hospital/clinic pharmacist. Study vaccine will be administered only to participants participating in the study. Returned study vaccine must not be dispensed again, even to the same participant. Study vaccine may not be relabeled or reassigned for use by other participants. The investigator agrees neither to dispense the study vaccine from, nor store it at, any site other than the study sites agreed upon with the sponsor. Further guidance and information for the final disposition of unused study vaccine are provided in the SIPPM.

# 6.3. Measures to Minimize Bias: Randomization and Blinding

#### **Intervention Allocation**

### Procedures for Randomization and Stratification

Central randomization will be implemented in this study in the double-blind phase. Participants will be randomly assigned to 1 of 2 vaccination groups (active vaccine [Group 1] versus placebo [Group 2]). This will be based on a computer-generated randomization schedule prepared before the study by or under the supervision of the sponsor. The randomization will be balanced by using randomly permuted blocks and will be stratified by vaccination unit (eg, site, mobile unit), age group ( $\geq$ 18 to <60 years of age versus  $\geq$ 60 years of age), and absence/presence of comorbidities that are or might be associated with an increased risk of progression to severe COVID-19 as described in Exclusion Criterion 15.

The IWRS will assign a unique intervention code, which will dictate the intervention assignment for the participant. The requestor must use his or her own user identification and personal identification number when contacting the IWRS and will then give the relevant participant details to uniquely identify the participant.

### **Blinding: Double-blind Phase**

Blinding will be guaranteed by the preparation of the study vaccine by an unblinded pharmacist or other qualified study-site personnel with primary responsibility for study vaccine preparation and dispensing, and by the administration of vaccine in a masked syringe by a blinded study vaccine administrator. Participants will be randomly assigned to 1 of the groups based on a computer-generated randomization schedule prepared before the study by or under the supervision of the sponsor and using the IWRS.

The investigator will not be provided with randomization codes. The codes will be maintained within the IWRS, which has the functionality to allow the investigator to break the blind for an individual participant.

Data that may potentially unblind the study vaccine assignment (ie, immunogenicity data, study vaccine accountability data, study vaccine allocation, biomarker, or other specific laboratory data) will be handled with special care to ensure that the integrity of the blind is maintained and the potential for bias is minimized. This can include making special provisions, such as segregating the data in question from view by the investigators, clinical team, or others as appropriate until the time of database lock and unblinding.

Under normal circumstances, the blind should not be broken until all participants have attended the Month 6/Unblinding Visit. Note that sponsor personnel will be unblinded at the time of primary analysis. Sites and participants will remain blinded until the Month 6/Unblinding Visit. Details will be provided in the DSMB Charter. The investigator may in an emergency determine the identity of the intervention by contacting the IWRS. While the responsibility to break the intervention code in emergency situations resides solely with the investigator, it is recommended that the investigator contact the sponsor or its designee if possible, to discuss the particular situation, before breaking the blind. Telephone contact with the sponsor or its designee will be available 24 hours per day, 7 days per week.

In the event the blind is broken, the sponsor must be informed as soon as possible. The date, time, and reason for the unblinding must be documented in the IWRS and in the source document. The documentation received from the IWRS indicating the code break must be retained with the participant's source documents in a secure manner.

Participants who have had their intervention assignment unblinded should continue to return for scheduled safety evaluations.

In general, randomization codes will be disclosed fully only at the Month 6/Unblinding Visit.

In the double-blind phase of the study, investigators may receive requests to unblind study participants who become eligible to receive an authorized/licensed COVID-19 vaccine if/when these become available. In these cases, the investigator will discuss with the participant available options and ramifications. If the participant is eligible for an authorized/licensed vaccine according to local immunization guidelines or recommendation and if the participant wishes to proceed with the unblinding, the investigator will follow the unblinding procedures described above. The reason for the unblinding request should be documented. The name and date(s) of administration of the other COVID-19 vaccine should be recorded (see Section 6.10).

When unblinding, if it is determined that the participant received the Ad26.COV2.S vaccine (and not placebo), the participant will be informed that there are no data on the safety of receiving two different COVID-19 vaccines. Unblinded participants, both in the double-blind and open-label phase will be asked to continue to be followed in this study in line with the Schedule of Activities to the extent that they permit. Safety, efficacy, and immunogenicity evaluations will be identical for all participants, including participants that are unblinded to obtain an authorized/licensed COVID-19 vaccine and who remain in the study, including participants in the Safety Subset, if applicable and feasible. All data will be analyzed separately from the point of unblinding for safety, efficacy, and immunogenicity, as described in the Statistical Analysis Plan.

Prior to EUA, conditional licensure, or approval in any country, participants who opt for enrollment in an Expanded Access Program or a Phase 3b study (eg, Sisonke/TOGETHER in South Africa) may be unblinded upon their request and will be encouraged to continue in study VAC31518COV3001. Study investigators should query participants to elicit and document such participation in other studies in the VAC31518COV3001 study record.

Once protocol Amendment 4 is approved, participants who were previously unblinded because they were offered another approved/licensed vaccine will follow the procedures detailed in Section 6.4.

# 6.4. Unblinding and Open-label Phase

Following Ad26.COV2.S EUA, conditional licensure, or approval in any country for a single dose regimen based on the VAC31518COV3001 interim results, all participants from countries where Amendment 4 is approved by the local Health Authority and IEC/IRB will be unblinded on-site at the Month 6/Unblinding Visit.

Participants who received placebo at the start of the double-blind phase will be offered a single dose of Ad26.COV2.S vaccine, under the following conditions:

- Participants, who were already unblinded for any reason, might receive a single dose of Ad26.COV2.S vaccine at the investigator's discretion, provided they did not receive another licensed/authorized COVID-19 vaccine.
- Participants, who had met study discontinuation criteria under previous amendments, will be
  offered a single dose of Ad26.COV2.S vaccine at the discretion of the investigator, except the
  following participants (who are not eligible to receive the Ad26.COV2.S vaccine);

received another licensed/authorized COVID-19 vaccine or,

withdrew consent from the study or,

received any COVID-19-related experimental medication (including experimental vaccines other than the study vaccine) or,

previously experienced TTS or heparin-induced thrombocytopenia (HIT) or,

previously experienced capillary leak syndrome

- Participants who are pregnant and received placebo during the double-blind phase may be vaccinated with Ad26.COV2.S, if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus.
- Participants who use systemic corticosteroids (chronic or recurrent use) or received antineoplastic and immunomodulating agents or radiotherapy may receive a single dose of Ad26.COV2.S if allowed by local regulations and after being made aware that the safety and efficacy data in patients using/receiving these medications/treatments is limited.
- Participants who have become infected with SARS-CoV-2 during the double-blind phase of
  the study may receive a single dose of Ad26.COV2.S vaccine, even if they received steroid
  treatment, convalescent plasma, or monoclonal antibody treatment, after they have recovered
  from the acute illness and at least 1 month has passed. Such participants should be made aware
  that the safety and efficacy data on vaccinating a previously infected individual is limited.
- Vaccination should be deferred in case of any other illness, until the person has recovered from the acute illness (see Section 5.5).

Participants who may have missed visits after vaccination on Day 1 and subsequently request
the active vaccine may be offered single dose of the Ad26.COV2.S vaccine at the discretion
of the investigator.

Investigators will be encouraged to follow health authority guidelines on prioritization of immunization when feasible. Investigators are encouraged to consider current local public health guidance for determining the scheduling priority of participants when feasible, eg, participants with comorbidities and/or of specific age groups can be scheduled prior to participants without comorbidities if this is in line with local guidance. This should be done in a blinded way, ensuring that participants who were not previously unblinded for other reasons are not unblinded until the Month 6/Unblinding Visit. All participants will be counselled to continue practicing other public health/preventative measures that were introduced at the start of this pandemic (eg, social distancing, face masks, frequent hand washing), in compliance with local and national guidelines. Participants who receive a single dose of Ad26.COV2.S will continue to follow the Schedule of Activities in Section 1.3.

### 6.5. Booster Vaccination

All ongoing participants in the study who have received primary vaccination with the Ad26.COV2.S vaccine, or an mRNA vaccine or another authorized COVID-19 vaccine including protein, inactivated, and adenovector based vaccines and who have subsequently remained in the study will be offered to receive a 1-dose booster vaccination with Ad26.COV2.S at the 5x10<sup>10</sup> vp dose level. Participants who have only received one dose of a two dose primary immunization regimen are also eligible to receive the booster vaccination with Ad26.COV2.S in this study. Participants in the study who have already received an additional COVID-19 vaccination after the primary regimen outside the study with any vaccine as described above will also be eligible for the Ad26.COV2.S booster in this study. Booster vaccination should occur preferably 6 months but at least 3 months after the last COVID-19 vaccination, but no later than the expiry date of the Ad26.COV2.S vials available at your site. Participants are free to choose when to receive the booster vaccination within the window of the booster vaccination visit, to receive booster vaccination outside the study, or not to receive booster vaccination. Participants who choose to receive a booster vaccination with the Ad26.COV2.S vaccine (if recommended and available) or another authorized COVID-19 vaccine outside the study or choose not to receive a booster vaccination will not be withdrawn from the study and will be encouraged to remain in the study.

Participants may be offered the single booster dose of Ad26.COV2.S vaccine under the following special conditions:

Participants, who had met study discontinuation criteria under previous amendments, will be
offered a single booster dose of Ad26.COV2.S vaccine at the discretion of the investigator,
except the following participants (who are not eligible to receive the Ad26.COV2.S vaccine);

withdrew consent from the study or,

received any COVID-19-related experimental medication (including any experimental vaccines other than the study vaccine) or,

previously experienced TTS or heparin-induced thrombocytopenia (HIT) or,

previously experienced capillary leak syndrome or,

are planning to receive another COVID-19 vaccine within the 3 months after the booster vaccination.

- Participants who are pregnant may receive booster vaccination with Ad26.COV2.S, if allowed
  by local regulations and if the investigator considers that the potential benefits outweigh the
  potential risks to the mother and fetus.
- Participants who use systemic corticosteroids (chronic or recurrent use) or received antineoplastic and immunomodulating agents or radiotherapy may receive booster vaccination with Ad26.COV2.S if allowed by local regulations and after being made aware that the safety and efficacy data in patients using/receiving these medications/treatments is limited.
- Participants who have become infected with SARS-CoV-2 during the study may receive
  booster vaccination with Ad26.COV2.S vaccine, even if they received steroid treatment,
  convalescent plasma, or monoclonal antibody treatment, after they have recovered from the
  acute illness and at least 1 month has passed. Such participants should be made aware that the
  safety and efficacy data on vaccinating a previously infected individual is limited.
- Vaccination should be deferred in case of any other illness, until the person has recovered from the acute illness (see Section 5.5).

Investigators will be encouraged to follow health authority guidelines on prioritization of immunization when feasible. Investigators are encouraged to consider current local public health guidance for determining the scheduling priority of participants when feasible, eg, participants with comorbidities and/or of specific age groups can be scheduled prior to participants without comorbidities if this is in line with local guidance. Based on operational considerations, the investigators at their discretion may prioritize those participants who had their priming regimen at a more distant time prior to the booster vaccination.

All participants will be counselled to continue practicing other public health/preventative measures that were introduced at the start of this pandemic (eg, social distancing, face masks, frequent hand washing), in compliance with local and national guidelines. Participants who receive booster vaccination with Ad26.COV2.S will continue to follow the Schedule of Activities in Section 1.3.

As of Protocol Amendment 7, no further booster doses will be administered, except if there was a medical reason that prevented a participant to receive the Ad26COV2.S vaccine prior to acceptance of amendment 7 or if there is a non-availability of other vaccines to the participant. The investigator should inform participants on the availability of other COVID-19 vaccines.

## 6.6. Study Vaccine Compliance

Study vaccines will be administered intramuscularly by a study vaccine administrator a trained and qualified study nurse, medical doctor, or otherwise qualified HCP. The date and time of study vaccine administration and the location used will be recorded in the eCRF.

#### 6.7. Dose Modification

Dose modification is not applicable in this study.

# 6.8. Continued Access to Study Vaccine After the End of the Study

Prior to EUA, conditional licensure, or approval in any country, participants who opt for enrollment in an Expanded Access Program or a Phase 3b study (eg, Sisonke/TOGETHER in South Africa) may be unblinded upon their request and will be encouraged to continue in study VAC31518COV3001. Study investigators should query participants to elicit and document such participation in other studies in the VAC31518COV3001 study record.

Following EUA, conditional licensure, or approval in any country and approval of protocol Amendment 4 by the local Health Authority and IEC/IRB, participants who initially received placebo will be offered a single dose of Ad26.COV2.S study vaccine at no cost, as described in Section 6.4.

With approval of Amendment 6 by the local Health Authority and IEC/IRB, ongoing participants who have previously received any COVID-19 vaccination(s) (as primary regimen or additional dose) with the Ad26.COV2.S vaccine, and/or an mRNA vaccine or another COVID-19 vaccine authorized for primary vaccination including protein, inactivated, and adenovector based vaccines will be offered a single booster dose of Ad26.COV2.S study vaccine at no cost, as described in Section 6.5.

At the time when another COVID-19 vaccine is determined to be efficacious and authorized/licensed for use, some participants may become eligible to receive such vaccine, country-specific registration depending conditions (eg local on status. recommendations/regulations, vaccine availability or the specific target group for vaccination). The investigator will discuss with the participants the available information and options to allow the participant to make an informed choice as to whether they qualify to receive the authorized/licensed vaccine and whether they should request individual unblinding to take up the offer of an authorized/licensed COVID-19 vaccine. Safety evaluations will be identical for all participants, including participants that are unblinded to obtain an authorized/licensed COVID-19 vaccine and who remain in the study. Access to Ad26.COV2.S vaccine for participants already unblinded will be under the conditions delineated in Section 6.4. All data will be analyzed from the point of unblinding for safety, efficacy, and immunogenicity, as described in the SAP.

### 6.9. Treatment of Overdose

For this study, any dose of Ad26.COV2.S greater than the assigned dose will be considered an overdose. The sponsor does not recommend specific treatment for an overdose.

In the event of a known overdose, the investigator should:

• Contact the medical monitor immediately.

- Closely monitor the participant for AE/SAE/MAAE (ie, the participant will remain at the study site for at least 1 hour and will be closely monitored for allergic or other reactions by study staff. Follow-up telephone calls 12 hours and 24 hours post-dose will be made).
- Document the quantity of the excess dose in the source document.
- Report as a special reporting situation.

# 6.10. Prestudy and Concomitant Therapy

Prestudy therapies are only to be recorded for participants with relevant comorbidities and participants aged ≥60 years. For these participants, all prestudy therapies (excluding vitamins, herbal supplements; non-pharmacologic therapies such as electrical stimulation, acupuncture, special diets, and exercise regimens) administered up to 30 days before the vaccination must be recorded at screening.

For all participants, concomitant therapies associated with an SAE or suspected AESI meeting the criteria outlined in Section 10.4.1 and Section 8.3.7, respectively, will be collected and recorded in the eCRF from the moment of vaccination (or from the time of local approval of protocol Amendment 5 for suspected AESIs) through the end of the study. Concomitant therapies associated with MAAEs will be collected and recorded in the eCRF from the moment of vaccination until 6 months after (double-blind or open-label) Ad26.COV2.S. Concomitant therapies associated with MAAEs leading to study discontinuation will be recorded in the eCRF during the entire study.

For all participants, concomitant therapies associated with COVID-19 will be captured in the electronic eCRF for the duration of the study. This will still be applicable after implementation of Protocol Amendment 7. Hence, under protocol amendment 7, concomitant medication in case of COVID-19 (S)AEs and COVID-19 MAAEs need to be recorded, as well any confirmatory laboratory result, if available (eg positive COVID-19 PCR results, positive nasal swab). The assay methodology should be mentioned.

For participants in the Safety Subset, concomitant therapies associated with unsolicited AEs will be collected and recorded in the eCRF from the time of vaccination through 28 days after double-blind vaccination. Concomitant therapies associated with solicited AEs will be collected by the participants and recorded in the eCRF from the time of vaccination through 7 days after double-blind vaccination.

Antipyretics are recommended post-vaccination for symptom relief as needed. Prophylactic antipyretic use is not encouraged; however, in some instances, it could be considered for participants with special circumstances and/or comorbidities.

Participants may not have received an investigational drug (including investigational drugs for prophylaxis of COVID-19) within 30 days or used an invasive investigational medical device within 30 days or received investigational Ig or monoclonal antibodies within 3 months, or received convalescent serum for COVID-19 treatment within 4 months or received an investigational vaccine (including investigational Adenoviral-vectored vaccines) within 6 months

before the planned administration of the study vaccine. During the study, the use of investigational vaccines other than the study vaccine is not allowed, and the use of investigational drugs is only allowed if medically indicated. Treatment with investigational COVID-19 drugs after diagnosis of a COVID-19 case is allowed during the follow-up period and needs to be recorded in the COVID-19 episode description.

Licensed live attenuated vaccines should be given at least 28 days before or at least 28 days after a study vaccination. Other licensed (not live) vaccines (eg, influenza, tetanus, hepatitis A, hepatitis B, rabies) should be given more than 14 days before (or more than 14 days after, as per exclusion criterion 6) administration of study vaccine in order to avoid potential confusion of adverse reactions and potential immune interference. The use of any coronavirus vaccine (licensed or investigational) other than Ad26.COV2.S is disallowed at any time prior to vaccination and during the study except under the conditions described in Sections 6.3 and 6.8. If a vaccine is indicated in a post-exposure setting (eg, rabies or tetanus), it must take priority over the study vaccine. Receipt of another licensed/authorized COVID-19 vaccine by a study participant at any timepoint during the study must be recorded. The name and date(s) of administration of the COVID-19 vaccine should be recorded in the eCRF.

Chronic or recurrent use of systemic corticosteroids<sup>a</sup> at immunosuppressive dose and administration of antineoplastic and immunomodulating agents or radiotherapy are prohibited during the study and within 6 months before the planned administration of the study vaccine. If any of these agents are indicated in a disease setting, these must take priority over the study vaccine.

Refer to Section 5.2 for further details of prohibited therapy.

The sponsor must be notified in advance (or as soon as possible thereafter) of any instances in which prohibited therapies are administered. The participant should remain in the study. Depending on the time of the occurrence, any participant who receives a prohibited concomitant therapy will not be included in the immunogenicity analyses.

# 6.11. Study Vaccination Pausing Rules for Stages 1a and 2a

A committee consisting of the representatives of the sponsor and collaboration partners, along with the principal investigator (the protocol safety review team [PSRT]) and the Janssen Medical Safety Council will monitor safety in a blinded manner, including the study vaccination pausing rules (applicable to Stages 1a and 2a only). Adverse events that may lead to the study vaccination pausing rules (applicable to Stages 1a and 2a only) are described below and will be assessed by the Janssen Medical Safety Council to confirm that the study pause is warranted.

The occurrence of any of the following events in Stages 1a and 2a will lead to a pause in further study vaccination:

<sup>&</sup>lt;sup>a</sup> Note: Ocular, topical or inhaled steroids are allowed.

- 1. Death of a participant, considered related to study vaccine or if the causal relationship to the study vaccine cannot be excluded; OR
- 2. One or more participants experience an SAE (solicited or unsolicited) that is determined to be related to study vaccine; OR
- 3. One or more participants experience anaphylaxis or generalized urticaria, clearly not attributable to other causes than vaccination with study vaccine.

To enable prompt response to a situation that could trigger pausing rules, the investigator should notify the sponsor's medical monitor or designee (AND fax or email the SAE form to Global Medical Safety Operations, if applicable), immediately and no later than 24 hours after becoming aware of any related SAE AND update the eCRF with relevant information on the same day the SAE information is collected (see also Section 8.3.1). Based on the pausing criteria, the sponsor's medical monitor or designee, in consultation with the Janssen Medical Safety Council, then decides whether a study pause is warranted and informs the DSMB of the decision. All sites will be notified immediately in the event of a study pause. The sponsor's medical monitor or designee is responsible for the immediate notification of DSMB members and coordination of a DSMB meeting in the event of a study pause.

The DSMB will review unblinded data and will make recommendations regarding the continuation of the study to the sponsor study team. Resumption of vaccinations will start only upon receipt of written recommendations by the DSMB. The clinical site(s) will be allowed to resume activities upon receipt of a written notification from the sponsor. The formal recommendation from the DSMB will be forwarded by the investigator to the IRB/IEC and by the sponsor to the relevant health authorities, according to local standards and regulations.

Vaccinations for an individual participant may be suspended for safety concerns other than those described in the pausing criteria, at the discretion of the investigator if he/she feels the participant's safety may be threatened. The sponsor's medical monitor or designee or the investigator(s) (upon consultation with the sponsor's medical monitor or designee) may initiate DSMB review for any single event or combination of multiple events which, in their professional opinion, could jeopardize the safety of the participants or the reliability of the data.

Vaccinations for the study may be suspended for safety concerns other than those described above, or before pausing rules are met, if, in the judgement of the DSMB, participant safety may be threatened.

# 7. DISCONTINUATION OF STUDY VACCINATION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 7.1. Discontinuation of Study Vaccination

Not applicable.

# 7.2. Participant Discontinuation/Withdrawal From the Study

A participant will be withdrawn from the study for any of the following reasons:

- Lost to follow-up
- Withdrawal of consent
- Death
- Repeated failure to comply with protocol requirements

When a participant withdraws before study completion, the reason for withdrawal is to be documented in the eCRF and in the source document. If the reason for withdrawal from the study is withdrawal of consent then no additional assessments are allowed.

#### Withdrawal of Consent

A participant declining to return for scheduled visits does not necessarily constitute withdrawal of consent. Alternate follow-up mechanisms that the participant agreed to when signing the consent form apply as local regulations permit.

# 7.2.1. Withdrawal From the Use of Research Samples

## Withdrawal From the Use of Samples in Future Research

The participant may withdraw consent for use of samples for research (refer to Long-Term Retention of Samples for Additional Future Research in Section 10.3.5 in Appendix 3). In such a case, samples will be destroyed after they are no longer needed for the clinical study. Details of the sample retention for research are presented in the main ICF.

### 7.3. Lost to Follow-up

To reduce the chances of a participant being deemed lost to follow-up, prior to randomization attempts should be made to obtain contact information from each participant, eg, home, work, and mobile telephone numbers and email addresses for both the participant as well as appropriate family members.

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. A participant cannot be deemed lost to follow-up until all reasonable efforts made by the study-site personnel to contact the participant are deemed futile. The following actions must be taken if a participant fails to return to the study site for a required study visit:

- The study-site personnel must attempt to contact the participant to reschedule the missed visit as soon as possible, to counsel the participant on the importance of maintaining the assigned visit schedule, to ascertain whether the participant wishes to or should continue in the study.
- Before a participant is deemed lost to follow-up, the investigator or designee must make every reasonable effort to regain contact with the participant (where possible, 3 telephone calls, e-mails, fax, and, if necessary, a certified letter to the participant's last known mailing address,

or local equivalent methods). Locator agencies may also be used as local regulations permit. These contact attempts should be documented in the participant's medical records.

• Should the participant continue to be unreachable, they will be considered to have withdrawn from the study.

Should a study site close, eg, for operational, financial, or other reasons, and the investigator cannot reach the participant to inform them, their contact information will be transferred to another study site.

### 8. STUDY ASSESSMENTS AND PROCEDURES

#### Overview

The Schedules of Activities summarize the frequency and timing of all measurements applicable to this study.

Up to Amendment 7, all participants will be provided access to an eCOA digital tool. This eCOA will be used to collect COVID-19 signs and symptoms surveillance info for all participants, ePRO (Symptoms of infection with Coronavirus-19 [SIC], including body temperature, and pulse oximetry results) for all participants at baseline and in case of COVID-19-like signs and symptoms, and e-Diary data on 7-day reactogenicity (solicited signs and symptoms, including body temperature) in the Safety Subset and all participants who receive booster vaccination at the Year 1/Booster Visit, if feasible. All eCOA assessments should be conducted/completed before any tests, procedures, or other consultations to prevent influencing participant responses. Refer to the PRO completion guidelines for instructions on the administration of ePROs.

As of Amendment 7, the number of on-site visits for participants who are not part of the Immunogenicity or Booster Subsets is reduced. For these participants, any outstanding Visits 8 and 9 are cancelled. In addition, any outstanding Visits 10 and 11 are replaced by a phone call. No further booster vaccination will be provided in the protocol. In addition, requirements for COVID-19 episodes reporting are changed (ie, a passive follow-up approach is adopted, defined as safety follow-up by the site at Month 18 and Month 24 to document COVID-19 participant-reported events as SAE, AE, or MAAE until end of study). All participants will be reconsented at an unscheduled visit and as per local informed consent process guidelines.

If multiple assessments are scheduled for the same timepoint, it is recommended that procedures be performed in the following sequence: vital signs before blood draws. If needed, assessments may be performed on another day within the applicable visit window. Actual dates and times of assessments will be recorded in the source document, the eCRF, or the sample requisition form.

Up to Amendment 7, all participants will be provided a thermometer to measure body temperature if they experience COVID-19-like signs and symptoms. Participants in the Safety Subset and all participants who receive booster vaccination at the Year 1/Booster Visit will be provided a ruler (to measure local injection site reactions) and a participant e-Diary in the eCOA digital tool to record body temperature and solicited local (at injection site) and systemic signs and symptoms. The e-Diary includes instructions on how to capture the data and grading scales to assess severity

of the signs and symptoms post-vaccination (reactogenicity). The study staff is responsible for providing appropriate training to the participant to avoid missing or incorrect data. The e-Diary from participants in the Safety Subset (double-blind phase) and a subset of participants who received booster vaccination at the Year 1/Booster Visit, ie, participants included in the Safety Subset of the double-blind phase and all participants who received a heterologous prime or heterologous additional COVID-19 vaccination outside the study, if feasible, will be reviewed by the study personnel at visits indicated in the Schedules of Activities. If the e-Diary review is missed, the diary will be reviewed during the following visit. All participants will also be provided with a kit to collect nasal swabs samples and recipients to collect saliva (see Section 8.1.2).

The total blood volume to be collected over the course of the study from each participant will be approximately a maximum of 168.5 mL for participants in the immunogenicity subsets and a maximum of 72.0 mL for the other participants. Additional blood samples (up to 35 mL) will be collected from participants that experience COVID-19-like signs and symptoms meeting prespecified criteria for suspected COVID-19. For participants who experience a suspected AESI, an additional 30 mL of blood will be collected. Refer to the Schedules of Activities for the total blood volume (serum and, as applicable, whole blood samples) to be collected at each visit, over the complete course of the study, and in the event of a suspected COVID-19 episode. Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.

If allowed by local regulation, study visits may take place at the participant's home or other location in the event of ongoing SARS-CoV-2 transmission in the area of the participant. If possible and allowed per local regulation, visits, except screening and vaccination visits, can be performed by a phone call or a telemedicine contact, provided that assessments requiring a face-to-face interaction between the participant and a trained health care professional (including but not limited to blood sampling) are performed by a site staff member or a designee at the participant's home or other location, whichever is applicable. Conversely, in case of home visit, assessments that cannot be delegated to a designee must be performed by an appropriate site staff member via a phone call or telemedicine.

### **Visit Windows**

Visit windows are provided in the Schedules of Activities. The participant should be encouraged to come on the exact day planned and use the visit window only if absolutely necessary.

If the Month 6/Unblinding Visit or vaccination window is missed due to a study/vaccination pause (see Section 6.11), efforts will be made to still vaccinate the participant as soon as possible after the pause has been lifted, even if out of the visit window.

### **Screening**

The study will consist of a screening phase of up to 28 days. Screening may also be performed prior to randomization on the day of vaccination. In that case, Visits 1 and 2 will coincide on Day 1. Screening must be completed, and all eligibility criteria must be fulfilled prior to randomization and vaccination.

Screening may be conducted in part via a sponsor- and IRB/IEC-pre-approved non-study-specific screening consent process, but only if the relevant pre-screening tests are identical to the per-protocol screening tests and are within 28 days prior to vaccination. However, no study-specific procedures, other than these pre-approved pre-screening assessments, will be performed until the participant has signed the study-specific ICF. The study-specific ICF date will be collected for the study database. The non-study-specific ICF will be considered source data.

# Long term follow-up

Until 1 year after the Month 6/Unblinding Visit, each participant will be asked at least twice a week, through the eCOA, if they have experienced any new symptoms or health concerns that could be related to infection with SARS-CoV-2. As of 1-year after the Month 6/Unblinding Visit, until the end of the 2-year follow-up period, the frequency of this (suspected) COVID-19 surveillance (symptom check) through the eCOA may decrease to once every 2 weeks depending on epidemiology. All participants will be monitored for safety (including enhanced disease) for approximately 1 year after the Year 1/Booster Visit, ie, until the last study visit. Sites should monitor participant compliance with (suspected) COVID-19 surveillance (symptom check) and SIC completion on a daily basis and reach out to a participant if the participant fails to complete the surveillance question upon any of these reminders. Every effort will be made to document the status of all participants that are lost to follow-up due to not completing the eCOA and for whom hospitalization has not been recorded. The questionnaire will be accessible on the eCOA platform in between scheduled reminders and participants will be encouraged to answer the surveillance question in the eCOA as soon as possible after the onset of COVID-19-like symptoms. Procedures to be followed in case of (suspected) COVID-19 are outlined in Section 8.1.1. As of Amendment 7, active follow-up of suspected COVID-19 episodes will be replaced by a passive surveillance and eCOA will be stopped.

## Sample Collection and Handling

The actual dates and times of sample collection must be recorded in the eCRF or laboratory requisition form. Refer to the Schedules of Activities for the timing and frequency of all sample collections.

Instructions for the collection, handling, storage, and shipment of samples are found in the laboratory manual that will be provided. Collection, handling, storage, and shipment of samples must be under the specified, and where applicable, controlled temperature conditions as indicated in the laboratory manual.

# **Study-Specific Materials**

The investigator will be provided with the following supplies:

- IB for Ad26.COV2.S
- Thermometer
- Ruler (to measure diameter of any erythema and swelling)

- A pulse oximeter
- Pharmacy manual/SIPPM
- IPPI
- IWRS Manual
- Sample ICF
- Laboratory manual and laboratory supplies
- Nasal swab kits, saliva recipients, and participant instructions
- eCOA platform access and participant instructions. Participants may use their own eDevice using an application if their device (smartphone or tablet) is compatible, or a web portal. Provisioned devices will be available on a limited basis.
- Tablet for eConsent, if applicable
- Contact information page(s)
- eCRF completion guidelines

# 8.1. Efficacy and Immunogenicity Assessments

No generally accepted immunological correlate of protection has been demonstrated for SARS-CoV-2 to date.

# 8.1.1. Prespecified Criteria for Suspected COVID-19 Prior to Protocol Amendment 7

The criteria for suspected COVID-19 (ie, the triggers to proceed with home-collection of the nasal swabs on COVID-19 Day 1-2 and to proceed with the COVID-19 Day 3-5 visit) are prespecified as follows:

• A positive RT-PCR result for SARS-CoV-2, through a private or public laboratory independent of the study, whether symptomatic or asymptomatic

OR

- New onset or worsening of any 1 of the symptoms, which lasts for at least 24 hours, not otherwise explained:
  - Headache
  - o Malaise (appetite loss, generally unwell, fatigue, physical weakness)
  - Myalgia (muscle pain)
  - Chest congestion
  - o Cough
  - o Runny nose

- Shortness of breath or difficulty breathing (resting or on exertion)
- Sore throat
- Wheezing
- o Eye irritation or discharge
- Chills
- o Fever ( $\geq 38.0$ °C or  $\geq 100.4$ °F)
- o Pulse oximetry value ≤95%, which is a decrease from baseline
- o Heart rate ≥90 beats/minute at rest, which is an increase from baseline
- o Gastrointestinal symptoms (diarrhea, vomiting, nausea, abdominal pain)
- Neurologic symptoms (numbness, difficulty forming or understanding speech)
- o Red or bruised looking toes
- Skin rash
- Taste loss or new/changing sense of smell
- O Symptoms of blood clots: pain/cramping, swelling or redness in your legs/calves
- Confusion
- Bluish lips or face
- Clinical suspicion/judgement by investigator of symptoms suggestive for COVID-19

As several of the prespecified criteria for suspected COVID-19 overlap with vaccine-related reactogenicity, investigators' clinical judgement is required to exclude vaccine-related events when assessing suspected COVID-19.

# 8.1.2. Procedures in the Event of (Suspected) COVID-19

# 8.1.2.1. Passive Follow-up (As of Amendment 7)

As of Amendment 7, active follow-up of suspected COVID-19 episodes will be replaced by a passive follow-up approach. For COVID-19 events that are ongoing at the time of informed consent:

- a. Participant will be instructed to stop using the eCOA.
- b. Any outstanding activities planned for the follow-up of COVID-19 events will end as of the consent.
- c. No further sampling for participants and no Day 1-2, Day 3-4, and Day 29 visit will be performed
- d. MRU and MA-COV forms are no longer to be completed

The eCOA will be stopped based on approval of protocol Amendment 7 at each study site. From that point onwards, active participants are no longer able to use eCOA.

For new suspected COVID-19 episodes no samples will be collected in the context of the study. Site staff will collect information on new COVID-19 episodes at scheduled time points and report these as SAEs, AEs, or MAAEs, as applicable. Participants may contact the site at any time in between scheduled visits to report COVID-19 episodes. Concomitant medications for each COVID-19 episode are to be reported into the eCRF as well as any laboratory confirmation of COVID-19, if available.

# 8.1.2.2. Active Follow-up (Until Amendment 7)

Procedures to be performed in the event a participant experiences signs or symptoms suggesting possible COVID-19 or a participant became aware of a positive RT-PCR test result for SARS-CoV-2 outside the study site context, whether symptomatic or asymptomatic, are detailed in the Schedules of Activities. A high-level schematic overview is presented in Figure 2.

Figure 2: Decision Tree for COVID-19 Procedures



If the participant no longer meets the prespecified criteria at Day 3 5 and results from the nasal sample at Day 1 2 and/or Day 3 5 are latently positive (i.e.  $\geq$ 14 days to result), the participant will be contacted and asked to proceed with COVID 19 procedures (2 day cycles).

If signs and symptoms are still ongoing on COVID-19 Day 3-5, collection of SIC will be continued until at least 14 days after onset unless both COVID-19 Day 1-2 and COVID-19 Day 3-5 are both negative. If either of the swabs is positive or the result is unknown AND the participant is beyond 14 days after onset of symptoms, the SIC can be stopped after 2 days without signs and symptoms.

If 2 consecutive nasal swabs negative for SARS CoV 2 are not available due to operational reasons (eg, delays in results availability), participants may cease collection of nasal swabs and saliva samples after COVID 19 Day 29, provided they have 2 consecutive days with no COVID 19 related signs and symptoms. In these cases, participants may be asked to resume sample collection if nasal sample results once available do not present with 2 consecutive negative swabs for SARS CoV 2.

COVID 19 coronavirus disease 2019; eCOA electronic clinical outcome assessment; PCR polymerase chain reaction; SARS CoV 2 severe acute respiratory syndrome coronavirus 2; SIC Symptoms of Infection with Coronavirus 19.

For all medical visits for COVID-19 or COVID-19 complications, including those resulting in hospitalization, a standard list of questions will be provided (MA-COV form [Appendix 8]), with the aim to collect additional information on any other diagnostics (eg, chest X-rays, spirometry, pulmonary function tests) or interventions during the clinical course of COVID-19. The MA-COV form will be provided to the participant at the vaccination visit and should be completed by the medical care provider or the study site personnel during medical visits for COVID-19 or COVID-19 complications.

*Note*: if for any reason a site visit per the procedures described below is not feasible, a member of the study staff can visit the participant at home (or at the hospital or other location, if needed), if allowed by local regulations.

# Day 1-2 procedures in case of signs and symptoms

If a participant records in the eCOA or informs the site that he/she experienced any signs or symptoms suggesting possible COVID-19, this will be considered **COVID-19 Day 1** (day of onset of signs and symptoms). The participant will be asked to complete the ePROs (ie, the SIC [Appendix 6], including body temperature) in the eCOA.

#### Notes:

The SIC questionnaire asks the participant if he/she had any of the prespecified signs or symptoms (see Appendix 6) during the past 24 hours, and (when applicable) to rate the severity. The SIC questionnaire takes approximately 5 minutes to complete.

The participant should record the highest temperature in the last 24 hours in the SIC.

The participant should record at least 1 of the 3 pulse oximetry readings in the last 24 hours in the eCOA.

If a participant is unable to complete the SIC in the eCOA, a study staff member can collect information on the participant's symptoms and body temperature, by contacting the participant by telephone (or visit the participant at home), reading the questions aloud to the participant and entering the participant's responses on the participant's behalf. If the participant requires assistance, the participant's caregiver can help the participant to complete the SIC in the eCOA by reading the questions aloud to the participant and recording the participant's responses in the eCOA using the caregiver's unique identifier and PIN on the participant's behalf. Procedures for caregivers to collect and report the participant's responses to the eCOA questions will be detailed in instructions for caregiver assessment of COVID-19 episodes. More details are provided in the PRO completion guidelines.

Based on the information collected through the SIC, the site will reach out to the participant at the latest on COVID-19 Day 2 (the day after the day of symptom onset) to assess whether the reported signs and symptoms qualify as a suspected COVID-19 episode using prespecified criteria (Section 8.1.1). As several of the prespecified criteria for suspected COVID-19 overlap with vaccine-related reactogenicity, investigators' clinical judgement is required to exclude vaccine-related events when assessing suspected COVID-19. If the participant would actively reach out to

the site already on COVID-19 Day 1, the site should already make a first assessment on COVID-19 Day 1 to check whether the reported signs and symptoms qualify as a suspected COVID-19 episode using prespecified criteria (Section 8.1.1). As soon as the prespecified criteria for suspected COVID-19 are met (COVID-19 Day 1-2), the participant will be asked to undertake the COVID-19 procedures. In particular:

The participant will be asked to continue to complete the ePROs in the eCOA as specified above for COVID-19 Day 1:

- SIC (including body temperature): every day, preferably in the evening around the same time each day.
- O Blood oxygen saturation and pulse rate using a pulse oximeter 3 times a day, preferably in the morning, at lunch time, and in the evening.

*Note*: the ePROs do not have to be completed if special circumstances occur, such as hospitalization or ventilation, in which case the reason for not completing the ePROs should be recorded by site staff in the eCRF.

The participant will be asked to collect a nasal swab at home on **COVID-19 Day 1-2**, as soon as possible after it has been confirmed that the prespecified criteria for suspected COVID-19 are met. If the participant requires assistance, a trained HCP can help the participant to collect the nasal swab. The study site should arrange transfer of the nasal swab to the study site as soon as possible after collection, preferably within 24 hours. The COVID-19 Day 1-2 nasal swab can also be collected at the study site (or hospital or other location, if needed), if preferred by the participant.

### Day 1-2 procedures in case of a positive RT-PCR test outside the study site context

If a participant becomes aware of a positive RT-PCR test for SARS-CoV-2 he/she should contact the site as soon as possible. The day the participant became aware of the positive RT-PCR test will be considered **COVID-19 Day 1**. Regardless of whether the participant is symptomatic or asymptomatic, they will be asked to:

Complete the (suspected) COVID-19 surveillance (symptom check) in the eCOA. In case of COVID-like signs and symptoms they will need to complete the SIC (Appendix 6, including body temperature) in the eCOA.

The participant will be asked to collect a nasal swab at home on **COVID-19 Day 1-2**, as described for the participants with signs and symptoms (see above).

These precautionary measures are to ensure that site staff who come into physical contact with a participant deemed to be a COVID-19 case undertake the proper safety procedures such as wearing of personal protective equipment.

# Day 3-5 procedures for all participants who have met the prespecified criteria for (suspected) COVID-19

The participant will be asked to come to the site on **COVID-19 Day 3-5** (between 2 and 4 days after symptom onset/becoming aware of a positive RT-PCR test).

If a site visit is not feasible, a member of the study staff or designee could visit the participant at home (or at the hospital or other location, if needed), if allowed by local regulations. The study staff or designee visiting participants at home will use personal protective equipment according to local regulations. The COVID-19 Day 3-5 assessments may also be performed by a trained HCP, if allowed per local regulations.

During Part 1 of the COVID-19 Day 3-5 visit, if the participant has experienced COVID-19 like signs and symptoms, the site will interview the participant to assess whether the reported signs and symptoms still qualify as a suspected COVID-19 episode using prespecified criteria (Section 8.1.1). In addition, for all participants with (suspected) COVID-19, a qualified member of the study site will measure vital signs (body temperature, blood pressure, heart rate, and respiratory rate) and pulse oximetry. A targeted physical examination will be performed based on the judgement of the investigator. A nasal swab will be collected for detection of SARS-CoV-2 by a qualified member of the study site.

If the signs and symptoms still meet the prespecified criteria for suspected COVID-19 on COVID-19 Day 3-5 or if at least one nasal sample from COVID-19 Day 1-2 or Day 3-5 visits is positive for SARS-CoV-2 (tested by RT-PCR), the following assessments and procedures are to be performed during **Part 2** of the **COVID-19 Day 3-5** visit: a blood sample for exploration of biomarkers that correlate with SARS-CoV-2 infection and COVID-19 severity will be collected by a qualified member of the study site. A saliva sample will be taken by the participant during the study visit. The MRU questionnaire will be completed based on a clinical interview (Appendix 7). The medical history and description of COVID-19 episode will be collected by interview with the participant.

If signs and symptoms are still ongoing on **COVID-19 Day 3-5**, collection of SIC will continue as specified in the next section (*Closure of the COVID-19 episode* 

If allowed by local regulations and if the participant consents, he/she will be interviewed on characteristics related to their current work situation, living situation, and community interactions (See Appendix 12). These data will be used for risk factor analysis.

If the signs and symptoms no longer meet the prespecified criteria for suspected COVID-19 on COVID-19 Day 3-5 and no result from nasal swabs collected on Day 1-2 and/or Day 3-5 visits is available, the participant will not undertake any further COVID-19 procedures. He/she will fall back to the default Schedule of Activities, until the end of the study/early withdrawal.

# Procedures during the 2-day cycles

If a participant has signs and symptoms that still meet the prespecified criteria for suspected COVID-19 (Section 8.1.1) at COVID-19 Day 3-5 visit or has at least one positive nasal sample for SARS-CoV-2 at COVID-19 Day 1-2 or COVID-19 Day 3-5 visits, he or she will be asked to undertake the COVID-19 procedures, in particular:

All participants will be asked to collect a nasal swab and a saliva sample at home once every 2 days (daily alternating between nasal swabs and saliva samples). If the participant

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

requires assistance, a trained HCP can help the participant to collect the nasal swabs and/or saliva samples. The study site should arrange transfer of the nasal swabs and saliva samples to the study site within 3 days after collection. Details are provided in the laboratory manual.

In case of signs and symptoms: The participant will be reminded to further complete the ePROs in the eCOA as described for COVID Day 1-2:

In case the nasal swabs collected on Day 1-2 or Day 3-5 visits are tested positive for SARS-CoV-2 and the participant is asymptomatic: The participant will be reminded to further complete (suspected) COVID-19 surveillance (symptom check).

If, on COVID-19 Day 3-5, the participant stopped the COVID-19 procedures and returned to default Schedule of Activities, due to lack of signs and symptoms and unavailability of results from nasal swabs collected on Day 1-2 and/or Day 3-5 visits, the participant will be contacted as soon as at least one of these samples is found to be positive for SARS-CoV-2 presence. The participant will be asked to resume COVID-19 procedures, until 14 days after symptom onset (COVID-19 Day 15) or until **resolution of the COVID-19 episode**, whichever comes last.

#### *Notes*:

o Participants should be encouraged by the site to collect nasal swabs and saliva samples as indicated in the Schedules of Activities. If the participant is unable or unwilling to collect all samples as requested, the participant should still complete the other COVID-19 assessments, including the visit at COVID-19 Day 29.

## Day 29 procedures

If a participant has at least 1 SARS-CoV-2 positive nasal swab collected on COVID-19 Day 1-2 or Day 3-5, then he or she will be asked to return to the site on COVID-19 Day 29 (±7 days) where a blood sample will be drawn for sero-confirmation and exploration of biomarkers that correlate with SARS-CoV-2 infection and COVID-19 severity. A qualified member of the study site will measure vital signs (body temperature, blood pressure, heart rate, and respiratory rate) and pulse oximetry. A targeted physical examination will be performed based on the judgement of the investigator. The MRU questionnaire will be completed based on a clinical interview (Appendix 7). The medical history and description of COVID-19 episode will be collected by interview with the participant. If the participant is still symptomatic, he/she will complete the SIC (Appendix 6) in the eCOA. Asymptomatic participants will complete the (suspected) COVID-19 surveillance (symptom check).

*Notes*: COVID-19 Day 29 should still be performed even if the nasal swabs results are still pending. The COVID-19 Day 29 assessments may also be performed by a trained HCP at the participant's home, if allowed per local regulations.

This visit can be combined with a regular study visit if within the applicable visit windows.

## Closure of the COVID-19 episode

The participant should continue the COVID-19 procedures until any of the following occurs, based on molecular test results:

If both nasal swabs (collected on COVID-19 Day 1-2 and COVID-19 Day 3-5) are **negative** for SARS-CoV-2, the participant will not undertake any further COVID-19 procedures and will fall back to the default Schedule of Activities, until the end of the study/early withdrawal.

If the participant has at least 1 SARS-CoV-2 positive nasal swab collected on COVID-19 Day 1-2 or Day 3-5 visits, then the participant will be asked to undertake the COVID-19 procedures (2-day cycles) until 14 days after symptom onset (COVID-19 Day 15) or until **resolution of the COVID-19 episode**, whichever comes last<sup>a</sup>. Resolution of the COVID-19 episode is defined as having 2 consecutive SARS-CoV-2 negative nasal swabs and 2 consecutive days with no COVID-19-related signs or symptoms. Once past COVID-19 Day 15, participants should stop the collection of nasal swabs and saliva samples as soon as 2 consecutive nasal swabs are SARS-CoV-2 negative, but (if still symptomatic at that time) should continue completing the ePROs (including SIC, body temperature, and pulse oximetry) in the eCOA until 2 consecutive days with no COVID-19-related signs or symptoms.

*Note*: for participants who have signs and symptoms present at baseline (assessed pre-vaccination), only signs and symptoms that are associated with COVID-19 and that developed during the COVID-19 episode are to be taken into account.

If signs and symptoms are still ongoing on **COVID-19 Day 3-5**, collection of SIC will be continued until at least 14 days after onset unless both **COVID-19 Day 1-2** and **COVID-19 Day 3-5** are both negative. If either of the swabs is positive or the result is unknown AND the participant is beyond 14 days after onset of symptoms, the SIC can be stopped after 2 days without signs and symptoms.

If 2 consecutive nasal swabs negative for SARS-CoV-2 are not available due to operational reasons (eg, delays in results availability), participants may cease collection of nasal swabs and saliva samples after COVID-19 Day 29, provided they have 2 consecutive days with no COVID-19-related signs and symptoms. In these cases, participants may be asked to resume sample collection if nasal sample results once available do not present with 2 consecutive negative swabs for SARS-CoV-2.

Upon closure of the COVID-19 episode and procedures, all participants will fall back to the default Schedules of Activities, until the end of the study/early withdrawal.

<sup>&</sup>lt;sup>a</sup> long-term sequelae of COVID-19 will not be followed until their resolution if not resolved within a month.

All confirmed COVID-19 episodes will be communicated to the respective participant and to other authorities according to local regulations.

If the participant experiences new signs or symptoms suggesting possible COVID-19 at a later point in time, the participant would re-start the COVID-19 procedures from COVID-19 Day 1 onwards.

With regards to the ePRO (ie, the SIC, including body temperature):

- The ePRO instrument will be provided in the local language in accordance with local guidelines.
- The ePRO instrument must be available for regulators and for IRB/ERC submissions, therefore the ePRO instrument or screen shots need to be attached to the protocol or provided in a companion manual with the instruments that will be submitted with the protocol.
- The ePRO and AE data will not be reconciled with 1 another.

# 8.1.3. Efficacy Assessments

Up to Amendment 7, identification and molecular confirmation of SARS-CoV-2 infection and symptomatic COVID-19 will be performed throughout the study as described in Section 8.1.2.2. Up to Amendment 7, the ePRO to evaluate VE parameters will be the SIC. See Section 8.1.3.1 for Case Definition of Moderate to Severe/Critical COVID-19 and Section 8.1.3.2 for Case Definition of Mild COVID-19. As of Amendment 7, no identification or molecular confirmation of SARS-CoV-2 infection and symptomatic COVID-19 will be done.

Molecular confirmation of SARS-CoV-2 infection by a central laboratory will be used for the analysis of the case definition.

All COVID-19 cases will be assessed independently by a Clinical Severity Adjudication Committee (see Section 8.1.3.6). Classification of severity will be based on the highest degree of severity during the observation period (see Sections 8.1.3.1 and 8.1.3.2).

As several of the prespecified criteria for suspected COVID-19 overlap with vaccine-related reactogenicity, investigators' clinical judgement is required to exclude vaccine-related events when assessing suspected COVID-19.

The occurrence of COVID-19-related hospitalization and COVID-19-related complications (such as but not limited to hyperinflammatory syndrome, pneumonia, neurological or vascular complications, severe pneumonia, severe neurological or vascular events, acute respiratory distress syndrome, renal complications, sepsis, septic shock, death)<sup>71</sup> will be monitored throughout the study (up to protocol amendment 7).

As a secondary objective, VE in the prevention of asymptomatic SARS-CoV-2 infection and mild COVID-19 will be analyzed. For samples collected prior to implementation of Amendment 7: an immunologic test for SARS-CoV-2 seroconversion (ELISA and/or SARS-CoV-2 immunoglobulin assay) based on SARS-CoV-2 N protein, may be performed to identify cases of asymptomatic

infection. This assay will be performed on samples obtained (if prior to Amendment 7) at Day 1 (pre-vaccination), Day 71, Month 6/Unblinding Visit, and Month 18.

#### 8.1.3.1. Case Definition for Moderate to Severe/Critical COVID-19

For the co-primary endpoints (see Section 3), all moderate and severe/critical COVID-19 cases will be considered.

# **Case Definition for Moderate COVID-19**

• A SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample

# AND at any time during the course of observation<sup>a</sup>:

# Any 1 of the following new or worsening signs or symptoms:

- Respiratory rate ≥20 breaths/minute
- Abnormal saturation of oxygen (SpO<sub>2</sub>) but still >93% on room air at sea level\*
- Clinical or radiologic evidence of pneumonia
- Radiologic evidence of deep vein thrombosis (DVT)
- Shortness of breath or difficulty breathing

# Any 2 of the following new or worsening signs or symptoms:

- Fever ( $\ge 38.0^{\circ}$ C or  $\ge 100.4^{\circ}$ F)
- Heart rate ≥90 beats/minute
- Shaking chills or rigors
- Sore throat
- Cough
- Malaise as evidenced by 1 or more of the following\*\*:
  - Loss of appetite
  - Generally unwell
  - Fatigue
  - Physical weakness
- Headache
- Muscle pain (myalgia)
- Gastrointestinal symptoms (diarrhea, vomiting, nausea, abdominal pain)\*\*
- New or changing olfactory or taste disorders
- Red or bruised looking feet or toes

OR

<sup>\*</sup> SpO2 criteria will be adjusted according to altitude per the investigator judgement.

<sup>\*\*</sup> Having 2 or more elements of a symptom (eg, vomiting and diarrhea or fatigue and loss of appetite) is counted only as 1 symptom for the case definition. To meet the case definition, a participant would need to have at least 2 different symptoms.

<sup>&</sup>lt;sup>a</sup> Until Amendment 7: Participants will be asked to undertake the COVID-19 procedures until 14 days after symptom onset (COVID-19 Day 15) or until **resolution of the COVID-19 episode**, whichever comes last (see Section 8.1.2).

## Case Definition for Severe/Critical COVID-19

 A SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample

## AND any 1 of the following at any time during the course of observation<sup>q</sup>:

- Clinical signs at rest indicative of severe systemic illness (respiratory rate ≥30 breaths/minute, heart rate ≥125 beats/minute, oxygen saturation (SpO<sub>2</sub>) ≤93% on room air at sea level\*, or partial pressure of oxygen/fraction of inspired oxygen (PaO<sub>2</sub>/FiO<sub>2</sub>) <300 mmHg)
  - \* SpO<sub>2</sub> criteria will be adjusted according to altitude per the investigator judgement.
- Respiratory failure (defined as needing high-flow oxygen, non-invasive ventilation, mechanical ventilation, or extracorporeal membrane oxygenation [ECMO])
- Evidence of shock (defined as systolic blood pressure <90 mmHg, diastolic blood pressure <60 mmHg, or requiring vasopressors)
- Significant acute renal, hepatic, or neurologic dysfunction
- Admission to the ICU
- Death

All cases meeting the severe/critical criteria will be adjudicated by the Clinical Severity Adjudication Committee to determine if the case is severe/critical in their judgement.

All cases meeting the moderate case definition and that include  $\geq 3$  signs and/or symptoms from the list of signs and symptoms will be evaluated by the Clinical Severity Adjudication Committee to determine if the case is severe/critical in their judgement.

Classification of a case as severe/critical by the Clinical Severity Adjudication Committee is considered definitive.

#### 8.1.3.2. Case Definition for Mild COVID-19

 A SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample;

## AND at any time during the course of observationa:

• One of the following symptoms: fever (≥38.0°C or ≥100.4°F), sore throat, malaise (loss of appetite, generally unwell, fatigue, physical weakness), headache, muscle pain (myalgia), gastrointestinal symptoms, cough, chest congestion, runny nose, wheezing, skin rash, eye

-

Until Amendment 7: Participants will be asked to undertake the COVID-19 procedures until 14 days after symptom onset (COVID-19 Day 15) or until **resolution of the COVID-19 episode**, whichever comes last (see Section 8.1.2).

irritation or discharge, chills, new or changing olfactory or taste disorders, red or bruised looking feet or toes, or shaking chills or rigors.

A case is considered mild when it meets the above case definition but not the moderate to severe/critical definition in Section 8.1.3.1. All cases will be evaluated by the Clinical Severity Adjudication Committee. Classification by the Clinical Severity Adjudication Committee is considered definitive.

#### 8.1.3.3. US FDA Harmonized Case Definition for COVID-19

If a participant presents with symptoms as those listed by the US FDA harmonized case definition <sup>14</sup> (see Appendix 10), the investigator (or designated medically trained clinician) should assess if these are suggestive of COVID-19:

- A SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample; AND
- COVID-19 symptoms consistent with those defined by the US FDA harmonized case definition <sup>14</sup> at the time of finalization of this protocol: fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea.

All cases will be evaluated by the Clinical Severity Adjudication Committee. Classification by the Clinical Severity Adjudication Committee is considered definitive.

# 8.1.3.4. Case Definition for Asymptomatic or Undetected COVID-19

If a participant does not fulfil the criteria for suspected COVID-19 based on signs and symptoms which would classify them as mild, moderate, or severe by the protocol definitions per Section 8.1.1,

#### **AND**

• has a SARS-CoV-2 positive RT-PCR or molecular test result from any available respiratory tract sample (eg, nasal swab sample, sputum sample, throat swab sample, saliva sample) or other sample

#### OR

• develops a positive serology (non-S protein) test

Then, the participant will be considered to have experienced asymptomatic or undetected COVID-19.

A molecularly confirmed positive RT-PCR for SARS-CoV-2 will need to be captured in the eCRF.

Cases will be classified as being an "Asymptomatic SARS-CoV-2 infection" by the Clinical Severity Adjudication Committee utilizing the following guidelines, which are described in more detail in the charter for the committee.

- The definition of any case that is either RT-PCR positive that was previously RT-PCR negative or seropositive for N protein specific antibodies that was previously seronegative for N protein specific antibodies and is clinically asymptomatic will be considered as an asymptomatic COVID-19 case.
- The definition of clinically asymptomatic COVID-19 is defined as no clinical symptoms that
  would be classified as mild, moderate, or severe COVID-19 by the protocol case definition
  for symptoms independent of the SARS-CoV-2 N protein specific antibody seroconversion or
  RT-PCR results.

Potential asymptomatic cases that are identified by N-serology seroconversion will all be examined by the Clinical Severity Adjudication Committee for the presence of any signs or symptoms and if found, to determine if they would still be classified as asymptomatic COVID-19. Moderate, severe, hospitalized, or fatal cases that are found by SARS-CoV-2 N protein specific antibody seroconversion will be utilized in a sensitivity analysis to determine if any conclusions would be changed by adding the primary case definition of a positive RT-PCR, with appropriate signs and symptoms, to those cases which were identified by SARS-CoV-2 N protein specific antibody seroconversion with appropriate signs and symptoms.

As of Amendment 7, severity assessment by the CSAC may still be performed and will be based on the data collected through the passive follow-up (eg, hospitalization reported in the context of SAEs). The scope of the severity review may change and will be described in the charter.

## 8.1.3.5. SARS-CoV-2 Seroconversion Assessment

An immunologic test for SARS-CoV-2 seroconversion (ELISA and/or SARS-CoV-2 immunoglobulin assay) based on SARS-CoV-2 N protein may be performed to identify cases of asymptomatic infection on samples obtained at Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, Year 1 + 28 days for participants who received booster vaccination, Year 1 + 72 days for participants who received booster vaccination, and Month 18 (24 weeks after Year 1 Visit). (see Section 8.1.4).

# 8.1.3.6. Clinical Severity Adjudication Committee

The Clinical Severity Adjudication Committee will review all cases in the study, except for cases already adjudicated as severe, as a supplement to the algorithm described in the SAP, as well as those requiring medical intervention (such as a composite endpoint of hospitalization, ICU admission, mechanical ventilation, and ECMO, linked to objective measures such as decreased oxygenation, X-ray or CT findings), including onset of cases, taking into account all available relevant information at the time of adjudication. As of Amendment 7, Clinical Severity Adjudication Committee may review all cases based on available data from the passive follow-up (eg, limited to COVID-19 AE/SAE data, CIOMS forms, local laboratory results). More details will be provided in the revised charter of the Clinical Severity Adjudication Committee. Readjudication will occur if new information becomes available. The last adjudication for a given case will determine the status of the case for analysis. The Clinical Severity Adjudication Committee's assessment will be considered the definitive classification of the case. The case review including

severity assessments after implementation of Protocol Amendment 7 may change and will be reflected in the charter of the committee.

# 8.1.4. Immunogenicity Assessments

Blood will be collected from all non-Immunogenicity Subset participants for humoral immunogenicity assessments at Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, and Year 1 (if Year 1 visit occurred prior to implementation of protocol amendment 7).

For a total of approximately 400 participants in the Immunogenicity Subset (ie, participants at sites with access to appropriate processing facilities), blood will be collected for analysis of humoral immune responses on Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, Year 1, Month 18, and Year 2 visit after double-blind vaccination, and additionally 28 days and 72 days after booster vaccination, if applicable.

Note: Those participants in the Immunogenicity Subset that transfer to the Homologous Booster Subset at the Year 1/Booster Visit (see below) will from that visit onwards follow the humoral immunogenicity sample schedule of the Homologous Booster Subset and discontinue the schedule of the Immunogenicity Subset.

Participants in the Immunogenicity Subset will be divided into 4 groups as presented in Table 3.

Table 3: Sample Size and Distribution of the Immunogenicity Subset Between Active and Placebo Groups

| Study Vaccine<br>(Double-blind) | Subgroup 1a | Subgroup 1b | Subgroup 2a | Subgroup 2b |
|---|---|---|---|---|
| 5×10 <sup>10</sup> vp | 50 | 50 | 50 | 50 |
| Placebo | 50 | 50 | 50 | 50 |
| Total | 100 | 100 | 100 | 100 |

vp virus particles

Subgroup 1a: healthy ≥18 to <60 year old adults without relevant comorbidities, enrolled during Stage 1a.

Subgroup 1b: ≥18 to <60 year old adults with relevant comorbidities, enrolled during Stage 1b.

Subgroup 2a: healthy ≥60 year old adults without relevant comorbidities, enrolled during Stage 2a.

Subgroup 2b: ≥60 year old adults with relevant comorbidities, enrolled during Stage 2b.

Up to Amendment 7, during a COVID-19 episode, blood will be collected on COVID-19 Day 3-5 and on COVID-19 Day 29 for immunogenicity assessments, including the assays summarized in Table 6. As from Amendment 7, active follow-up will no longer be pursued and blood sampling for this purpose will no longer be performed.

#### **Booster Vaccination**

Up to Amendment 7, blood will be collected from all non-Subset participants who received booster vaccination for humoral immunogenicity assessments at the Year 1/Booster Visit and 28 days, 72 days, and 6 months after booster vaccination. A blood sample for transcriptomics will be collected from all participants 28 days after booster vaccination.

<u>Homologous Booster Subset</u>: The Homologous Booster Subset will include approximately 200 participants, as described in Table 4. This subset will include participants from the Immunogenicity Subset (Table 3), who received Ad26.COV2.S in the double-blind phase or after cross-over, and subsequently received an Ad26.COV2.S booster vaccination in the study. This group may be augmented by other participants to replace participants who are not available. Participants in the Homologous Booster Subset will have a blood sample collected pre-booster vaccination, and 28 days, 72 days, 6 months, and 1 year post booster vaccination for humoral immunogenicity assessment (see Section 1.3).

Table 4: Sample Size and Distribution of the Homologous Booster Subset Age Groups

| Study Vaccine | Subgroup 1a | Subgroup 1b | Subgroup 2a | Subgroup 2b |
|---|---|---|---|---|
| 5×10 <sup>10</sup> vp | 50 | 50 | 50 | 50 |

vp virus particles

Subgroup 1a: healthy ≥18 to <60 year old adults without relevant comorbidities.

Subgroup 1b: ≥18 to <60 year old adults with relevant comorbidities.

Subgroup 2a: healthy ≥60 year old adults without relevant comorbidities.

Subgroup 2b: ≥60 year old adults with relevant comorbidities.

Heterologous Booster Subset: The Heterologous Booster Subset will include approximately 400 participants, as described in Table 5. This subset will include participants in the study who received placebo in the double-blind phase and have received primary vaccination with an mRNA vaccine or another authorized COVID-19 vaccine including protein, inactivated, and adenovector based vaccines outside the study, who subsequently remained in the study and subsequently received an Ad26.COV2.S booster vaccination in the study. Participants who already received an additional COVID-19 vaccination after the primary regimen outside the study will not be included in the Heterologous Booster Subset. Participants will be selected out of countries where these vaccines were authorized for emergency use or are licensed. Participants in the Heterologous Booster Subset will have blood collected pre booster vaccination, and 28 days, 72 days, 6 months, and 1 year post booster vaccination for humoral immunogenicity assessment (see Section 1.3).

Table 5: Sample Size and Distribution of the Heterologous Booster Subset Primary Vaccination Groups

| Age group for participants who received a booster dose | mRNA vaccine subgroup | Protein vaccine subgroup | Adenovector vaccine subgroup | Inactivated vaccine subgroup |
|---|---|---|---|---|
| 18-59 years old | 50 | 50 | 50 | 50 |
| ≥60 years old | 50 | 50 | 50 | 50 |
| Total | 100 | 100 | 100 | 100 |

vp virus particles

Enrollment into the Homologous Booster Subset and Heterologous Booster subset will start once operationally feasible.

Additionally, approximately the first 60 eligible participants once operationally feasible of the Homologous Booster Subset (approximately 15 per subgroup [1a, 1b, 2a, and 2b]) and

15 A ....:1 2022

approximately the first 60 eligible participants once operationally feasible of the Heterologous Booster Subset (approximately 15 per subgroup [primary vaccination with mRNA vaccine, protein vaccine, adenovector vaccine, and inactivated vaccine]) will have blood collected pre-booster and 1 day and 28 days post booster vaccination for transcriptomics and cytokine/chemokine assessment (see Section 1.3).

Table 6: Immunogenicity and Transcriptomic Assays

| Humoral Assays | Purpose |
|---|---|
| Supportive of Secondary Objectives | |
| SARS-CoV-2 binding antibodies | Analysis of antibodies binding to SARS-CoV-2 S protein |
| to S protein (ELISA) | |
| SARS-CoV-2 seroconversion | Analysis of antibodies binding to SARS-CoV-2 N protein |
| based on antibodies to N protein | |
| (ELISA and/or SARS-CoV-2 | |
| immunoglobulin assay) | |
| Supportive of Secondary and Exp | |
| SARS-CoV-2 neutralization | Analysis of neutralizing antibodies against SARS-CoV-2 original |
| (VNA) | strain and/or variants, using a live VNA and/or pseudovirion |
| | expressing S protein neutralization assay |
| SARS-CoV-2 binding antibodies | Analysis of antibodies binding to the original and/or variants |
| to S protein (MSD) | SARS-CoV-2 S protein (different than the assays supportive of the |
| | secondary objectives) and the receptor-binding domain (RBD) of |
| | SARS-CoV-2 S protein |
| Functional and molecular | Analysis of antibody characteristics including, but not limited to, |
| antibody characterization | avidity, Fc-mediated viral clearance, Fc characteristics, Ig |
| | subclass, IgG isotype, antibody glycosylation, and assessment of |
| | antibody repertoire |
| Adenovirus neutralization (VNA) | Adenovirus neutralization assay to evaluate neutralizing antibody |
| | responses against the Ad26 vector |
| Binding antibodies to other | Analysis of antibodies binding to coronaviruses other than SARS- |
| coronaviruses (MSD) | CoV-2 |
| Cytokine profiling | Analysis of cytokines, chemokines, and other proteins of the |
| | innate or adaptive immune response in the serum or plasma |
| Transcriptomic Assay | Purpose |
| | Supportive of Exploratory Objectives |
| Gene expression analysis | Analysis of gene expression by RNA transcript profiling in |
| | unstimulated cells or whole blood |

Ad26 adenovirus type 26; ELISA enzyme linked immunosorbent assay; Fc crystallizable fragment; Ig(G) immunoglobulin (G); MSD Meso Scale Discovery; N nucleocapsid; RBD receptor binding domain; RNA ribonucleic acid; S spike; SARS CoV 2 severe acute respiratory syndrome coronavirus 2; VNA virus neutralization assay.

In areas where seroprevalence is predicted to be high, a screening serologic test for past or current infection with SARS-CoV-2 may be performed (in a local laboratory), at the discretion of the sponsor, to restrict the proportion of seropositive participants in the study. This does not apply to the open-label phase of the study.

A serologic test for past or current infection with SARS-CoV-2 may be performed for all participants at Day 1 (pre-vaccination), Day 29, Day 71, Month 6/Unblinding Visit, Year 1/Booster Visit (prior to vaccination, if applicable), Year 1 + 28 days for participants who received booster vaccination, Year 1 + 72 days for participants who received booster vaccination, and Month 18
(24 weeks after Year 1 Visit). Samples for the serologic tests will be sent to a central laboratory for testing.<sup>a</sup> Participants who test positive will be informed of the result by the study staff.

# 8.2. Safety Assessments

Details regarding the DSMB are provided in Section 9.8 and in Appendix 3.

Adverse events will be reported and followed by the investigator as specified in Section 8.3 and Appendix 4.

Any clinically relevant changes occurring during the study must be recorded on the AE section of the eCRF.

Any clinically significant abnormalities persisting at the end of the study/early withdrawal will be followed by the investigator until resolution or until a clinically stable condition is reached.

The study will include the following evaluations of safety and reactogenicity according to the timepoints provided in the Schedules of Activities.

As of Amendment 7, active follow-up of new suspected COVID-19 episodes will be replaced by a passive follow-up approach.

The PSRT and the Janssen Medical Safety Council will monitor safety in a blinded manner in the double-blind phase (see Section 6.11) as well as in the open-label phase.

# 8.2.1. Physical Examinations (Until Amendment 7)

Height and body weight will be assessed at screening. To obtain the actual body weight, participants must be weighed lightly clothed. The height should be measured without footwear.

A targeted physical examination will be performed during a COVID-19 episode by the investigator or designated medically trained clinician (or a trained HCP, if allowed per local regulations). Any clinically relevant abnormalities or changes in severity observed during the review of body systems should be documented in the eCRF.

# 8.2.2. Vital Signs

At all on-site visits, body temperature (oral route preferred, or in accordance with the local standard of care) will be assessed.

<sup>&</sup>lt;sup>a</sup> Vaccination with Ad26.COV2.S may interfere with some serologic assays utilized at local community health clinics/commercial laboratories, by seeking and identifying the spike protein in the vaccine and rendering a false positive result. For this reason, participants will be encouraged to not seek testing outside the study. If a participant requires testing outside of the protocol-mandated testing schedule, the site will guide them on the appropriate assay that identifies the viral nucleocapsid protein (and not the spike protein).

Participants in the Safety Subset (double-blind phase) will utilize an e-Diary to record body temperature measurements from the time of vaccination until 7 days post-vaccination in the eCOA (see Section 8).

Up to Amendment 7, all participants with COVID-19 signs and symptoms should measure body temperature daily (oral route preferred, or in accordance with the local standard of care) and record the highest temperature in the last 24 hours each day in the ePRO in the eCOA, for the duration of follow-up of COVID-19 episodes (as defined in Section 8.1.2).

Up to Amendment 7, vital signs will be measured during a COVID-19 episode by a qualified member of the study site. This includes measurement of preferably supine systolic and diastolic blood pressure, heart rate, respiratory rate, oxygen saturation, and body temperature. It is recommended that vital signs are measured before collection of nasal swabs and blood draws.

Blood pressure and pulse/heart rate measurements will be assessed in a supine position (preferably) with a completely automated device. Manual techniques will only be used if an automated device is not available.

Blood pressure and pulse/heart rate measurements should be performed before blood draws and preceded by at least 5 minutes of rest in a quiet setting without distractions (eg, television, cell phones).

Under special circumstances such as high altitude, the investigator should assess baseline respiratory rate and other vital signs, as appropriate.

Any vital signs measurements taken at home that may trigger the severe/critical case definition will be confirmed as soon as possible by qualified medical staff and participants will be referred for care, if needed.

### 8.2.3. Pregnancy Testing

A urine pregnancy test for participants of childbearing potential will be performed at screening, before double-blind vaccination, before open-label vaccination, and before the booster vaccination. Participants of childbearing potential who originally received placebo and will not be receiving the Ad26.COV2.S vaccine under EUA do not need to complete a pregnancy test.

Additional serum or urine pregnancy tests may be performed for participants of childbearing potential, as determined necessary by the investigator or required by local regulation, to establish the absence of pregnancy at any time during the participation in the study.

# 8.2.4. Clinical Laboratory Assessments

Blood samples for clinical laboratory assessments (as detailed in Section 10.2, Appendix 2) will be collected as described in the Schedules of Activities in Section 1.3.

In case of a thrombotic event or TTS, every effort should be made to collect local hospital/laboratory test results obtained by the treating physician to allow rapid diagnosis and

treatment. This information should be reported through the TTS AESI form (see Section 10.13, Appendix 13) electronically per instructions in the eCRF completion guidelines. In addition, every effort should be made to collect blood samples from the participant for a platelet count (local laboratory or substitute for local laboratory) and other applicable testing (central laboratory) (see the Schedule of Activities in Section 1.3.5 and Section 10.2, Appendix 2). The Investigator will review the laboratory test results to assist the investigation of the AESI.

See Section 8.3.7.1 for details on laboratory test details to be reported for an AE of thrombocytopenia.

# 8.3. Adverse Events, Serious Adverse Events, Medically-attended Adverse Events, Adverse Events of Special Interest, and Other Safety Reporting

Timely, accurate, and complete reporting and analysis of safety information, including AEs, SAEs, suspected AESIs, MAAEs, and product quality complaints (PQCs), from clinical studies are crucial for the protection of participants, investigators, and the sponsor, and are mandated by regulatory agencies worldwide. The sponsor has established Standard Operating Procedures in conformity with regulatory requirements worldwide to ensure appropriate reporting of safety information; all clinical studies conducted by the sponsor or its affiliates will be conducted in accordance with those procedures.

AEs will be reported by the participant (or, when appropriate, by a caregiver or surrogate) during the reporting periods detailed below.

Further details on AEs, SAEs, suspected AESIs, MAAEs, and PQCs can be found in Appendix 4.

# 8.3.1. Time Period and Frequency for Collecting Adverse Event, Medicallyattended Adverse Event, Adverse Events of Special Interest, and Serious Adverse Event Information

#### **All Adverse Events**

For all participants (throughout the study regardless of any protocol amendment)<sup>a</sup>:

- (S)AEs that are related to study procedures or that are related to non-investigational sponsor products will be reported from the time a signed and dated ICF is obtained until the end of the study/early withdrawal.
- Clinically relevant medical events not meeting the above criteria and occurring between signing of the ICF and moment of vaccination in the double-blind phase of the study will be collected on the Medical History eCRF page as pre-existing conditions. This does not apply to the open-label phase.

\_

<sup>&</sup>lt;sup>a</sup> 90% of the participants who received a booster vaccination will be monitored for safety until 1 year post booster vaccination. The remaining 10% of the active participants who receive a booster vaccination will be monitored for safety at least for 6 months

- All SAEs and all AEs leading to study discontinuation (regardless of the causal relationship)
  are to be reported from the moment of vaccination until completion of the participant's last
  study-related procedure, which may include contact for safety follow-up. The sponsor will
  evaluate any safety information that is spontaneously reported by an investigator beyond the
  time frame specified in the protocol.
- MAAEs are defined as AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. Routine study visits will not be considered medically-attended visits. New onset of chronic diseases will be collected as part of the MAAEs. MAAEs are to be reported for all participants from the moment of each vaccination until 6 months after the vaccination (applicable for both the double-blind and open-label phases of the study), except for MAAEs leading to study discontinuation which are to be reported during the entire study.
- Special reporting situations, whether serious or non-serious, will be recorded from the time of each vaccination until 28 days post-vaccination (applicable for both the double-blind and open-label phases of the study).
- All AEs will be followed until resolution or until clinically stable.

### As of Amendment 7, for all participants:

- A passive follow-up approach is adopted, defined as follow-up by the site at Month 18 and Month 24 to document new COVID-19 participant-reported episodes as SAEs, AEs, or MAAEs. Participants may contact the site at any time in between scheduled visits to report COVID-19 episodes.
- Concomitant medications for these events should be reported.
- If a COVID-19 confirmatory laboratory or assay read-out is available, this should be reported in the eCRF (self-reported or as part of CIOMS form).
- Participants may contact the site at any time in between scheduled visits to report COVID-19 episodes.
- Events ongoing at time of informed consent do not need to be reported as AEs, SAE, or MAAEs, only new onset of COVID-19 events need to be reported.
- 90% of the participants who received a booster vaccination will be monitored for safety until 1 year post booster vaccination. The remaining 10% of the active participants who receive a booster vaccination will be monitored for safety at least for 6 months.

For participants in the Safety Subset (double-blind phase):

- Solicited AEs, collected through an e-Diary, will be recorded from the time of vaccination until 7 days post-vaccination.
- All other unsolicited AEs, whether serious or non-serious, will be recorded from the time of vaccination until 28 days post-vaccination.

Up to Amendment 7: For all participants who received booster vaccination at the Year 1/Booster Visit:

• Solicited AEs, collected through an e-Diary, will be recorded from the time of vaccination until 7 days post-vaccination. All participants will collect signs and symptoms in the e-Diary, if feasible. For a subset of participants, ie, participants included in the Safety Subset of the double-blind study phase and all participants who received a heterologous COVID-19 vaccination outside the study, the e-Diary will be reviewed by the study personnel and solicited AEs recorded in the eCRF, if feasible. All other unsolicited AEs, whether serious or non-serious, will be recorded from the time of vaccination until 28 days post-vaccination for all participants who received the booster at Year 1/Booster Visit.

As of Amendment 7, solicited and unsolicited AE reporting will stop for all participants.

#### **Adverse Events of Special Interest**

Suspected AESIs (thrombotic events and thrombocytopenia [defined as platelet count below  $150,000/\mu L^9$ ]) will be recorded from the moment of vaccination until the end of the study/early withdrawal (see Section 8.3.7). An AESI Adjudication Committee with appropriate expertise will be established to evaluate each suspected AESI and determine whether it is a case of TTS. From the time of local approval of protocol Amendment 5 onwards, TTS is considered an AESI.

#### **Serious Adverse Events**

All SAEs, as well as PQCs, occurring during the study must be reported to the appropriate sponsor contact person by study-site personnel within 24 hours of their knowledge of the event.

SAEs, including those spontaneously reported to the investigator before the end of the study, must be reported using an SAE form. The sponsor will evaluate any safety information that is spontaneously reported by an investigator beyond the time frame specified in the protocol.

Up to Amendment 7, participants will be reminded once a month to contact the study site in case of an SAE. As from Protocol Amendment 7, this is replaced by the passive follow-up approach.

All study participants will be monitored for SAEs for up to 2 years after their double-blind vaccination.

Information regarding SAEs will be transmitted to the sponsor using the SAE Form and Safety Report Form of the eCRF, which must be completed and reviewed by a physician from the study site and transmitted to the sponsor within 24 hours. The initial and follow-up reports of an SAE should be transmitted electronically or by facsimile (fax). Telephone reporting should be the exception and the reporter should be asked to complete the appropriate form(s) first.

### Overview of Safety Reporting in the Main Study



- (a) Refer to Section 10.4.4; eg, this includes AEs related to study procedures which are procedures related to interventions (eg, blood drawn for immunogenicity sampling) that may result in an AE (eg, bruise).
- (b) Adverse events of special interest (AESIs that require reporting to the sponsor within 24 hours).

# 8.3.2. Method of Detecting Adverse Events, Medically-attended Adverse Events, Adverse Events of Special Interest, and Serious Adverse Events

Care will be taken not to introduce bias when detecting AEs, MAAEs, suspected AESIs, or SAEs. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about AE occurrence.

# **Solicited Adverse Events (Applicable for Double-blind phase only)**

Solicited AEs are used to assess the reactogenicity of the study vaccine and are predefined local (at injection site) and systemic events for which the participant is specifically questioned, and which are noted by participants in their e-Diary.

The first 2,000 participants in each of the 2 age groups will remain under observation at the study site for at least 30 minutes post-vaccination to monitor for the development of acute reactions. If at the time of the Day 3 safety review of the initial 2,000 participants no acute reactions have been observed in the age groups, the observation period at the study site may be reduced to at least 15 minutes post-vaccination for the remaining participants in the study.

In addition, participants in the Safety Subset (double-blind phase) will record solicited signs and symptoms in an e-Diary from time of double-blind vaccination until 7 days post-vaccination. Participants in the Safety Subset will be provided with an e-Diary and instructions on how to complete the diary (see Overview in Section 8). Electronic diary information will be transferred

from the e-Diary source to the sponsor. After review and verbal discussion of the initial e-Diary entries with the participant, the investigator will complete his/her own assessment in the relevant sections of the eCRF/eCOA. Once a solicited sign or symptom from an e-Diary is considered to be of severity Grade 1 or above, it will be recorded as a solicited AE.

#### Solicited Injection Site (Local) Adverse Events

Participants will be asked to note in the e-Diary occurrences of injection site pain/tenderness, erythema, and swelling at the study vaccine injection site daily for 7 days post-vaccination (day of vaccination and the subsequent 7 days). The extent (largest diameter) of any erythema and swelling should be measured (using the ruler supplied) and recorded daily. The case definitions for solicited injection site events can be found in the references.<sup>37,47</sup>

### Solicited Systemic Adverse Events

Participants will be instructed on how to record daily temperature using a thermometer provided for home use. Participants should record the temperature in the e-Diary in the evening of the day of vaccination, and then daily for the next 7 days approximately at the same time each day. If more than 1 measurement is made on any given day, the highest temperature of that day will be recorded in the e-Diary.

Fever is defined as endogenous elevation of body temperature  $\ge 38.0^{\circ}$ C or  $\ge 100.4^{\circ}$ F, as recorded in at least 1 measurement.<sup>51</sup>

Participants will also be instructed on how to note signs and symptoms in the e-Diary on a daily basis for 7 days post-vaccination (day of vaccination and the subsequent 7 days), for the following events: fatigue, headache, nausea, myalgia.

#### **Unsolicited Adverse Events (Applicable for Double-blind phase only)**

Unsolicited AEs are all AEs for which the participant is not specifically questioned.

#### **Medically-attended Adverse Events**

MAAEs are AEs with medically-attended visits including hospital, emergency room, urgent care clinic, or other visits to or from medical personnel for any reason. New onset of chronic diseases will be collected as part of the MAAEs. Routine study visits will not be considered medically-attended visits.

For details about AESIs, refer to Section 8.3.7.

# 8.3.3. Follow-up of Adverse Events, Medically-attended Adverse Events, Adverse Events of Special Interest, and Serious Adverse Events

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and evaluations as medically indicated to elucidate the nature and causality of the AE, suspected AESI, MAAE, SAE, or PQC as fully as possible. This may include laboratory tests or investigations, histopathological examinations, or consultation with other HCPs.

AEs, including pregnancy, will be followed by the investigator as specified in Appendix 4.

# 8.3.4. Regulatory Reporting Requirements for Serious Adverse Events

The sponsor assumes responsibility for appropriate reporting of AEs to the regulatory authorities. The sponsor will also report to the investigator (and the head of the investigational institute where required) all suspected unexpected serious adverse reactions (SUSARs). The investigator (or sponsor where required) must report SUSARs to the appropriate IEC/IRB that approved the protocol unless otherwise required and documented by the IEC/IRB. A SUSAR will be reported to regulatory authorities unblinded. Participating investigators and IEC/IRB will receive a blinded SUSAR summary, unless otherwise specified.

# 8.3.5. Pregnancy

All initial reports of pregnancy in participants or partners of male participants must be reported to the sponsor by the study-site personnel within 24 hours of their knowledge of the event using the appropriate pregnancy notification form. Abnormal pregnancy outcomes (eg, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs and must be reported using an SAE reporting form. Any participant who becomes pregnant during the study will remain in the study and will continue to undergo all procedures for surveillance and follow-up of COVID-19 and all safety follow-up as outlined in the protocol for all participants. Participants who are pregnant and received placebo during the double-blind phase may be vaccinated with Ad26.COV2.S if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (See Section 6.4). Participants who are pregnant may receive booster vaccination with Ad26.COV2.S if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus (See Section 6.5).

Follow-up information regarding the outcome of the pregnancy and any postnatal sequelae in the infant will be required.

# 8.3.6. Disease-related Events and Disease-related Outcomes Not Qualifying as Adverse Events or Serious Adverse Events

(S)AEs caused by molecularly confirmed SARS-CoV-2 infection will be removed at the analysis level from the (S)AE listings and tables and presented separately.

All events that meet the definition of an SAE will be reported as SAEs, regardless of whether they are protocol-specific assessments.

#### 8.3.7. Adverse Events of Special Interest

Adverse events of special interest are significant AEs that are judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Adverse events of special interest will be carefully monitored during the study by the sponsor.

Adverse events of special interest must be reported to the sponsor within 24 hours of awareness irrespective of seriousness (ie, serious and non-serious AEs) or causality following the procedure described above for SAEs.

Specific requirements for the AESI are described below.

#### 8.3.7.1. Thrombosis with Thrombocytopenia Syndrome

As described in Section 2.3.1, Risks Related to Study Participation, TTS has been observed very rarely following vaccination with Ad26.COV2.S and is considered an AESI in this study. TTS is a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia.<sup>2,9</sup>

Because this syndrome is rare and not completely understood, all cases of thrombosis and/or thrombocytopenia will be considered a suspected case of TTS until further adjudication can be performed. An AESI Adjudication Committee with appropriate expertise will be established to evaluate each suspected AESI and determine whether it is a case of TTS. The investigator shall be responsible for reporting any suspected AESI of TTS using the SAE form and the form detailed in Section 10.13, Appendix 13. A suspected TTS case is defined as:

Thrombotic events: suspected deep vessel venous or arterial thrombotic events as detailed in Section 10.14, Appendix 14

Thrombocytopenia, defined as platelet count below  $150,000/\mu L^9$  as per the Brighton Collaboration.

Symptoms, signs, or conditions suggestive of a thrombotic event should be recorded and reported as a suspected AESI even if the final or definitive diagnosis has not yet been determined, and alternative diagnoses have not yet been eliminated or shown to be less likely. Follow-up information and final diagnoses, if applicable, should be submitted to the sponsor as soon as they become available.

In the event of thrombocytopenia, study site personnel should report the absolute value for the platelet count and the reference range for the laboratory test used.

For either a thrombotic event or thrombocytopenia, testing for anti-PF4 should be performed at the local laboratory or substitute local laboratory; repeat testing may be requested for confirmation upon sponsor discretion.

Suspected AESIs will require enhanced data collection and evaluation (see Section 1.3.5). Every effort should be made to report as much information as possible about the AESI to the sponsor in a reasonable timeframe.

If an event meets the criteria for an SAE (Section 10.4.1), it should be reported using the same process as for other SAEs.

The form detailed in Section 10.13, Appendix 13 is intended as a guide for assessment of the AESIs to facilitate diagnosis and determine treatment options. If the investigator is not the treating

physician, every effort should be made to collect the information requested in the form from the treating physician and enter the available information in the eCRF.

The sponsor will also attempt to collect information from any thrombotic event /thrombocytopenia/ TTS reported prior to protocol Amendment 5.

#### 8.4. Virology Assessments

Nasal swabs will be used to detect and/or quantify SARS-CoV-2. Exploratory quantification of the SARS-CoV-2 viral load in saliva samples may also be performed.

Gene sequencing may be performed to detect changes in the S gene and potentially also other parts of the viral genome, if a sample is available.

Up to Amendment 7, nasal swabs collected during a confirmed COVID-19 episode may also be tested at a central laboratory for the presence of other respiratory pathogens using a broad respiratory pathogens panel.

All confirmed COVID-19 episodes will be communicated to the respective participant and to other authorities according to local regulations.

Participants, with stable/well-controlled HIV infection, will be encouraged to have HIV RNA viral load and CD4 cell count assessed at least twice a year and to provide these data for inclusion in the eCRF.

#### 8.5. Biomarkers

Up to Amendment 7, during a COVID-19-episode, blood will be collected on COVID-19 Day 3-5 and on COVID-19 Day 29 for evaluation of biomarkers (eg, those associated with severe COVID-19).

#### 8.6. Medical Resource Utilization

As of Amendment 7, this is no longer applicable.

Medical resource utilization data over the last 3 months, associated with medical encounters, will be collected by interview with the participant and recorded in the eCRF by the investigator and study-site personnel at baseline (for all participants, concerning MRU within the last 3 months before double-blind vaccination), and on COVID-19 Day 3-5 and COVID-19 Day 29 (for all participants during a COVID-19 episode; which is defined to be resolved after having 2 consecutive SARS-CoV-2 negative nasal swabs and 2 consecutive days with no COVID-19-related signs or symptoms; see Section 8.1.2]) (Appendix 7). Medical resource utilization data will also be collected through the MA-COV form (Appendix 8). This form will be provided to the participant at the double-blind vaccination visit and should be completed by the medical care provider or the study site personnel during medical visits for COVID-19 or COVID-19 complications. Protocol-mandated procedures, tests, and encounters are excluded. The data collected may be used to conduct exploratory economic analyses and will include:

- Number and duration of medical care encounters, including selected procedures (inpatient and outpatient)
- Duration and type of mechanical ventilation and ECMO use
- Duration of hospitalization (total days length of stay, including duration by wards; eg, ICU)
- Number and character of diagnostic and therapeutic tests and procedures
- Outpatient medical encounters and treatments (including physician or emergency room visits, tests and procedures, and medications)

#### 8.7. Risk Factor Assessment

As of Amendment 7, this is no longer applicable.

If allowed by local regulations and if the participant consents, he/she will be interviewed on characteristics related to his/her current work situation, living situation, and community interactions (See Appendix 12) prior to double-blind vaccination on Day 1 and, at other timepoints, on changes compared to Day 1. These characteristics can potentially be useful to identify the risk of individual participants in acquiring COVID-19 and will be used in several analyses including the correlate analysis.

Risk factor data initially collected from participants at screening prior to implementation of protocol Amendment 3 will also be used for the planned risk-factor analysis.

# 8.8. Participant Medical Information Prior to, During and After the Study (Realworld Data)

For consenting participants in the US, medical data from 5 years prior to study enrollment until 5 years after study completion, such as electronic health records, claims and laboratory data from other care settings may be accessed utilizing tokenization and matching procedures. These data, together with data collected as part of the study as specified in the Schedules of Activities, may be used to conduct exploratory analyses to enhance our understanding of the impact of prior medical history on the response to immunization and the impact of immunization on efficacy and duration of efficacy as well as adverse events that may occur during and after completion of the study (see Section 9.5.4). The utilization of tokenization and matching procedures allows for the medical data to be obtained without violation of participant confidentiality (Section 4.2 and 4.2.1). The real-world medical data, which are not collected as part of the study, will not be part of the clinical study database.

# 8.9. Assessment and Procedures After EUA or Approval/Licensure and Implementation of Protocol Amendment 4

Following EUA, conditional licensure, or approval in any country for a single dose regimen based on the VAC31518COV3001 study interim results, all participants from countries where Amendment 4 is approved by the local Health Authority and IEC/IRB will be unblinded at the onsite Month 6/Unblinding Visit. The study will then be conducted in an open-label fashion. A final analysis of the double-blind phase will be performed, using the data collected prior to unblinding,

when all participants have completed the Month 6/Unblinding Visit or discontinued earlier. Depending on the operational implementation of the Month 6/Unblinding Visit, as well as the stage of the pandemic, this analysis may be conducted when a minimum of 90% of the study population has been unblinded.

Participants in the Ad26.COV2.S group will be assured they received at a minimum the dose level that was submitted for EUA approval (single-dose regimen of  $5x10^{10}$  vp Ad26.COV2.S) and will be asked to continue to be followed in this study in line with the Schedules of Activities.

A Month 6/Unblinding Visit will take place for all participants. A nasal swab and blood sample for serology will be collected from all participants. In addition, body temperature and urine pregnancy test (for participants of childbearing potential) will be collected from participants who will be vaccinated at this visit. Participants from placebo group will be offered to receive 1 dose of Ad26.COV2.S vaccine under the conditions delineated in Section 6.4. After vaccination, participants should remain under observation at the study site for at least 15 minutes for the presence of any acute reactions after vaccination and will be followed for SAEs until 1 year after Ad26.COV2.S administration.

The importance to continue practicing other public health or preventative measures that were introduced at the start of this pandemic (eg, social distancing, face masks, frequent hand washing), in compliance with local and national guidelines, will be emphasized.

# 8.10. Assessment and Procedures Related to Booster Vaccination

#### **As of Protocol Amendment 7:**

No further booster doses will be administered after implementation of Protocol Amendment 7, except if there is a medical reason that prevented a participant to receive the Ad26COV2.S vaccine prior to acceptance of amendment 7 or if there is a non-availability of other vaccines to the participant. The investigator should inform participants on the availability of other COVID-19 vaccines.

#### **Up to Protocol Amendment 7:**

The Year 1/Booster Visit will take place for all ongoing participants. Participants who have previously received any COVID-19 vaccination(s) (as primary regimen or additional dose) with the Ad26.COV2.S vaccine, and/or an mRNA vaccine or another COVID-19 vaccine authorized for primary vaccination including protein, inactivated, and adenovector based vaccines will be offered to receive a 1-dose booster vaccination with Ad26.COV2.S at the 5x10<sup>10</sup> vp dose level. Participants who choose not to receive booster vaccination at this time will be informed that they can still choose to receive the booster vaccination at a later date within the visit window. In addition, body temperature and urine pregnancy test (for participants of childbearing potential) will be collected from participants who will be vaccinated at this visit. After vaccination, participants should remain under observation at the study site for at least 15 minutes for the presence of any acute reactions after vaccination and will be followed for SAEs until 1 year after Ad26.COV2.S administration.

Participants who choose to receive a booster vaccination outside of the study are encouraged to schedule their Year 1/Booster Visit prior to their booster vaccination, if feasible, and come in for the Year 1 + 28 Days and Year 1 + 72 Days visits within the specified visit window, if feasible, or as close as possible to the visit window.

During the Year 1/Booster Vaccination visit, the investigator should ask the participant if he/she received any other COVID-19 vaccines and record type and date of administration.

The importance to continue practicing other public health or preventative measures that were introduced at the start of this pandemic (eg, social distancing, face masks, frequent hand washing), in compliance with local and national guidelines, will be emphasized.

#### 9. STATISTICAL CONSIDERATIONS

Statistical analysis will be done by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be used to analyze the efficacy and safety data is outlined below. Specific details will be provided in the SAP.

Sections 9.1 to 9.7 are applicable to the double-blind phase of the study. Considerations for the analysis of the open-label booster vaccination phase (introduced with Amendment 6) of the study are described in Section 9.8; details will be provided in a separate SAP.

### 9.1. Statistical Hypotheses

Refer to Section 3 for the statistical hypotheses.

The study will have the following timepoints for analysis:

- 1. The evaluation of the primary objective will be performed as soon as the target number of events (TNE) has been reached in the double-blind phase for both co-primary endpoints, or earlier based on sequential monitoring of both co-primary endpoints (details in Section 9.5.1). Sponsor unblinding will occur but investigator and participants remain blinded until implementation of Amendment 4 (see Section 6.4).
- 2. If an efficacy signal is triggered before the required 8-week follow-up after double-blind vaccination of 50% of participants is reached, an additional analysis will be performed when that follow-up timepoint is reached (8-week median follow-up timepoint). If the time between the efficacy signal and the required 8-week median follow-up is too short to make a difference in terms of preparing two analyses, then a single analysis will take place at the time of the 8-week median follow-up. The analysis at the time of the 8-week median follow-up is considered the primary analysis.
- 3. After the primary analysis, additional analyses to support health authority interactions will be planned, as deemed appropriate.
- 4. A final analysis of the double-blind phase of the study, including all double-blind data, will be performed when all participants have completed the Month 6/Unblinding Visit or

discontinued earlier. Depending on the operational implementation of the Month 6/Unblinding Visit, as well as the stage of the pandemic, this analysis may be conducted when a minimum of 90% of the study population has been unblinded.

During the open-label phase 2 possible analysis timepoints will be foreseen:

- 5. The open-label cross-over and booster analysis (active follow-up) can be triggered when a minimum of 90% of participants consented to Amendment 7. The timing of this analysis may be once all study sites have approved Amendment 7 or later.
- 6. An end-of-study analysis is planned 1 year after a minimum of 90% of the enrolled study population have reached the Year 1/Booster Visit or discontinued earlier (31 March 2023) and will be conducted upon completion of the last participant visit. Depending on the timing of approval of Amendment 7 across study sites, the 2 analysis timepoints may be combined. At the end-of-study analysis, 90% of participants will have completed one year safety follow-up; the remaining 10% of participants will have at least 6 months of safety follow-up.

Additional analyses may be conducted to support health authority interactions and/or based on public health demand in case of emerging variants.

# 9.2. Sample Size Determination

### 9.2.1. Efficacy (Total Sample Size)

The study TNE is determined using the following assumptions:

- a VE for molecularly confirmed, moderate to severe/critical SARS-CoV-2 infection of 60%.
- approximately 90% power to reject a null hypothesis of H0: VE < 30%.
- type 1 error rate α 2.5% to evaluate VE of the vaccine regimen (employing the sequential probability ratio test [SPRT] to perform a fully sequential design analysis; detailed in Section 9.5.1).
- a randomization ratio of 1:1 for active versus placebo

Events are defined as first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to the case definition in Section 8.1.3.1 in the PP population. The two co-primary endpoints will evaluate the events at least 14 days after double-blind vaccination (Day 15) and at least 28 days after double-blind vaccination (Day 29) with study vaccine.

Under the assumptions above, the TNE to compare the active vaccine versus placebo equals 154, based on events in the active vaccination and placebo group, according to the primary endpoints case definition of moderate to severe/critical COVID-19 (Section 8.1.3.1).

If the co-primary hypothesis testing is successful for both co-primary endpoints, secondary objectives will be evaluated against a null hypothesis employing a lower limit VE>0%. The

method to perform hypothesis testing of primary and secondary objectives preserving the FWER will be specified in the SAP. The FWER will be controlled at 2.5%.

### **Sample Size Justification**

Based on epidemiological modeling for the targeted study countries, province/states of the various site locations, the annualized incidence of moderate to severe/critical COVID-19 cases meeting the primary endpoints definitions has been predicted to be 1.4% for the October-November timeframe. The estimate incorporates that real-world-evidence data and literature data only detected and reported a fraction of SARS-CoV-2 infections.

Furthermore, it includes that, based on literature and real-world-evidence data, only a fraction of all infections meets the moderate and severe/critical COVID-19 case definition and the fraction varies by age as well (increasing with higher ages). Moreover, projections for the selected study regions indicate that incidences will decline over time. Finally, seroprevalence rates are expected to vary between 5-15%.

For the purpose of sample size evaluation, an incidence assumption of moderate to severe/critical COVID-19 cases meeting the primary endpoints definition of 1.4% during the first 3 months of the study, with a 50% reduction in Month 4, and 62% reduction in the months thereafter is assumed in combination with a seroprevalence rate of 10%.

At the time of protocol planning, the epidemiological situation was uncertain: actual seroprevalence rates, degree of social distancing and use of personal protective equipment during the study, local regulations (eg, potential lockdowns, other vaccines if available) potentially becoming in effect during the course of the study and potential drop-outs from the study could impact the disease incidence rate.

To that end, the maximum sample size of approximately 60,000 participants was selected. This sample size was selected, based on the uncertainty of the epidemiological situation in combination with the ability to provide a high probability (approximately 90%) to reach a time to signal within 8 months of the study for a vaccine with an assumed 60% VE.

Based on an estimated case-hospitalization ratio of 2.5% and estimates obtained from reported real-world-evidence data of 3-10% of all SARS-CoV-2 infections meeting the severe/critical COVID-19 definition, this would provide a reasonable likelihood of observing 5 severe cases in the placebo group within the same time frame (8 months).

At the time of writing protocol Amendment 3, the incidence of moderate to severe COVID-19 seen in the US and reported in other COVID-19 vaccine studies is significantly higher than assumed at the time of protocol planning as described above. Furthermore, based on that incidence and modeling there is a high degree of probability that an efficacy signal meeting the prespecified criteria in this amendment will be reached at, or prior to, the time when approximately 40,000 participants will have been followed for a median of 8 weeks from the time of vaccination. Therefore, the sample size is reduced from 60,000 to approximately 40,000.

The operating characteristics of the study design, statistical methods, study monitoring rules and efficacy evaluations specified in this protocol with the chosen event and sample sizes will be described in a separate modeling and simulation report and will be added to the SAP before the first participant is vaccinated.

No additional participants will be recruited for the open-label phase.

# 9.2.2. Immunogenicity Subset (Double-blind Phase)

All participants included in the Immunogenicity Subset (N 400) will be added randomly at each stage of the enrollment. Healthy adults (Subset 1a) will be enrolled in Stage 1a, adults with comorbidities (Subset 1b) in Stage 1b, healthy elderly (Subset 2a) in Stage 2a, and elderly with comorbidities (Subset 2b) in Stage 2b, with approximately 100 participants per group as displayed in Table 3. Although Stage 1b and 2b will also enroll participants without comorbidities, only participants with comorbidities will be included in Immunogenicity Subset 1b and Subset 2b.

A sample size of 400 participants, distributed as described in Table 3, is estimated to be sufficient to allow robust description of immune responses to Ad26.COV2.S vaccine. These numbers are expected to provide a solid understanding of the magnitude and kinetics of the humoral response induced by the Ad26.COV2.S vaccine.

# 9.2.3. Immunogenicity Correlates (Correlates Subset)

Correlates will be assessed in a subset where immune responses and transcriptome modifications are measured in all vaccine recipients who experience a SARS-CoV-2 event, and in random samples of vaccine recipients who have not been infected, in a 1:5 ratio. The goal of this case control study is to assess correlates of risk of SARS-CoV-2 infection (and potential other secondary endpoints) in the vaccine group by comparing vaccine-induced immune responses and transcriptome modifications associated with COVID-19. Also, placebo participants will be included in this subset (placebo infected, seropositive [based on N protein] non-infected and seronegative non-infected), if feasible.

Correlates will also be investigated via a case-cohort design, including measurement of immunological markers in a random subcohort augmented by infected and symptomatic cases.

Controls will be matched with cases from the same stage (age, comorbidities) and other co-factors as deemed appropriate. These will be detailed in the Correlates SAP.

#### 9.2.4. Safety

### 9.2.4.1. Safety Subset

While mild to moderate reactogenicity (local injection site and systemic reactions) are expected, AEs that preclude further vaccine administration (if applicable) are not anticipated.

Unsolicited AEs will be captured for a period of 28 days after double-blind vaccination. Solicited and unsolicited AEs will be captured in the Safety Subset, ie, approximately 6,000 participants

( $\sim$ 3,000 from the active group,  $\sim$ 3,000 from the placebo group; and including at least 2,000 from the older age group [ $\geq$ 60 years of age] if feasible).

# 9.2.4.2. All Participants

Adverse events of special interest (from protocol Amendment 5 onwards) and SAEs will be captured in all participants and throughout the study. MAAEs (including new onset of chronic diseases) will be captured in all participants until 6 months after (double-blind or open-label) vaccination with Ad26.COV2.S, except for MAAEs leading to study discontinuation which are to be reported during the entire study. Based on a sample size of approximately 40,000 participants, and approximately 20,000 in the active vaccination group, for SAEs, the observation of 0 events in the database would be associated with 95% confidence that the true rate is less than 0.015%. Table 7 shows the probabilities of observing at least 1 event (solicited, unsolicited, or SAE) in 1 of the groups at given true AE rates.

Table 7: Probability of Observing at Least 1 Adverse Event or Serious Adverse Event at a Given True Adverse Event Rate in the Active Group (With a Total Sample Size of 40,000 Participants)

| _ | Probability of Observing at Least 1 Adverse Event in the Active Group in N Participants | |
|---|---|---|
| True AE<br>Rate | Solicited/Unsolicited AEs<br>N=3,000 | SAEs<br>N=20,000 |
| 0.01% | 26% | 86% |
| 0.1% | 95% | 100% |
| ≥0.5% | 100% | 100% |

AE adverse event; N number of participants receiving study vaccine (Ad26.COV2.S or placebo); SAE serious adverse events

As of Amendment 7, a passive follow-up approach is adopted: the investigator will place a phone call at Month 18 and Month 24 to collect information on any protocol-required safety assessment (see Section 8.3.1).

In addition, SAEs, AEs, and MAAEs related to COVID-19 need to be reported together with the concomitant medications related to these events until study end. Any confirmatory COVID-19 laboratory information should be reported in the eCRF. Note that 90% of the participants who receive a booster vaccination will be monitored for safety until 1 year post booster vaccination as mentioned in Section 8.3. The remaining 10% of the participants who receive a booster vaccination will be monitored for safety at least for 6 months.

# 9.3. Populations for Analysis Sets

For purposes of analysis, the following populations are defined:

**Full Analysis Set (FAS):** All randomized participants with a documented study vaccine administration, regardless of the occurrence of protocol deviations and serostatus at enrollment. Analyses of safety will be performed on the FAS. Vaccine efficacy analyses can be repeated using the FAS.

**Safety Subset**: subset of the FAS for the analysis of solicited and unsolicited AEs.

**Per-protocol Efficacy (PP) population:** Participants in the FAS who receive double-blind study vaccine and who are seronegative at the time of double-blind vaccination and who have no other major protocol deviations that were judged to possibly impact the efficacy of the vaccine. Participants who became aware of their study vaccine allocation will cease to be part of the PP population. The PA of VE will be based on the PP population. The PP will be the main analysis population for efficacy analyses.

**Per-protocol Immunogenicity (PPI) population:** All randomized and vaccinated participants, including those who are part of the Immunogenicity Subset and for whom immunogenicity data are available, excluding participants with major protocol deviations expected to impact the immunogenicity outcomes. In addition, for participants who experience a SARS-CoV-2 event (molecularly confirmed), samples taken after the event and samples taken outside protocol windows will not be taken into account in the assessment of the immunogenicity. The PPI population is the primary immunogenicity population. For key tables, sensitivity immunogenicity analyses will also be performed on the FAS, including participants who are part of the Immunogenicity Subset for whom immunogenicity measures are available. Excluded samples might be taken into account as well in the sensitivity analysis. Analyses of vaccine immunogenicity and immune correlates of risk will be based on PPI.

The populations for the open-label cross-over, booster and passive follow-up phase are described in the SAP.

The list of major protocol deviations to be excluded from the efficacy for the double-blind analysis and/or immunogenicity analyses will be specified in the SAP and/or this list will be reported into the protocol deviation dataset of the clinical database before database lock and unblinding.

#### 9.4. Participant Information

For all participants, descriptive statistics of demographic (eg, gender, age, height, weight, BMI, race, and other baseline characteristics) will be provided by vaccination group. Additional characteristics related to current work situation, living situation, and community interactions will be collected for risk factor analysis, if allowed per local regulations. Risk factor data initially collected from participants at screening prior to implementation of protocol Amendment 3 will also be used for the planned risk-factor analysis. See also Section 9.5.3.

#### 9.5. Efficacy Analyses

The SAP will be finalized prior to first participant in and it will include a more technical and detailed description of the statistical analyses described in this section. This section is a summary of the planned statistical analyses of the most important endpoints including primary and key secondary endpoints.

#### 9.5.1. Primary Endpoints Evaluation

The study is designed to test the co-primary hypotheses of VE in the PP population. For both co-primary endpoints the following hypothesis will be tested:

H0: VE  $\leq$ 30% versus H1: VE >30% and each hypothesis will be evaluated at a 2.5% one-sided significance level.

The co-primary endpoints will evaluate:

- the first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to the case definition in Section 8.1.3.1, with onset at least 14 days after double-blind vaccination (Day 15) with Ad26.COV2.S versus placebo, in the PP population, including all events from both age groups, with and without comorbidities.
- the first occurrence of molecularly confirmed, moderate to severe/critical COVID-19 according to the case definition in Section 8.1.3.1, with onset at least 28 days after double-blind vaccination (Day 29) with Ad26.COV2.S versus placebo, in the PP population, including all events from both age groups, with and without comorbidities.

Participants included in the seronegative analysis set are those participants with a negative SARS-CoV-2 serology test result at (double-blind) baseline.

Considering the current COVID-19 pandemic, early detection of VE will be very important. The proposed current analysis setup is designed for continuous sequential analyses (see Section 9.5.1.1), where statistical hypothesis testing is conducted repeatedly on accumulating data, generating an earliest possible signal if and when the splits between the number of events in placebo recipients are much larger compared to the Ad26.COV2.S-vaccinated group for both co-primary endpoints and in such a way that they are unlikely to be due to chance alone using a truncated SPRT. A successful primary efficacy conclusion will require:

- Establishing the hypothesis H1: VE>30% for each co-primary endpoint AND
- 2. A favorable split vaccine:placebo for the subset of primary endpoints meeting the severe/critical COVID-19 case definition (expressed as a VE point estimate against severe/critical COVID-19 molecularly confirmed endpoints ≥50%) and a minimum of 5 events in the placebo group. This requirement needs to be met for severe/critical events with onset at least 14 days after double-blind vaccination and for severe/critical events with onset at least 28 days after double-blind vaccination.

**AND** 

3. A VE of at least 50% for each co-primary endpoint.

To evaluate the primary null hypotheses: H0:  $VE \le 30\%$  versus H1: VE > 30% for the co-primary endpoints, the truncated sequential probability ratio test will be used based on accumulating event data for each co-primary endpoint. This boundary is set up using the fully sequential design and is derived in such a way to have approximately 90% power to detect a VE = 60% using a one-sided alpha 0.025 against H0: $VE \le 30\%$ . For the evaluation of the favorable ratio against the severe/critical COVID-19 endpoints a sequential boundary corresponding to a VE = 10% point estimate

≥50% and a minimum of 5 events in the placebo group will be prespecified. The specific boundaries will be detailed in the SAP.

The monitoring can start as soon as the following conditions are met:

- 1. A minimum of 6 COVID-19 cases for the ≥60 years age group with onset at least 28 days after double-blind vaccination
- 2. At least 42 cases meeting the primary endpoints definition of moderate to severe/critical COVID-19 with onset at least 28 days after double-blind vaccination
- 3. A subset of at least 5 cases meeting the primary endpoints definition of severe/critical COVID-19 with onset at least 28 days after double-blind vaccination

No interim evaluation will be done, until those conditions are fulfilled. Monitoring for efficacy will not start before the above conditions 1-3 are met and will occur at least once a week by the SSG of the DSMB until the prespecified boundaries have been crossed.

The efficacy analysis will be triggered by either:

1. a) An interim evaluation if all prespecified efficacy boundaries have been met OR if 154 cases meeting the primary endpoints definition of moderate to severe/critical COVID-19 are observed for events with onset at least 28 days after double-blind vaccination

**AND** 

b) The above 3 conditions are met.

OR, alternatively,

2. If the prespecified non-efficacy boundary has been met (evaluating events with start 28 days after double-blind vaccination) or when the harm boundary has been crossed. The decision rules for harm and non-efficacy are detailed in Section 9.5.1.1.

If an efficacy signal is triggered before the required 8-week follow-up after double-blind vaccination of 50% of participants is reached, an additional analysis will be performed when that follow-up timepoint is reached. If the time between the efficacy signal and the required 8-week median follow-up is too short to make a difference in terms of preparing two analyses, then a single analysis will take place at the time of the 8-week median follow-up. The analysis at the time of the 8-week median follow-up is considered the primary analysis.

If more than 154 primary endpoints are observed for events with onset at least 28 days after double-blind vaccination before the 3 conditions above are met, a single analysis will take place as soon as the conditions are met, using the full 2.5% one-sided significance level.

If the prespecified boundaries and above conditions are met, the SSG will inform the DSMB and, if deemed appropriate by the DSMB, a meeting with the DSMB and the Oversight Group will be set up to discuss the efficacy signal. Upon this meeting the sponsor representative on the Oversight Group can trigger internal decision procedures to initiate health authority interactions based on the

outcome of the study. However, the study sites and participants will remain blinded to allow for evaluation of durability of VE. Sponsor personnel will be unblinded at the time of the primary analysis. If an efficacy signal is triggered before the required 8-week follow-up after double-blind vaccination of 50% of participants is reached (defined as "snapshot analysis"), selected sponsor personnel will be unblinded at the time of the snapshot analysis.

A positive RT-PCR or other molecular diagnostic test result obtained from a central laboratory will be utilized to define a molecularly confirmed case of COVID-19. Sensitivity analysis comparing cases also including a positive RT-PCR test result from any source, including external to the study, will be performed for each diagnostic category individually (mild, moderate, severe, moderate+severe, and medical utilization [hospitalization, ICU care, mechanical ventilation, ECMO]).

The primary efficacy analysis will pool data across populations (both age groups with and without comorbidities) to evaluate the primary and secondary objectives. In addition, these will be supplemented with a subgroup analysis for age group (18 to <60 years,  $\geq$ 60 years) and comorbidities employing a descriptive summary including 95% confidence intervals to describe the VE in each subpopulation. Depending on the recruited study population, the  $\geq$ 60 years subgroup may be further subcategorized ( $\geq$ 70 years,  $\geq$ 80 years).

In addition, to assess potential time-effects of VE, the Kaplan-Meier method will be used to plot the estimated cumulative incidence rates over time for the vaccine and placebo groups. This method will be used to estimate cumulative VE over time, defined as [(1 minus ratio (vaccine/placebo) of cumulative incidence by time t) ×100%]. Divergence of vaccine and placebo curves may be utilized to estimate onset of efficacy following immunization.

Furthermore, VE will be evaluated in seronegative participants, counting primary endpoints since onset after double-blind vaccination.

At the time of unblinding, one additional analysis will be performed to assess the VE of Ad26.COV2.S vaccination versus placebo repeating analyses on all primary and secondary endpoints for the blinded portion of the study.

For the statistical analysis, individual data will be included up to the Month 6/Unblinding Visit for the double blind, placebo-controlled period. For the analysis of the open-label phase for an individual subject, data as of the Month 6/Unblinding Visit will be included in the analysis. For the evaluation of the durability of vaccine efficacy, the analyses of the open label part of the study will employ methods as described in Follmann (2020).<sup>34</sup> Details will be provided in the SAP.

### 9.5.1.1. Study Monitoring

**Table 8:** Specification of Sequential Statistical Analyses

| Parameter | Population | Hypothesis | Statistical Method | Criterion | Monitoring Plan |
|---|---|---|---|---|---|
| Potential Harm <sup>a</sup> of Symptomatic Cases | FAS | H <sub>0</sub> : VE ≥0%<br>vs.<br>H <sub>1</sub> : VE <0% | Exact 1 sided binomial test of the fraction of infections assigned to who receive the vaccine. | Constant p value cut off controlling α at 5% | After every event starting from the 12 <sup>th</sup> event <sup>b</sup> |
| Potential Harm <sup>a</sup> of Severe Cases | FAS | H <sub>0</sub> : VE ≥0%<br>vs.<br>H <sub>1</sub> : VE <0% | Exact 1 sided binomial test of the fraction of infections assigned to who receive the vaccine. | Unadjusted p value α at 5% | After every event starting from the 5 <sup>th</sup> event |
| Non efficacy | PP | H <sub>0</sub> : VE ≥40%<br>vs.<br>H <sub>1</sub> : VE <40% | Exact 95% CI | Upper limit of the 95%CI <40% | Every 2 weeks, starting<br>from the 20 <sup>th</sup> event after<br>14 days following double<br>blind vaccination<br>(Day 15) <sup>b</sup> |
| Efficacy | PP | H <sub>0</sub> : VE ≤50%<br>vs.<br>H <sub>1</sub> : VE >50% | Sequential probability ratio test | Controlling the family wise error rate α at 2.5% | Starting from the 42 <sup>nd</sup><br>event <sup>c</sup> 14 days following<br>double blind vaccination<br>(Day 15), <b>then at least</b><br><b>once a week</b> |
| Efficacy | PP | $\begin{array}{c} H_0 \hbox{: VE} \le & 30\% \\ vs. \\ H_1 \hbox{: VE} > & 30\% \end{array}$ | Sequential probability ratio test | Controlling the family wise error rate α at 2.5% | Starting from the 42 <sup>nd</sup><br>event <sup>c</sup> 28 days following<br>double blind vaccination<br>(Day 29), <b>then at least</b><br><b>once a week</b> |

CI confidence interval; FAS full analysis set; PP per protocol; VE vaccine efficacy.

All boundaries will be monitored by an SSG. Once a boundary has been crossed, the SSG will inform the DSMB and a DSMB meeting will be organized. The statistical details of the decision rules and the frequency of evaluation and operational implementation will be fully detailed in the SAP and DSMB Charter.

#### **Sequential Probability Ratio Test**

Following the notation of Dragalin et al. (2002) and Dragalin and Fedorov (2006),  $^{30,31}$  consider,  $X_1$  and  $X_2$  the number of events in respectively the placebo group and the vaccine group. The distribution of  $X_1$  and  $X_2$  can be approximated by a Poisson distribution with the following parameters:  $\lambda_i = n_i p_i$  (with i = 1,2). Thus, the conditional distribution of  $X_2$  given  $T = X_1 + X_2 = t$  approximately follows a binomial distribution with parameters  $(t,\pi)$ , where  $\pi = \frac{\lambda_2}{(\lambda_1 + \lambda_2)} = \frac{n_2 p_2}{n_1 p_1 + n_2 p_2} = \frac{1 - VE}{2 - VE}$ , with VE 1-RR,  $RR = \frac{p_2}{p_1}$ , assuming a vaccine group allocation ratio of 1:1. Consequently, testing the null hypothesis  $H0: VE = VE_0$  against  $H1: VE = VE^*$  is equivalent to testing  $H0: \pi = \pi_0$  against  $H1: \pi$   $\pi^*$  the conditional binomial test.

Consider  $\alpha = P(reject \ H0 | VE = VE0)$  and  $\beta = P(accept \ H0 | VE = VE^*)$ . Rejecting H0 occurs when  $X_2 <= C_\alpha$  with  $C_\alpha$  and  $C_\alpha$  calculated to preserve  $C_\alpha$  over all the sequential looks such that

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

<sup>&</sup>lt;sup>a</sup> Harm in the form of an increased rate of symptomatic COVID 19 events due to vaccination (which meet the mild, moderate or severe/critical case definition).

<sup>&</sup>lt;sup>b</sup> Monitoring stops when the primary efficacy analysis is triggered.

<sup>&</sup>lt;sup>c</sup> The monitoring can only start as soon as the conditions outlined in Section 9.5.1 are met.

 $P(X_2 \le C_\alpha | \pi = \pi_0) = B(C_\alpha; T, \pi_0) \le \alpha$ . With  $B(.; T, \pi)$  the cumulative binomial distribution function with parameter T and  $\pi$ . The solution to the above equation,  $T^*$ , is the smallest T such that  $B(B^{-1}(\alpha; T, \pi_0); T, \pi^*) \ge 1 - \beta$ , with  $B^{-1}(\alpha; T; \pi)$  the  $\alpha$ -quantile of the cumulative binomial distribution function with parameters T and  $\pi$ .

The implemented critical boundaries for success are based on the truncated SPRT for which success boundaries are set based on observing  $X_2$  events on the vertical axis out of total T events on the horizontal axis.

### 9.5.2. Secondary Endpoints

All secondary endpoint analyses will occur in the PP analysis set, in seronegative participants unless otherwise indicated.

To evaluate the effect of the vaccine against symptomatic molecularly confirmed COVID-19, including mild infections, a BOD endpoint will be evaluated based on the first occurrence of molecularly confirmed COVID-19, including mild, moderate and severe/critical case definitions in Sections 8.1.3.1 and 8.1.3.2, with onset at least 14 days after double-blind vaccination (Day 15) and with onset at least 28 days after double-blind vaccination (Day 29) with Ad26.COV2.S versus placebo, in the PP population, including all events across age groups, with and without comorbidities. In this study, the BOD endpoint is defined as taking the value 1 for mild and moderate disease and the value 2 for severe disease (implicitly assigning a value of 0 for no disease [not infected or asymptomatic infection]). By assigning higher weight to severe infections, the BOD endpoint aims at providing higher statistical power for differentiating from placebo vaccines with increased protection against severe infections (but potentially lower vaccine efficacy against milder infections). The BOD evaluates the severity-adjusted VE against preventing symptomatic incidence. The hypothesis to evaluate the vaccine efficacy against symptomatic infection will be based on this method. In addition, the VE against each severity category according to the case definition (severe, moderate, mild) will be summarized separately. Statistical significance for the BOD endpoint will be tested using H0:VE≤0 at a one-sided α 2.5% according to multiplicity adjusted strategy.

Details on the calculation of VE for the BOD endpoint and its associated confidence interval (for testing) and hypothesis testing will be foreseen in the SAP.

VE against severe/critical infections with onset at least 14 days after double-blind vaccination (Day 15) and with onset 28 days after double-blind vaccination will be evaluated. Exact Poisson regression will be used to estimate the VE and associated confidence interval in seronegative participants in the PP analysis set.

The co-primary endpoints and BOD endpoint will be evaluated at the time of efficacy signal, and again at the time when the 8-week median follow-up requirement is reached (should the efficacy signal occur earlier).

VE against any SARS-CoV-2 infection and against asymptomatic infections will be evaluated as soon as a sufficient number of participants have data available. This timepoint will be detailed in

the Statistical Analysis Plan and may occur at any of the planned analysis timepoints. Available N-serology measurements will be incorporated to evaluate VE against any infection, including asymptomatic infection and against asymptomatic/undetected infection only. A participant will be defined as having any infection whether he/she had either a symptomatic infection (mild, moderate or severe according to the case definition) or an asymptomatic infection (as defined in Section 8.1.3.4). Poisson regression will be used to estimate the VE and associated confidence interval in seronegative participants in the PP analysis set for each of both analyses.

Among participants with SARS-CoV-2 infection, the effect of the study vaccine on the viral load levels at and after diagnosis as well as on the duration of SARS-CoV-2 viral load positivity will be evaluated.

The effect of the vaccine will be evaluated against molecularly confirmed COVID-19 infections requiring medical intervention once sufficient events are available for events with onset at least 14 days after double-blind vaccination and with onset at least 28 days after double-blind vaccination. Medical interventions are evaluated as a composite endpoint of hospitalization, ICU admission, mechanical ventilation and ECMO, linked to objective measures such as decreased oxygenation, X-ray or CT findings. Exact Poisson regression will be used to estimate the VE and the associated confidence interval in seronegative participants in the PP analysis set.

All VE evaluations will be repeated regardless of their serostatus.

Supportive and/or descriptive analysis will be reported with 95% confidence intervals; confirmatory endpoints will have an adjusted confidence interval reported at the time of hypothesis testing whereby the alpha level is determined according to the FWER-controlled testing strategy.

The statistical analysis for secondary endpoints, multiple testing strategy to evaluate the secondary objectives, and the timing of the hypothesis testing will be detailed in the SAP.

See also Section 9.5.1.

### 9.5.3. Exploratory Endpoints

Exploratory endpoint analyses will be detailed in the SAP.

If appropriate, subgroup or covariate-adjusted analyses may be performed. These subgroups/covariates may include baseline demographics and other characteristics.

### 9.5.4. Other Analyses

#### **Biomarkers Analyses**

Exploratory biomarker analyses will be part of a separate report.

### Participant Medical Information Prior to, During and After the Study (Real-world Data)

The exploratory analyses that may be conducted using the real-world data will be detailed in a SAP and results may, partially, be reported separately from the VAC31518 Clinical Study Report(s).

#### **Medical Resource Utilization Analyses**

Medical resource utilization will be descriptively summarized by intervention group.

# 9.6. Immunogenicity Analyses

No formal statistical testing of the immunogenicity data is planned. All immunogenicity analyses will be performed on the PPI set. Key tables might be repeated for the FAS (including samples that are excluded from the PPI analysis).

# 9.6.1. Immunogenicity Subset

No formal hypothesis on immunogenicity will be tested. Descriptive statistics (eg, geometric mean and 95% confidence interval for the neutralization assay and ELISA) will be calculated for continuous immunologic parameters at all timepoints. Geometric mean fold rises from baseline and corresponding 95% confidence intervals might additionally be calculated. Baseline is considered as the last available assessment before double-blind vaccination. For participants, who received vaccination with Ad26.COV2.S at the Month 6/Unblinding Visit in the open-label phase after having received placebo initially, descriptive statistics of available data after vaccination will be provided. Graphical representations of immunologic parameters will be made as applicable.

The impact of baseline factors on the humoral responses will be explored graphically or via descriptive statistics. In addition, in a subset of 400 participants (the Immunogenicity Subset; ~200 from the active group, ~200 from the placebo group), humoral immunogenicity samples are taken on more occasions.

#### 9.6.2. Correlates of Risk

If VE is demonstrated, correlates of risk will be explored. More details with appropriate methods will then be provided in a separate analysis plan.

#### 9.7. Safety Analysis

No formal statistical testing of safety data is planned. Safety data according to the vaccination schedules received and based on the FAS will be analyzed descriptively. The analysis of solicited and unsolicited AEs will be restricted to a subset of the FAS (ie, the Safety Subset).

For SAEs, AESIs, and MAAEs the full FAS is considered. New onset of chronic diseases will be collected as part of the MAAEs.

Subanalyses (descriptive) will be performed on participants with stable/well-controlled HIV infection to evaluate the effect of the vaccine on HIV RNA viral load and CD4 cell count.

Safety endpoints following the open-label cross-over vaccination and following the booster vaccination will be descriptively summarized. Pooled safety analyses with other studies may also be performed.

# **Adverse Events (Solicited and Unsolicited)**

The verbatim terms used in the eCRF by investigators to identify AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). All Reported AEs with onset during the active vaccination phase (ie, AEs occurring after double-blind vaccination up to 28 days post-vaccination), and all SAEs/AESIs/MAAEs will be included in the analysis. (S)AEs and MAAEs caused by molecularly confirmed SARS-CoV-2 infection will be removed at the analysis level from the (S)AE listings and tables and presented separately. For each AE, the percentage of participants who experience at least 1 occurrence of the given event will be summarized by study vaccine group.

Summaries, listings, datasets, or participant narratives may be provided, as appropriate, for those participants who die, who discontinue the study due to an AE or who experience a severe AE, an AESI, or an SAE.

Solicited local (at injection site) and systemic AEs will be summarized descriptively. The number and percentages of participants with at least 1 solicited local (at injection site) or systemic AE will be presented. Solicited AEs shown in the tables and listings will be based on the overall assessment of the investigator. The overall frequencies by vaccine group as well as frequencies according to severity and duration will be described for solicited AEs. Frequencies of unsolicited AEs, separately for all and vaccination-related only, will be presented by System Organ Class and preferred term, while those of solicited AEs will be presented only by preferred term. Solicited and unsolicited AEs collected following booster vaccination will be summarized descriptively, as of amendment 7, the collection of these AEs will stop.

#### **Clinical Laboratory Tests**

Laboratory data (abnormal or graded, when available) will be listed and/or tabulated by participant and time point.

#### **Vital Signs**

For all participants, weight and height (and BMI) at baseline will be summarized using descriptive statistics. Temperature will be measured at each scheduled timepoint and summarized using descriptive statistics. Other vital signs may be measured at the discretion of the investigator. Vital signs abnormalities will be listed.

For COVID-19 cases, temperature will be summarized over time from start of symptoms, using descriptive statistics and/or graphically. For systolic and diastolic blood pressure, heart rate, respiratory rate, oxygen saturation, and pulse oximetry, values and the percentage of participants with values beyond clinically relevant limits will be summarized at each scheduled timepoint. Descriptive statistics will be calculated for changes between COVID-19 Day 29 and COVID-19 Day 3-5.

#### **Physical Examinations**

For all participants, physical examinations can be performed at the discretion of the investigator. Physical examination abnormal findings will be listed.

For COVID-19 cases, physical examination findings and the percentage of participants with values beyond clinically relevant limits will be summarized at each scheduled timepoint. Descriptive statistics will be calculated for changes between COVID-19 Day 29 and COVID-19 Day 3-5, if available.

# 9.8. Analysis of the Open-label Cross-over Phase, Open-label Booster Vaccination Phase and Open-label Passive Follow-up Phase

No additional participants will be recruited for the open-label phase.

Safety, immunogenicity, and efficacy endpoints following cross-over and/or booster vaccination will be descriptively summarized by the different cohorts for the different phases (ie, for the open-label phase: early vaccinated cohort and late vaccinated cohort; ie, for the booster phase: 1-dose cohort, homologous booster cohort and the heterologous booster cohort).

Additional analyses may be conducted to support health authority interactions and/or based on public health demand in case of emerging variants.

# 9.8.1. Sample Size Determination of Immunogenicity Subset (Open-label Booster Vaccination Phase)

<u>Homologous Booster Subset:</u> The Homologous Booster Subset will include approximately 200 participants. This subset will include participants from the Immunogenicity Subset, who received Ad26.COV2.S in the double blind phase or after cross-over, and subsequently received an Ad26.COV2.S booster vaccination in the study. This group may be augmented by other participants to replace participants who are not available. Participants in the Homologous Booster Subset will have a blood sample collected pre-booster vaccination, and 28 days, 72 days, 6 months, and 1 year post booster vaccination for humoral immunogenicity assessment.

Heterologous Booster Subset: The Heterologous Booster Subset will include approximately 400 participants. This subset will include participants in the study who received placebo in the double-blind phase and have received primary vaccination with an mRNA vaccine or another authorized COVID-19 vaccine including protein, inactivated, and adenovector based vaccines outside the study, who subsequently remained in the study and subsequently received an Ad26.COV2.S booster vaccination in the study. Participants who already received an additional COVID-19 vaccination after the primary regimen outside the study will not be included in the Heterologous Booster Subset. Participants will be selected out of countries where these vaccines were authorized for emergency use or are licensed. Participants in the Heterologous Booster Subset will have blood collected pre booster vaccination, and 28 days, 72 days, 6 months, and 1 year post booster vaccination for humoral immunogenicity assessment.

A sample size of approximately 600 participants, distributed as described in Table 4 and Table 5, is estimated to be sufficient to allow robust description of immune responses to Ad26.COV2.S vaccine. These numbers are expected to provide a solid understanding of the magnitude and kinetics of the humoral response induced by a booster dose of Ad26.COV2.S vaccine in participants who received homologous Ad26.COV2.S primary vaccination or heterologous primary vaccination with an mRNA, protein, inactivated or adenovector based vaccine.

# 9.8.2. Immunogenicity Correlates (Correlates Subset)

Correlates for participants who received a booster dose will be assessed in a subset where immune responses and transcriptome modifications are measured in all vaccine recipients who experience a SARS-CoV-2 event, and in random samples of vaccine recipients who have not been infected, in a 1:5 ratio. The goal of this case control study is to assess correlates of risk of SARS-CoV-2 infection (and potential other secondary endpoints) in the vaccine group by comparing vaccine-induced immune responses and transcriptome modifications associated with COVID-19.

# 9.8.3. Efficacy Analyses

If deemed feasible, efficacy of the booster vaccination may be explored by comparing efficacy data after boosting to data in the absence of booster, on the same primary regimen.

Feasibility will be assessed based on data availability as well as adjustments for potential confounding in the statistical analysis.

The following data sources will be explored:

- 1. If available, data of participants in the study who did not receive a booster and/or available data prior to boosting.
- 2. Data of individuals outside the study who received a similar primary regimen but did not receive a booster. It will be explored if external data (eg, real world evidence data, and/or published literature data) is available to that end for the countries enrolled in this study.

For the statistical analysis, it will be explored if adjustment for potential confounding factors is feasible (based on risk factors identified in the analysis of the double-blind phase/and or literature) in each comparison. This may include, but not limit to age, presence of co-morbidities as well as the spatiotemporal evolution of variants and the epidemic. It is anticipated that comparative evaluation of efficacy against asymptomatic infections using real world evidence of data of individuals outside the study will not be feasible due to the difficulty of detecting asymptomatic infections in real world evidence.

Efficacy data may be compared following homologous versus heterologous booster vaccination. Efficacy data after primary vaccination until booster vaccination may be summarized (as immediate, early versus delayed, late vaccination).

All of the above will be detailed in an SAP prior to conducting the analysis.

# 9.9. Interim Analysis and Committees

The study will be formally monitored by a DSMB (also known as an IDMC). In general, the DSMB will monitor safety data on a regular basis to ensure the continuing safety of the participants. Enrollment will not be paused during these safety reviews, except after Stage 1a (2,000 participants) and stage 2a (2,000 participants). The DSMB will review unblinded data. The DSMB responsibilities, authorities, and procedures will be documented in the DSMB Charter.

The DSMB will also review Day 3 safety data (ie, from Day 1 to Day 3; including safety data from the ongoing clinical studies) from participants enrolled in Stage 1a and Stage 2a, before enrollment of participants in Stage 1b and Stage 2b, respectively. Vaccination of participants in the respective age groups will be paused during these safety reviews.

Continuous monitoring for vaccine-associated enhanced disease will be performed through the SSG who will look at each of the diagnosed FAS COVID-19 events. Vaccine harm monitoring will be performed for the severe/critical COVID-19/death endpoint based on the FAS. As these events will be monitored in real-time, and, after each confirmed respective case, the SSG will assess if a stopping boundary is reached. Specifically, monitoring for a higher rate of severe/critical disease or death in the vaccine group compared to the placebo group starts at the 5<sup>th</sup> event and at each additional event until the harm boundary is reached or until the primary analysis is triggered. If the stopping boundary is met, then the SSG immediately informs the Chair of the DSMB through secure communication procedures. At this point the DSMB will convene and provide a recommendation to the Oversight Group, which includes a sponsor representative as a core member. As such, the potential harm monitoring is in real-time, resulting in the earliest indication of harm possible as soon as data come in. In addition, the DSMB will formally monitor the SARS-CoV-2 events to conclude both non-efficacy and efficacy (for more details on the evaluation of and monitoring for efficacy, see section 9.5.1 and 9.5.1.1, respectively). The DSMB will evaluate in an unblinded fashion whether superiority is established for the primary endpoints or whether non-efficacy is shown based on a report provided by the SSG, when the prespecified boundaries have been crossed.

The study will also be monitored for operational non-efficacy to evaluate whether enough events to perform the PA can be collected within reasonable time. For that purpose, a monitoring rule will be set up to assess the probability that the minimal needed target number of primary endpoints events to be able to perform the PA in the PP set will be reached. For the double-blind phase of the study, two versions of the non-efficacy monitoring report will be generated. A report provided to the DSMB will contain unblinded events and a report provided to the sponsor will contain blinded events. While it is the primary responsibility of the sponsor to make decisions regarding study operations and modifications based on monitoring of study vaccine-blinded primary events from the study, the DSMB can evaluate the progress towards primary endpoints targets in the context of the study vaccine-unblinded data, and based on this review may recommend to the Oversight Group, which includes a sponsor representative as a core member, to complete the study early due to reaching the boundaries for efficacy or non-efficacy to assess VE (see Section 9.5.1). During the open-label phase, the DSMB will continue to monitor safety.

The monitoring rules will be detailed in the DSMB Charter, with the statistical details in the SAP.

A final analysis of the double-blind phase will be performed when all participants have completed the Month 6/Unblinding Visit. Depending on the operational implementation of the Month 6/Unblinding Visit, as well as the stage of the pandemic, this analysis may be conducted when a minimum of 90% of the study population has been unblinded. This will provide an analysis of all endpoints for the blinded portion of the study. This analysis will incorporate data collected after the EUA submission to the FDA. All data generated after the unblinding will be considered as part of an analytic plan devoted to the open-label phase. This analysis may be supplemented by independent measures of incidence and efficacy with real world data obtained in separate studies, to be described in a separate protocol. More details will be provided in the SAP.

The SAP will describe the planned analyses in greater detail.

# 9.10. Analyses for Cohort Unblinded Due to Administration of an Authorized/Licensed COVID-19 Vaccine

In the double-blind phase of the study, investigators may receive requests to unblind study participants who become eligible to receive an authorized/licensed COVID-19 vaccine if/when these become available. In these cases, the investigator will discuss with the participant available options and ramifications. If the participant is eligible for an authorized/licensed vaccine according to local immunization guidelines or recommendation and if the participant wishes to proceed with the unblinding, the investigator will follow the unblinding procedures. The reason for the unblinding request should be documented.

When unblinding, if it is determined that the participant received the Ad26.COV2.S vaccine (and not placebo), the participant will be informed that there are no data on the safety of receiving 2 different COVID-19 vaccines. Unblinded participants, both in the double-blind and open-label phase, will be asked to continue to be followed in this study in line with the Schedule of Activities to the extent that they permit. Safety, efficacy, and immunogenicity evaluations will be identical for all participants, if applicable and feasible, including participants who are unblinded to obtain an authorized/licensed COVID-19 vaccine and who remain in the study, including participants in the Safety Subset, if applicable and feasible. All data will be analyzed separately from the point of unblinding for safety, efficacy, and immunogenicity, as described in the Statistical Analysis Plan.

#### 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

#### 10.1. Appendix 1: Abbreviations

Ad26 adenovirus type 26 AdVac® adenoviral vaccine AE adverse event

AESI adverse event of special interest

ART anti-retroviral treatment

BIDMC Beth Israel Deaconess Medical Center

BMI body mass index BOD burden of disease

CDC Centers for Disease Control and Prevention COPD chronic obstructive pulmonary disease

COVID-19 coronavirus disease-2019
CT computed tomographic
DNA deoxyribonucleic acid
DSMB Data Safety Monitoring Board

DVT deep vein thrombosis

ECMO extracorporeal membrane oxygenation eCOA electronic clinical outcome assessment

eCRF electronic case report form eDC electronic data capture

ePRO electronic patient-reported outcomes ELISA enzyme-linked immunosorbent assay

ERD enhanced respiratory disease EUA Emergency Use Authorization

FAS Full Analysis Set
FC crystallizable fragment
FDA Food and Drug Administration

FIH first-in-human

FiO<sub>2</sub> fraction of inspired oxygen
FOIA Freedom of Information Act
FWER family-wise error rate
GCP Good Clinical Practice
GLP Good Laboratory Practice
HCP health care professional

HIPAA Health Insurance Portability and Accountability Act

HIT heparin-induced thrombocytopenia HIV human immunodeficiency virus

IB Investigator's Brochure ICF informed consent form

ICH International Council for Harmonisation of Technical Requirements for Pharmaceuticals for

Human Use

ICMJE International Committee of Medical Journal Editors

ICU intensive care unit

IDMC independent Data Monitoring Committee

IEC Independent Ethics Committee

IFN-γ interferon gamma Ig immunoglobulin IM intramuscular(ly)

IPPI Investigational Product Preparation Instructions

IRB Institutional Review Board
IWRS interactive web response system
MAAE medically-attended adverse event
MA-COV medically-attended COVID-19

MedDRA Medical Dictionary for Regulatory Activities

MERS Middle East respiratory syndrome

MERS-CoV Middle East respiratory syndrome coronavirus

multisystem inflammatory syndrome MIS

**MRU** medical resource utilization MSD Meso Scale Discovery

nucleocapsid N NHP non-human primate

National Institute of Allergy and Infectious Diseases **NIAID** 

OL open-label primary analysis PA

partial pressure of oxygen PaO<sub>2</sub> Per-protocol (efficacy) PP Per-protocol Immunogenicity PPI product quality complaint POC

**PSRC** Prevention Science Review Committee

**PSRT** protocol safety review team **RBD** receptor-binding domain

ribonucleic acid **RNA** 

**RSV** respiratory syncytial virus

reverse-transcriptase polymerase chain reaction RT-PCR

S spike

SAE serious adverse event SAP Statistical Analysis Plan

SARS severe acute respiratory syndrome

severe acute respiratory syndrome coronavirus(-2) SARS-CoV(-2) Symptoms of Infection with Coronavirus-19 SIC **SIPPM** site investigational product and procedures manual

 $SpO_2$ oxygen saturation

**SPRT** sequential probability ratio test SSG statistical support group

**SUSAR** suspected unexpected serious adverse reaction

T-helper cell (type 1/2) Th(1/2)target number of events TNE tumor necrosis factor alpha TNF-α

TTS thrombosis with thrombocytopenia syndrome

United States US vaccine efficacy VE

**VNA** virus neutralization assay

virus particles vp

WHO World Health Organization

#### **Definitions of Terms**

COVID-19 COVID-19 is the disease caused by the virus SARS-CoV-2. COVID-19 refers to SARS-

> CoV-2 infection with symptoms, and can range from mild to severe disease, the latter including pneumonia, severe acute respiratory syndrome, multi-organ failure, and death. 66,67

eCOA An umbrella term encompassing different types of outcomes assessments, in particular, the

COVID-19 signs and symptoms surveillance question, the ePRO and the e-Diary.

ePRO The electronic technology used to collect the patient-reported outcome data. PROs are

> reports that come directly from the participant without interpretation by clinician or anyone else. This includes the SIC questionnaire (Symptoms of Infection with Coronavirus-19) and

the recording of pulse oximetry results.

The electronic technology used to record solicited signs and symptoms by the participants e-Diary

in the Safety Subset.

Electronic source

Contains data traditionally maintained in a hospital or clinic record to document medical care or data recorded in a CRF as determined by the protocol. Data in this system may be system

considered source documentation.

Unblinding Visit The Month 6 visit will be used as an unblinding visit when all participants will be called in

for an on-site visit and will be made aware of their study vaccine allocation, upon

implementation of protocol Amendment 4.

Cross-over Term used when the participants who initially received placebo will be administered a single

dose of Ad26.COV2.S vaccine (only upon EUA, conditional licensure or approval in any

country).

# 10.2. Appendix 2: Clinical Laboratory Tests

The following tests will be performed according to the Schedules of Activities:

# **Protocol-Required Laboratory Assessments**

As of Amendment 7, the number of on-site study visits will be reduced for participants who are not part of the Immunogenicity Subset and who are not part of the Booster Subset. In addition, no more laboratory samples will be collected in the context of a COVID-19 episode.

Text in italics below will no longer be applicable after implementation of Amendment 7.

| Laboratory | Parameters | Timepoints |
|---|---|---|
| Assessments Testing done locally or substitute of a local laboratory | Urine pregnancy testing for participants of childbearing potential only | At screening and before each vaccination At additional timepoints as determined necessary by the investigator or required by local regulation |
| | Serum pregnancy testing for participants of childbearing potential only | At timepoints as determined necessary by the investigator or required by local regulation |
| | Nasal swabs for virology testing (molecular confirmation of SARS CoV 2 infection using a test approved by FDA EUA or equivalent) | On COVID 19 Day 1 2 (nasal swab collected by the participant at home) |
| | | On COVID 19 Day 3 5 (nasal swab collected by qualified study staff) |
| | | Once every 2 days following COVID 19 Day 3 5, until closure of the COVID 19 procedures (nasal sample collected by the participant at home) |
| | Serology blood sample for sero-confirmation of SARS-CoV-2 infection using a test approved by FDA-EUA or equivalent | At screening (prior to vaccination) (at the discretion of the sponsor) |
| | As of Amendment 7, any local COVID-19 confirmatory laboratory finding | At all visits after protocol amendment 7 (Month 12, 18, 24 or exit visit) |
| | Whole blood sample for platelet count which at some sites may be part of a complete blood count with differential | Pre-vaccination with Ad26.COV2.S: • At Month 6/Unblinding Visit (if applicable) |
| | | At Year 1/Booster Visit, if applicable |
| | | At the 28 days post Year 1/Booster Visit, if applicable |
| | | As part of a suspected AESI investigation, if applicable |

| Laboratory<br>Assessments | Parameters | Timepoints |
|---|---|---|
| Testing done centrally | Nasal swab for virology testing (molecular confirmation of SARS-CoV-2 infection and viral load testing) | At baseline (nasal swab collected by qualified study staff) |
| Nota: samples | | At Month 6/Unblinding Visit |
| Note: samples<br>for molecular<br>confirmation of | | On COVID 19 Day 1 2 (nasal swab collected by the participant at home) |
| SARS CoV 2 infection will be | | On COVID 19 Day 3 5 (nasal swab collected by qualified study staff) |
| tested if the<br>participant met<br>the prespecified<br>criteria for<br>suspected | | Once every 2 days following COVID 19 Day 3 5, until closure of the COVID 19 procedures (nasal sample collected by the participant at home) |
| COVID 19 on<br>COVID 19 Day<br>1 2 or Day 3 5,<br>as determined | Serum sample for sero-confirmation of past SARS-CoV-2 infection | On Day 1 (pre-vaccination), Day 29, Day 71,<br>Month 6/Unblinding Visit, Year 1/Booster<br>Visit (pre-vaccination, if applicable) |
| locally. | | At 28 days and 72 days post Year 1/Booster<br>Visit only for participants who received<br>booster vaccination |
| | | At Month 18 (24 weeks after Year 1/Booster visit) |
| | | COVID 19 Day 29 |
| | Nasal swab for virology testing (other respiratory pathogens using a broad respiratory pathogens panel) | May be performed on samples collected during a confirmed COVID 19 episode and in a subset of samples from participants with a symptomatic infection. |
| | | All participants during the open label phase. |
| | Saliva samples for virology testing (molecular confirmation of SARS CoV 2 infection and viral load testing) | On COVID 19 Day 3 5 (saliva sample collected by the participant at the study site or at home) |
| | | Once every 2 days following COVID 19 Day 3 5, until closure of the COVID 19 procedures (saliva sample collected by the participant at home) |
| | Serum samples for humoral immunogenicity | Non-Immunogenicity Subset: on study visits 2 (Day 1; pre-vaccination), 3 (Day 29), 4 (Day 71), 5 (Month 6/Unblinding), 6 (Year 1/Booster; pre-vaccination, if applicable), 8 (Year 1 + 28 days, if applicable), 9 (Year 1 + 72 days, if applicable), 10 (Month 18; 24 weeks after Year 1/Booster), and the early exit visit (if applicable) |
| | | Immunogenicity Subset: on study visits 2 (Day 1), 3 (Day 29), 4 (Day 71), 5 (Month 6/Unblinding), 6 (Year 1/Booster), 10 |

| Laboratory<br>Assessments | Parameters | Timepoints |
|---|---|---|
| Assessments | | (Month 18; 24 weeks after Year 1/Booster), and 11 (Year 2; 52 weeks after Year 1 Visit), and the early exit visit (if applicable), and additionally Visit 8 (Year 1 + 28 days, if applicable) and 9 (Year 1 + 72 days, if applicable). |
| | | Homologous and Heterologous Booster<br>Subsets: Visits 6 (Year 1/Booster), 8 (Year 1<br>+ 28 days); 9 (Year 1 + 72 days);10 (Month<br>18; 24 weeks after Year 1/Booster), and 11<br>(Year 2; 52 weeks after Year 1 Visit), and the<br>early exit visit (if applicable) |
| : | Serum sample for humoral immunogenicity | On COVID 19 Day 3 5 and COVID 19<br>Day 29 |
| | Serum/plasma samples for coagulation- related assays such as but not limited to: O Activated partial thromboplastin time O Prothrombin time O International normalized ratio O Fibrinogen O D-dimer O Lupus anticoagulant O Anti-cardiolipin antibody O Beta-2 glycoprotein O Heparin Induced Thrombocytopenia (HIT)/PF4 Ab, IgG·(HIT assay) O Platelet activation assay (if HIT/PF4 is positive) O Homocysteine O ADAMTS13 Activity and Inhibitor Profile | Based on the clinical evaluation of the suspected AESI (eg, whether thrombocytopenia is observed with a thrombotic event), all or some of these tests may be conducted on the stored pre-vaccination sample (retrospective test) and on the samples obtained as part of the AESI investigation, upon discretion of the sponsor. Similar samples from appropriate controls within the study may be used as part of investigation of any AESI's. |
| | Blood for cytokine/chemokine assessment | Subset of Homologous and Heterologous<br>Booster Subsets: At Year 1/Booster (pre-<br>vaccination), Year 1 + 1 day and Year 1 + 28<br>days |
| | RNAseq blood sample (transcriptomics) for exploration of biomarkers correlating with SARS-CoV-2 infection and COVID-19 severity (PAXgene tubes, whole blood) | On Day 1, Day 29, Year 1 + 28 days (only for participants who received booster vaccination). On COVID 19 Day 3 5, and Day 29, if applicable. |
| | | Subset of Homologous and Heterologous<br>Booster Subsets: At Year 1/Booster (pre-<br>vaccination), Year 1 + 1 day and Year 1 + 28<br>days |
## 10.3. Appendix 3: Regulatory, Ethical, and Study Oversight Considerations

## 10.3.1. Regulatory and Ethical Considerations

# **Investigator Responsibilities**

The investigator is responsible for ensuring that the study is performed in accordance with the protocol, current International Council for Harmonisation (ICH) guidelines on Good Clinical Practice (GCP), and applicable regulatory and country-specific requirements.

Good Clinical Practice is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human participants. Compliance with this standard provides public assurance that the rights, safety, and well-being of study participants are protected, consistent with the principles that originated in the Declaration of Helsinki, and that the study data are credible.

#### **Protocol Amendments**

Neither the investigator nor the sponsor will modify this protocol without a formal amendment by the sponsor. All protocol amendments must be issued by the sponsor, and signed and dated by the investigator. Protocol amendments must not be implemented without prior IEC/IRB approval, or when the relevant competent authority has raised any grounds for non-acceptance, except when necessary to eliminate immediate hazards to the participants, in which case the amendment must be promptly submitted to the IEC/IRB and relevant competent authority. Documentation of amendment approval by the investigator and IEC/IRB must be provided to the sponsor. When the change(s) involve only logistic or administrative aspects of the study, the IEC/IRB (where required) only needs to be notified.

During the course of the study, in situations where a departure from the protocol is unavoidable, the investigator or other physician in attendance will contact the appropriate sponsor representative listed in the Contact Information page(s), which will be provided as a separate document. Except in emergency situations, this contact should be made <u>before</u> implementing any departure from the protocol. In all cases, contact with the sponsor must be made as soon as possible to discuss the situation and agree on an appropriate course of action. The data recorded in the eCRF and source documents will reflect any departure from the protocol, and the source documents will describe this departure and the circumstances requiring it.

## Regulatory Approval/Notification

This protocol and any amendment(s) must be submitted to the appropriate regulatory authorities in each respective country, if applicable. A study may not be initiated until all local regulatory requirements are met.

## **Required Prestudy Documentation**

The following documents must be provided to the sponsor before shipment of study vaccine to the study site:

• Protocol and amendment(s), if any, signed and dated by the principal investigator

- A copy of the dated and signed (or sealed, where appropriate per local regulations), written IEC/IRB approval of the protocol, amendments, ICF, any recruiting materials, and if applicable, participant compensation programs. This approval must clearly identify the specific protocol by title and number and must be signed (or sealed, where appropriate per local regulations) by the chairman or authorized designee.
- Name and address of the IEC/IRB, including a current list of the IEC/IRB members and their function, with a statement that it is organized and operates according to GCP and the applicable laws and regulations. If accompanied by a letter of explanation, or equivalent, from the IEC/IRB, a general statement may be substituted for this list. If an investigator or a member of the study-site personnel is a member of the IEC/IRB, documentation must be obtained to state that this person did not participate in the deliberations or in the vote/opinion of the study.
- Regulatory authority approval or notification, if applicable
- Signed and dated statement of investigator (eg, Form FDA 1572), if applicable
- Documentation of investigator qualifications (eg., curriculum vitae)
- Completed investigator financial disclosure form from the principal investigator, where required
- Signed and dated Clinical Trial Agreement, which includes the financial agreement
- Any other documentation required by local regulations

The following documents must be provided to the sponsor before enrollment of the first participant:

- Completed investigator financial disclosure forms from all subinvestigators
- Documentation of subinvestigator qualifications (eg., curriculum vitae)
- Name and address of any local laboratory conducting tests for the study, and a dated copy of current laboratory normal ranges for these tests, if applicable
- Local laboratory documentation demonstrating competence and test reliability (eg, accreditation/license), if applicable

## **Independent Ethics Committee or Institutional Review Board**

Before the start of the study, the investigator (or sponsor where required) will provide the IEC/IRB with current and complete copies of the following documents (as required by local regulations):

- Final protocol and amendments
- Sponsor-approved ICF (and any other written materials to be provided to the participants)
- IB (or equivalent information) and amendments/addenda
- Sponsor-approved participant recruiting materials

- Information on compensation for study-related injuries or payment to participants for participation in the study, if applicable
- Investigator's curriculum vitae or equivalent information (unless not required, as documented by the IEC/IRB)
- Information regarding funding, name of the sponsor, institutional affiliations, other potential conflicts of interest, and incentives for participants
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after the IEC/IRB has given full approval of the final protocol, amendments (if any, excluding the ones that are purely administrative, with no consequences for participants, data or study conduct, unless required locally), the ICF, applicable recruiting materials, and participant compensation programs, and the sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the IEC/IRB and the documents being approved.

During the study the investigator (or sponsor where required) will send the following documents and updates to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments (excluding the ones that are purely administrative, with no consequences for participants, data or study conduct)
- Revision(s) to ICF and any other written materials to be provided to participants
- If applicable, new or revised participant recruiting materials approved by the sponsor
- Revisions to compensation for study-related injuries or payment to participants for participation in the study, if applicable
- New edition(s) of the IB and amendments/addenda
- Summaries of the status of the study at intervals stipulated in guidelines of the IEC/IRB (at least annually)
- Reports of AEs that are serious, unlisted/unexpected, and associated with the study vaccine
- New information that may adversely affect the safety of the participants or the conduct of the study
- Deviations from or changes to the protocol to eliminate immediate hazards to the participants
- Report of deaths of participants under the investigator's care
- Notification if a new investigator is responsible for the study at the site
- Development Safety Update Report and Line Listings, where applicable
- Any other requirements of the IEC/IRB

For all protocol amendments (excluding the ones that are purely administrative, with no consequences for participants, data or study conduct), the amendment and applicable ICF revisions

must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will be asked to review and reapprove this study, where required.

At the end of the study, the investigator (or sponsor where required) will notify the IEC/IRB about the study completion.

## **Country Selection**

This study will only be conducted in those countries where the intent is to launch or otherwise help ensure access to the developed product if the need for the product persists, unless explicitly addressed as a specific ethical consideration in Section 4.2.1.

#### **Other Ethical Considerations**

For study-specific ethical design considerations, refer to Section 4.2.1.

#### 10.3.2. Financial Disclosure

Investigators and subinvestigators will provide the sponsor with sufficient, accurate financial information in accordance with local regulations to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

Refer to Required Prestudy Documentation (above) for details on financial disclosure.

## 10.3.3. Informed Consent Process

Consent of each participant must be obtained according to local requirements after the nature of the study has been fully explained. The informed consent(s) must be obtained before performance of any study-related procedure. Downloading of an application to the participant's eDevice, to access materials for enrollment and study information, is not considered a study-related procedure. The ICF can be signed remotely prior to the Screening Visit.

The ICF(s) that is/are used must be approved by both the sponsor and by the reviewing IEC/IRB and be in a language that the participant can read and understand. The informed consent should be in accordance with principles that originated in the Declaration of Helsinki, current ICH and GCP guidelines, applicable regulatory requirements, and sponsor policy.

Before enrollment in the study, the investigator or an authorized member of the study-site personnel must explain to potential participants the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort participation in the study may entail. Participants will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the participant will receive. Finally, they will be told that the investigator will maintain a participant identification register for the purposes of long-term follow-up if needed and

that their records may be accessed by health authorities and authorized sponsor personnel without violating the confidentiality of the participant, to the extent permitted by the applicable law(s) or regulations. By signing the ICF the participant is authorizing such access. It also denotes that the participant agrees to allow his or her study physician to recontact the participant for the purpose of obtaining consent for additional safety evaluations, if needed.

The participant will be given sufficient time to read the ICF and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the participant's personally dated signature. After having obtained the consent, a copy of the ICF must be given to the participant.

Participants who are rescreened are required to sign a new ICF. Participants entering the open-label phase are required to sign a new ICF at the Month 6/Unblinding Visit or at an unscheduled visit beyond the Month 6/Unblinding Visit if this visit has already been conducted. All participants are required to sign a new ICF at the Year 1/Booster Visit.

As described in Section 8.1.2, a caregiver may assist a participant who is unable to complete the SIC in the eCOA, by reading the questions aloud and recording the responses in the eCOA on the participant's behalf (using the caregiver's unique identifier and PIN). For this purpose, a caregiver consent form has been developed. Consent must be obtained according to local requirements and must be obtained from the caregiver before he or she is allowed to complete the eCOA on behalf of the participant. After having obtained the caregiver's consent, a copy of the consent form must be given to the caregiver. Of note, the caregiver is not intended to be a Legally Authorized Representative who can provide informed consent for study participation on behalf of the participant. It is also not the intent that the caregiver collects nasal swabs or other samples from the participant unless he or she is specifically qualified to perform these tasks and can document the use of appropriate personal protective equipment during the performance of such tasks.

#### 10.3.4. Data Protection

## **Privacy of Personal Data**

The collection and processing of personal data from participants enrolled in this study will be limited to those data that are necessary to fulfill the objectives of the study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of participants confidential.

The informed consent obtained from the participant includes explicit consent for the processing of personal data and for the investigator/institution to allow direct access to his or her original medical records (source data/documents) for study-related monitoring, audit, IEC/IRB review, and

regulatory inspection. This consent also addresses the transfer of the data to other entities and to other countries.

The participant has the right to request through the investigator access to his or her personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps will be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Exploratory biomarker and immunogenicity research is not conducted under standards appropriate for the return of data to participants. In addition, the sponsor cannot make decisions as to the significance of any findings resulting from exploratory research. Therefore, exploratory research data will not be returned to participants or investigators, unless required by law or local regulations. Privacy and confidentiality of data generated in the future on stored samples will be protected by the same standards applicable to all other clinical data.

## 10.3.5. Long-term Retention of Samples for Additional Future Research

Samples collected in this study may be stored for up to 15 years (or according to local regulations) for additional research. Samples will only be used to understand Ad26.COV2.S, to understand SARS-CoV-2 infection, to understand differential vaccine responders, and to develop tests/assays related to Ad26.COV2.S and SARS-CoV-2 infection. The research may begin at any time during the study or the post-study storage period.

Stored samples will be coded throughout the sample storage and analysis process and will not be labeled with personal identifiers. Participants may withdraw their consent for their samples to be stored for research (refer to Section 7.2.1).

## 10.3.6. Committees Structure

#### **Independent Data Monitoring Committee**

A DSMB (also known as an IDMC) will be established to monitor safety data on an ongoing basis to ensure the continuing safety of the participants enrolled in this study. Enrollment will not be paused during these safety reviews, except after stage 1a (2,000 participants) and stage 2a (2,000 participants). This committee will consist of at least 1 medical expert in the relevant therapeutic area and at least 1 statistician; committee membership responsibilities, authorities, and procedures will be documented in its charter.

The DSMB will also review Day 3 safety data (ie, from Day 1 to Day 3; including safety data from the ongoing clinical studies) from participants enrolled in Stage 1a and Stage 2a, before enrollment of participants in Stage 1b and Stage 2b, respectively. Vaccination of participants in the respective age groups will be paused during these safety reviews.

Ad hoc review may be performed further to the occurrence of any SAE leading to a study pausing situation as outlined in Section 6.11, or at request of the sponsor's medical monitor or designee. The principal investigator and sponsor's study responsible physician will inform the DSMB of any AE of concern.

If the SSG assesses that the stopping boundary is met (see below), the Chair of the DSMB will immediately be informed through secure communication procedures. At this point, the DSMB will convene and provide a recommendation to the Oversight Group, which includes a sponsor representative as a core member.

In addition, the DSMB will formally monitor the infections in all groups to conclude both non-efficacy and efficacy. The DSMB will evaluate in an unblinded fashion whether superiority is established for the primary endpoints or whether non-efficacy is shown (see Section 9.8) based on a report provided by the SSG, when the prespecified boundaries have been crossed. The boundaries are based on the SPRT. Following the EUA and treatment group unblinding, the DSMB will continue to monitor participant safety during the open-label phase.

The PSRT and the Janssen Medical Safety Council review all clinical and laboratory safety data during the course of the study.

# **Statistical Support Group**

The SSG is the statistical support group to the DSMB; they are unblinded and provide the DSMB with the statistical analysis based on unblinded data. As the DSMB, they are independent to the company. They will continuously monitor for vaccine-associated enhanced disease by looking at each diagnosed COVID-19 case in the FAS (and also SARS-CoV-2 infections in participants requiring hospitalization; and SARS-CoV-2 infections in participants being admitted to the ICU [or equivalent]; and SARS-CoV-2 infections resulting in death [with death being at least probably related to COVID-19]). As these infections will be monitored in real-time, and, after each confirmed respective case, the SSG will assess if a stopping boundary is reached. If the stopping boundary is met, then the SSG immediately informs the Chair of the DSMB through secure communication procedures. At this point the DSMB will convene and provide a recommendation to the Oversight Group, which includes a sponsor representative as a core member. As such, the potential harm monitoring is in real-time, resulting in the earliest indication of harm possible as soon as data come in.

## **Clinical Severity Adjudication Committee**

The Clinical Severity Adjudication Committee will review all cases in the study, except for cases already adjudicated as severe, as a supplement to the algorithm described in the SAP, as well as those requiring medical intervention (such as a composite endpoint of hospitalization, ICU admission, mechanical ventilation, and ECMO, linked to objective measures such as decreased oxygenation, X-ray or CT findings), including onset of cases, taking into account all available relevant information at the time of adjudication. As of Amendment 7, Clinical Severity Adjudication Committee may review all cases based on available data from the passive follow-up (eg, limited to COVID-19 AE/SAE data, CIOMS forms, local laboratory results). More details will be provided in the revised charter of the Clinical Severity Adjudication Committee. Readjudication will occur if new information becomes available. The last adjudication for a given case will determine the status of the case for analysis. The Clinical Severity Adjudication Committee's assessment will be considered the definitive classification of the case. The case review including

severity assessments after implementation of Protocol Amendment 7 may change and will be reflected in the charter of the committee.

## **Oversight Group**

The Oversight Group's responsibilities, authorities, procedures and their interactions with the DSMB will be documented in the Oversight Group charter.

## **AESI Adjudication Committee**

An AESI Adjudication Committee with appropriate expertise will be established to evaluate each suspected AESI and determine whether it is a case of TTS (see Section 8.3.7). A Charter will be developed to describe the roles and responsibilities of the Committee.

# 10.3.7. Publication Policy/Dissemination of Clinical Study Data

All information, including but not limited to information regarding Ad26.COV2.S or the sponsor's operations (eg, patent application, formulas, manufacturing processes, basic scientific data, prior clinical data, formulation information) supplied by the sponsor to the investigator and not previously published, and any data generated as a result of this study, are considered confidential and remain the sole property of the sponsor. The investigator agrees to maintain this information in confidence and use this information only to accomplish this study and will not use it for other purposes without the sponsor's prior written consent.

The investigator understands that the information developed in the study will be used by the sponsor in connection with the continued development of Ad26.COV2.S, and thus may be disclosed as required to other clinical investigators or regulatory agencies. To permit the information derived from the clinical studies to be used, the investigator is obligated to provide the sponsor with all data obtained in the study.

The results of the study will be reported in a Clinical Study Report generated by the sponsor and will contain data from all study sites that participated in the study as per-protocol. Recruitment performance or specific expertise related to the nature and the key assessment parameters of the study will be used to determine a coordinating investigator for the study. Results of analyses performed after the Clinical Study Report has been issued will be reported in a separate report and will not require a revision of the Clinical Study Report.

Study participant identifiers will not be used in publication of results. Any work created in connection with performance of the study and contained in the data that can benefit from copyright protection (except any publication by the investigator as provided for below) shall be the property of the sponsor as author and owner of copyright in such work.

Consistent with Good Publication Practices and International Committee of Medical Journal Editors (ICMJE) guidelines, the sponsor shall have the right to publish such primary (multicenter) data and information without approval from the investigator. The investigator has the right to publish study site-specific data after the primary data are published. If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for

review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application. In the event that issues arise regarding scientific integrity or regulatory compliance, the sponsor will review these issues with the investigator. The sponsor will not mandate modifications to scientific content and does not have the right to suppress information. For multicenter study designs and sub-study approaches, secondary results generally should not be published before the primary endpoints of a study have been published. Similarly, investigators will recognize the integrity of a multicenter study by not submitting for publication data derived from the individual study site until the combined results from the completed study have been submitted for publication, within 18 months after the study end date, or the sponsor confirms there will be no multicenter study publication. Authorship of publications resulting from this study will be based on the guidelines on authorship, such as those described in the ICMJE Recommendations for the Conduct, Reporting, Editing and Publication of Scholarly Work in Medical Journals, which state that the named authors must have made a significant contribution to the conception or design of the work; or the acquisition, analysis, or interpretation of the data for the work; and drafted the work or revised it critically for important intellectual content; and given final approval of the version to be published; and agreed to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

## Registration of Clinical Studies and Disclosure of Results

The sponsor will register and disclose the existence of and the results of clinical studies as required by law. The disclosure of the final study results will be performed after the end-of-study in order to ensure the statistical analyses are relevant.

## 10.3.8. Data Quality Assurance

## **Data Quality Assurance/Quality Control**

Steps to be taken to ensure the accuracy and reliability of data include the selection of qualified investigators and appropriate study sites, review of protocol procedures with the investigator and study-site personnel before the study, and periodic monitoring visits by the sponsor. Written instructions will be provided for collection, handling, storage, and shipment of samples.

Guidelines for eCRF completion will be provided and reviewed with study-site personnel before the start of the study.

The sponsor will review the eCRF for accuracy and completeness after transmission to the sponsor; any discrepancies will be resolved with the investigator or designee, as appropriate. After upload of the data into the study database they will be verified for accuracy and consistency with the data sources.

## 10.3.9. Case Report Form Completion

Case report forms are prepared and provided by the sponsor for each participant in electronic format. All data relating to the study will be recorded in the eCRF or eCOA. All eCRF entries, corrections, and alterations must be made by the investigator or authorized study-site personnel. The investigator must verify that all data entries in the eCRF are accurate and correct.

The study data will be transcribed by study-site personnel from the source documents onto an eCRF, if applicable. Study-specific data will be transmitted in a secure manner to the sponsor.

Worksheets may be used for the capture of some data to facilitate completion of the eCRF. Any such worksheets will become part of the participant's source documents. Data must be entered into the eCRF in English. The eCRF must be completed as soon as possible after a participant visit and the forms should be available for review at the next scheduled monitoring visit.

If necessary, queries will be generated in the electronic data capture (eDC) tool. If corrections to an eCRF are needed after the initial entry into the eCRF, this can be done in either of the following ways:

- Investigator and study-site personnel can make corrections in the eDC tool at their own initiative or as a response to an auto query (generated by the eDC tool).
- Sponsor or sponsor delegate can generate a query for resolution by the investigator and studysite personnel.

#### 10.3.10. Source Documents

At a minimum, source documents consistent in the type and level of detail with that commonly recorded at the study site as a basis for standard medical care must be available for the following: participant identification, eligibility (including relevant medical history, including anything related to footnotes h and i to the Schedules of Activities in Section 1.3.3), and study identification; study discussion and date of signed informed consent; dates of visits; results of safety and efficacy parameters as required by the protocol; record of all AEs and follow-up of AEs; concomitant therapy; study vaccine receipt/dispensing/return records; study vaccine administration information; and date of study completion and reason withdrawal from the study, if applicable.

The author of an entry in the source documents should be identifiable. Given that PROs are reports of a patient's health condition that come directly from the patient, without interpretation by a clinician or anyone else, the responses to ePRO measures entered by study participants into source records cannot be overridden by site staff or investigators.

Up to protocol amendment 7, participant- and investigator-completed scales and assessments designated by the sponsor (ie, SIC) will be recorded directly into an eDevice and will be considered source data. The participant's e-Diary used to collect information regarding solicited signs and symptoms after vaccination will be considered source data. The documentation of the positive RT-PCR result that serves as a trigger to start procedures for COVID-19 follow-up, will be considered source data.

Specific details required as source data for the study and source data collection methods will be reviewed with the investigator before the study and will be described in the monitoring guidelines (or other equivalent document).

An eSource system may be utilized, which contains data traditionally maintained in a hospital or clinic record to document medical care (eg, electronic source documents) as well as the clinical study-specific data fields as determined by the protocol. This data is electronically extracted for use by the sponsor. If eSource is utilized, references made to the CRF in the protocol include the eSource system but information collected through eSource may not be limited to that found in the eCRF.

# 10.3.11. Monitoring

The sponsor will use a combination of monitoring techniques (central, remote, or on-site monitoring) to monitor this study.

The sponsor will perform on-site monitoring visits as frequently as necessary, if allowed per local regulations. If on-site monitoring visits are not possible due to local regulations, restrictions and guidance, the monitor will conduct site monitoring visits and activities remotely. Additional on-site monitoring visits may be needed at a later moment in time to catch up on source data review. Remote source data review of electronic records might be performed if possible and if allowed by local/national regulations, restrictions and guidance.

The monitor will record dates of the visits in a study site visit log that will be kept at the study site. The first post-initiation visit will be made as soon as possible after enrollment has begun. At these visits, the monitor will review the source documents (eg, hospital/clinic/physician's office medical records) to ensure adherence to the protocol. The nature and location of all source documents will be identified to ensure that all sources of original data required to complete the eCRF are known to the sponsor and study-site personnel and are accessible for review by the sponsor study-site contact. If electronic records are maintained at the study site, the method of review must be discussed with the study-site personnel.

Direct access to source documents (medical records) must be allowed for the purpose of source document review and may be needed to ensure that the recorded data are consistent with the original source data. Findings from this review will be discussed with the study-site personnel. The sponsor expects that during monitoring visits, the relevant study-site personnel will be available, the source documents will be accessible, and a suitable environment will be provided for review of study-related documents. The monitor will meet with the investigator on a regular basis during the study to provide feedback on the study conduct.

In addition to on-site monitoring visits, remote contacts can occur. It is expected that during these remote contacts, study-site personnel will be available to provide an update on the progress of the study at the site.

Central monitoring will take place for data identified by the sponsor as requiring central review.

#### 10.3.12. On-Site Audits

Representatives of the sponsor's clinical quality assurance department may visit the study site at any time during or after completion of the study to conduct an audit of the study in compliance with regulatory guidelines and company policy. Remote auditing techniques may also be utilized, if necessary. These audits will require access to all study records, including (electronic) source documents as allowed per local regulations, for inspection. Participant privacy must, however, be respected. The investigator and study-site personnel are responsible for being present and available for consultation during routinely scheduled study-site audit visits conducted by the sponsor or its designees.

Similar auditing procedures may also be conducted by agents of any regulatory body, either as part of a national GCP compliance program or to review the results of this study in support of a regulatory submission. The investigator should immediately notify the sponsor if he or she has been contacted by a regulatory agency concerning an upcoming inspection.

#### 10.3.13. Record Retention

In compliance with the ICH/GCP guidelines, the investigator/institution will maintain all eCRF and all source documents that support the data collected from each participant, as well as all study documents as specified in ICH/GCP Section 8, Essential Documents for the Conduct of a Clinical Trial, and all study documents as specified by the applicable regulatory requirement(s). The investigator/institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the sponsor. It is the responsibility of the sponsor to inform the investigator/institution as to when these documents no longer need to be retained.

If the responsible investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the investigator relocate or dispose of any study documents before having obtained written approval from the sponsor.

If it becomes necessary for the sponsor or the appropriate regulatory authority to review any documentation relating to this study, the investigator/institution must permit access to such reports.

#### 10.3.14. Study and Site Start and Closure

## First Act of Recruitment

The first site open is considered the first act of recruitment and it becomes the study start date.

## **Study/Site Termination**

The sponsor reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IEC/IRB or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of participants by the investigator
- Discontinuation of further study vaccine development

10.4. Appendix 4: Adverse Events, Serious Adverse Events, Adverse Events of Special Interest, Medically-attended Adverse Events, Product Quality Complaints, and Other Safety Reporting: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### 10.4.1. Adverse Event Definitions and Classifications

#### **Adverse Event**

An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the vaccine. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. (Definition per ICH).

This includes any occurrence that is new in onset or aggravated in severity or frequency from the baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.

For the Safety Subset, any respiratory tract infection will be reported as an AE if it occurs between the time of any vaccination through the following 28 days. Any respiratory tract infection recorded as an AE in the eCRF will be excluded from the AE analysis if the molecular test is subsequently found to be positive for SARS-CoV-2. Respiratory tract infections arising from SARS-CoV-2 infection will not be reported as (S)AEs in the Clinical Study Report but will be tabulated separately.

As of Protocol Amendment 7, COVID-19 will be reported as SAE, AE, or MAAE.

*Note*: For time period of sponsor's AE collection, see All Adverse Events under Section 8.3.1.

#### **Serious Adverse Event**

An SAE based on ICH and EU Guidelines on Pharmacovigilance for Medicinal Products for Human Use is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening
  (The participant was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect
- Is a suspected transmission of any infectious agent via a medicinal product

## Is Medically Important\*

\*Medical and scientific judgement should be exercised in deciding whether expedited reporting is also appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent 1 of the other outcomes listed in the definition above. These should usually be considered serious.

If a serious and unexpected AE occurs for which there is evidence suggesting a causal relationship between the study vaccine and the event (eg, death from anaphylaxis), the event must be reported as a SUSAR even if it is a component of the study endpoint (eg, all-cause mortality).

Any respiratory tract infection fulfilling the criteria of an SAE will be reported as such during the entire study. If the molecular test is positive for SARS-CoV-2, the SAE will be excluded from the SAE analysis in the Clinical Study Report, and will be tabulated separately.

As of Amendment 7, a passive follow-up approach is adopted: the investigator will place a phone call at Month 18 and Month 24 to collect information on any protocol required safety information (see Section 8.3.1). In addition, SAEs, AEs, and MAAEs related to COVID-19 need to be reported together with the concomitant medications related to these events until study end. Any confirmatory COVID-19 laboratory finding should be reported in the eCRF.

## Unlisted (Unexpected) Adverse Event/Reference Safety Information

An AE is considered unlisted if the nature or severity is not consistent with the applicable product reference safety information. For Ad26.COV2.S, the expectedness of an AE will be determined by whether or not it is listed in the IB.

## 10.4.2. Attribution Definitions

## **Assessment of Causality**

The causal relationship to study vaccine is determined by the investigator. The following selection should be used to assess all AEs.

#### Related

There is a reasonable causal relationship between study vaccine administration and the AE.

#### **Not Related**

There is not a reasonable causal relationship between study vaccine administration and the AE.

The term "reasonable causal relationship" means there is evidence to support a causal relationship.

By definition, all solicited AEs at the injection site (local) will be considered related to the study vaccine administration.

## 10.4.3. Severity Criteria

All AEs and laboratory data will be coded for severity using a modified version of the FDA grading table, based on version of September 2007<sup>63</sup>, included in Appendix 9.

The AESI definition includes thrombocytopenia, defined as platelet count  $<150,000/\mu$ L as per the Brighton Collaboration (Section 8.3.7.1).

For the purpose of severity grading, an AE of thrombocytopenia based on platelet counts  $>140,000/\mu L$  and  $<150,000~\mu L$  should be considered Grade 1.

For AEs not identified in the grading table, the following guidelines will be applied:

| Grade 1 | Mild | Symptoms causing no or minimal interference with usual social and functional activities |
|---|---|---|
| Grade 2 | Moderate | Symptoms causing greater than minimal interference with usual social and functional activities |
| Grade 3 | Severe | Symptoms causing inability to perform usual social and functional activities and requires medical intervention |
| Grade 4 | Potentially life-threatening | Symptoms causing inability to perform basic self-care functions OR medical or operative intervention indicated to prevent permanent impairment, persistent disability OR ER visit or hospitalization |

For participants in the Safety Subset, the severity of solicited signs and symptoms will be graded in the e-Diary by the participant based on the severity assessment provided in the diary as well as assessed by the investigator using the toxicity grading scale in Appendix 9. (*Note*: severity of the measured events will be derived from the diameter [for erythema and swelling] and the temperature measurements [for fever]). See also Section 8.3.2.

## 10.4.4. Special Reporting Situations

Safety events of interest on a sponsor study vaccine in an interventional study that may require expedited reporting or safety evaluation include, but are not limited to:

- Known overdose of a sponsor study vaccine
- Suspected abuse/misuse of a sponsor study vaccine
- Accidental or occupational exposure to a sponsor study vaccine
- Medication error, intercepted medication error, or potential medication error involving a
  Johnson & Johnson medicinal product (with or without patient exposure to the Johnson &
  Johnson medicinal product, eg, product name confusion, product label confusion, intercepted
  prescribing or dispensing errors)

Special reporting situations should be recorded in the eCRF. Any special reporting situation that meets the criteria of an SAE should be recorded on the Safety Report Form of the eCRF.

#### 10.4.5. Procedures

#### **All Adverse Events**

All AEs, regardless of seriousness, severity, or presumed relationship to study vaccine, must be recorded using medical terminology in the source document and the eCRF. Whenever possible, diagnoses should be given when signs and symptoms are due to a common etiology (eg, cough, runny nose, sneezing, sore throat, and head congestion should be reported as "upper respiratory infection"). Investigators must record in the eCRF their opinion concerning the relationship of the AE to study therapy. All measures required for AE management must be recorded in the source document and reported according to sponsor instructions.

For all studies with an outpatient phase, including open-label studies, the participant must be provided with a "wallet (study) card" and instructed to carry this card with them for the duration of the study indicating the following:

- Study number
- Statement, in the local language(s), that the participant is participating in a clinical study
- Investigator's name and 24-hour contact telephone number
- Local sponsor's name and 24-hour contact telephone number (for medical personnel only)
- Site number
- Participant number
- Any other information that is required to do an emergency breaking of the blind

#### **Serious Adverse Events**

All SAEs that have not resolved by the end of the study, or that have not resolved upon the participant's discontinuation from the study, must be followed until any of the following occurs:

- The event resolves
- The event stabilizes
- The event returns to baseline, if a baseline value/status is available
- The event can be attributed to agents other than the study vaccine or to factors unrelated to study conduct
- It becomes unlikely that any additional information can be obtained (participant or health care practitioner refusal to provide additional information, lost to follow-up after demonstration of due diligence with follow-up efforts)

Suspected transmission of an infectious agent by a medicinal product will be reported as an SAE.

Any event requiring hospitalization (or prolongation of hospitalization) that occurs during participation in the study must be reported as an SAE, except hospitalizations for the following:

- Hospitalizations not intended to treat an acute illness or AE (eg, social reasons such as pending placement in long-term care facility)
- Surgery or procedure planned before entry into the study (must be documented in the eCRF). *Note*: Hospitalizations that were planned before the signing of the ICF, and where the underlying condition for which the hospitalization was planned has not worsened, will not be considered SAEs. Any AE that results in a prolongation of the originally planned hospitalization is to be reported as a new SAE.

The cause of death of a participant in a study, whether or not the event is expected or associated with the study vaccine, is considered a SAE.

Information regarding SAEs will be transmitted to the sponsor using a SAE Form and Safety Report Form of the eCRF, which must be completed and reviewed by a physician from the study site, and transmitted in a secure manner to the sponsor within 24 hours. The initial and follow-up reports of an SAE should be transmitted in a secure manner electronically or by facsimile (fax). Telephone reporting should be the exception and the reporter should be asked to complete the appropriate form(s) first.

#### **Adverse Events of Special Interest**

AESIs will be carefully monitored during the study by the sponsor. Suspected AESIs must be reported to the sponsor within 24 hours of site awareness irrespective of seriousness (ie, serious and non-serious AEs) or causality assessment, following the procedure described above for SAEs and will require enhanced data collection.

## 10.4.6. Product Quality Complaint Handling

#### **Definition**

A PQC is defined as any suspicion of a product defect related to manufacturing, labeling, or packaging, ie, any dissatisfaction relative to the identity, quality, durability, reliability, or performance of a distributed product, including its labeling, drug delivery system, or package integrity. A PQC may have an impact on the safety and efficacy of the product. In addition, it includes any technical complaints, defined as any complaint that indicates a potential quality issue during manufacturing, packaging, release testing, stability monitoring, dose preparation, storage or distribution of the product or the drug delivery system.

#### **Procedures**

All initial PQCs must be reported to the sponsor by the study-site personnel within 24 hours after being made aware of the event.

A sample of the suspected product should be maintained under the correct storage conditions until a shipment request is received from the sponsor.

# 10.4.7. Contacting Sponsor Regarding Safety, Including Product Quality

The names (and corresponding telephone numbers) of the individuals who should be contacted regarding safety issues, PQC, or questions regarding the study are listed in the Contact Information page(s), which will be provided as a separate document.

# 10.5. Appendix 5: Contraceptive Guidance and Collection of Pregnancy Information

Participants must follow contraceptive measures as outlined in Section 5.1. Pregnancy information will be collected and reported as noted in Section 8.3.5.

## **Definition of a Person of Childbearing Potential**

## A Person of Childbearing Potential

A person is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

# A Person Not of Childbearing Potential

## premenarchal

A premenarchal state is 1 in which menarche has not yet occurred.

## postmenopausal

A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

# • permanently sterile (for the purpose of this study)

Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

*Note*: If the childbearing potential changes after start of the study (eg, a premenarchal person experiences menarche) or the risk of pregnancy changes (eg, a person who is not heterosexually active becomes active), a person must begin an acceptable effective method of contraception, as described throughout the inclusion criteria.

# 10.6. Appendix 6: Symptoms of Infection with Coronavirus-19 (SIC)

As of Amendment 7, this is no longer applicable.

The following questions ask about symptoms people with coronavirus-19 infection may experience. Answer each question carefully by choosing 'yes' if you have experienced the symptom or 'no' if you have not experienced the symptom in the last 24 hours. If you choose 'yes,' select the rating that best matches your experience.

| n the last 24 hours,<br>have you<br>experienced | Please rate | the sev | erity of | each sy | mpton | ı you e | xperier | iced. | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Feeling generally | How severe | was you | ır feelin | g (gene | rally ur | well o | r run do | <b>own)</b> in | the last | 24 hou | rs? |
| unwell (run down) ☐ Yes ☐ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Fatigue (tiredness) | How severe was your fatigue (tiredness) in the last 24 hours? | | | | | | | | | | |
| □ Yes □ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | □<br>7 | 8 | 9 | 10<br>Worst<br>possible |
| Physical weakness | How severe | was you | ır feeling | of <b>phy</b> | sical w | eaknes | s in the | last 24 | hours? | • | |
| □ <b>Yes</b> □ <b>No</b> If yes, → | 0<br>None | 1 | □<br>2 | □<br>3 | 4 | □<br>5 | 6 | □<br>7 | 8 | 9 | 10<br>Worst<br>possible |
| Cough | How severe | was you | ır cough | in the | ast 24 l | nours? | | | | | |
| □ <b>Yes</b> □ <b>No</b> If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Shortness of breath | How severe | was you | ır <b>shortı</b> | ness of | breath | (difficu | ılty bre | athing) | in the I | ast 24 h | ours? |
| (difficulty breathing) □ Yes □ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | □<br>7 | 8 | 9 | 10<br>Worst<br>possible |
| Sore throat | How severe | was you | ır <b>sore t</b> | <b>hroat</b> ir | the las | t 24 ho | urs? | | | | |
| □ <b>Yes</b> □ <b>No</b> If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Nasal congestion | How severe | was you | ır nasal | conges | tion (s | tuffy no | ose) in t | the last | 24 hou | rs? | |
| (stuffy nose) ☐ Yes ☐ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |

| In the last 24 hours,<br>have you<br>experienced | Please rate | the sev | erity of | each sy | ympton | n you e | xperier | nced. | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Wheezing | How severe was your wheezing (whistling sound while breathing) in the last 24 hours? | | | | | | | | | | |
| (whistling sound while breathing) ☐ Yes ☐ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Runny nose | How severe | How severe was your <b>runny nose</b> in the last 24 hours? | | | | | | | | | |
| □ Yes □ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Sneezing | How severe | was you | ır sneez | ing in t | ne last 2 | 24 hour | s? | | | | |
| □ Yes □ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Chest congestion | How severe was your chest congestion (mucus in chest) in the last 24 hours? | | | | | | | | | | |
| (mucus in chest) □ Yes □ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Chest pain/ | How severe | was you | ır chest | pain/pı | essure | /tightn | ess in t | he last 2 | 24 hour | s? | |
| pressure/tightness ☐ Yes ☐ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Muscle aches/pains | How severe | were yo | ur musc | cle ache | es or pa | ains in t | the last | 24 hour | rs? | | |
| □ Yes □ No If yes, → | 0<br>None | □<br>1 | 2 | 3 | 4 | □<br>5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Joint aches/pains | How severe | were the | aches | or pair | ıs in yo | ur join | ts in the | last 24 | hours | ? | |
| ☐ Yes ☐ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | □<br>5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |

| In the last 24 hours,<br>have you<br>experienced | Please rate | the seve | erity of | each sy | mptom | ı you e | xperier | iced. | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Headache | How severe | was you | r <b>heada</b> | che in t | he last | 24 houi | rs? | | | | |
| □ Yes □ No | | | | | | | | | | | |
| If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Feeling faint | How severe | was you | r feelin | g of fail | ntness | in the la | ast 24 h | ours? | | | |
| ☐ Yes ☐ No | | | | | | | | | | | |
| If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Problems thinking clearly/brain fog | How severe | were you | ır <b>prob</b> l | ems th | inking | clearly/ | brain f | og in th | e last 2 | 4 hours? | • |
| ☐ Yes ☐ No | 0 | □<br>1 | 2 | □<br>3 | □<br><b>4</b> | □<br>5 | □<br>6 | □<br>7 | □<br>8 | 9 | □<br>10 |
| If yes, → | None | ı | 2 | 3 | 4 | 3 | O | , | 0 | 9 | Worst<br>possible |
| Chills | How severe | were you | ur <b>chills</b> | in the l | ast 24 h | nours? | | | | | |
| □ Yes □ No | | | | | | | | | | | |
| If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Skin rash | How severe | was you | r skin r | <b>ash</b> in t | he last 2 | 24 hour | s? | | | | |
| □ Yes □ No | | | | | | | | | | | |
| If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Eye | How severe | was you | r <b>eye ir</b> ı | ritation | /discha | <b>rge</b> in t | he last : | 24 hour | s? | | |
| irritation/discharge | | | | | | | | | | | |
| □ <b>Yes</b> □ <b>No</b> If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Diarrhea | How severe | was you | r <b>diarrh</b> | ea in th | e last 2 | 4 hours | ? | | | | |
| ☐ Yes ☐ No | | | | | | | | | | | |
| If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |

| In the last 24 hours, have you experienced | Please rate | e the sev | erity of | each s | ympton | n you e | xperie | nced. | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Vomiting | How severe | e was you | ur <b>vomit</b> | ing in th | ne last 2 | 24 hours | s? | | | | |
| □ Yes □ No | | | | | | | | | | | |
| If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Nausea | How severe | e was yo | ur <b>naus</b> e | a in the | last 24 | hours? | , | | | | |
| □ Yes □ No | | | | | | | | | | | |
| If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| Abdominal/ | | | | | | | | | 0 | | |
| stomach pain | How severe | e was yo | ur <b>abdo</b> i | minai/si | omacn | pain in | i the las | st 24 no | urs? | | |
| □ Yes □ No If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst possible |
| Loss of appetite | How severe | e was yo | ur loss d | of appe | t <b>ite</b> in th | ne last 2 | 24 hours | s? | | | |
| □ Yes □ No | | | | | | | | | | | |
| If yes, → | 0<br>None | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Worst<br>possible |
| What was your <b>highe</b> What method did you | use to take | your tem | nperatur | | ? | °C/°F | | | | | |
| In the last 24 hours, | have you e | xperien | ced | | | | | | | | |
| Uncontrollable body ☐ Yes ☐ No | / shaking/sh | nivering | * | | | | | | | | |
| Degrees de como | | | | | | | | | | | |
| Decreased sense of<br>☐ Yes ☐ No | smeii* | | | | | | | | | | |
| Decreased sense of ☐ Yes ☐ No | taste* | | | | | | | | | | |
| Dad an books at 1 | | * | | | | | | | | | |
| Red or bruised look ☐ Yes ☐ No | ing leet of t | ues" | | | | | | | | | |

| Please rate the severity of your symptoms in the last 24 hours? |
|-----------------------------------------------------------------|
| □ No Symptoms |
| □ Mild |
| □ Moderate |
| □ Severe |

# 10.7. Appendix 7: MRU Questionnaire

As of Amendment 7, this is no longer applicable since the MRU questionnaire will be decommissioned in view of passive follow-up.

#### **Baseline Version**

Participant ID:

Date (dd-mmm-yyyy):

## 1. Medical consultations

In the last 3 months, how many times have you had medical consultations?

| | No | Yes | Type of contact<br>(personal consultation<br>/telemedicine) | If yes,<br>specify the number of<br>visits | Indicate a reason<br>for each visit |
|---|---|---|---|---|---|
| General Practitioner/Nurse practitioner | | | | | |
| Internal Medicine/Medical<br>Outpatient Department | | | | | |
| Other Specialist (Please specify): | | | | | |
| Other (eg Physiotherapy,<br>Pharmacist for a consultation<br>Please specify): | | | | | |

## 2. Professional home care

Please indicate the need for professional care at home in the last 3 months.

| | No | Yes | Type of contact<br>(personal consultation<br>/telemedicine) | If yes,<br>specify the number of<br>visits | Indicate a reason<br>for each type of<br>professional care |
|---|---|---|---|---|---|
| General Practitioner | | | | | |
| Nurse/ Nurse practitioner | | | | | |
| Internal Medicine/Medical<br>Outpatient Department | | | | | |
| Other Specialist (Please | | | | | |
| Other (eg Physiotherapy,<br>Pharmacist Please specify:) | | | | | |
| Supplemental oxygen | | | | | |

## 3. Hospital Services

In the last 3 months, did you visit the hospital?

Yes: No:

| | No | Yes | If yes,<br>specify the number<br>of visits/admissions | If yes,<br>specify the length of<br>each stay/use (days) | Indicate a reason for each hospital visit |
|---|---|---|---|---|---|
| Emergency Department* | | | | | |
| Short-term hospital visit (<24 hours admission) | | | | | |
| Hospitalization in general ward <sup>#</sup> | | | | | |
| Hospitalization in intensive/critical care | | | | | |
| Mechanical ventilation use | | | | | |

<sup>\*</sup>Please count Emergency Department visits only if the visit did not result in a hospital admission.

## 4. Institutional care admission(s) other than hospital

Yes:

No:

Please indicate if there has been any need for admission for care in a long-term facility, in the last 3 months.

| | No | Yes | If yes,<br>specify number of<br>admissions | If yes,<br>specify the length<br>of stay (days) | Indicate a reason for each institutional care admission |
|---|---|---|---|---|---|
| Long-term facilities | | | | | |
| Rehabilitation facility | | | | | |
| Supplemental oxygen | | | | | |

<sup>\*</sup>Please capture type of ward and length of stay in each ward.

## **Version for Confirmed COVID-19 Cases**

Participant ID:

Date (dd-mmm-yyyy):

## 1. Medical consultations

Since onset of the confirmed COVID-19 episode, how many times have you had medical consultations?

| | No | Yes | Type of contact<br>(personal<br>consultation/<br>telemedicine) | If yes,<br>specify the<br>number of visits | Specify number of<br>visits related to<br>COVID-19 or its<br>complications | Indicate a<br>reason for each<br>visit |
|---|---|---|---|---|---|---|
| General Practitioner | | | | | | |
| Internal<br>Medicine/Medical<br>Outpatient Department | | | | | | |
| Other Specialist (Please specify): | | | | | | |
| Other (eg Physiotherapy,<br>Pharmacist for a<br>consultation Please<br>specify:) | | | | | | |

## 2. Professional home care

Please indicate the need for professional care at home since onset of the confirmed COVID-19 episode

| | No | Yes | Type of contact<br>(personal<br>consultation/<br>telemedicine) | If yes,<br>specify the<br>number of<br>visits | Specify number of<br>visits related to<br>COVID-19 or its<br>complications | Indicate a<br>reason for each<br>type of<br>professional<br>care at home |
|---|---|---|---|---|---|---|
| General Practitioner | | | | | | |
| Nurse/ Nurse<br>practitioner | | | | | | |
| Internal<br>Medicine/Medical<br>Outpatient Department | | | | | | |
| Other Specialist (Please specify): | | | | | | |
| Other (eg<br>Physiotherapy,<br>Pharmacist Please<br>specify:) | | | | | | |
| Supplemental oxygen | | | | | | |

#### 3. Hospital Services

Since onset of the confirmed COVID-19 episode, did you visit the hospital?

Yes:

No:

| | No | Yes | of | Specify number of visits/admissions related to COVID-19 or its complications | stay/yea (days) | Indicate a<br>reason for each<br>hospital visit |
|---|---|---|---|---|---|---|
| Emergency Department* | | | | | | |
| Short-term hospital visit (<24 hours admission) | | | | | | |
| Hospitalization in general ward# | | | | | | |
| Hospitalization in intensive/critical care | | | | | | |
| Mechanical ventilation use | | | | | | |

<sup>\*</sup>Please count Emergency Department visits only if the visit did not result in a hospital admission.

## 4. Institutional care admission(s) other than hospital

Please indicate if there has been any need for admission for care in a long-term facility, since onset of the confirmed COVID-19 episode.

Yes:

No:

| | No | Yes | If yes,<br>specify number<br>of admissions | Specify number of admissions related to COVID-19 or its complications | Specify the length of each stay (days) | Indicate a<br>reason for each<br>institutional<br>care admission |
|---|---|---|---|---|---|---|
| Long-term facilities | | | | | | |
| Rehabilitation facility | | | | | | |
| Supplemental oxygen | | | | | | |

<sup>\*</sup>Please capture type of ward and length of stay in each ward.

# 10.8. Appendix 8: Medically-attended COVID-19 (MA-COV) Form

As of Amendment 7, this is no longer applicable since the MA-COV form will be decommissioned in view of passive follow-up.

<u>Section 1</u>: To be completed in all healthcare settings<sup>a</sup> (eg, family doctor, nurse practitioner, outpatient clinic, emergency department visits, and hospitalizations).

| outpatient clinic, emergency department visits, and hospitalization | 18). |
|---|---|
| Participant ID (to be completed by study staff): | |
| Date of visit: | |
| Name and role of healthcare professional completing form: | |
| Contact details for healthcare professional: | |
| DIAGNOSIS/DIAGNOSES | |
| Please list diagnosis/ diagnoses made during the patient's clinical interactions at this facility. | |
| MEDICATIONS | |
| Please list any new medications prescribed or changes in medication dosing. | |
| CLINICAL NARRATIVE INCLUDING COURSE OF INFECTION | |
| COVID-19 DIAGNOSTIC TEST | |
| COVID-19 DIAGNOSTIC TEST | |
| Was a COVID-19 diagnostic test performed? If 'yes' selected, please fill out remaining questions below | □ Yes □ No |
| Specify diagnostic method: | |
| Specify test name and manufacturer: | |
| Date performed: | |
| Type of sample taken:_ | |
| □ Nasal swab sample □ Saliva sample | |
| □ Sputum sample □ Other (specify): | |
| Specify results: | |

<sup>&</sup>lt;sup>a</sup> The MA-COV form should be completed by the medical care provider or study site personnel during medical visits for COVID-19 or COVID-19 complications.

| VITAL SIGNS | | | | |
|---|---|---|---|---|
| Has vital sign assessment been performed? | | | | |
| □ Yes □ No | | | | |
| l les l No | | | | |
| Temperature (°C/°F): | | | | |
| Posnivatowy votos | | | | |
| Respiratory rate: | | | | |
| Pulse: | | | | |
| Systolic and Diastolic Blood Pressure: | | | | |
| Oxygen saturation: | | | | |
| Does the subject have a clinically abnormal oxygen saturation? | | | | |
| □ Yes □ No | | | | |
| If yes, is the oxygen saturation adjusted for altitude per the investigator judgement: | | | | |
| □ ≤93% □ >93% | | | | |
| 253/0 1 253/0 | | | | |
| | | | | _ |
| DIAGNOSTIC TESTING Was a real flow massworment mode? | _ | Yes | | No |
| Was a peak flow measurement made? | Ш | res | Ц | NO |
| If yes, please indicate date performed: | | | | |
| Peak flow (L/min): | | | | |
| Teak now (Limin). | | | | |
| Was a chest X-ray and/or CT performed? | | Yes | | No |
| If yes, please indicate date performed: | | | | |
| What percentage of the lung was involved? | | | | |
| . 12 9 | | | | 027 |
| Was an arterial blood gas measured? | | Yes | | No |
| If yes, please indicate date performed: | | | | |
| South Miles Miles | | | | |
| Specify results:<br>pH:; pCO <sub>2</sub> (mmHg):; pO <sub>2</sub> (mmHg):; HCO <sub>3</sub> (mEq/L):; O <sub>2</sub> satur | ation | (%). | | |
| ри, реодининду, родининду, неозиници, одзаки | auon | (/0). | | |
| Were additional diagnostic tests performed? | | Yes | | No |
| If yes, please specify diagnostic method: | | | | |
| Date performed: | | | | |

Specify results:

| SIGNS | SIGNS AND SYMPTOMS | | | |
|---|---|---|---|---|
| In case | In case the severity and/or start and/or end date of any of the experienced signs and symptoms are known, please | | | |
| indicate | | | | |
| Did the | patient experience any of these ever | nts, signs or symptoms? | | |
| • | | | 0.000 | rate ≥30 breaths/minute or heart rate |
| | ≥125 beats/minute or SpO2 ≤93%<br>□ Yes □ No | on room air at sea level <sup>a</sup> or Pa | aO2/ | FiO2 <300 mmHg) |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | -20 | |
| • | Respiratory failure requiring high | h-flow oxygen, non-invasive ve | ntila | tion, mechanical ventilation, or ECMO |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | | |
| • | Respiratory rate ≥20 breaths/min □ Yes □ No | ute | | |
| | Severity: Mild | □ Moderate | | Severe |
| | Start date: | □ End date: | | |
| • | Shortness of breath Yes No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | 21 | |
| • | Heart rate ≥90 beats/minute □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | -22 | |
| | Shock (systolic blood pressure <90 | 0 mm Hg, or diastolic blood pr | essu | re <60 mm Hg or requiring vasopressors) |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | | |
| • | Radiologic evidence of DVT Ves No | | | |
| | No. | □ Moderate | | Severe |
| | □ Start date: | □ End date: | - | |
| • | Significant acute renal or hepatic □ Yes □ No | dysfunction | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | -0 | |
| • | Hyperinflammatory Syndrome | | | |
| | □ Yes □ No | = Madaust | 0.000 | Savana |
| | Severity: Mild | | | Severe |
| | □ Start date: | □ End date: | =0 | |

| SIGNS | AND SYMPTOMS | | | |
|-------|-----------------------------------|---------------|-----|--------|
| • | Symptoms or signs of stroke | | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | Start date: | □ End date: | _ | |
| | Numbness, tingling, or weakness | face or limbs | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | | |
| - | Difficulty speaking or forming sp | eech | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | | |
| | Difficulty understanding speech | | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | | |
| • | Feelings of confusion | | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | -0 | |
| • | Clinical or radiological evidence | of pneumonia | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | 5.1 | |
| | Fever (≥38.0°C or ≥100.4°F) | | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | -> | |
| • | Shaking chills or rigors | | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | Start date: | □ End date: | - | |
| • | Cough | | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | Start date: | □ End date: | •) | |
| • | Sore throat | | | |
| | □ Yes □ No | | | |
| | Severity: Mild | □ Moderate | | Severe |
| | □ Start date: | □ End date: | | |

 $^{\text{a}}$   $\text{SpO}_2$  criteria will be adjusted according to altitude per investigator judgement.

| SIGNS | AND SYMPTOMS | | | | · |
|---|---|---|---|---|---|
| • | Malaise | | | | |
| | □ Yes □ No | | | | |
| | Severity: Mild | □ Moderate | | Severe | |
| | Start date: | □ End date: | | | |
| | Headache | | | | |
| | □ Yes □ No | | | | |
| | Severity: Mild | □ Moderate | | Severe | |
| | □ Start date: | □ End date: | | | |
| • | Myalgia | | | | |
| | □ Yes □ No | | | | |
| | Severity: Mild | □ Moderate | | Severe | |
| | □ Start date: | □ End date: | | | |
| • | Gastrointestinal symptoms | | | | |
| | □ Yes □ No | | | | |
| | Severity: Mild | □ Moderate | | Severe | |
| | □ Start date: | □ End date: | | | |
| • | Chilblains/pernio (red or bruise | ed looking feet or toes) | | | |
| | □ Yes □ No | | | | |
| | Severity: Mild | □ Moderate | | Severe | |
| | □ Start date: | □ End date: | | | |
| • | Anosmia (olfactory or taste disc | orders) | | | |
| | □ Yes □ No | | | | |
| | Severity: Mild | □ Moderate | | Severe | |
| | □ Start date: | □ End date: | | | |
| MANA | GEMENT | | | | |
| ANY T | YPE OF MANAGEMENT OTHE | ER THAN MEDICATION? | | | □ Yes □ No |
| If yes, p | please specify: | | | | |
| | Nebulizer treatments | | | | |
| | □ Yes □ No | | | | |
| | IV fluids | | | | |
| | □ Yes □ No | | | | |
| | Intubation | | | | |
| | □ Yes □ No | | | | |
| 18. | | | | | |
| Section | 2: COVID-19-related Pro | ocedures completed du | ring the | event. | |
| | | | - | | |

| SUPPLEMENTAL OXYGEN | | | |
|---|---|---|---|
| Was supplemental oxygen administered? | | Yes | □ No |
| If 'yes' selected, please fill out remaining questions in this section. | | | |
| Type of supplemental oxygen administration: | | | |
| □ Invasive Mechanical Ventilation | □ Venturi Mask | | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| SUPPLEMENTAL OXYGEN | |
|---|---|
| □ Non-Invasive Mechanical Ventilation | □ Simple Face Mask |
| Nasal Cannula | Reservoir Cannulas |
| □ Nonrebreathing Face Mask with Reservoir and One-Way Valve | Reservoir Camillas |
| Nonrepreaching Pace Mask with Reservoir and One-way valve | |
| Other: | |
| If invasive mechanical ventilation, specify: | |
| ☐ Through endotracheal tube ☐ Through tracheostomy | v tube |
| If non-invasive mechanical ventilation, specify: | |
| □ Continuous positive airway pressure □ Bilevel positive airway | pressure |
| Oxygen concentration and units: | |
| Start data and times | |
| Start date and time: | |
| End date and time (if applicable): | |
| End date and time (if applicable). | |
| Has supplemental oxygen administration returned to that level provided p | rior to the current respiratory illness? |
| □ Yes □ No | Harder 1 - State (Anthon Control of the State (Anthon Sta |
| DIALYSIS | |
| Was dialysis performed? | □ Yes □ No |
| was dialysis per for med: | □ 1es □ No |
| If yes, please specify: | |
| Tryes, preuse speen, | |
| ANY OTHER PROCEDURES PERFORMED | |
| Were any other procedures for COVID-19 performed? | |
| Yes No | |
| 163 U NO | |
| If yes, please specify: | |
| Procedure: | |
| Reason performed: | |

# 10.9. Appendix 9: Toxicity Grading Scale

Adapted from the FDA Guidance document "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" (September 2007)

| Local Reaction to<br>Injectable Product | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Pain/Tenderness# | Aware of symptoms<br>but easily tolerated;<br>Does not interfere<br>with activity;<br>Discomfort only to<br>touch | Notable symptoms;<br>Requires modification<br>in activity or use of<br>medications;<br>Discomfort with<br>movement | Incapacitating<br>symptoms;<br>Inability to do work,<br>school, or usual<br>activities; Use of<br>narcotic pain reliever | Hospitalization;<br>Pain/tenderness<br>causing inability to<br>perform basic self-<br>care function |
| Erythema# | 25 – 50 mm | 51 – 100 mm | >100 mm | Hospitalization;<br>Necrosis or<br>exfoliative dermatitis |
| Swelling <sup>#</sup> | 25 – 50 mm | 51 – 100 mm | >100 mm | Hospitalization;<br>Necrosis |

<sup>#</sup> Revised by the sponsor.

| Vital Signs * | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Fever (°C) **<br>(°F)** | 38.0 - 38.4<br>100.4 - 101.1 | 38.5 - 38.9<br>101.2 - 102.0 | 39.0 - 40.0<br>102.1 - 104.0 | >40<br>>104.0 |
| Tachycardia - beats<br>per<br>minute | 101 – 115 | 116 – 130 | >130 | Hospitalization for arrhythmia <sup>#</sup> |
| Bradycardia - beats<br>per<br>minute*** | 50 – 54 | 45 – 49 | <45 | Hospitalization for arrhythmia <sup>#</sup> |
| Hypertension<br>(systolic) - mm Hg | 141 – 150 | 151 – 155 | >155 | Hospitalization for malignant hypertension# |
| Hypertension<br>(diastolic) - mm Hg | 91 – 95 | 96 – 100 | >100 | Hospitalization for malignant hypertension# |
| Hypotension<br>(systolic) – mm Hg | 85 – 89 | 80 – 84 | <80 | Hospitalization for hypotensive shock <sup>#</sup> |
| Respiratory Rate – breaths per minute | 17 – 20 | 21 – 25 | >25 | Intubation |

<sup>\*</sup> Participant should be at rest for all vital sign measurements.

<sup>\*\*</sup> For oral temperature: no recent hot or cold beverages or smoking.

<sup>\*\*\*</sup> When resting heart rate is between 60 - 100 beats per minute. Use clinical judgement when characterizing bradycardia among some healthy participant populations, for example, conditioned athletes.

<sup>#</sup> Revised by the sponsor.
| Systemic (General) | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Vomiting <sup>#</sup> | No interference with activity or 1 – 2 episodes/24 hours | Some interference with activity or >2 episodes/24 hours | Prevents daily<br>activity, requires<br>outpatient IV<br>hydration | Hospitalization;<br>Hypotensive shock |
| Nausea <sup>#</sup> | Minimal symptoms;<br>causes minimal or no<br>interference with<br>work, school, or self-<br>care activities | Notable symptoms;<br>Requires modification<br>in activity or use of<br>medications;<br>Does NOT result in<br>loss of work, school,<br>or cancellation of<br>social activities | Incapacitating<br>symptoms;<br>Requires bed rest<br>and/or results in loss<br>of work, school, or<br>cancellation of social<br>activities | Hospitalization;<br>Inability to perform<br>basic self-care<br>functions |
| Diarrhea# | 2 – 3 loose stools or<br><400 gms/24 hours | 4 – 5 stools or<br>400 – 800 gms/24<br>hours | 6 or more watery<br>stools or<br>>800 gms/24 hours or<br>oral rehydration<br>necessary | Hospitalization;<br>Hypotensive shock<br>OR IV fluid<br>replacement indicated |
| Headache# | Minimal symptoms;<br>causes minimal or no<br>interference with<br>work, school, or self-<br>care activities | Notable symptoms;<br>Requires modification<br>in activity or use of<br>medications;<br>Does NOT result in<br>loss of work, school,<br>or cancellation of<br>social activities | Incapacitating symptoms; Requires bed rest and/or results in loss of work, school, or cancellation of social activities; Use of narcotic pain reliever | Hospitalization;<br>Inability to perform<br>basic self-care<br>functions |
| Fatigue# | Minimal symptoms;<br>causes minimal or no<br>interference with<br>work, school, or self-<br>care activities | in activity or use of medications; Does NOT result in loss of work, school, | Incapacitating symptoms; Requires bed rest and/or results in loss of work, school, or cancellation of social activities; Use of narcotic pain reliever | Hospitalization;<br>Inability to perform<br>basic self-care<br>functions |
| Myalgia <sup>#</sup> | Minimal symptoms;<br>causes minimal or no<br>interference with<br>work, school, or self-<br>care activities | Notable symptoms;<br>Requires modification<br>in activity or use of<br>medications;<br>Does NOT result in<br>loss of work, school,<br>or cancellation of<br>social activities | Incapacitating symptoms; Requires bed rest and/or results in loss of work, school, or cancellation of social activities; Use of narcotic pain reliever | Hospitalization;<br>Inability to perform<br>basic self-care<br>functions |

<sup>#</sup> Revised by the sponsor.

| Systemic Illness | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Illness or clinical<br>adverse<br>event (as defined<br>according to<br>applicable<br>regulations) | No interference with activity | Some interference<br>with activity not<br>requiring medical<br>intervention | Prevents daily<br>activity and<br>requires medical<br>intervention | Hospitalization <sup>#</sup> |

<sup>#</sup> Revised by the sponsor.

# 10.10. Appendix 10: Symptoms of Coronavirus (US Centers for Disease Control and Prevention)

The following extract shows symptoms of coronavirus infection as listed on the US CDC website (https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html) dated 13 May 2020:

# Watch for symptoms

People with COVID-19 have had a wide range of symptoms reported – ranging from mild symptoms to severe illness. Symptoms may appear **2-14 days after exposure to the virus.** People with these symptoms may have COVID-19:

- · Fever or chills
- Cough
- · Shortness of breath or difficulty breathing
- Fatigue
- · Muscle or body aches
- Headache
- · New loss of taste or smell
- · Sore throat
- · Congestion or runny nose
- · Nausea or vomiting
- Diarrhea

This list does not include all possible symptoms. CDC will continue to update this list as we learn more about COVID-19.

# 10.11. Appendix 11: Summary of Guidance from CDC Website on Underlying Medical Conditions That Lead or Might Lead to Increased Risk for Severe Illness From COVID-19

People of any age with **certain underlying medical conditions** are at increased risk for severe illness from COVID-19:

People of any age with the following conditions **are at increased risk** of severe illness from COVID-19:

- Cancer
- Chronic kidney disease
- COPD (chronic obstructive pulmonary disease)
- Immunocompromised state (weakened immune system) from solid organ transplant
- Obesity (body mass index [BMI] of 30 or higher)
- Serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies
- Sickle cell disease
- Type 2 diabetes mellitus

COVID-19 is a new disease. Currently there are limited data and information about the impact of underlying medical conditions and whether they increase the risk for severe illness from COVID-19. Based on what we know at this time, people with the following **conditions might be at an increased risk** for severe illness from COVID-19:

- Asthma (moderate to severe)
- Cerebrovascular disease (affects blood vessels and blood supply to the brain)
- Cystic fibrosis
- Hypertension or high blood pressure
- Immunocompromised state (weakened immune system) from blood or bone marrow transplant, immune deficiencies, HIV, use of corticosteroids, or use of other immune weakening medicines
- Neurologic conditions, such as dementia
- Liver disease
- Pregnancy
- Pulmonary fibrosis (having damaged or scarred lung tissues)
- Smoking
- Thalassemia (a type of blood disorder)
- Type 1 diabetes mellitus

Source: https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/people-with-medical-conditions.html?CDC AA refVal=https%3A%2F%2Fwww.cdc.gov%2 Fcoronavirus% 2F2019-ncov%2Fneed-extra-precautions%2Fgroups-at-higher-risk.html. Accessed: 19 July 2020.

# 10.12. Appendix 12: Risk Factor Assessment

As of Amendment 7, this is no longer applicable since risk factor assessment will be terminated in view of passive follow-up.

| Are you a student? ☐ Yes ☐ No |
|---|
| If Yes Are you likely to return to school in person in the near future? |
| Are you retired? |
| How often do you go in person to your main workplace (other than work from home)? □ 0 days/week □ 1 day/week □ 2 4 days/week □ 5 or more days/week |
| Does your main workplace have social distancing measures in place? |
| ☐ Yes ☐ No ☐ I don't know ☐ Not applicable |
| Is your main workplace cleaned on a regular basis? |
| ☐ Yes ☐ No ☐ I don't know ☐ Not applicable |
| Do people in your main workplace use personal protection equipment (such as masks)? ☐ Yes ☐ No ☐ I don't know ☐ Not applicable |
| How do you get to work? (Check all that apply) |
| ☐ Drive own car ☐ Carpool ☐ Rideshare (Taxi, Uber, Lyft, others) |
| ☐ Bus ☐ Train / Subway ☐ Walk / Bike |
| ☐ Frequent Air Travel ☐ Not applicable |
| On a typical day, how many people do you interact with in person at work? |
| ☐ No one ☐ Between 1 and 10 people ☐ Between 11 and 30 people ☐ Between 31 and 50 people |
| ☐ More than 50 people ☐ Between 31 and 30 people |
| On a typical day, how many people do you interact with in person outside of work? |
| □ No one □ Between 1 and 10 people |
| ☐ Between 11 and 30 people ☐ Between 31 and 50 people |
| ☐ More than 50 people |
| Living Situation Decree Virginia and 6th of Hamilton (all and all the translation) |
| Do you live in any of the following (choose all that apply): ☐ Single family home ☐ Multi family housing (apartment building, condo) |
| ☐ Long term care facility ☐ Assisted living facility |
| ☐ Dormitory ☐ RV / Trailer |
| ☐ Single room in a hotel ☐ Shelter |
| ☐ Other adult group setting ☐ Staying with friends / Couch surfing |
| ☐ No residence ☐ Tribal Lands / Reservation |
| □ Other |
| How many people do you live with (other than yourself)? |
| Total people under 18 years of age Total people between 18 64 years of age |
| Total people over 65 years of age |
| Are any of the people you live with expected to return to school in person in the near future? |
| ☐ Yes ☐ No ☐ I don't know |
| Community Interactions In the last 2 weeks, have you attended any gatherings with more than 10 people? (e.g., church, party, concert, wedding, funeral, demonstration |
| or other event). Yes No Not applicable / Don't want to tell |
| If yes, approximately how many people were at the largest gathering? |
| □ less than 10 □ 10 20 □ 21 50 □ 51 250 □ More than 250 |
| Was this gathering an indoor or outdoor event? |
| ☐ Indoor ☐ Outdoor ☐ Both |
| How frequently do you have <u>visitors</u> in your residence including people completing work inside? □ Daily |
| □ Weekly |
| ☐ Monthly |
| Rarely |
| □ Never |
| □ N/A |
| Over the past month, have you been in close contact with anyone that tested positive for COVID 19? |
| ☐ Yes ☐ No ☐ I don't know ☐ Not applicable / Don't want to tell If yes, is this person someone that you live with? |
| ☐ Yes ☐ No ☐ Not applicable / Don't want to tell |
| 11 |

# 10.13. Appendix 13: TTS AESI Form

The form below represents the type of information that may be collected in case of a suspected AESI to help adjudicate whether the event is a case of TTS. Additional data may be requested by the sponsor for investigation of the event.

Adverse Event of Special Interest Questionnaire (AESIQ) for Thromboembolism with Thrombocytopenia Syndrome

| Date of Report: | [dd-MMM | -уууу] | |
|---|---|---|---|
| 1. Adverse Event De | escription | | |
| Participant's cli | nical signs | s and symptoms | |
| Leg/Calf Oed | ema | ☐ Pain in Leg/Calf | ☐ Haemoptysis |
| ☐ Dyspnoea | | ☐ Chest Pain/Discomfort | ☐ Syncope |
| ☐ Tachypnoea | | ☐ Tachycardia | ☐ Cough |
| Loss of consc | ciousness | Headache | ☐ Seizure |
| ☐ Visual impairr | ment | ☐ Weakness | Impaired speech |
| ☐ Confusional s | tate | ☐ Paresthesia | ☐ Gait disturbance |
| ☐ Other sympto | ms: | | |
| Was patient on V | /TE prophy | laxis? | ails: |

#### 2. Medical History and Concurrent Conditions

| Provide details: | |
|---|---|
| Is the participant overweight or have obesity? If available, please provide: Does the participant have a sedentary lifestyle <sup>a</sup> ? Has the participant been in a sitting position for long periods of time prior to the event? | ☐ No ☐ Yes Weight BMI ☐ No ☐ Yes – details: ☐ No ☐ Yes – details: |
| Is there a current history of smoking (active or passive)? Is there a prior history of smoking (active or passive)? | No Yes – details: No Yes – details: |
| | To Tos – details. |
| Does the participant have a prior history of: Cancer | ☐ No ☐ Yes – details: |
| Autoimmune disease (ie, collagen-vascular disease, inflammatory bowel disease) or myeloproliferative disease? | ☐ No ☐ Yes – details: |
| Clotting disorder or a hypercoagulable state Varicose veins | □ No □ Yes – details: |
| Trauma to the involved leg or pelvis | <ul><li>No ☐ Yes – details:</li><li>No ☐ Yes – details:</li></ul> |
| DVT/PE or other VTE | ☐ No ☐ Yes – details: |
| Blood transfusion | ☐ No ☐ Yes – details: |
| Cardiovascular disease | ☐ No ☐ Yes – details: |
| If the participant has experienced a previous thrombotic ever 1. Date (or estimate) 2. Provide brief description of the nature of the event 3. Provide brief description of the treatment of the event 4. Note any residual manifestations of the event. | nt, address the following: |
| If the participant has experienced more than one previous the events. | rombotic event, please list other |
| Was the (female) participant pregnant at the time of event? | ☐ No ☐ Yes – details: |
| Does the participant have any genetic risk factors: | |
| □ Dysfibrinogenemia □ Antiphospholipid syndrome □ Factor V Leiden mutation □ Protein C or S deficiency □ Elevated factor VIII levels □ Anti-thrombin deficiency □ Hyperhomocysteinemia □ Prothrombin gene mutation □ Blood-clotting disorder □ Thrombophilia | |
| Does the participant have any acquired risk factors: | |
| <ul> <li>☐ Reduced mobility (paralysis, paresis, travel etc.)</li> <li>☐ Recent surgery</li> <li>☐ Indwelling central venous catheters</li> <li>☐ Recent trauma</li> <li>☐ Recent discontinuation of anticoagulants (eg, heparin, warfarin, DOACs)</li> <li>☐ Hormone replacement therapy (including contraceptives)</li> <li>☐ Phlebitis</li> <li>☐ Lupus</li> </ul> | |

<sup>&</sup>lt;sup>a</sup> Any waking behavior characterized by an energy expenditure less than or equal to 1.5 metabolic equivalents (METs), while in a sitting, reclining, or lying posture

| VAC31518 (JNJ-78436735) | Clinical Protocol VAC31518COV3001 Amendment 7 |
|---|---|
| ☐ Inflammatory bowel disease | ☐ Myeloproliferative disorders |
| ☐ Diabetes mellitus | ☐ Hyperlipidemia |
| Hypertension | ☐ Dehydration |
| Other significant medical comorbidities or risk fac | ctors for DVT, specify: |
| If yes to any of the above, provide details: | |
| Provide Well's score, if calculated: | |

3. Relevant results of diagnostic tests including laboratory tests, imaging, biopsies, etc. (Note the levels/conclusion, date performed, normal ranges as well as any other details. Alternatively, attach full reports of the diagnostic tests).

| Diagnostic Test | Results at baseline or prior to use of product (Include date and value/details) | Test results after use of<br>product (Include date<br>and value/details) |
|---|---|---|
| CBC with smear (microscopic evaluation) | | |
| ESR | | |
| Platelet count | | |
| Antibodies to platelet factor 4 (PF4) | | |
| Fibrinogen levels | | |
| Clauss fibrinogen assay | | |
| D-Dimer | | |
| Clotting Profile (PT, aPTT- prior to an anticoagulation treatment) | | |
| Thrombin time (Bovine) Plasma | | |
| Prothrombin | | |
| Antithrombin activity | | |
| Factor V Leiden | | |
| Protein C activity | | |
| Protein S activity | | |
| C-reactive protein | | |
| Homocystein levels | | |
| Dilute Russells Viper Venom<br>Time (DRVVT), Plasma | | |
| Activated Protein C Resistance V (APCRV), Plasma | | |
| Thrombophilia interpretation | | |
| Anticardiolipin antibodies (IgG and IgM) or beta-2 glycoproteins antibodies | | |

| Diagnostic Test | Results at baseline or prior<br>to use of product (Include<br>date and value/details) | Test results after use of<br>product (Include date<br>and value/details) |
|---|---|---|
| Antiphospholipid antibodies (IgG and IgM) | | |
| Lupus anticoagulant | | |
| Heparin antibodies | | |
| ANA and ANCA | | |
| IL6 levels | | |
| ADAMTS13 Activity Assay | | |
| Ceruloplasmin | | |
| Direct Coombs test | | |
| Complement C3, C4 | | |
| MethylenetetraHydrofolate reductase gene mutation | | |
| Prothrombin gene mutation (G20210A) | | |
| Occult blood in stool | | |
| COVID-19 test | | |
| Troponins | | |
| Brain Natriuretic Peptide | | |
| Arterial Blood Gases | | |
| Chest X-Ray | | |
| Electrocardiography | | |
| Echocardiography | | |
| Duplex Ultrasonography | | |
| MRI scan | | |
| CT scan | | |
| Contrast Venography | | |
| Pulmonary Angiography | | |
| Ventilation-Perfusion Scanning | | |

Provide details of any additional diagnostic results:

#### 10.14. Appendix 14: Thrombotic Events to be Reported as AESIs

At the time of protocol Amendment 5 writing, the list of thrombotic events to be reported to the sponsor as suspected AESIs is provided below. Further guidance may become available on thrombotic events of interest.

- MedDRA PTs for large vessel thrombosis and embolism:
  - Aortic embolus, aortic thrombosis, aseptic cavernous sinus thrombosis, brain stem embolism, brain stem thrombosis, carotid arterial embolus, carotid artery thrombosis, cavernous sinus thrombosis, cerebral artery thrombosis, cerebral venous sinus thrombosis, cerebral venous thrombosis, superior sagittal sinus thrombosis, transverse sinus thrombosis, mesenteric artery embolism, mesenteric artery thrombosis, mesenteric vein thrombosis, splenic artery thrombosis, splenic embolism, splenic thrombosis, thrombosis mesenteric vessel, visceral venous thrombosis, hepatic artery embolism, hepatic artery thrombosis, hepatic vein embolism, hepatic vein thrombosis, portal vein embolism, portal vein thrombosis, portosplenomesenteric venous thrombosis, splenic vein thrombosis, spontaneous heparin-induced thrombocytopenia syndrome, femoral artery embolism, iliac artery embolism, jugular vein embolism, jugular vein thrombosis, subclavian artery embolism, subclavian vein thrombosis, obstetrical pulmonary embolism, pulmonary artery thrombosis, pulmonary thrombosis, pulmonary venous thrombosis, renal artery thrombosis, renal embolism, renal vein embolism, renal vein thrombosis, brachiocephalic vein thrombosis, vena cava embolism, vena cava thrombosis, truncus coeliacus thrombosis
- MedDRA PTs for more common thrombotic events:
  - Axillary vein thrombosis, deep vein thrombosis, pulmonary embolism, MedDRA PTs for acute myocardial infarction\*, MedDRA PTs for stroke\*

Source: Shimabukuro T. CDC COVID-19 Vaccine Task Force. Thrombosis with thrombocytopenia syndrome (TTS) following Janssen COVID-19 vaccine. Advisory Committee on Immunization Practices (ACIP). April 23, 2021. https://www.cdc.gov/vaccines/acip/meetings/slides-2021-04-23.html.

\*Vaccine Adverse Event Reporting System (VAERS) Standard Operating Procedures for COVID-19 (as of 29 January 2021) https://www.cdc.gov/vaccinesafety/pdf/VAERS-v2-SOP.pdf

#### 10.15. Appendix 15: Protocol Amendment History

The Protocol Amendment Summary of Changes Table for the current amendment is located directly before the Table of Contents (TOC).

### Amendment 6 (04 September 2021)

Overall Rationale for the Amendment: The main purpose of this amendment is to offer a 1-dose booster vaccination with Ad26.COV2.S at the 5x10<sup>10</sup> vp dose level to all ongoing participants in the study, regardless of their primary vaccination regimen (Ad26.COV2.S vaccine or a single or two dose regimen of an mRNA vaccine or another authorized COVID-19 vaccine including protein, inactivated, and adenovector based vaccines). The booster vaccination will be administered in the open-label phase of the study. The combination of homologous or heterologous prime/boost vaccination will not be randomized, but depend on what participants received during the double-blind phase of the study as described in this protocol. Booster vaccination should occur preferably 6 months but at least 3 months after the primary vaccination regimen. Participants in the study who have already received an additional COVID-19 vaccination after the primary regimen outside the study with any vaccine as described above will also be eligible for the Ad26.COV2.S booster in this study preferably 6 months but at least 3 months after their last COVID-19 vaccination. Participants are free to choose when to receive the booster vaccination within the window of the booster vaccination visit, to receive booster vaccination outside the study, or not to receive booster vaccination. Participants who choose to receive a booster vaccination with the Ad26.COV2.S vaccine (if recommended and available) or another authorized COVID-19 vaccine outside the study or choose not to receive a booster vaccination will not be withdrawn from the study and will be encouraged to remain in the study. All participants who received a booster vaccination within the study or received a booster vaccination outside the study and remained in the study will be monitored for safety, immunogenicity, and efficacy. Immunogenicity will be assessed with blood draws on the day of booster vaccination (prior to booster vaccination, if feasible), and 28 days, 72 days, and 6 months post booster vaccination. In addition, immunogenicity subsets with more extensive blood draws for immunogenicity assessments will be included. Safety blood draws will include a platelet count at Baseline (prior to booster vaccination, if feasible), and 28 days after booster vaccination and extra blood, aside from that required for immunogenicity and N serology for determination of infection, to assess relevant parameters in case of an adverse event of interest. With implementation of this amendment, the start date of the first cross-over unblinding visit (implemented with Amendment 4) and the date of first booster vaccine administration until 1-year follow-up of the last booster vaccination define the open-label booster vaccination phase of the study. This phase will be utilized to describe safety, immunogenicity, and efficacy during the time participants have and have not been boosted.

Rationale: A single dose of Ad26.COV2.S vaccine is immunogenic and highly efficacious against severe COVID-19 disease and COVID-19 related hospitalization and death for at least 8 months. Despite this durability, signs of waning immunity in terms of the numbers of participants with undetectable antibody have been observed, especially in the older population, where as many as 28% have no detectable neutralizing antibody at 6 months post vaccination. Furthermore, while protection against variants of concern such as the Beta variant, the Gamma variant, and the B.1.621

variant in this study<sup>24</sup> and the Delta variant in the Sisonke study remains high against serious disease, hospitalization, and death, this protection is somewhat lower against, for example, the Delta variant compared to the reference Wuhan strain.<sup>38</sup> Protection against mild to moderate disease against the Delta variant is very low at the late time points when measured in the Sisonke study, although it is unknown if this is due to waning immunity or biologic factors related to the Delta variant. Waning immune responses and less protection against moderate to severe disease against the Delta variant has also been observed for mRNA vaccines. Based on these findings, regulatory and advisory bodies including the FDA are planning to recommend booster doses for vaccines when data supports such recommendations. Therefore, based on this recommendation for a booster vaccination and the availability of booster vaccinations outside the study, this amendment will permit boosting of all ongoing participants in this study who have previously received any COVID-19 vaccine(s) (either as part of a primary regimen or as an additional dose administered after the primary regimen). All participants who received vaccination with Ad26.COV2.S, an mRNA vaccine and/or another COVID-19 vaccine authorized for primary vaccination, if the last vaccination was preferably 6 months but at least 3 months ago, and who subsequently remained in the study will be eligible to receive the booster.

These and other changes made to the clinical protocol of study VAC31518COV3001 are listed below, including the rationale for each change and a list of all applicable sections.

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | |
| 1.1 Synopsis | At the 1 Year visit, all ongoing | See overall rationale for |
| 1.2 Schema | participants who have previously | amendment. |
| 1.3.1 Schedule of Activities "All | received any COVID-19 vaccination(s) | |
| Participants" | (as primary regimen or additional dose) | |
| 2.1 Study Rationale | with Ad26.COV2.S, an mRNA vaccine | |
| 2.3.3 Benefit-Risk Assessment of | and/or another for primary vaccination | |
| Study Participation | authorized protein, inactivated, or | |
| 4.1 Overall Design | adenovector based vaccine will be offered | |
| 5 STUDY POPULATION | a single booster dose of Ad26.COV2.S | |
| 5.5 Criteria for Temporarily Delaying | vaccine $(5 \times 10^{10} \text{ vp})$ if the last vaccination | |
| Administration of Study Vaccination | was preferably 6 months but at least | |
| 6.1 Study Vaccines Administered | 3 months ago. | |
| 6.2 Preparation/Handling/Storage/ | | |
| Accountability | The window of the 1 Year visit has been | |
| 6.8 Continued Access to Study Vaccine | widened to allow booster vaccination as | |
| After the End of the Study | of approximately $\geq 3$ months following | |
| 8 STUDY ASSESSMENTS AND | the last previous COVID-19 vaccination. | |
| PROCEDURES | | |
| 8.1.3 Efficacy Assessments | A visit 28 days post booster vaccination | |
| 8.1.3.5 SARS-CoV-2 Seroconversion | has been added for all participants who | |
| Assessment | received a booster vaccination at the | |
| 8.1.4 Immunogenicity Assessments | Year 1/Booster Visit for follow up of | |
| 8.2.3 Pregnancy Testing | safety and immunogenicity, and 72 days | |
| 8.3.1 Time Period and Frequency for | post booster vaccination for follow up of | |
| Collecting Adverse Event, Medically- | immunogenicity. Immunogenicity | |
| attended Adverse Event, Adverse | subsets (a total of 600 participants) with | |
| Events of Special Interest, and Serious | more extensive blood draws for | |
| Adverse Event Information | immunogenicity assessments were added. | |
| 8.3.5 Pregnancy | | |

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| 8.10 Assessments and Procedures Related to Booster Vaccination 9.2.2 Immunogenicity Subset (Double-blind Phase and Booster Vaccination 10.1 Appendix 1: Abbreviations 10.2 Appendix 2: Clinical Laboratory | A visit 1 day post booster vaccination has been added for additional immunogenicity and safety assessment for a subgroup of the immunogenicity subsets (120 participants). | |
| Test 10.3.3 Informed Consent Process | The timing of the Month 18 and Year 2 visits have been adjusted to accommodate 6- and 12-months follow-up for participants who received booster vaccination at the Year 1/Booster Visit. | |
| | An additional urine pregnancy test at the Year 1/Booster Visit was added for participants of childbearing potential who choose to receive booster vaccination. | |
| | Added that a new ICF needs to be signed at the Year 1/Booster Visit. | |
| 1.1 Synopsis 3.2 Booster Vaccination | Objectives & Endpoints were added for the open-label booster vaccination phase of the study. | To obtain information regarding the safety, immunogenicity, and efficacy of a booster vaccination. |
| 6.5 Booster Vaccination | Describes the conditions under which participants may receive booster vaccination. | To provide appropriate guidance. |
| 1.1 Synopsis 1.3.1 Schedule of Activities "All Participants" 8.1.4 Immunogenicity Assessments 9.8.1 Immunogenicity Subset (Openlabel Booster Vaccination Phase) | Immunogenicity subsets (Homologous Booster Subset and Heterologous Booster Subset) were added for the open-label booster vaccination phase of the study. Of the total 600 participants with extensive blood draws for immunogenicity, 200 participants will be from the Homologous Booster Subset and 400 from the Heterologous Booster Subset. | To investigate the magnitude and kinetics of the humoral response induced by a booster dose of Ad26.COV2.S vaccine in participants who received homologous Ad26.COV2.S primary vaccination or heterologous primary vaccination with an mRNA, protein, inactivated or adenovector based vaccine. |
| | Of the 120 participants with additional immunogenicity and safety assessment at the visit 1 day post booster vaccination 60 will be from the Homologous Booster Subset and 60 from the Heterologous Booster Subset. | |
| 1.1 Synopsis 9 STATISTICAL CONSIDERATIONS 9.2.1 Efficacy (Total Sample Size) 9.8 Analysis of the Open-label Booster Vaccination Phase 9.8.1 Immunogenicity Subset (Open-label Booster Vaccination Phase) 9.8.2 Immunogenicity Correlates | Statistical considerations for the analysis of the open-label booster vaccination phase were added. It was clarified that Sections 9.1 to 9.7 are only applicable to the double-blind phase of the study. Text was added to indicate that details of | To describe the statistical considerations of the open-label booster vaccination phase. |
| (Correlates Subset) 9.8.3 Efficacy Analyses | the statistical analysis of the open-label | |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | booster vaccination phase will be specified in a separate SAP. It was clarified that no additional participants will be recruited for the open- | |
| | label phase. It was clarified that analysis of the open-label booster vaccination phase data is planned to be performed 6 months and 1 year after all participants were offered the booster vaccination. Additional analyses may be conducted to support health authority interactions and/or based on public health demand in case of emerging variants. | |
| 2.3.1 Risks Related to Study Participation | It was added that no clinical data are available for Ad26.COV2.S administration after previous vaccination with a COVID-19 vaccine other than Ad26.COV2.S. Available clinical information on the administration of an Ad26.COV2.S booster vaccination following a single dose Ad26.COV2.S was added. | To update the potential risks. |
| | Text was added that participants who are pregnant may receive booster vaccination with Ad26.COV2.S, if allowed by local regulations and if the investigator considers that the potential benefits outweigh the potential risks to the mother and fetus. | |
| 1.3.1 Schedule of Activities "All<br>Participants"<br>8 STUDY ASSESSMENTS AND<br>PROCEDURES | Blood volumes to be collected in the study were updated to include additional blood samples added for the open-label booster vaccination phase. | Update |
| 1.3.3 Participants with a Suspected<br>AESI<br>8 STUDY ASSESSMENTS AND<br>PROCEDURES | The volume of the clinical laboratory blood sample (whole blood) taken at AESI Day 1 and Day 29 has been corrected; 15 mL instead of 12 mL of blood will be collected at each of the visits. | Correction |
| 1.1 Synopsis<br>11 REFERENCES | The reference to the Brighton Collaboration case definition of thrombotic events and thrombocytopenia was updated. | Update |
| 6.4 Unblinding and Open-label Phase | Text was added that participants with a history of capillary leak syndrome are not eligible for cross-over vaccination with Ad26.COV2.S at the Month 6/Unblinding Visit (nor are they eligible to receive a booster vaccination at the Year 1/Booster Visit). | Update |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | |
| 10.2 Appendix 2: Clinical Laboratory | Added that, as part of investigation of any | Clarification |
| Test | AESI, samples from appropriate controls | |
| | within the study could be used for | |
| | coagulation-related assays. | |
| Throughout the protocol | Minor errors and inconsistencies were | Correction of minor errors and |
| | corrected, and minor clarifications were | inconsistencies. Addition of |
| | added throughout the protocol. | minor clarifications. |
| | _ | Alignment across sections in |
| | | the protocol. |

#### **Amendment 5 (07 May 2021)**

Overall Rationale for the Amendment: This amendment has been created to include additional safety measures due to reports of adverse events following use of the Ad26.COV2.S vaccine under Emergency Use Authorization (EUA) in the United States (US), suggesting an increased risk of thrombosis combined with thrombocytopenia. Based on this, thrombosis with thrombocytopenia syndrome (TTS), which is a very rare event, will be followed in this protocol as an adverse event of special interest (AESI) that needs to be reported to the sponsor within 24 hours of awareness. In addition, anaphylaxis has been added as an important identified risk.

In addition, this amendment has been created to reinstate the use of a central laboratory for RT-PCR tests or other molecular diagnostic test to confirm cases of SARS-CoV-2 infection upon health authority (HA) request.

These and other changes made to the clinical protocol of study VAC31518COV3001 are listed below, including the rationale for each change and a list of all applicable sections.

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | |
| 1.1 Synopsis | Thrombosis with thrombocytopenia | Emerging data following use of the |
| 1.3.1 All Participants | syndrome (TTS) will be considered | Ad26.COV2.S vaccine under |
| 1.3.3 Participants with a Suspected | an AESI. Follow-up assessments will | Emergency Use Authorization in |
| AESI | be performed in the event of a | the US suggest an increased risk of |
| 2.3.1 Risks Related to Study | suspected AESI. | thrombosis combined with |
| Participation | In addition, blood samples will be | thrombocytopenia, with onset of |
| 2.3.3 Benefit-Risk Assessment of | collected for a baseline assessment of | symptoms approximately 1 to |
| Study Participation | platelet count and storage for future | 2 weeks after vaccination. |
| 3. OBJECTIVES AND ENDPOINTS | coagulation-related testing. | Therefore, additional reporting and |
| 4.1 Overall Design | | data collection procedures are |
| 6.4 Unblinding and Open-label Phase | | implemented to follow-up |
| 6.9 Prestudy and Concomitant Therapy | | thrombotic events and |
| 8. STUDY ASSESSMENTS AND | | thrombocytopenia and identify |
| PROCEDURES | | cases of TTS. |
| 8.2.4 Clinical Laboratory Assessments | | |
| 8.3 Adverse Events, Serious Adverse | | |
| Events, Medically-attended Adverse | | |
| Events, Adverse Events of Special | | |
| Interest, and Other Safety Reporting | | |
| 8.3.1 Time Period and Frequency for | | |
| Collecting Adverse Event, Medically- | | |
| attended Adverse Event, Adverse | | |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| Event of Special Interest, and Serious Adverse Event Information 8.3.2 Method of Detecting Adverse Events, Medically-attended Adverse Events, Adverse Events of Special Interest, and Serious Adverse Events 8.3.3 Follow-up of Adverse Events, Medically-attended Adverse Events, Adverse Events of Special Interest, and Serious Adverse Events 8.3.7 Adverse Events of Special Interest, and Serious Adverse Events of Special Interest 8.3.7 Adverse Events of Special Interest 8.3.7.1 Thrombosis with Thrombocytopenia Syndrome 9.2.4.2 All Participants 9.7 Safety Analysis 10.2 Appendix 2: Clinical Laboratory Tests 10.3.6 Committees Structure 10.4 Appendix 4: Adverse Events, Serious Adverse Events, Adverse Events of Special Interest, Medically-attended Adverse Events, Product Quality Complaints, and Other Safety Reporting: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting 10.4.5 Procedures 10.13 Appendix 13: TTS AESI Form | Description of Change | Brief Rationale |
| 10.14 Appendix 14: Thrombotic Events to be Reported as AESIs 11 REFERENCES 1.1 Synopsis 1.3.1 Schedule of Activities "All Participants" 1.3.2 Schedule of Activities "Participants With (Suspected) COVID-19" 3 OBJECTIVES AND ENDPOINTS 4.1 Overall Design 8.1.3 Efficacy Assessments 9.5.1 Primary Endpoint Evaluation 10.2 Appendix 2: Clinical Laboratory Test | Reinstated text to use a central laboratory for RT-PCR tests or other molecular diagnostic test to confirm cases of SARS-CoV-2 infection. | Changed upon HA request. |
| 2.3.1 Risks Related to Study<br>Participation | Side effects were updated to include injection site pain and nausea. It has been clarified that anaphylaxis is considered an important identified risk. | To align with the vaccine's identified risks. Added anaphylaxis as identified risk. |
| 1.3.1 All Participants 2.3.1 Risks Related to Study Participation 5.5 Criteria for Temporarily Delaying Administration of Study Vaccination 6.4 Unblinding and Open-label Phase | It has been further clarified that participants who are pregnant at the Month 6/unblinding visit and previously received placebo during the double-blind phase may be vaccinated with Ad26.COV2.S, if the | For clarification purposes. |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | |
| 8.2.3 Pregnancy Testing<br>8.3.5 Pregnancy | investigator considers that the potential benefits outweigh the potential risks. | |
| | Participants who originally received placebo and will not be receiving the Ad26.COV2.S vaccine under EUA, do not need to complete a pregnancy test. | |
| 6.1 Study Vaccines Administered | Placebo is now correctly classified as an Investigational Medicinal Product instead of a Non-Investigational Medicinal Product. | Correction of an error. |
| 8.3.1 Time Period and Frequency for<br>Collecting Adverse Event, Medically-<br>attended Adverse Event, Adverse<br>Event of Special Interest, and Serious<br>Adverse Event Information | A diagram on the safety reporting process is added for clarity. | Additional clarification per health authority request. |
| 1.1 Synopsis 4.1 Overall Design 8.9 Assessment and Procedures after EUA or Approval/Licensure and Implementation of Protocol Amendment 4 9.1 Statistical Hypotheses 9.8 Interim Analysis and Committees | Clarified that the final analysis of the double-blind phase may be conducted when a minimum of 90% of the study population has been unblinded depending on the operational implementation of Month 6 unblinding visit, as well as the stage of the pandemic. | To update the analysis as appropriate for the change to an open-label design. |
| Throughout the protocol | Minor errors and inconsistencies were corrected, and minor clarifications were added throughout the protocol. | Correction of minor errors and inconsistencies. Addition of minor clarifications. Alignment across sections in the protocol. |

#### Amendment 4 (22 February 2021)

Overall Rationale for the Amendment: The main purpose of this amendment is to outline the procedures to be followed after Emergency Use Authorization (EUA), conditional licensure, or approval in any country and approval of the protocol Amendment 4 by both Health Authority and Independent Ethics Committee (IEC)/Institutional Review Board (IRB) where a single dose of Ad26.COV2.S vaccine will be offered to enrolled participants who initially received placebo, resulting in de facto unblinding of participants and investigators. All participants will be encouraged to remain in the study and continue to be followed for efficacy/effectiveness, safety and immunogenicity as originally planned for up to 2 years post-vaccination on Day 1. This will allow assessment of the duration of protection and immunogenicity of a single dose of Ad26.COV2.S by comparing 2 groups vaccinated approximately 4 to 6 months apart.

In addition, clarification is provided that RT-PCR test results obtained from any source (including local laboratories) may be used for analyses and that confirmation by the central laboratory will no longer be required as part of the case definitions.

These and other changes made to the clinical protocol of study VAC31518COV3001 are listed below, including the rationale of each change and a list of all applicable sections.

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | |
| and Name 1.1 Synopsis 1.2 Study Schema 1.3.1 Schedule of Activities 2 Introduction 2.1 Study Rationale 2.3.3 Benefit-Risk Assessment of Study Participation 3 Objectives and endpoints 4.1 Overall Design 4.2 Scientific Rationale for Study Design 5. Study Population 5.5 Criteria for Temporarily Delaying Administration of Study Vaccination 6.1 Study Vaccines Administered 6.2 Preparation/Handling/Storage/ Accountability 6.3 Measures to Minimize Bias: Randomization and Blinding 6.4 Unblinding and Open-label Phase (added) 6.7 Continued Access to Study Vaccine After the End of the Study 8.9 Assessment and Procedures After EUA or Approval/Licensure and Implementation of protocol Amendment 4 10.2 Appendix 2: Clinical Laboratory Test 10.3.3 Informed Consent Process | At the 6 Month/unblinding visit, all participants who initially received placebo will be offered a single dose of Ad26.COV2.S vaccine (5×10 <sup>10</sup> vp), starting an open-label phase of the study. This is to occur as soon as possible after the Day 71 visit. All participants at the Month 6/unblinding visit will have a blood draw and nasal swab. Relevant sections were updated regarding the open-label phase. Participants to be reminded there is no data on the safety of receiving 2 different COVID-19 vaccines. Removed the following sentence at the end of Section 6.6: "At such time, an amendment will be submitted to permit individual unblinding and to determine the approach to this situation in the Statistical Analysis Plan." | As the vaccine is highly efficacious against severe disease, hospitalization and death, it is considered ethical to offer the active vaccine to the placebo controls in this study. Hereby, an unblinding visit will be scheduled to inform all participants about their study vaccine allocation as well as to offer all placebo recipients Ad26.COV2.S after EUA, conditional licensure or approval in any country. Taking blood samples and nasal swabs from all participants will allow the comparison of efficacy and immunogenicity results in a placebo-controlled manner up to the point of the Month 6/unblinding visit, as well as having a new baseline read-out for the remainder of the study. The 6 Month visit with a broadened visit window will be used as an unblinding visit to allow for rapid cross-over in the context of logistic issues. Investigators will be encouraged to follow health authority guidelines on prioritization of immunization when feasible. All participants will be counselled to continue practicing other public health/preventative measures that were introduced at the start of this pandemic (eg, social distancing, face masks, frequent hand washing), in compliance with local and national guidelines. |

| Section Number and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 1.1 Synopsis 6.3 Measures to Minimize Bias: Randomization and Blinding 6.7 Continued Access to Study Vaccine After the End of the Study | Additional changes needed to allow unblinding prior to authorization/licensure and simultaneous participation in an Expanded Access Program or a Phase 3B study (eg, Sisonke/TOGETHER in South Africa). | To allow participants in an Expanded Access Program for Ad26.COV2.S prior to EUA, conditional licensure or approval in any country to continue to be followed in VAC31518COV3001. |
| 6.4 Unblinding and Open-label<br>Phase (added) | Describes the conditions under which participants who received placebo initially may be vaccinated with Ad26.COV2.S. | To provide guidance on the appropriate vaccination of participants at the start of the open-label phase. |
| 1.1 Synopsis 9.5.1 Primary Endpoint Evaluation | Text has been added describing a final analysis of the double-blind phase which will be performed when all participants will have completed the Month 6/unblinding visit and will provide an analysis of all endpoints for the blinded portion of the study. | To provide an analysis on all data that can be considered part of the double-blind phase of the study. |
| 3 Objectives and endpoints | Reference to "post-vaccination" in objectives and endpoints has been updated to "after double-blind." | To clarify changes required by adding the open-label phase of the study. |
| 3 Objectives and endpoints 9.5.1 Primary Endpoint Evaluation | The following secondary endpoint was added: - Asymptomatic infection detected by RT-PCR at the time of the Month 6/unblinding visit. The following exploratory objectives were added: - To evaluate the long term durability of the efficacy of Ad26.COV2.S in the prevention of molecularly confirmed, moderate to severe/critical COVID-19, in adults by comparing 2 groups of participants vaccinated approximately 4 to 6 months apart. - To examine efficacy for moderate/severe and severe disease as well as medical utilization or death in the vaccine and placebo groups for variant strains that have been identified. | To gather information regarding long term efficacy and efficacy against variants. |
| 1.1 Synopsis 9 Statistical Considerations | Added text describing analysis of the data once EUA, conditional licensure or approval in any country is obtained and all participants are unblinded. | To ensure assessment of the duration of protection and immunogenicity of a single dose of Ad26.COV2.S by comparing 2 groups vaccinated approximately 4 to 6 months apart. |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name 1.1 Synopsis 1.3.1 Schedule of Activities 3 Objectives and Endpoints 4.1 Overall Design 8.1.3 Efficacy Assessments 9.5.1 Primary Endpoint Evaluation 10.2 Appendix 2: Clinical Laboratory Test | Added text to clarify that a RT-PCR test obtained from any source will be used for all analyses. These include RT-PCR tests performed by local laboratories that have utilized RT-PCR testing devices approved by the COVID-19 Response Team (formerly known as OWS), laboratories that are designated as substitutes for local laboratories within the context of the study or any PCR test utilized for a hospitalized study participant for diagnosis and treatment of COVID-19. In addition, any RT-PCR test not meeting the above criteria can only be used for determination of an asymptomatic case. Confirmation by the central laboratory will not be required as part of any of the case definitions. | Based on data seen thus far, there was a high concordance of results between the central and local laboratories, therefore it is deemed reasonable to use RT-PCR results from local laboratories to confirm cases of SARS-CoV-2 infection. |
| 1.1 Synopsis 8.1.3.6 Clinical Severity Adjudication Committee 10.3.6 Committees Structure | Added text describing adjudication of asymptomatic, mild, moderate, severe, and cases requiring hospitalization, ICU, ventilator support or ECMO and death including date of onset and reasons for the classification. As new information becomes available, cases may be readjudicated. | The role of the Clinical Severity Adjudication Committee is being expanded to improve the classification of the cases. The SAP will be amended to include the new adjudication process in the efficacy assessment of the vaccine (endpoint selection for the analysis). |
| 1.1 Synopsis 8.1.3.4 Case Definition for Asymptomatic or Undetected COVID-19 9.5.1 Primary Endpoints Evaluation | Clarification about the definition of asymptomatic infection. | The current definition does not clearly eliminate cases that are SARS-CoV-2 N antibody sero-converters but RT-PCR negative and have symptoms consistent with COVID-19. |
| 1.1 Synopsis 1.3.1 Schedule of Activities 4.1 Overall Design 8 Study Assessments and Procedures | Updated the twice weekly eCOA assessments to occur 1 year following the Month 6/unblinding visit. | To ensure that all participants have 1 year of eCOA assessments following the Month 6/unblinding visit. |
| 6.9 Prestudy and Concomitant<br>Therapy | A statement was added that receipt of another COVID-19 vaccine by a study participant at any time during the study should be recorded along with the name and date(s) of the vaccine. | This was added so receipt of another COVID-19 vaccine can be accounted for in determining efficacy, duration of efficacy calculations and safety evaluations. Participants that have received another COVID-19 vaccine will not be allowed to receive a single dose of Ad26.COV2.S |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name 1.1 Synopsis 9.5.1 Primary Endpoints Evaluation | Include the study success criterion of the point estimate of VE being >50% for both co-primary endpoints. | A consequence of using a VE of 30% in the hypothesis testing is that the null hypothesis could be rejected with a result for either co-primary VE of less than 50%. It is specified that this would not be considered a successful study. |
| 6.3 Measures to Minimize Bias: Randomization and Blinding 9.9 Analyses for Cohort Unblinded Due to Administration of an Authorized/Licensed COVID-19 Vaccine | Changed SARS-COV-2 to<br>Ad26.COV2.S | Consistency |
| 1.3.1 Schedule of Activities<br>8.1.4 Immunogenicity Assessments | Blood draw at the 1-Year visit will<br>be replaced by Month 18 visit for<br>non-immunogenicity subset<br>participants (10 mL). | To evaluate the levels of immunogenicity 1 year after beginning of the open label phase of the study. |
| 1.3.1 Schedule of Activities 2.3.1 Risks Related to Study Participation 6.3 Measures to Minimize Bias: Randomization and Blinding 8.2.3 Pregnancy Testing | Added an additional urine pregnancy test at the time of Month 6/unblinding visit for cross-over participants who initially received placebo. | In order to be aware of potential pregnancy before administering Ad26 vaccine. Vaccination of pregnant may be allowed depending on local guidelines. |
| 1.1 Synopsis 8.1.4 Immunogenicity Assessments 8.2 Safety Assessments 8.3.1 Time Period and Frequency for Collecting Adverse Event, Medically-attended AdverseEvent, and Serious Adverse Event Information 8.3.2 Method of Detecting Adverse Events, Medically-attended Adverse Events, and Serious Adverse Events 9.2.4 Safety | Clarified that the Safety and Immunogenicity Subsets are applicable for the double-blind phase only, but special reporting situations will be recorded until 28 days as well as MAAEs will be reported until 6 months after (double-blind or open-label) vaccination with Ad26.COV2.S and SAEs will be reported until end-of-study. | To be consistent with the safety reporting requirements following administration of an investigational vaccine. |
| 1.1 Synopsis 9 Statistical Considerations | Added statement to indicate that samples from open-label phase will be analyzed separately. | The double-blind and the open-<br>label phases will be analyzed<br>separately and will be described in<br>separate SAPs. |
| Synopsis 9.8Interim Analysis and Committees | Text was added to describe the final analysis of the double-blind data and the open-label data, supplemented by real-world data. | The double-blind and the open-<br>label phases will be analyzed<br>separately. Interpretation of the<br>open-label data may be<br>supplemented by real-world data<br>from other studies if applicable. |
| 8.1.2 Procedures in Event of (Suspected) COVID-19 | Clarified procedures around suspected COVID-19 cases. | Clarification |
| 2.3.2 Benefits of Study Participation | Added statement about recent data suggesting efficacy/safety of Ad26.COV2.S from primary analysis of COV3001. | Updated text |
| 10.12 Appendix 12: Risk Factor<br>Assessment | Updated the assessment form to change any references to "2020" to "the near future." | To extend the data collection period, as the study is still ongoing. |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| Throughout the protocol | Specified "double-blind" vaccination throughout as applicable | This was done to clarify that the timing of follow-up (except for MAAEs and special reporting situations) is relative to the first vaccination for participants who cross-over to open-label active vaccine. |
| | Updated terminology from "COVID-19 infection" to "SARS-CoV-2 infection" | To differentiate the disease from its causative agent. |
| | Minor errors and inconsistencies were corrected, and minor clarifications were added throughout the protocol. | Correction of minor errors and inconsistencies. Addition of minor clarifications. Alignment across sections in the protocol. |

#### Amendment 3 (14 December 2020)

Overall Rationale for the Amendment: The main purpose of this amendment is to add first occurrence of molecularly confirmed, moderate to severe/critical COVID-19, with onset at least 28 days post double-blind vaccination as a co-primary endpoint in addition to the current primary endpoint counting as of 14 days post double-blind vaccination. The applicable secondary and exploratory endpoints were updated similarly to also include COVID-19 cases with onset at least 28 days post double-blind vaccination. In addition, the total sample size was reduced from 60,000 to approximately 40,000 participants. The protocol is further amended to change the conditions for monitoring whether efficacy greater than 30% is achieved using the sequential monitoring algorithm: (1) The minimum number of COVID-19 cases meeting the primary case definition needed to start the efficacy monitoring was modified to at least 42 instead of 20, (2) The need for a follow-up of 8 weeks for 50% of the participants prior to an initial look at an efficacy signal if the other conditions are met was removed.

These and other changes made to the clinical protocol of study VAC31518COV3001 are listed below, including the rationale of each change and a list of all applicable sections.

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | |
| 1.1 Synopsis 3 OBJECTIVES AND ENDPOINTS 4.1 Overall Design 8.1.3.1 Case Definition for Moderate to Severe/Critical COVID-19 8.1.3.6 Clinical Severity Adjudication Committee 9.1 Statistical Hypotheses 9.2.1 Efficacy (Total Sample Size) 9.5.1 Primary Endpoints Evaluation 9.5.1.1 Study Monitoring 9.5.2 Secondary Endpoints 9.8 Interim Analysis and Committees 10.3.6 Committees Structure | A co-primary endpoint was added counting COVID-19 cases from 28 days post-vaccination (Day 29), in addition to from 14 days post-vaccination (Day 15). The applicable secondary and exploratory endpoints were updated to also include COVID-19 cases with onset at least 28 days post-vaccination, in addition to from 14 days post-vaccination. | This change will allow for formal testing and reporting of the primary endpoint counting cases from 28 days post-vaccination as an additional condition for success along with the 14 days post-vaccination endpoint results. Maintaining the original primary endpoint will preserve trial integrity. This approach will allow to provide the most accurate description of the vaccine efficacy and to assess vaccine efficacy as early as 14 days post-vaccination. |
| 3 OBJECTIVES AND ENDPOINTS | Deletion of the exploratory endpoint relating to evaluation of the occurrence, severity and duration of COVID-19 episodes in participants who received Ad26.COV2.S, as compared to placebo, by the Clinical Severity Adjudication Committee, previously known as the Clinical Evaluation Committee. | The Clinical Severity Adjudication<br>Committee only exists to determine<br>severe/critical cases of COVID-19. |

| Section Number and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 9.2.1 Efficacy (Total Sample Size) 9.2.4 Safety Subset | The total sample size was reduced from 60,000 to approximately 40,000. The paragraph on the operational futility was removed. | The incidence of moderate to severe COVID-19 seen in the US and reported in other COVID-19 vaccine studies is significantly higher than assumed at the time of protocol planning. Furthermore, based on that incidence and modeling, there is a high degree of probability that an efficacy signal meeting the prespecified criteria in this amendment will be reached at, or prior to, the time when 50% of participants will have been followed for 8 weeks from the time of vaccination. |
| 1.1 Synopsis 9.5.1 Primary Endpoints Evaluation | The conditions for monitoring whether efficacy greater than 30% is achieved using the sequential monitoring algorithm were changed: (1) The minimum number of COVID-19 cases with onset at least 28 days after vaccination meeting the primary case definition needed to start the efficacy monitoring was modified to at least 42 instead of 20. (2) The need for a follow-up of 8 weeks for 50% of participants prior to an initial look at an efficacy signal if the other conditions are met, was removed. In addition, text was added to clarify the timing of primary and | (1) The minimum number of COVID-19 cases was increased to have a more robust signal at the time of the efficacy declaration. (2) This change was made to expedite submissions to ensure the vaccine is made available to the public as soon as possible. Following 50% of participants for 8 weeks from the day of vaccination meets the sponsor's understanding of the requirement for 8 weeks median follow-up for a 40,000-participant study. |
| 1.1 Synopsis 3 OBJECTIVES AND ENDPOINTS 9.5.2 Secondary Endpoints | interim analyses. A secondary objective and endpoint were added assessing the efficacy of the vaccine in the prevention of molecularly confirmed, severe/critical COVID-19 with onset at least 14 days post-vaccination and 28 days post-vaccination. | With the increased incidence of disease that is being observed, the likelihood of having enough severe cases of COVID-19 to examine vaccine efficacy against this endpoint has increased. Vaccine efficacy against severe disease is considered an important endpoint for a 1-dose vaccine. |
| 1.1 Synopsis 1.3.1 All Participants 3 OBJECTIVES AND ENDPOINTS 8.1.3 Efficacy Assessments 8.1.3.5 SARS-CoV-2 Seroconversion Assessment 8.1.4 Immunogenicity Assessments 10.2 Appendix 2: Clinical Laboratory Tests | An exploratory objective and endpoint were added assessing the effect of the vaccine on confirmed asymptomatic or undetected infections by testing serologic conversion between baseline and 28 days post-vaccination. | This change allows the evaluation of the effect of the vaccine on asymptomatic infections up to Day 29, in line with other efficacy endpoints. |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name 3 Objectives and Endpoints OBJECTIVES AND ENDPOINTS | An exploratory objective and endpoint to examine the degree of frailty were added. | The vaccine will be especially useful in the elderly population with co-morbidities. The frailty index has been utilized as a tool to summarize the degree of frailty that a participant has. |
| 1.1 Synopsis 2.3.1. Risks Related to Study Participation 3 OBJECTIVES AND ENDPOINTS 8.1.3 Efficacy Assessments 8.1.3.6 Clinical Severity Adjudication Committee 10.3.6 Committees Structure | The Clinical Evaluation Committee was replaced by the Clinical Severity Adjudication Committee. | The standard case definition of severe/critical disease may not cover all situations where clinical judgement would disagree with the classification on clinical grounds. |
| 1.1 Synopsis<br>8.1.3.1 Case Definition for<br>Moderate to Severe/Critical<br>COVID-19 | Addition of text defining the definitive role of the Clinical Severity Adjudication Committee in determining whether cases are severe/critical cases of COVID-19. | Clarification of the definitive role of the Clinical Severity Adjudication Committee in defining the severity of cases of COVID-19. |
| 1.1 Synopsis 1.3.1 All Participants 3 OBJECTIVES AND ENDPOINTS 4.1 Overall Design 4.2 Scientific Rationale for Study Design 4.2.1 Study-Specific Ethical Design Considerations 8.8 Participant Medical Information Prior to, During and After the Study (Real-world Data) 9.5.4 Other Analyses 10.1 Appendix 1: Abbreviations 11 References | Addition of the utilization of tokenization and matching procedures to obtain medical data 5 years prior to enrollment of the participant until 5 years after the participant completed the study from consenting participants in the United States (US). | Participant medical data (electronic health records, claims, laboratory data from other care settings) prior to, during and following participation in the study (realworld data) is important to obtain in order to better understand the impact of prior medical history on the response to immunization and the impact of immunization on efficacy and duration of efficacy as well as adverse events that may occur during and after completion of the study. The technique proposed to obtain this data, ie, tokenization and matching procedures, allows for such data to be obtained without violation of participant confidentiality. This collection of real-world data will only be conducted for consenting participants from the US where this technique is feasible. |
| 1.1 Synopsis 3 OBJECTIVES AND ENDPOINTS 8.1.4 Immunogenicity Assessments | psVNA was removed from the protocol. wtVNA will be used to support the exploratory immunogenicity endpoint. | Due to lack of sensitivity of the evaluated psVNA, the assay has been removed from the protocol wtVNA is currently only qualified and not validated and can therefore not be used to support a secondary immunogenicity endpoint unless validated. |
| 1.3.1 All Participants 1.3.2 Participants With (Suspected) COVID-19 | Further clarifications are made to the procedures to be followed in case of (suspected) COVID-19. | Alignment across the protocol and clarifications on the procedures to |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| 4.1 Overall Design<br>8.1.2 Procedures in the Event of<br>(Suspected) COVID-19 | | be followed in case of (suspected) COVID-19. |
| 5.1 Inclusion Criteria | Inclusion criterion 4 was updated to clarify that all comorbidities need to be stable and well-controlled, those that are associated with severe COVID-19 AND those that are not associated with severe COVID-19. In addition, a time frame was added for criteria a and b for stable/well-controlled HIV infection. | Clarification |
| 5.1 Inclusion Criteria | In inclusion criterion 4, it was clarified that participants with stable/well-controlled HIV infection that are on stable ART are included if nationwide guidelines require transition from one ART regimen to another, within a period of less than 6 months. | Clarification |
| 5.1 Inclusion Criteria | It was clarified in inclusion criterion 9 that participants with visual impairment are eligible and may have caregiver assistance in completing the eCOA questionnaires. | Clarification |
| 5.2 Exclusion Criteria | In exclusion criterion 3, "Patients on hemodialysis" has been added to the examples of clinical conditions expected to have an impact on the immune response of the study vaccine. | There is evidence that hemodialysis has a negative impact on the immune response elicited by the vaccination. |
| 5.2 Exclusion Criteria | In exclusion criterion 4, it was clarified that autologous blood transfusions are not excluded. | Clarification |
| 1.1 Synopsis<br>8.1.4 Immunogenicity Assessments | The list of immunoassays used in support of exploratory endpoints has been completed. | Addition of missing assay. |
| 1.1 Synopsis 6.3 Measures to Minimize Bias: Randomization and Blinding 6.7 Continued Access to Study Vaccine After the End of the Study 9.9 Analyses for Cohort Unblinded Due to Administration of an Authorized/Licensed COVID-19 Vaccine | Clarification of procedures for unblinding of study participants who may become eligible to receive an authorized/licensed COVID-19 vaccine during the course of the study. | To ensure that if participants become eligible to receive an authorized/licensed COVID-19 vaccine, they are aware of the potential options and ramifications, including the lack of safety data of the authorized/licensed vaccine. |
| 10.8 Appendix 8: Medically-<br>attended COVID-19 (MA-COV)<br>Form | The MA-COV form has been updated to also capture hyperinflammatory syndrome. | To ensure collection of all necessary information in order to determine the severity of COVID-19 per the case definitions and clarification purposes. |
| 2.3.1 Risks Related to Study<br>Participation | It was clarified that the use of condoms is not considered an | Clarification |

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| 5.1 Inclusion Criteria | acceptable contraceptive barrier method due to the failure rate of female and male condoms. | |
| 8 STUDY ASSESSMENTS AND PROCEDURES | It was clarified that in case of home visits, assessments that cannot be delegated to a designee must be performed by an appropriate site staff member via a phone call or telemedicine. | Clarification |
| 8.7 Risk Factor Assessment 9.4 Participant Information | It was clarified that the risk factor data initially collected at screening from the participants, before the implementation of this amendment will also be used for the planned risk factor analysis. | Clarification |
| 6.3 Measures to Minimize Bias:<br>Randomization and Blinding<br>9.5.1 Primary Endpoints Evaluation | The timepoints of analyses at which the sponsor will be unblinded were clarified. | Clarification |
| Throughout the protocol | Minor errors and inconsistencies were corrected, and minor clarifications were added throughout the protocol. | Correction of minor errors and inconsistencies. Addition of minor clarifications. Alignment across sections in the protocol. |

#### Amendment 2 (29 October 2020)

**Overall Rationale for the Amendment:** This amendment is written to clarify that all participants that have a reverse-transcriptase polymerase chain reaction (RT-PCR) positive finding for SARS-CoV-2 from any source, even if asymptomatic, will be followed until there are two consecutive negative PCRs. Also, some errors, have been corrected, including the clarification that blood will be drawn on Day 29 for biomarker RNAseq analyses (PAXgene tube), which is needed in order to assess the current objectives. Finally, some minor errors have been corrected.

The changes made to the clinical protocol of study VAC31518COV3001 are listed below, including the rationale of each change and a list of all applicable sections.

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name 1.1 Synopsis 1.3.2 Participants With (Suspected) COVID-19 4.1 Overall Design 8 STUDY ASSESSMENTS AND PROCEDURES 8.1.1 Prespecified Criteria for Suspected COVID-19 8.1.2 Procedures in the Event of (Suspected) COVID-19 8.1.3.4 Case Definition for Asymptomatic or Undetected COVID-19 10.3.10 Source Documents | Clarified that all participants that have a RT-PCR positive finding for SARS-CoV-2 from outside the study, even if asymptomatic, will be followed until there are two consecutive negative PCRs. | To ensure safety of staff and other persons coming in contact with the infected participant. |
| 1.3.1 All Participants 8 STUDY ASSESSMENTS AND PROCEDURES 10.2 Appendix 2: Clinical Laboratory Tests | It has been clarified that at Day 29 2.5 mL blood will be collected from participants for biomarker RNAseq analyses (PAXgene tube). | Correction. In order to assess<br>the objectives as currently stated<br>in the protocol, a blood<br>sampling for biomarker<br>RNAseq (PAXgene) performed<br>after the participants have<br>received the vaccination is<br>required. |
| 1.1 Synopsis 2.1 Study Rationale 2.3.3 Benefit-Risk Assessment of Study Participation 4.1 Overall Design 9.2.2 Immunogenicity Subset | It has been clarified that Stage 1b and Stage 2b will enroll participants with and without comorbidities. However, participants in the Immunogenicity Subset 1b and 2b will be participants with comorbidities. | Clarification |
| 5.2 Exclusion Criteria 6.8 Prestudy and Concomitant Therapy | The specification of '(>10 days)' when referring to the chronic use of systemic corticosteroids has been removed from the exclusion criterion 3. | To remove ambiguity as within the same exclusion criterion 3 a substantial immunosuppressive steroid dose is defined as ≥2 weeks of daily receipt of 20 mg of prednisone or equivalent |
| 1.3.1 All Participants 1.3.2 Participants With (Suspected) COVID- 19 8.6 Medical Resource Utilization | The MA-COV form has been updated to also capture if a participant has clinical or radiological evidence of pneumonia and if the oxygen | To ensure collection of all necessary information in order to determine the severity of COVID-19 per the case |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

| Section Number | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| and Name | Description of Change | Diei Kationale |
| 10.8 Appendix 8: Medically-attended COVID-19 (MA-COV) Form | saturation for a participant is considered clinically abnormal but >93% (corrected for altitude). In addition, some clarifications were added to the form and it is clarified that the form may also be completed by the study site personnel. | definitions and clarification purposes. |
| 10.3.11 Monitoring | Source data verification has been replaced by review of the source data. | Source document review will be done instead of source document data verification. |
| 2.3.1 Risks Related to Study Participation 10.4.4 Special Reporting Situations | It is stated more clearly that breastfeeding women are allowed to participate in the study. In alignment with this, exposure to a sponsor study vaccine from breastfeeding has been removed from the list of special reporting situations. | Breastfeeding is allowed in the current study VAC31518COV3001. |
| 1.1 Synopsis 5.1 Inclusion Criteria 5.2 Exclusion Criteria | Gestational diabetes has been removed from the list of comorbidities (or risk factors) that might be associated with increased risk of progression to severe COVID-19. | Gestational diabetes is not applicable in the current study VAC31518COV3001 as pregnant women are not allowed to participate in the study. |
| 9.5.1.1 Study Monitoring | Clarified that there will be no adjustment for multiple testing for the potential harm monitoring of severe cases, ie, an exact 1-sided binomial test of the fraction of infections assigned to who receive the vaccine will be used with an unadjusted p-value $\alpha$ at 5%. | Adjusted in line with HA feedback to start monitoring of severe events as soon as 5 events and subsequently after every new event without adjustment for multiple testing |
| 1.1 Synopsis 1.3.1 All Participants 1.3.2 Participants With (Suspected) COVID- 19 4.1 Overall Design 8.7 Risk Factor Assessment 9.4 Participant Information 10.12 Appendix 12: Risk Factor Assessment | It is clarified that, besides being interviewed on characteristics related to current work situation, living situation, and community interactions, as specified in Appendix 12, prior to vaccination on Day 1, they will be asked about any changes related to these characteristics at Day 71 and 6 months and 1 year post vaccination and at COVID-19 Day 3-5. | Clarification on when participants will be interviewed on additional characteristics that will be used for risk factor analysis. |
| <ul><li>5.2 Exclusion Criteria</li><li>6.8 Prestudy and Concomitant Therapy</li></ul> | Exclusion criterion 7 was adjusted to exclude participants who received investigational | Alignment across Ad26.COV2.S Phase 3 study protocols |

| Section Number<br>and Name | Description of Change | Brief Rationale |
|---|---|---|
| and Ivanic | immunoglobulin or<br>monoclonal antibodies within | |
| | 3 months, or received convalescent serum for COVID-19 treatment within 4 | |
| 5.2 Exclusion Criteria | months. Chronic kidney disease (with dialysis) has been removed from the examples of clinical | There is no evidence that dialysis has an impact on antibody concentration in the |
| | conditions expected to have an impact on the immune response of the study vaccine. | blood. |
| 1.1 Synopsis<br>5.2 Exclusion Criteria | It is clarified Parkinson's disease, seizures, ischemic strokes, intercranial hemorrhage encephalopathy, meningoencephalitis are not part of the CDC list of | Clarification |
| | comorbidities that are associated with increased risk of progression to severe COVID-19. | |
| 5.2 Exclusion Criteria | It is clarified that participants with Guillain-Barré syndrome are excluded from the study altogether and not only in Stage 1a and Stage 2a of the study. | Correction |
| 5.1 Inclusion Criteria | Clarifications have been made to the inclusion criterion 4, indicating that for Stages 1a and 2a participants can have a condition that is stable and well controlled except the ones listed in exclusion criterion 15 which are associated with increased risk of progression to severe COVID-19. In addition, medication dose for allowed stable conditions (in all stages of the study) cannot have been increased within 12 weeks | Clarification |
| 5.4 Screen Failures | prior to vaccination. It has been clarified that participants can be rescreened once, also when they meet all in- and exclusion criteria but the 28-day screening period was exceeded. | To allow participants who were found eligible to be enrolled in the study but were not randomized within the 28-day screening window to still participate in the study. |
| 1.1 Synopsis 9.8 Interim Analysis and Committees | Reference to a possible sample size adjustment has been deleted. | Correction; per the VAC31518COV3001 Amendment 1, the sample size of approximately 60,000 participants was selected based |

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | on available epidemiology data at the time of Amendment 1 writing. |
| 1.3.1 All Participants | It is clarified that the diagnostic molecular RT-PCR test for SARS-CoV-2 infection (from nasal swab taken at baseline) will be performed at a central laboratory on a retrospective basis. These baseline results are not available in real time, and thus cannot be used to inform participants at time of enrollment. | Clarification |
| 1.1 Synopsis 3 OBJECTIVES AND ENDPOINTS 4.1 Overall Design | It is clarified that molecularly confirmed COVID-19 is defined as a positive SARS-CoV-2 viral RNA result <b>by a central laboratory</b> using a PCR-based or other molecular diagnostic test. | For clarification purposes and to align information included in Section 8.1.3 which states that molecular confirmation of SARS-CoV-2 infection by a central laboratory will be used for the analysis of the case definition. |
| 10.3.10 Source Documents | It has been clarified that source documents for any relevant medical history and prestudy therapies determining eligibility (ie, as specified in the footnotes to the Schedule of Activities) of the participants needs to be collected | To ensure that all necessary information to properly assess SAEs (relatedness) is collected. |
| 1.1 Synopsis<br>5.2 Exclusion Criteria | The list of comorbidities (or risk factors) that are or might be associated with an increased risk of progression to severe COVID-19 has been corrected from 'uncontrolled human immunodeficiency virus (HIV) infection' to 'HIV infection' | Correction |
| 1.1 Synopsis 8.1.3.1 Case Definition for Moderate to Severe/Critical COVID-19 10.8 Appendix 8: Medically-attended COVID-19 (MA-COV) Form | It has been clarified that the adjustment according to altitude for the SpO2 criteria is per the investigator judgement. | Clarification |
| 8.3.6 Disease-related Events and Disease-related Outcomes Not Qualifying as Adverse Events or Serious Adverse Events | It has been clarified that (S)AEs caused by molecularly confirmed SARS-CoV-2 infection will be removed at the analysis level from the (S)AE listings and tables and presented separately. | Alignment across different sections of the protocol. |

# VAC31518 (JNJ-78436735)

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| Title page | Prepared by line removed | To align with internal guidelines on legal entity to be mentioned on title page |
| Throughout the protocol | Minor errors and inconsistencies were corrected, and minor clarifications were added throughout the protocol. | Correction of minor errors and inconsistencies. Addition of minor clarifications. Alignment across sections in the protocol. |

#### Amendment 1 (15 September 2020)

Overall Rationale for the Amendment: The amendment is written to adjust the dose level for Ad26.COV2.S from 1×10<sup>11</sup> virus particles (vp) to 5×10<sup>10</sup> vp based on data from the first-in-human (FIH) study VAC31518COV1001, including safety and immunogenicity data from Cohort 1a, safety data from Cohort 3 and immunogenicity data from the sentinel group of Cohort 3. Additional changes such as the determination of the sample size, further fine tuning of the case definitions for COVID-19, and the addition of target percentages (min/max) for enrollment of certain age groups are made based on emerging epidemiology information and advancing insights. Furthermore, throughout the protocol changes are made in response to the feedback received from Health Authorities, partners, and the community. Finally, minor errors and inconsistencies were corrected throughout the protocol.

The changes made to the clinical protocol of study VAC31518COV3001 are listed below, including the rationale of each change and a list of all applicable sections.

| Section Number | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| and Name | | |
| 1.1 Synopsis 2.1 Study Rationale 2.2 Background 4.1 Overall Design 4.4 End-of-study Definition 4.3 Justification for Dose 6.1 Study Vaccines Administered 8.1.4 Immunogenicity Assessments | The Ad26.COV2.S dose level has been lowered from 1×10 <sup>11</sup> vp to 5×10 <sup>10</sup> vp. | Immunogenicity data from Cohort 1a and a sentinel group of Cohort 3 of study VAC31518COV1001 have become available. The data demonstrated that a single dose of Ad26.COV2.S at a dose level of 5×10¹⁰ vp is sufficient to induce an acceptable immune response that meets prespecified minimum criteria: (1) wild-type virus neutralization assay (wtVNA)³ response rate (28 days post-Dose 1): lower limit of 95% confidence interval (CI) ≥65%; (2) T-helper cell type 1 (Th1)/T-helper cell type 2 (Th2) response magnitude ratio: Th1>Th2 within responder population and (3) pseudovirus (ps)VNA magnitude associated with protection in non-human primate (NHP) studies is induced by vaccination in humans: estimated population mean protection probability ≥40% and lower limit of 95% CI of estimated population mean protection probability ≥20%. This finding was |

<sup>&</sup>lt;sup>a</sup> psVNA was to be used for the seroconversion criterion, however, the psVNA was not sensitive enough to cover the range of human responses, hence wtVNA was used instead.

\_

| Section Number and Name | Description of Change | Brief Rationale |
|---|---|---|
| 1.1 Synopsis 2.1 Study Rationale 4.1 Overall Design 9.2.1 Efficacy (Total Sample Size) | The protocol has been adjusted to reflect the selected sample size of approximately 60,000 participants. A | supplemented with several sensitivity analyses utilizing ELISA, a more sensitive psVNA, and statistical evaluation of attributed values below the level of sensitivity of the original psVNA. The safety data from Cohort 1a and Cohort 3 of the FIH study with the Ad26.COV2.S 5×10 <sup>10</sup> vp dose level were deemed acceptable. Since all criteria for proceeding to Phase 3 were met by the 5x10 <sup>10</sup> vp dose, the sponsor decided to use this dose for further evaluation in the Phase 3 study VAC31518COV3001. Based on epidemiological modeling and currently available data (further explained in Section 9.2.1), the maximum |
| 9.2.4 Safety (Safety Subset) | detailed rationale for the sample size selection has been added to Section 9.2 Sample Size Determination of the protocol. | sample size of 60,000 participants was selected. |
| 1.1 Synopsis 9.5.1 Primary Endpoint Evaluation | The trigger for the evaluation of the primary endpoint has been modified, adding 3 conditions, one related to available follow-up information, one related to the number of severe/critical COVID-19 cases and one related to the number of cases meeting the primary endpoint definition of moderate to severe/critical COVID-19 in the elderly population, that need to be met. | In order to ensure the evaluation of the primary endpoint provides sufficient information to assess the benefit/risk and potentially support an Emergency Use Authorization. |
| 1.1 Synopsis 1.3.1 All Participants 3 OBJECTIVES AND ENDPOINTS 8 STUDY ASSESSMENTS AND PROCEDURES 8.1.4 Immunogenicity Assessments 9.2.1 Efficacy (Total Sample Size) 9.5.1 Primary Endpoint Evaluation 9.5.2 Secondary Endpoints 9.5.1.1 Study Monitoring 10.2 Appendix 2: Clinical Laboratory Tests | The time to begin counting COVID-19 cases after vaccination with Ad26.COV2.S has been decreased from at least 28 days post-vaccination to at least 14 days post-vaccination (Day 15). | Based on preliminary data from Cohort 1b of study VAC31518COV1001, showing robust immunology data 14 days after vaccination that are similar to the data seen 28 days after vaccination. |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name 1.1 Synopsis 2.1 Study Rationale 4.1 Overall Design 9.2.1 Efficacy (Total Sample Size) 9.5.1 Primary Endpoint Evaluation | The assumed vaccine efficacy (VE) has been adjusted from a VE=65% VE to a 60%=VE. The target number of events (TNE) has been adjusted accordingly from 104 to 154 events | The study power was adjusted to have approximately 90% power to detect an assumed vaccine efficacy as low as 60%, in line with Health Authority guidance. The target number of events has been adjusted accordingly. |
| 1.1 Synopsis 1.2 Schema 2.1 Study Rationale 2.3.3 Benefit-Risk Assessment of Study Participation 4.1 Overall Design 9.2.2 Immunogenicity Subset | It has been clarified that Stage 2a (adults ≥60 years of age) can start in parallel to Stage 1a (adults ≥18 to <60 years of age) unless this is not allowed per local Health Authority guidance. | After a review of the currently available safety and immunogenicity data from Cohort 1a and Cohort 3 of study VAC31518COV1001 (see above), staggered enrollment of Stage 2 is no longer deemed necessary. |
| 5.1 Inclusion Criteria 5.2 Exclusion Criteria | A clarification was added to<br>the eligibility criteria on blood<br>pressure for Stage 1a and<br>Stage 2a. | Following discussion with the agency on the VAC31518COV1001 protocol, it was agreed that the blood pressure criteria from the CDC list of comorbidities associated with COVID-19 progression could be modified. The VAC31518COV3001 protocol has been harmonized with the VAC31518COV1001 protocol. |
| 1.1 Synopsis 5.1 Inclusion Criteria 5.2 Exclusion Criteria 10.10 Appendix 10: Symptoms of Coronavirus (US Centers for Disease Control and Prevention) | It has been clarified that the current list of CDC comorbidities applicable to the in- and exclusion criteria will not be adjusted during the conduct of the study even if the source CDC list is updated. | Changing the CDC list of comorbidities during the study would be operationally very difficult and should not be required since they are only used in the initial part of the study, ie, in enrollment of the first 2,000 participants in each of the age groups, which will occur only a few weeks apart. |
| <ul><li>1.3.1 All Participants</li><li>5.1 Inclusion Criteria</li><li>5.2 Exclusion Criteria</li><li>8.4 Virology Assessments</li><li>9.7 Safety Analysis</li></ul> | The eligibility criteria, HIV RNA viral load and CD4 cell count assessment and subanalyses of the data related to HIV positive participants in this study has been updated. | To provide objective criteria for stable/well-controlled HIV infection and details regarding this subpopulation on various other study aspects. |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | 2 | |
| 1.1 Synopsis 3 OBJECTIVES AND ENDPOINTS 9.2.3 Immunogenicity Correlates (Correlates Subset) 9.5.2 Secondary Endpoints | The endpoint used to assess the effect of Ad26.COV2.S on all molecularly confirmed symptomatic COVID-19, as compared to placebo was adjusted to the Burden of Disease endpoint. | Following a Health Authority question on how the different groups of mild, moderate and severe COVID-19 cases will be analyzed, the Burden of Disease (BOD) secondary endpoint has been added to the protocol. The BOD endpoint will be evaluated based on the first occurrence of molecularly confirmed COVID-19, including mild, moderate and severe/critical case definitions. |
| 1.1 Synopsis 9.5.1 Primary Endpoint Evaluation 9.5.1.1 Study Monitoring 9.8 Interim Analysis and Committee(s) | The severe harm monitoring rule has been modified to indicate that monitoring will start from the 5 <sup>th</sup> severe event onwards instead of the 8 <sup>th</sup> severe event and monitoring will be done until the primary analysis is triggered instead of until the end of the study. In addition, monitoring for efficacy will start from the 20 <sup>th</sup> event onward at least once a week instead of after each event. | Based on Health Authority request to start monitoring earlier. |
| 1.1 Synopsis 3 OBJECTIVES AND ENDPOINTS 9.5.2 Secondary Endpoints | It has been clarified that all secondary endpoint analyses will occur in the per protocol analysis set, in seronegative participants unless otherwise indicated. | To clarify the analysis set used to evaluate the secondary endpoints. |
| 1.1 Synopsis 8.1.3.1 Case Definition for Moderate to Severe/Critical COVID-19 8.1.3.2 Case Definition for Mild COVID-19 | The case definitions of both mild and moderate COVID-19 have been modified and terminology has been aligned across case definitions. | To incorporate additional key conditions in the case definition of mild disease and for clarification purposes. |
| 1.1 Synopsis 1.3.2 Participants With COVID-19-like Signs and Symptoms 4.1 Overall Design 8.1.1 Prespecified Criteria for Suspected COVID-19 8.1.2 Procedures in the Event of COVID-19-like Signs and Symptoms 4.2.1 Study-Specific Ethical Design Considerations | It has been clarified that because several of the prespecified criteria for suspected COVID-19 overlap with vaccine-related reactogenicity, investigators' clinical judgement is required to exclude vaccine-related events. It has been clarified that the sponsor will also look into the | To ensure that vaccine-related events do not trigger the COVID-19 related follow-up procedures for mild disease, to be able to include cases of moderate disease that were not classifiable by the definition and for simplification and clarification purposes. Based on a partner request to clarify the plans of providing |
| 6.6 Continued Access to Study Vaccine After the End of the Study | possibility of offering placebo recipients the study vaccine, if this vaccine is determined to be efficacious, considering country-specific conditions and ethical considerations. | vaccine, if it is determined to be efficacious, to participants who received placebo. |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.
| Section Number<br>and Name | Description of Change | Brief Rationale |
|---|---|---|
| 5.2 Exclusion Criteria | It has been clarified that every effort will be made to avoid inclusion of participants who have been previously enrolled in coronavirus studies and to prevent subsequent enrollment of a participant in other coronavirus studies during their participation in this study. | To ensure that co-enrollment in other efficacy studies is avoided. |
| 1.1 Synopsis 8.1.3.4 Case Definition for Asymptomatic or Undetected COVID 19 8.1.3.5 SARS-CoV-2 Seroconversion Assessment | A subsection on case definition of asymptomatic or undetected COVID-19 and SARS-CoV-2 seroconversion assessment has been added to the Efficacy Assessment section. | To clarify what is considered an asymptomatic infection. |
| 5.2 Exclusion Criteria | It has been clarified that planning to become pregnant within 3 months after study vaccine administration will lead to exclusion from participation in the study. | For clarification purposes. |
| 1.1 Synopsis 8.1.4 Immunogenicity Assessments | It has been added that serology testing outside the study is discouraged and if testing would be needed, the site will guide the participant to an appropriate assay. | Vaccination with Ad26.COV2.S may interfere with some serologic assays utilized at local community health clinics/commercial laboratories and may result in unblinding the participant. |
| 2.3.1 Risks Related to Study Participation<br>6.8 Prestudy and Concomitant Therapy | Guidance on the use of antipyretics during the study has been added in the prestudy and concomitant therapy section of the protocol. | To clarify that antipyretics are recommended post-vaccination for symptom relief, as needed. Prophylactic antipyretic use is not encouraged. |
| 1.1 Synopsis 1.3.1 All Participants 2.3.1 Risks Related to Study Participation 2.3.3 Benefit-Risk Assessment of Study Participation 4.1 Overall Design 8.3.2 Method of Detecting Adverse Events, Medically-attended Adverse Events, and Serious Adverse Events | It has been clarified that the post-vaccination observation period at the study site will be at least 30 minutes for the first 2,000 participants in each of the 2 age groups and may be decreased to 15 minutes for the remaining participants, if no acute reactions are observed. | To decrease the burden for the participant and for clarification purposes. |
| 1.1 Synopsis 4.1 Overall Design 8.1.4 Immunogenicity Assessments | It has been clarified that the participant will be notified of a confirmed positive SARS-CoV-2 infection and positive serology test. | For clarification purposes. |
| 6.2<br>Preparation/Handling/Storage/Accountability<br>6.4 Study Vaccine Compliance | It has been clarified that the unblinded pharmacist cannot vaccinate participants. | Administration of the vaccine by an unblinded pharmacist is not permitted. |

| Section Number and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 8.1.2 Procedures in the Event of COVID-19-like Signs and Symptoms | It has been clarified that the study staff visiting participants at home will use personal protective equipment according to local regulations. | Based on partner recommendations to include protective measures for site staff visiting participants at home. |
| 8.2.2 Vital Signs | It has been clarified that any vital signs measures taken at home that may trigger the severe/critical case definition will be confirmed as soon as possible by qualified medical staff and participants will be referred for care, if needed. | Based on a partner request to clarify if a participant with a positive test will be referred to a health care provider. |
| 1.1 Synopsis 1.3.1 All Participants 4.1 Overall Design 8.7 Baseline and Longitudinal Risk Factor Assessment 9.4 Participant Information 9.5.3 Exploratory Endpoints 10.12 Appendix 12: Baseline Risk Factor Assessment | It has been added that additional baseline and longitudinal characteristics related to current work situation, living situation, and community interactions, from participants who consent to this, will be collected for risk factor analysis, if allowed per local regulations. | To assess baseline and longitudinal characteristics that are potentially useful to identify the risk of acquiring COVID-19 which will be used for the correlates of protection analysis. |
| 5.2 Exclusion Criteria | Exclusion of participants with drug or alcohol abuse has been removed from exclusion criterion 12. | To avoid redundancy as this is also covered in exclusion criterion 14. |
| 1.1 Synopsis 9.1 Statistical Hypotheses | It has been clarified that additional analyses after the primary analysis can be planned, if deemed appropriate. | For clarification purposes. |
| 1.1 Synopsis 3 Objectives and Endpoints 8.1.4 Immunogenicity Assessments | An exploratory immunogenicity objective/endpoint and respective assays have been added to assess other coronavirus immune responses at baseline. | To assess the impact of pre-<br>existing humoral immunity<br>against coronaviruses other than<br>SARS-CoV-2 at baseline on<br>Ad26.COV2.S vaccine<br>immunogenicity. |
| 2.3.1 Risks Related to Study Participation 5.2 Exclusion Criteria | It has been clarified that breastfeeding women can participate in the study. | To allow the enrollment of breastfeeding women in the study, as the risk of getting infected outweighs the risk of exposing the child to vaccine induced antibodies. |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name 1.1 Synopsis 1.2 Schema 2.1 Study Rationale 4.1 Overall Design | In Stages 1a and 1b combined, the enrollment of participants aged ≥18 to <40 years will be limited to approximately 20% of the total study population. The aim of having a minimum of approximately 25% of recruited participants ≥60 years of age has been adjusted to 30%. | The sponsor believes that Ad26.COV2.S is more likely to protect against more severe disease and progression of infection is age related with twice the level of severity in 50-year-olds compared to 20-year-olds. The cap of approximately 20% of participants 18-40 years and the aim to enroll a minimum of approximately 30% elderly participants, will allow to enroll a more representative population at highest risk of severe disease per the protocol case definition. |
| 5.2 Exclusion Criteria 6.8 Prestudy and Concomitant Therapy 1.1 Synopsis 1.3.1 All Participants 3 OBJECTIVES AND ENDPOINTS 8 STUDY ASSESSMENTS AND PROCEDURES 8.1.3 Efficacy Assessments 8.1.4 Immunogenicity Assessments | In the exclusion criteria and the concomitant medication section, it has been further clarified that the use of any investigational or approved COVID-19 vaccine (other than Ad26.COV2.S) is disallowed at any time prior to and during the study. Blood draws for immunologic testing for SARS-CoV-2 seroconversion (ELISA and/or SARS-CoV-2 immunoglobulin assay) based on SARS-CoV-2 N protein, have been added on Day 71 | Clarification of an inconsistency and alignment across sections within the protocol. To allow for the identification of a possible signal for the prevention of asymptomatic infection at earlier timepoints. |
| 1.3.1 All Participants 1.3.2 Participants With COVID-19-like Signs and Symptoms 2.3.1 Risks Related to Study Participation 8 Study Assessments and Procedures 8.1.2 Procedures in the Event of COVID-19-like Signs and Symptoms 10.2 Appendix 2: Clinical Laboratory Tests 10.8 Medically-attended COVID-19 (MA-COV) Form | and 6 months in order to identify cases of asymptomatic infection. Visit 4 has therefore become a mandatory visit for all participants. The term "mid-turbinate" in relation to the nasal swabs collection has been removed throughout the protocol. | To remove any confusion around the type of swabs used during the study as the swabs currently used are not mid turbinate swabs but their performance can be considered equivalent. |

| Section Number and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| 1.3.2 Participants With COVID-19-like<br>Signs and Symptoms<br>8.1.2 Procedures in the Event of COVID-19-<br>like Signs and Symptoms<br>10.2 Appendix 2: Clinical Laboratory Tests | The sample for sero-<br>confirmation of SARS-CoV-2<br>infection to be collected on<br>Day 3-5 in participants with<br>COVID-19 like signs and<br>symptoms has been removed | It is unlikely to detect antibodies 3-5 days post signs and symptoms or a positive PCR for SARS-COV-2 infection. Antibodies will likely be observed from 7 days post signs and symptoms onwards. |
| 1.1 Synopsis 1.3.1 All Participants 4.1 Overall Design | It has been clarified that enrolled participants will be counselled on SARS-COV-2 infection prevention. In addition, it is clarified that at the time of study entry, each participant will need to indicate to the study site where, in case they would get infected with SARS-CoV-2 the identity and location of their routine medical care physician and/or facility and the identity and location of where they would obtain emergency care and hospitalization if necessary. If this information is not available, a plan for where such care could be obtained should be developed. | For clarification purposes. |
| 1.3.2 Participants With COVID-19-like<br>Signs and Symptoms<br>8.1.2 Procedures in the Event of COVID19-<br>like Signs and Symptoms<br>10.3.3 Informed Consent Process | It has been clarified that the caregiver can only assist with the eCOA. | To provide clarity on the roles and responsibilities of the caregiver. |
| 1.3.2 Participants With COVID-19-like<br>Signs and Symptoms<br>8.1.2 Procedures in the Event of COVID19-<br>like Signs and Symptoms | Term "episode" was added to include all aspects of the COVID-19 illness. | For clarification purposes. |
| 5.1 Inclusion Criteria 8.3 Adverse Events, Serious Adverse Events, Medically-attended Adverse Events, and Other Safety Reporting 10.3.3 Informed Consent Process 10.3.4 Data Protection | References to a legally Acceptable Representative being allowed to provide consent instead of the potential participant has been removed from the protocol. | A participant needs to fully understand and be able to provide consent themselves given there may be no benefit to participation. Participants unable to consent for themselves should not be enrolled in the study. |
| 1.1 Synopsis 2.1 Study Rationale 2.3.3 Benefit-Risk Assessment of Study Participation 4.1 Overall Design 9.8 Interim Analysis and Committee(s) 10.3.6 Committees Structure | Reference to Grade 4 AEs and SAEs in the context of Day 3 safety review by the DSMB has been deleted from the protocol. | The DSMB review of the Day 3 safety data from Stage 1a and 2a prior to enrollment of Stage 1b and 2b, respectively, will not be limited to Grade 4 AEs and SAEs. All available safety data will be reviewed. |

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | |
| <ul> <li>1.1 Synopsis</li> <li>2.1 Study Rationale</li> <li>4.1 Overall Design</li> <li>9.5.1 Primary Endpoint Evaluation</li> <li>9.8 Interim Analysis and Committee(s)</li> <li>10.3.6 Committees Structure</li> </ul> | The role of the Sponsor<br>Committee has been replaced<br>either by the role of the<br>Oversight Group (as described<br>in the Oversight Group<br>Charter) or the role of the | For clarification purposes. |
| | sponsor. | |
| 2.3.1 Risks Related to Study Participation | Influenza will not be used as a control in the surveillance system for detection of COVID-19. | Influenza may not serve as a good positive control due to social distancing measures and the need for significant sampling to have a valid comparison. |
| 6.10 Study Vaccination Pausing Rules for Stages 1a and 2a | It has been clarified that based on the pausing criteria, the sponsor's medical monitor or designee decides whether a study pause is warranted and informs the DSMB of the decision, instead of the PSRT deciding whether a pausing rule is warranted. | For clarification purposes. |
| 9.5.2 Secondary Endpoints | It has been clarified that among participants with SARS-CoV-2 infection, the effect of vaccination on the viral load levels at and after diagnosis as well as on the duration of SARS-CoV-2 viral load positivity will be evaluated. | For clarification purposes. |
| 1.1 Synopsis 3 OBJECTIVES AND ENDPOINTS | The exploratory efficacy objective assessing both symptomatic and asymptomatic infections combined, (that are serologically and/or molecularly confirmed) compared to placebo has been moved to the secondary objectives. | This endpoint was moved to secondary as it will be included in the inferential testing strategy. |
| 3 OBJECTIVES AND ENDPOINTS | An exploratory objective to assess the impact of the vaccine on other respiratory diseases has been added. | To obtain epidemiology data of other important respiratory infections that may be affected by COVID-19 circulation. |
| 1.1 Synopsis<br>8.1.4 Immunogenicity Assessments | Analysis of neutralizing antibodies to SARS-CoV-2 using a reporter SARS-CoV-2 virus has been added. | To add a new assay that may become available. |
| 10.7 Appendix 7: MRU Questionnaire | Clarifications were made in the MRU Questionnaire. | For clarification purposes |

## VAC31518 (JNJ-78436735)

| Section Number | Description of Change | Brief Rationale |
|---|---|---|
| and Name | | |
| Throughout the protocol | Minor errors and | Correction of minor errors and |
| | inconsistencies were | inconsistencies. Addition of |
| | corrected, and minor | minor clarifications. |
| | clarifications were added | |
| | throughout the protocol. | |

## 11. REFERENCES

- 1. Agrawal AS, Tao X, Algaissi A, et al. Immunization with inactivated Middle East Respiratory Syndrome coronavirus vaccine leads to lung immunopathology on challenge with live virus. Hum Vaccin Immunother. 2016;12(9):2351-2356.
- 2. American Society of Hematology. COVID-19 resources. Thrombosis with Thrombocytopenia Syndrome (also termed Vaccine-induced Thrombotic Thrombocytopenia). https://www.hematology.org/covid-19/vaccine-induced-immune-thrombotic-thrombocytopenia. Accessed: 27 April 2021.
- 3. Anywaine Z, Whitworth H, Kaleebu P, et al. Safety and Immunogenicity of a 2-Dose Heterologous Vaccination Regimen With Ad26.ZEBOV and MVA-BN-Filo Ebola Vaccines: 12-Month Data From a Phase 1 Randomized Clinical Trial in Uganda and Tanzania. J Infect Dis. 2019;220(1):46-56.
- 4. Barouch DH, Liu J, Peter L, et al. Characterization of humoral and cellular immune responses elicited by a recombinant adenovirus serotype 26 HIV-1 Env vaccine in healthy adults (IPCAVD 001). J Infect Dis. 2013:207(2);248-256.
- 5. Barouch DH, Tomaka FL, Wegmann F, et al. Evaluation of a mosaic HIV-1 vaccine in a multicentre, randomised, double-blind, placebo-controlled, phase 1/2a clinical trial (APPROACH) and in rhesus monkeys (NHP 13-19). Lancet. 2018;392(10143):232-243.
- 6. Berry JD, Jones S, Drebot MA, et al. Development and characterisation of neutralising monoclonal antibody to the SARS-coronavirus. J Virol Methods. 2004;120(1):87-96.
- 7. Bisht H, Roberts A, Vogel L, et al. Severe acute respiratory syndrome coronavirus spike protein expressed by attenuated vaccinia virus protectively immunizes mice. Proc Natl Acad Sci USA. 2004;101(17):6641-6646.
- 8. Bolles M, Deming D, Long K, et al. A double-inactivated severe acute respiratory syndrome coronavirus vaccine provides incomplete protection in mice and induces increased eosinophilic proinflammatory pulmonary response upon challenge. J Virol. 2011;85(23):12201-12215.
- 9. Updated Proposed Brighton Collaboration process for developing a standard case definition for study of new clinical syndrome X, as applied to Thrombosis with Thrombocytopenia Syndrome (TTS). 18 May 2021. https://brightoncollaboration.us/wp-content/uploads/2021/05/TTS-Interim-Case-Definition-v10.16.3-May-23-2021.pdf .Accessed: 02 September 2021.
- British Society for Haematology. Guidance produced from the Expert Haematology Panel (EHP) focussed on Covid-19 Vaccine induced Thrombosis and Thrombocytopenia (VITT). https://b-sh.org.uk/media/19530/guidance-version-13-on-mngmt-of-thrombosis-with-thrombocytopenia-occurring-afterc-19-vaccine 20210407.pdf. Version 1.3; 7 April 2021. Accessed: 27 April 2021.
- 11. Buchholz UJ, Bukreyev A, Yang L, et al. Contributions of the structural proteins of severe acute respiratory syndrome coronavirus to protective immunity. Proc Natl Acad Sci USA. 2004;101(26):9804-9809.
- 12. Bukreyev A, Lamirande EW, Buchholz UJ, et al. Mucosal immunisation of African green monkeys (Cercopithecus aethiops) with an attenuated parainfluenza virus expressing the SARS coronavirus spike protein for the prevention of SARS. Lancet. 2004;363(9427):2122-2127.
- Center for Disease Control and Prevention. Multisystem Inflammatory Syndrome in Children (MIS-C)
   Associated with Coronavirus Disease 2019 (COVID-19). Available at:
   https://emergency.cdc.gov/han/2020/han00432.asp. Accessed: 15 May 2020.
- 14. Center for Disease Control and Prevention. Symptoms of Coronavirus. https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html. Accessed on 22 July 2020.
- 15. Centers for Disease Control and Prevention (CDC). Cases of cerebral venous sinus thrombosis with thrombocytopenia after receipt of the Johnson & Johnson COVID-19 Vaccine. 13 April 2021. https://emergency.cdc.gov/han/2021/han00442.asp. Accessed: 27 April 2021.
- Centers for Disease Control and Prevention. Coronavirus Disease 2019 (COVID-19) Symptoms and Complications. https://www.cdc.gov/coronavirus/2019-ncov/about/symptoms.html. Accessed 15 February 2020.

- 17. Centers for Disease Control and Prevention. Coronavirus Disease 2019 (COVID-19) Groups at Higher Risk for Severe Illness. https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/groups-at-higher-risk.html. Accessed 19 July 2020.
- 18. Centers for Disease Control and Prevention. COVID-19 Response Team. Coronavirus disease 2019 in children United States, February 12–April 2, 2020. Morb Mortal Wkly Rep 2020;69:422–426.
- 19. Centers for Disease Control and Prevention. Reproductive Health: Contraception. https://www.cdc.gov/reproductivehealth/contraception/index.htm. Accessed 23 November 2020.
- 20. Chan JF, Lau SK, To KK, Cheng VC, Woo PC, Yuen KY. Middle East respiratory syndrome coronavirus: another zoonotic betacoronavirus causing SARS-like disease. Clin. Microbiol. Rev. 2015; 28(2):465–522.
- 21. Chen N, Zhou M, Dong X, et al. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020;395(10223):507-513.
- 22. Chen Z, Zhang L, Qin C, et al. Recombinant modified vaccinia virus Ankara expressing the spike glycoprotein of severe acute respiratory syndrome coronavirus induces protective neutralizing antibodies primarily targeting the receptor binding region. J Virol. 2005;79(5):2678-2688.
- 23. Chin J, Magoffin RL, Shearer LA, Schieble JH, Lennette EH. Field evaluation of a respiratory syncytial virus vaccine and a trivalent parainfluenza virus vaccine in a pediatric population. Am J Epidemiol. 1969;89(4);449-463.
- 24. Clinical Study Report VAC31518COV1002. Cohort 1 and Cohort 2 Interim Clinical Study Report. A Randomized, Double-blind, Placebo-controlled Phase 1 Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Ad26.COV2.S in Adults. Janssen Pharmaceutical K.K. (04 August 2021).
- 25. Colby DJ, Sarnecki M, Barouch DH, et al. Safety and immunogenicity of Ad26 and MVA vaccines in acutely treated HIV and effect on viral rebound after antiretroviral therapy interruption. Nat Med. 2020;26(4):498-501.
- 26. Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020;5(4):536-544.
- 27. Cyranoski D. The biggest mystery: what it will take to trace the coronavirus source. Nature news; 5 June 2020. doi: 10.1038/d41586-020-01541-z.
- 28. Deming D, Sheahan T, Heise M, et al. Vaccine efficacy in senescent mice challenged with recombinant SARS-CoV bearing epidemic and zoonotic spike variants. PLoS Med. 2006;3(12):e525.
- 29. Dong Y, Mo X, Hu Y, et al. Epidemiological Characteristics of 2143 Pediatric Patients With 2019 Coronavirus Disease in China. Pediatrics. 2020 Mar 16. pii: e20200702. [Epub ahead of print]
- 30. Dragalin V, Fedorov V, Cheuvart B. Statistical approaches to establishing vaccine safety. Statistics in Medicine. 2002;21, 877–893.
- 31. Dragalin V. and Fedorov V. (2006) 'Multistage Designs for Vaccine Safety Studies', Journal of Biopharmaceutical Statistics. 2006;16:4:539-553.
- 32. European Centre for Disease Prevention and Control. Factsheet for health professionals on coronaviruses. https://www.ecdc.europa.eu/en/factsheet-health-professionals-coronaviruses. Accessed 15 February 2020.
- 33. Faber M, Lamirande EW, Roberts A, et al. A single immunization with a rhabdovirus-based vector expressing severe acute respiratory syndrome coronavirus (SARS-CoV) S protein results in the production of high levels of SARS-CoV-neutralizing antibodies. J Gen Virol. 2005;86(Pt 5):1435-1440.
- 34. Follmann D, Fintzi J, Fay MP, Janes HE, Baden L, El Sahly H, et al. Assessing Durability of Vaccine Effect Following Blinded Crossover in COVID-19 Vaccine Efficacy Trials. medRxiv 2020. https://doi.org/10.1101/2020.12.14.20248137
- 35. Fulginiti VA, Eller JJ, Sieber OF, Joyner JW, Minamitani M, Meiklejohn G. Respiratory virus immunization. I. A field trial of two inactivated respiratory virus vaccines; an aqueous trivalent parainfluenza virus vaccine and an alum-precipitated respiratory syncytial virus vaccine. Am J Epidemiol. 1969:89(4);435-448.

- Garg S, Kim L, Whitaker M, et al. Hospitalization rates and characteristics of patients hospitalized with laboratory-confirmed coronavirus disease 2019 — COVID-NET, 14 States. Morb Mortal Wkly Rep 2020;69:458–464.
- 37. Gidudu JK, Walco GA, Taddio A, et al./The Brighton Immunization Site Pain Working Group. Immunization site pain: Case definition and guidelines for collection, analysis, and presentation of immunization safety data. Vaccine. 2012:30(30);4558-4577.
- 38. Gray G, Bekker L-G. Sisonke Update on the Janssen®(JNJ) Ad26.COV2.S vaccine. https://sacoronavirus.co.za/wp-content/uploads/2021/08/Sisonke-Provisional-Results-6-August-2021GG2.pdf (accessed August 23, 2021).
- Honda-okubo Y, Barnard D, Ong CH, Peng BH, Tseng CT, Petrovsky N. Severe acute respiratory syndromeassociated coronavirus vaccines formulated with delta inulin adjuvants provide enhanced protection while ameliorating lung eosinophilic immunopathology. J Virol. 2015;89(6):2995-3007.
- 40. Houser KV, Broadbent AJ, Gretebeck L, et al. Enhanced inflammation in New Zealand white rabbits when MERS-CoV reinfection occurs in the absence of neutralizing antibody. PLoS Pathog. 2017;13(8):e1006565.
- 41. Investigator's Brochure: Ad26COVS1 (VAC31518), Edition 1.0. Addendum 1. Janssen Vaccines & Prevention B.V. (July 2020).
- 42. Investigator's Brochure: VAC31518 (JNJ-78436735), Edition 4.0. Janssen Vaccines & Prevention B.V. (February 2021).
- 43. Janssen Vaccines & Prevention B.V. Data on file.
- Johns Hopkins CSSE. Coronavirus COVID-19 Global Cases. https://gisanddata.maps.arcgis.com/apps/opsdashboard/index.html#/bda7594740fd40299423467b48e9ecf6. Accessed 2 Jun 2020.
- 45. Kapikian AZ, Mitchell RH, Chanock RM, Shvedoff RA, Stewart CE. An epidemiologic study of altered clinical reactivity to respiratory syncytial (RS) virus infection in children previously vaccinated with an inactivated RS virus vaccine. Am J Epidemiol. 1969:89;405-421.
- 46. Kim HW, Canchola JG, Brandt CD, et al. Respiratory syncytial virus disease in infants despite prior administration of antigenic inactivated vaccine. Am J Epidemiol. 1969:89(4);422-434.
- 47. Kohl KS, Walop W, Gidudu J, et al./The Brighton Collaboration Local Reaction Working Group for Swelling at or near Injection Site. Swelling at or near injection site: Case definition and guidelines for collection, analysis and presentation of immunization safety data. Vaccine 2007:31;5858-5874.
- 48. Letko M, Marzi A, Munster V. Functional assessment of cell entry and receptor usage for SARS-CoV-2 and other lineage B betacoronaviruses. Nat Microbiol. 2020;5:562–569.
- 49. Li Q, Guan X, Wu P, et al. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020;382(13):1199-1207.
- 50. Lu R, Zhao X, Li J, et al. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Jan 30. pii: S0140-6736(20)30251-8.
- 51. Marcy SM, Kohl KS, Dagan R, et al./The Brighton Collaboration Fever Working Group. Fever as an adverse event following immunization: case definition and guidelines of data collection, analysis, and presentation. Vaccine 2004:22(5-6);551-556.
- 52. Mercado NB, Zahn R, Wegmann F, et al. Single-shot Ad26 vaccine protects against SARS-CoV-2 in rhesus macaques. Nature. 2020. https://doi.org/10.1038/s41586-020-2607-z.
- 53. Milligan ID, Gibani MM, Sewell R, et al. Safety and immunogenicity of novel adenovirus type 26- and modified vaccinia ankara-vectored ebola vaccines: a randomized clinical trial. JAMA. 2016:315;1610-1623.
- 54. Modjarrad K, Roberts CC, Mills KT, et al. Safety and immunogenicity of an anti-Middle East respiratory syndrome coronavirus DNA vaccine: a phase 1, open-label, single-arm, dose-escalation trial. Lancet Infect Dis. 2019;19(9):1013-1022.
- 55. Moghaddam A, Olszewska W, Wang B, et al. A potential molecular mechanism for hypersensitivity caused by formalin-inactivated vaccines. Nat Med. 2006:12(8);905-907.

- 56. Mutua G, Anzala O, Luhn K, et al. Safety and Immunogenicity of a 2-Dose Heterologous Vaccine Regimen With Ad26.ZEBOV and MVA-BN-Filo Ebola Vaccines: 12-Month Data From a Phase 1 Randomized Clinical Trial in Nairobi, Kenya. J Infect Dis. 2019;220(1):57-67.
- 57. Salisch NC, Izquierdo gil A, Czapska-casey DN, et al. Adenovectors encoding RSV-F protein induce durable and mucosal immunity in macaques after two intramuscular administrations. NPJ Vaccines. 2019;4:54.
- 58. Smatti MK, Al Thani AA, Yassine HM. Viral-Induced Enhanced Disease Illness. Front Microbiol. 2018;9:2991.
- 59. Stephenson KE, Wegmann F, Tomaka F, et al. Comparison of shortened mosaic HIV-1 vaccine schedules: a randomised, double-blind, placebo-controlled phase 1 trial (IPCAVD010/HPX1002) and a preclinical study in rhesus monkeys (NHP 17-22). Lancet HIV. 2020; Erratum in: Lancet HIV. 2020 Feb 28.
- 60. Subbarao K, Mcauliffe J, Vogel L, et al. Prior infection and passive transfer of neutralizing antibody prevent replication of severe acute respiratory syndrome coronavirus in the respiratory tract of mice. J Virol. 2004;78(7):3572-3577.
- 61. Sui J, Li W, Roberts A, et al. Evaluation of human monoclonal antibody 80R for immunoprophylaxis of severe acute respiratory syndrome by an animal study, epitope mapping, and analysis of spike variants. J Virol. 2005;79(10):5900-5906.
- 62. US Department of Health and Human Services Office of the Assistant Secretary for Planning and Evaluation. Health Insurance Portability and Accountability Act of 1996. Available at: https://aspe.hhs.gov/report/health-insurance-portability-and-accountability-act-1996. Accessed: 5 November 2020.
- 63. US Department of Health and Human Services, Food and Drug Administration, Center for Biologics Evaluation and Research. September 2007. Guidance for Industry. Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Available from: https://www.fda.gov/media/73679/download. Accessed: 19 Feb 2020.
- 64. US Department of Health and Human Services. Office for Human Research Protections OHRP Expedited Review Categories. 1998. https://www.hhs.gov/ohrp/regulations-and-policy/guidance/categories-of-research-expedited-review-procedure-1998/index.html. Accessed 24 February 2020.
- 65. US Food and Drug Administration. Conditions for IRB Use of Expedited Review. Federal Register: November 9, 1998 (Volume 63, Number 216). https://www.fda.gov/science-research/guidance-documents-including-information-sheets-and-notices/conditions-irb-use-expedited-review. Accessed 24 February 2020.
- 66. US Food and Drug Administration. COVID-19: Developing Drug and Biological Products for Treatment or Prevention. Guidance for Industry. May 2020. Accessed 20 July 2020.
- 67. US Food and Drug Administration. Development and Licensure of Vaccines to Prevent COVID-19. Guidance for Industry. June 2020. https://www.fda.gov/media/139638/download. Accessed 20 July 2020.
- 68. van der Fits L, Bolder R, Heemskerk-van der Meer M, et al. Adenovector 26 encoded prefusion conformation stabilized RSV-F protein induces long-lasting Th1-biased immunity in neonatal mice. NPJ Vaccines. 2020 [provisionally accepted for publication]
- 69. Verdoni L, Mazza A, Gervasoni A, Martelli L et al. An outbreak of severe Kawasaki-like disease at the Italian epicenter of the SARS-CoV-2 epidemic: an observational cohort study. The Lancet. Published Online May 13, 2020 https://doi.org/10.1016/S0140-6736(20)31103-X.
- Widjojoatmodjo MN, Bogaert L, Meek B, et al. Recombinant low-seroprevalent adenoviral vectors Ad26 and Ad35 expressing the respiratory syncytial virus (RSV) fusion protein induce protective immunity against RSV infection in cotton rats. Vaccine. 2015;33(41):5406-5414.
- World Health Organization. Clinical management of severe acute respiratory infection (SARI) when COVID-19 disease is suspected. Interim guidance, 13 March 2020. https://www.who.int/docs/defaultsource/coronaviruse/clinical-management-of-novel-cov.pdf. Accessed 12 May 2020.
- 72. World Health Organization. WHO Director-General's opening remarks at the media briefing on COVID-19 11 March 2020. https://www.who.int/dg/speeches/detail/who-director-general-s-opening-remarks-at-the-media-briefing-on-covid-19--11-march-2020. Accessed 12 March 2020.

- World Health Organization. WHO guidelines for the global surveillance of severe acute respiratory syndrome (SARS). Updated recommendations, October 2004. https://www.who.int/csr/resources/publications/WHO CDS CSR ARO 2004 1/en/. Accessed 15 February 2020.
- 74. Wu F, Zhao S, Yu B, et al. A new coronavirus associated with human respiratory disease in China. Nature. 2020;579(7798):265-269.
- 75. Yang ZY, Kong WP, Huang Y, et al. A DNA vaccine induces SARS coronavirus neutralization and protective immunity in mice. Nature. 2004;428(6982):561-564.
- 76. Zahn R, Gillisen G, Roos A, et al. Ad35 and Ad26 vaccine vectors induce potent and cross-reactive antibody and T-cell responses to multiple filovirus species. PLoS ONE. 2012;7(12):e44115.
- 77. Zhang H, Wang G, Li J, et al. Identification of an antigenic determinant on the S2 domain of the severe acute respiratory syndrome coronavirus spike glycoprotein capable of inducing neutralizing antibodies. J Virol. 2004;78(13):6938-6945.
- 78. Zhao J, Alshukairi AN, Baharoon SA, et al. Recovery from the Middle East respiratory syndrome is associated with antibody and T-cell responses. Sci Immunol. 2017;2(14). pii: eaan5393.
- 79. Zhou P, Yang XL, Wang XG, et al. A pneumonia outbreak associated with a new coronavirus of probable bat origin. Nature. 2020;579(7798):270-273.
- 80. Zhou T, Wang H, Luo D, et al. An exposed domain in the severe acute respiratory syndrome coronavirus spike protein induces neutralizing antibodies. J Virol. 2004;78(13):7217-7226.
- 81. Zumla A, Chan JF, Azhar EI, Hui DS, Yuen KY. Coronaviruses drug discovery and therapeutic options. Nat Rev Drug Discov. 2016;15(5):327-347.

## **INVESTIGATOR AGREEMENT**

I have read this protocol and agree that it contains all necessary details for carrying out this study. I will conduct the study as outlined herein and will complete the study within the time designated.

I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of this study. I will discuss this material with them to ensure that they are fully informed regarding the study intervention, the conduct of the study, and the obligations of confidentiality.

| Coordinating Investigato | r (where required): | | |
|---|---|---|---|
| Name (typed or printed): | | | |
| Institution and Address: | | | |
| Signature: | | Date: | |
| | | | (Day Month Year) |
| Principal (Site) Investiga | tor: | | |
| Name (typed or printed): | | | |
| Institution and Address: | | | |
| Telephone Number: | | | |
| Signature: | | Date: | |
| | | | (Day Month Year) |
| Sponsor's Responsible M | edical Officer: | | |
| Name (typed or printed): | Jerald Sadoff, MD | | |
| Institution: | Janssen Research & Development | | |
| Signature: electronic sig | nature appended at the end of the protocol | Date: | |
| | | | (Day Month Year) |

**Note:** If the address or telephone number of the investigator changes during the study, written notification will be provided by the investigator to the sponsor, and a protocol amendment will not be required.

## **Signature**

| User | Date | Reason |
|------------------|----------------------------------|-------------------|
| Sadoff Jerry PPD | 15-Apr-2022<br>16:19:00<br>(GMT) | Document Approval |